### 16.1.9 Documentation of Statistical Methods

### 16.1.9.1 Statistical Analysis Plans

Statistical Analysis Plan version 1.0 dated 22 December 2015 Statistical Analysis Plan version 2.0 dated 13 January 2017

### 16.1.9.2 Method for Analysis of Abuse Related Adverse Events

**Abuse Assessment Section Terms** 

Acorda Therapeutics, Inc. CVT-301-005





### Statistical Analysis Plan

| Document<br>Type: | Template | Document ID: |
|-------------------|-------------|-----------------------------|
| Issue Date: | 02 APR 2012 | Effective Date: 30 APR 2012 |

Sponsor Name: Civitas Therapeutics, Inc.

Protocol Number and Title: CVT-301-005

A Phase 3, Randomized Study Investigating the

Safety of CVT-301 (Levodopa Inhalation Powder) in Parkinson's Disease Patients With Motor Response Fluctuations (OFF Phenomena) Compared to an Observational Cohort Control

(SUPPORT-PD™)

**Protocol Version and Date:** Version 3.0, 19-Aug-2015

INC Research Project Code:

Author(s):

SAP Version: Final Version 1.0

SAP Version Date: 22-Dec-2015

### Notice of Confidential and Proprietary Information:

The information contained in this document is confidential belonging to Civitas Therapeutics, Inc. Acceptance of this document constitutes agreement by the recipient that no information contained herein will be published or disclosed without prior written authorization from an official of Civitas Therapeutics, Inc. However, this document may be disclosed to appropriate Institutional Review Board and Ethics Committees or duly authorized representatives of a national regulatory authority under the condition that they are requested to keep it confidential. In the event of an actual or suspected breach of this obligation, INC Research should be notified promptly.



### Statistical Analysis Plan

Version:

Final Version 1.0

**Version Date:** 

22-Dec-2015

I confirm that I have reviewed this document and agree with the content.



This document is proprietary and confidential to INC Research LLC. INC Research  $\Phi$  LLC

03.007A.00

Page 2 of 66



## **TABLE OF CONTENTS**

| 1. | GLOSSARY OF ABBREVIATIONS | 6 |
|------------|------------------------------------|----|
| 2. | PURPOSE | 9 |
| 2.1. | Responsibilities | 9 |
| 2.2. | Timings of Analyses | 9 |
| 3. | STUDY OBJECTIVES AND STUDY DESIGN | 10 |
| 3.1. | Primary Objective | 10 |
| 3.2. | Secondary Objectives | 10 |
| 3.3. | Exploratory Efficacy Objectives | 10 |
| • | Patient Selection | 12 |
| 3.5. | Determination of Sample Size | 14 |
| 3.6. | Treatment Assignment & Blinding | 15 |
| 3.7. | Administration of Study Medication | 15 |
| 3.8. | Study Procedures and Flowchart | 16 |
| 4. | ENDPOINTS | 19 |
| 4.1. | Primary Endpoint | 19 |
| 4.2. | Secondary Endpoints | 19 |
| 4.3. | Exploratory EffiCacy Endpoints | 20 |
| <b>5</b> . | ANALYSIS SETS | 24 |
| 5.1. | All Available Population (AAP) | 24 |



### Final Version 1.0

# Statistical Analysis Plan

| 5.2. | Safety population | 4 |
|---|---|---|
| 5.3. | Intent-to-Treat population (ITT)2 | 4 |
| 5.4. | Protocol Deviations | 4 |
| 6. | GENERAL ASPECTS FOR STATISTICAL ANALYSIS2 | 6 |
| 6.1. | General Methods2 | 6 |
| 6.2. | Key Definitions2 | 7 |
| 6.3. | Missing Data2 | 9 |
| 6.4. | Visit Windows | 0 |
| 6.5. | Pooling of sites | 1 |
| 6.6. | Subgroups | 1 |
| 7. | DEMOGRAPHIC, OTHER BASELINE CHARACTERISTICS AND MEDICATION3 | 2 |
| 7.1. | Patient Disposition and Withdrawals3 | 2 |
| 7.1.<br>7.2. | Patient Disposition and Withdrawals | |
| | | 2 |
| 7.2. | Demographic and Other Baseline Characteristics | 2 |
| 7.2.<br>7.3. | Demographic and Other Baseline Characteristics | 4 |
| <ul><li>7.2.</li><li>7.3.</li><li>7.4.</li></ul> | Demographic and Other Baseline Characteristics | 2<br>4<br>4<br>6 |
| <ul><li>7.2.</li><li>7.3.</li><li>7.4.</li><li>8.</li></ul> | Demographic and Other Baseline Characteristics | 4 4 6 |
| <ul><li>7.2.</li><li>7.3.</li><li>7.4.</li><li>8.</li><li>8.1.</li></ul> | Demographic and Other Baseline Characteristics | 2<br>4<br>4<br>6<br>8 |
| 7.2.<br>7.3.<br>7.4.<br>8.<br>8.1.<br>8.2. | Demographic and Other Baseline Characteristics | 2<br>4<br>4<br>6<br>6<br>8 |
| 7.2.<br>7.3.<br>7.4.<br>8.<br>8.1.<br>8.2.<br>8.3. | Demographic and Other Baseline Characteristics | 2<br>4<br>4<br>6<br>8<br>9 |




# Statistical Analysis Plan

| 8.7. | Electrocardiogram | 43 |
|---|---|---|
| 8.8. | Physical Examination | 44 |
| 8.9. | Columbia-Suicidality Severity Rating Scale | 44 |
| 8.10. | Epworth Sleepiness Scale | 45 |
| 8.11. | Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease | 45 |
| 8.12. | UPDRS part 4 | 46 |
| 8.13. | examiner-rated dyskinesia | 46 |
| 9. E | EXPLORATORY EFFICACY | 47 |
| 9.1. | Exploratory Efficacy Endpoint and Analysis | 47 |
| 10. | INTERIM ANALYSES | 50 |
| 11. | CHANGE FROM ANALYSIS PLANNED IN PROTOCOL | 51 |
| 12. | PROGRAMMING CONSIDERATIONS | 52 |
| 12.1. | General Considerations | 52 |
| 12.2.<br>12.2<br>12.2<br>12.2<br>12.2<br>12.2 | 2.2. Headers | 52<br>53<br>53 |
| 13. | QUALITY CONTROL | 56 |
| 14. | INDEX OF TABLES | 57 |
| 15. | INDEX OF LISTINGS | 64 |
| 16. | INDEX OF FIGURES | 66 |



## 1. GLOSSARY OF ABBREVIATIONS

| Abbreviation | Description |
|--------------|--------------------------------------------|
| AAP | All Available Population |
| ADL | Activities of Daily Living |
| AE | Adverse Event |
| ANCOVA | Analysis of Covariance |
| ATC | Anatomical Therapeutic Chemical |
| ATS | American Thoracic Society |
| BMI | Body Mass Index |
| BMS | Biomedical Systems |
| ВР | Blood Pressure |
| CI | confidence interval |
| СМН | Cochran-Mantel-Haenszel |
| COPD | Chronic Obstructive Pulmonary Disease |
| CRO | Contract Research Organization |
| C-SSRS | Columbia-Suicidality Severity Rating Scale |
| DBP | diastolic blood pressure |
| DDI | Dopamine Decarboxylase Inhibitor |
| DL | Dose Level |
| DLco | Carbon Monoxide Diffusion Capacity |
| DSMC | Data Safety Monitoring Committee |
| ECG | Electrocardiogram |
| ERS | European Respiratory Society |
| ET | Early Termination |
| FEV1 | Forced Expiratory Volume in 1 second |
| FVC | Forced Vital Capacity |
| Hb | hemoglobin |
| HR | Heart Rate |



| Abbreviation | Description |
|---|---|
| IEC | Independent Ethics Committee |
| IFU | Instructions for Use |
| IRB | Institutional Review Board |
| ITT | Intent-to-Treat |
| IWRS | Interactive Web Response System |
| LD | Levodopa |
| LS | least square |
| MAR | Missing At Random |
| MCMC | Markov Chain Monte Carlo |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MI | Multiple Imputation |
| MMSE | Mini Mental State Examination |
| MMRM | Mixed Model for Repeated Measures |
| PCS | potentially clinically significant values |
| PCSC | potentially clinically significant changes |
| PD | Parkinson's Disease |
| PDQ-39 | 39-Item Parkinson's Disease Questionnaire |
| PGI-C | Patient Global Impression of Change |
| PMM | Pattern Mixture Models |
| PRN | As needed |
| PT | Preferred Term |
| QUIP | Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease |
| QTcB | QT interval corrected using Bazett's formula |
| QTcF | QT interval corrected using Fridericia's formula |
| RR | Respiratory Rate |
| S&E | Schwab and England |
| SAP | Statistical Analysis Plan |



# Statistical Analysis Plan

| Abbreviation | Description |
|--------------|---------------------------------------------|
| SBP | systolic blood pressure |
| SD | Standard Deviation |
| SEM | Standard Error of the Mean |
| SI | International System of Units |
| SOC | System Organ Class |
| SV | Screening Visit |
| TEAE | Treatment-Emergent Adverse Event |
| TLF | tables, listings, figure |
| TV | Treatment Visit |
| UPDRS | RS Unified Parkinson's Disease Rating Scale |
| WHO-DD | World Health Organization Drug Dictionary |



### Statistical Analysis Plan

### 2. PURPOSE

The purpose of this statistical analysis plan (SAP) is to ensure that the data listings, summary tables and figures which will be produced, and the statistical methodologies that will be used, are complete and appropriate to allow valid conclusions regarding the study objectives.

This SAP describes the statistical analysis as it is foreseen at the time of planning the study. The SAP will serve as a compliment to the study protocol and supersedes it in case of differences. In case of major differences between the study protocol and SAP (e.g. changes in the analysis related to the primary endpoint) protocol amendment will be considered. The SAP may be updated during the conduct of the study and will be finalized before database lock. However, because this is an open-label study, the analyses defined after the first patient has been randomized to the study will be considered as exploratory.

#### 2.1. RESPONSIBILITIES

INC Research will perform the statistical analyses and are responsible for the production and quality control of all tables, figures and listings. Acorda (or it's designee) will review and approve all statistical work done by INC Research as agreed between INC Research and Acorda.

### 2.2. TIMINGS OF ANALYSES

The primary analysis of safety and efficacy is planned after all patients complete the final study visit or terminate early from the study, and database is cleaned and locked.



### 3. STUDY OBJECTIVES AND STUDY DESIGN

#### 3.1. PRIMARY OBJECTIVE

To characterize the pulmonary safety, as assessed by spirometry (forced expiratory volume in 1 second [FEV1], forced vital capacity [FVC], and FEV1/ FVC ratio), over a 12-month period within the CVT-301-treated patients.

#### 3.2. SECONDARY OBJECTIVES

- To characterize the pulmonary safety, as assessed by spirometry (FEV1, FVC and FEV1/FVC ratio), over a 12-month period in the observational ('standard of care') cohort.
- To estimate the difference between the CVT-301-treated patients and the observational cohort on measures of pulmonary safety.
- To characterize the effects of CVT-301 on safety over a 12-month period: safety will be assessed by adverse event (AE) reports, physical examination, standard and orthostatic vital signs (blood pressure [BP], heart rate [HR], and respiratory rate [RR]), clinical laboratory tests, 12-lead electrocardiograms (ECGs), the Parkinson's Disease Impulsive-Compulsive Disorders Questionnaire (QUIP), the Epworth Sleepiness Scale, and the Columbia-Suicide Severity Rating Scale (C-SSRS).
- To evaluate the effect of CVT-301 on mean change from baseline in the UPDRS Part 4 measures of motor fluctuations (dyskinesias [Q32-35] and wearing off [Q36-39]) measured at baseline and at 6 and 12 months after the initiation of CVT-301 treatment.
- To characterize the occurrence and severity of examiner-rated dyskinesia following treatment of patients experiencing an OFF episode in the clinic over a 12-month period.
- To describe the effects of CVT-301 on Carbon Monoxide Diffusion Capacity (DLco) over a 12-month period.

### 3.3. EXPLORATORY EFFICACY OBJECTIVES

The following exploratory objectives related to the efficacy endpoints will primarily be assessed for the CVT-301-treated patients. The same objectives will be explored for the pool of CVT-301-naïve patients and patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies, if feasible.



- Change from pre-dose in UPDRS Part 3 motor score at 10, 20, 30, and 60 minutes following treatment of patients experiencing an OFF episode.
- Time curves of the UPDRS response at 10, 20, 30 and 60 minutes will be evaluated descriptively
- Change from pre-dose in the average UPDRS Part 3 motor score at 10 to 60 minutes following treatment of patients experiencing an OFF episode.
- Proportion of patients with a ≥ 3, ≥ 6, and ≥ 11 point reduction in the UPDRS Part 3 motor score from pre-dose to post-dose, at 10, 20, 30, and 60 minutes.
- Proportion of patients achieving resolution of an OFF to an ON state within 60 minutes after study drug is administered in the clinic, maintaining the ON state at 60 minutes after study drug administration (per the examiner's subjective assessment).
- Total daily OFF time, total daily ON time without dyskinesia, total daily ON time with non-troublesome dyskinesia, and total daily ON time with troublesome dyskinesia, assessed by the patient and recorded in the patient diary.
- Change from baseline in 39-Item Parkinson's Disease Questionnaire (PDQ-39).
- Proportion of patients who improved based on the Patient Global Impression of Change (PGI-C) rating scale.
- Change from baseline in Schwab and England (S&E) Activities of Daily Living (ADL).
- Change from baseline in UPDRS Part 2 score.

#### 3.4. PATIENT SELECTION

The study population for this study is PD patients experiencing motor fluctuations (OFF episodes) that meet the following inclusion criteria and do not meet any of the following exclusion criteria.

Patients may have been previously enrolled in the CVT-301-002 or CVT-301-003 studies, or may be CVT-301-naïve i.e. no previous exposure to CVT-301. Patients previously enrolled in the CVT-301-002 and CVT-301-003 studies must have completed all of the CVT-301 study visits without any safety issues that would preclude participation in this study according to the investigator. Patients who withdrew from either of the CVT-301 studies prior to completion, for any reason, will not be eligible.



#### 3.4.1. Inclusion Criteria

In order to be eligible to enter the study, patients must meet all of the following criteria:

- Has signed and dated an IRB/IEC-approved informed consent form before any protocol-specific screening procedures are performed.
- Is a male or female aged 30 to 85 years, inclusive. Women of child-bearing potential must use protocol-defined contraceptive measures (see Section 11.1.5) and must have a negative serum human chorionic gonadotropin (hCG) test at screening. These patients must be willing to remain on their current form of contraception for the duration of the study.
- Patients who have idiopathic PD (i.e., not induced by drugs or other diseases) as defined by fulfilling Steps 1 and 2 of the UK Brain Bank criteria, diagnosed after the age of 30 years.
- Patients who are classified as Stage 1 to 3 (in the ON state) on the modified Hoehn and Yahr scale for staging of PD severity.
- Patients who have experienced motor fluctuations for a minimum of 2 hours of average daily OFF time per waking day (excluding early morning OFF time) by self-report and confirmed by the PD Diary (on 3 consecutive days) during the screening period.
- Patients who are on a LD-containing therapy, not including Rytary (or equivalent), must be stable on oral LD-containing therapy for at least 2 weeks prior to SV1 with a LD/dopamine decarboxylase inhibitor (DDI)-containing regimen.
- Patients who are on a LD containing therapy, when including Rytary (or equivalent), should be on a stable dose for at least 6 weeks prior to SV1
- The frequency of L-dopa administrations must be at least 3 times during the waking day and a total daily LD dose of ≤1600 mg (exclusive of PRN LD-containing medications).
- Patients should be stable on other PD medications for at least 4 weeks prior to SV1.



- Patients must have a ≥ 25% difference between UPDRS Part 3 scores recorded in their ON and OFF states at screening.
- Patients must have normal cognition as confirmed by a score of ≥ 25 on the MMSE.
- Patients must be able to perform a spirometry maneuver in the ON and OFF states, and must have a screening FEV1 ≥ 50% of predicted and an FEV1/FVC ratio >60% in the ON state at screening. (A pulmonologist will review the spirometry tracings/morphology of any patient with an FEV1 that is ≥ 50% to <60% of predicted or an FEV1/FVC ratio that is >60% to <70% in order to determine potential eligibility. All CVT-301-naïve patients with an FEV1/FVC ratio of >60% to <70% will be required to undergo a bronchodilator challenge and the results must be reviewed prior to entry into the study. Patients with an FEV1/FVC ratio that is >60% to <70% will complete spirometry before and after the administration of a bronchodilator in a pulmonary function laboratory. Testing will be performed in accordance with the 2005 ATS/European Respiratory Society [ERS] criteria prior to randomization. The results of the bronchodilator challenge will be reviewed by a pulmonologist prior to potential randomization.)

#### 3.4.2. Exclusion Criteria

Patients meeting any of the following exclusion criteria at screening will not be enrolled in the study:

- Patients who have dyskinesia of a severity that would significantly interfere with their ability to participate or perform study procedures.
- Pregnant or lactating females or females wishing to become pregnant.
- Patients who have any known contraindication to the use of LD, including a history of malignant melanoma or a history of narrow-angle glaucoma.
- Patients who have had previous surgery for PD (including but not limited to deep brain stimulation [DBS] or cell transplantation).
- Patients with a history of psychotic symptoms requiring treatment, or suicide ideation or attempt within the prior 12 months (stable regimens [for at least 4 weeks prior to SV1] of anti-depressant and certain low-dose atypical antipsychotic medications are permitted, in case they are indicated to treat symptoms other than psychotic symptoms).



- Patients who have cancer with the exception of the following: basal cell carcinoma or successfully treated squamous cell carcinoma of the skin; cervical carcinoma in situ; prostatic carcinoma in situ; or other malignancies curatively treated and with no evidence of disease recurrence for at least 3 years.
- Patients taking certain prohibited medications (see Section 9.4.2).
- Patients with a history of drug or alcohol abuse within the prior 12 months.
- Patients with chronic obstructive pulmonary disease (COPD), asthma, or other chronic respiratory disease within the last 5 years.
- Patients with any contraindication to performing routine spirometry or who are unable to perform a spirometry maneuver (see Appendix 20 for a list of contraindications).
- Patients with a current history of *symptomatic* orthostatic hypotension despite adequate treatment.
- Patients with any condition that in the investigator's opinion would make patients unsuitable or interfere with their participation in the study. Potential issues of concern should be raised to the medical monitor during eligibility review.
- Patients who have any clinically significant abnormality or finding from examination, tests, or history that may compromise patient safety.
- Patients who have been treated with an investigational drug within 4 weeks or 5 half-lives (whichever is longer) prior to the beginning of the screening period (this includes investigational formulations of marketed products).
- Prior exposure to CVT-301.

#### 3.5. DETERMINATION OF SAMPLE SIZE

Approximately 250 CVT-301 treatment patients and 115 control patients will be enrolled in this study. It is assumed that the drop-out rate will be approximately 25%.

The primary objective of this study will be to characterize the pulmonary safety within the CVT-301-treated patients and the differences between the groups will be estimated as a secondary objective. However, for the secondary comparison of FEV1 change



### Statistical Analysis Plan

#### 3.6. TREATMENT ASSIGNMENT & BLINDING

This study is a 12-month, open-label, randomized, multicenter study which will evaluate the safety and effects of CVT-301 for the treatment of up to 5 OFF episodes per day in PD patients experiencing motor fluctuations (OFF episodes) and will include a concurrent observational cohort of PD patients managed using the usual standards of care. Patients may have been previously enrolled in the CVT-301-002 or CVT-301-003 studies, or may be CVT-301-naïve. Patients who were previously enrolled in the CVT-301-002 and CVT-301-003 studies will be assigned to the CVT-301 treatment group (CVT-301 at a target nominal respirable dose of 50 mg LD fine particle dose [FPD]), in this study. Patients who are CVT-301-naïve will be randomized in a 2:1 ratio to the CVT-301 treatment group (CVT-301 at a target nominal respirable dose of 50 mg LD FPD) or the observational cohort. Randomization will be stratified by the patient's Hoehn and Yahr stage (<2.5 versus ≥2.5) to balance the severity of disease across each group and by screening spirometry (FEV1 <60% of predicted or FEV1/FVC ratio <70% versus FEV1 ≥60% of predicted and FEV1/FVC ratio ≥70%).

Following completion of SV2 and prior to randomization, the patients' eligibility criteria will be reviewed by delegated staff. Upon confirmation of eligibility, the site will randomize an eligible patient using the Interactive Web Response System (IWRS). The study is an open-label study, so patients and clinical staff will not be blinded to study group assignment.

#### 3.7. ADMINISTRATION OF STUDY MEDICATION

Prior to the self-administration of inhaled study treatment, study staff will ensure that patients are adequately trained on the use of the inhaler according to the Instructions for Use (IFU). The IFU will be provided to each patient and will be part of the permanent study record.

Since this is an open-label study, the patient, investigator, and study site personnel, the Sponsor, representatives of the Contract Research Organization (CRO) involved in



### Statistical Analysis Plan

monitoring, data management, or other aspects of the study, and Core Laboratories will be not blinded to the inhaled study treatment.

During inhaler training, patients will be instructed to use the inhalation system in accordance with the IFU which includes a breath hold of 5 seconds following each capsule inhalation. For the purposes of timing study assessments in the clinic, "Time 0" (T0) is defined as the time of completion of inhalation of the last capsule of inhaled study treatment administered (i.e., beginning of the final breath hold). In the event that a capsule needs to be reinhaled, T0 is at the end of the reinhalation administration.

During the treatment period, patients will self-administer inhaled study treatment (CVT-301 DL1, CVT-301 DL2) up to 5 times daily to treat OFF episodes during their waking day.

#### 3.8. STUDY PROCEDURES AND FLOWCHART

This study has 3 periods: screening period, treatment period, and follow-up period; and a total of 9 planned visits: 2 screening visits, 6 treatment visits, and 1 follow-up visit. For each patient, the planned treatment period will be approximately 52 weeks, and maximum anticipated study duration, including screening and follow-up, will be approximately 62 weeks.

The screening period, which takes place within 35 days prior to Day 1 of the treatment period, will have 2 separate visits: SV1 and SV2 must be separated by at least 4 days. The screening period may be extended an additional 7 days if repeat screening assessments are required.

Before patients return to the clinic for TV/OV1, they will be randomized to treatment. The treatment period includes 6 separate in-clinic visits over approximately 52 weeks. The first dose of study drug will be given in the clinic at TV/OV1. The subsequent visits during the treatment period take place as follows:

- TV/OV2: Week 4; 28±5 days after TV/OV1.
- TV/OV3: Week 12; 84±14 days after TV/OV1.
- TV/OV4: Week 24; 168±14 days after TV/OV1.
- TV/OV5: Week 36; 252±14 days after TV/OV1.
- TV/OV6: Week 52; 364±14 days after TV/OV1.



## Statistical Analysis Plan

Patients who terminate the study early will complete TV/OV6 and return for the Follow-up DLco visit 4-5 weeks after TV/OV6.

Refer to Protocol Appendices 1 to 15 for tables of study assessments at each visit.



## Statistical Analysis Plan

| | S | V1 | S' | V2 | TV/OV1 | TV/OV2 | TV/OV3 | TV/OV4 | TV/OV5 | TV/OV6 |
|---|---|---|---|---|---|---|---|---|---|---|
| In Clinic Assessments | ON | OFF | ON | OFF | ON* | ON | ON | ON | ON | ON |
| MMSE | Х | | | | | | | | | |
| UPDRS Part 1 | | | | | | | | | | |
| UPDRS Part 2 | | | | | х | | | х | | х |
| UPDRS Part 3 | Х | Х | | | | x** | x** | x** | x** | x** |
| UPDRS Part 4 | | | | | х | | | x*** | | x*** |
| C-SSRS | | | | | Х | Х | Х | х | х | х |
| Epworth Sleep Scale | | | | | Х | | | Х | | Х |
| QUIP | | | | | Х | | | Х | | х |
| PDQ-39 | | | | | Х | | | х | | х |
| PGI-C | | | | | | | | X*** | | X*** |
| S&E ADL | | | | | х | | | х | | х |
| At home for patients | | | | | | | | | | |
| PD Diary (only treatment after screening) | Х | Х | Х | Х | х | х | х | х | х | х |
| ON/OFF logs (both groups) | Х | Х | | | | | | | | |
| Inhaled dosing (CVT-301 only) | | | | | Х | х | Х | Х | Х | Х |

<sup>\*</sup> For the CVT 301 arm these assessments are performed pre-dose

<sup>\*\*</sup> Performed pre-dose, 10, 20, 30, and 60 min post dose (only performed in CVT 301 arm)

<sup>\*\*\*</sup> CVT 301 arm only




### Statistical Analysis Plan

### 4. ENDPOINTS

#### 4.1. PRIMARY ENDPOINT

The primary endpoints related to the primary objective of the study are the pulmonary safety measures, FEV1, FVC and FEV1/ FVC ratio, assessed over a 12 month period. FEV1, FVC and FEV1/FVC ratio will be recorded from the single "best test" (based on effort with highest summed FEV1 and FVC). Variables will include the absolute FEV1, FVC, and FEV1/FVC ratio and FEV1 and FVC expressed as % of predicted value. Changes from baseline (TV/OV1) for each variable will be calculated at each subsequent visit.

Percent Predicted = 100 \* (Observed) / Predicted, where predicted is calculated and provided to INC by Biomedical Systems (BMS).

#### 4.2. SECONDARY ENDPOINTS

The following endpoints related to the secondary objectives will be calculated.

- Standard safety endpoints; for definitions see Section 8 of this SAP
  - Adverse Event (AE) reports
  - Physical examination
  - Standard and orthostatic vital signs (BP, HR and RR)
  - Clinical laboratory tests (hematology, clinical chemistry, and additional laboratory parameters)
  - 12-lead ECGs (HR, PR, QRS, QT, QT interval corrected using Bazett's formula [QTcB] and QT interval corrected using Fridericia's formula [QTcF])
  - o Parkinson's Disease Impulsive-Compulsive Disorders Questionnaire (QUIP)
  - Epworth Sleepiness Scale
  - Columbia-Suicide Severity Rating Scale (C-SSRS)
- Change from TV/OV1 (baseline) in the UPDRS Part 4 sum scores of dyskinesias (UPDRS items 32-35) and wearing-off (UPDRS items 36-39). The dyskinesia score will be calculated as the sum of the individual items 32-35 and the wearing-off score as sum of 36-39. Missing individual items will not be imputed and the sum score will be missing in case of 1 or more missing items.
- Occurrence and severity of examiner-rated dyskinesia following treatment of
  patients experiencing an OFF episode in the clinic. The occurrence will be based on
  the examiner's subjective assessment and no further derivation will be performed.
  Among the patients with reported dyskinesia, the severity will be classified as mild,
  moderate, severe or missing based on the examiner's subjective assessment and no
  further derivation will be performed. Only observed cases will be used for this
  endpoint and the visits with missing data will not be included in the analysis.



### Statistical Analysis Plan

• Carbon Monoxide Diffusion Capacity (DLco) assessed over a 12 month period within the CVT 301 treated and the observational ('standard of care') cohorts. Variables will include the absolute DLco values and DLco expressed as % of predicted value.

#### 4.3. EXPLORATORY EFFICACY ENDPOINTS

The following endpoints related to the exploratory efficacy objectives will be calculated.

- Change from pre-dose in UPDRS Part 3 motor score at 10, 20, 30, and 60 minutes following treatment of patients experiencing an OFF episode.
  - The UPDRS Part 3 total score will be calculated as the sum of the individual items of the UPDRS Part 3 questionnaire (UPDRS items 18-31) separately at each time point, i.e. the scores will range from 0 to 108. Missing individual items will be imputed using the 2 non-missing values at time points adjacent to the missing item on the same date. The maximum of the 2 adjacent values will be assigned as the score for the missing item. However, pre-dose values will not be assigned as post-dose values and if one of the adjacent values for a post-dose value is a pre-dose value, only 1 adjacent value will be used. The total score for UPDRS Part 3 assessments will be calculated after imputation of the missing item(s). Missing items at screening will not be imputed. If a pre-dose value is missing, the pre-dose value at the prior visit will be used. A missing TV/OV1 pre-dose value will be imputed using the last screening value in OFF state.
- Time curve of the UPDRS response shown as change from pre-dose in UPDRS Part 3 motor score to 10, 20, 30 and 60 minutes following treatment of patients experiencing an OFF episode in the clinic. The UPDRS Part 3 scores will be derived as described above.
- Change from pre-dose in the average UPDRS Part 3 score at 10 to 60 minutes following treatment of patients experiencing an OFF episode in the clinic. The change from pre-dose to the average of the 4 UPDRS Part 3 total scores (assessments scheduled at 10, 20, 30 and 60 minutes) will be used as the response variable in the statistical analysis.
- A ≥3, ≥6, and ≥11 point reduction in the UPDRS Part 3 motor score from pre-dose to post-dose, at 10 to 60 minutes following treatment in the clinic (cumulative and non-cumulative). The non-missing UPDRS Part 3 motor scores at each time point (10, 20, 30 and 60 minutes post-dose) are classified as a reduction of ≥3 points or not, reduction of ≥6 points or not and reduction of ≥11 points or not. Furthermore,



### Statistical Analysis Plan

for the purpose of the cumulative analysis, the time point (10, 20, 30 and 60 minutes post-dose) when the reduction of  $\geq 3$ ,  $\geq 6$  or  $\geq 11$  points occurs for the first time will be defined. The categorical scheduled time point is used in this analysis. The missing assessment regarding single items will be managed similarly as describe above. The missing values regarding visits will be managed by considering the missing visits as non-responses.

- Proportion of patients achieving resolution of an OFF to an ON state within 60 minutes after study drug is administered in the clinic and maintaining the ON at 60 minutes after study drug administration (per the examiner's subjective assessment). This endpoint will be based on the examiner's subjective assessment. In case the assessment of turning on within 60 minutes is missing but the assessment of maintaining the ON at 60 minutes has been done, the patient will be classified based on the available assessment. In case the assessment of maintenance of ON at 60 minutes is missing, the patient will be classified as having missing data.
- Change from baseline (3 consecutive days prior to TV/OV1, or in case of missing data, the last 3 recorded days before TV/OV1) in patient-recorded total daily OFF time, assessed by the patient and recorded in the PD Diary for 3 consecutive days prior to in-clinic visits (or in case of missing data, the last 3 recorded days before the visit). The validity of the PD diary entries will be checked prior to including a diary day in the summary calculations. Only valid diary days will be included in the diary summarizations. Change from baseline in total daily ON time without dyskinesia, total daily ON time with non-troublesome dyskinesia, and total daily ON time with troublesome dyskinesia will be calculated similarly.
  - A day will be considered as being valid if at least 80% of the entries during the day have been completed per instructions. That is, for each half hour period, only one entry among the responses (Asleep, OFF, ON without dyskinesia, ON with non-troublesome dyskinesia, or ON with troublesome dyskinesia) has been checked. The entry will not be used if no responses are checked or more than one response is checked. However, if the proportion of entries rejected due to multiple checked responses is large, sensitivity analysis will be performed by using the worst case out of the entries that had been checked. The worst case will be defined in the following order: OFF, ON with troublesome dyskinesia, ON with non-troublesome dyskinesia, ON without dyskinesia, Asleep. In case there are duplicate entries (i.e., multiple entries recorded with same date and time interval), the worst entry will be used for the date and time interval in question. The worst entry will be selected in the order defined above.
  - All diary data will be normalized to 16 awake hours per day. The daily OFF time will be extrapolated to a 16 hour period by determining the percentage



of OFF time among accurately recorded entries, excluding Asleep time and missing/non-valid recordings, and by multiplying this percentage by 16 hours.

- Off Time / (Total time recorded Asleep Time missing time interval)
   x 16
- The mean daily OFF time prior to each visit will be calculated as mean value of the valid days documented in the patient's diary prior to that visit. In case there are gaps within the 3 days preceding the visit, the last 3 recorded days before the visit will be used regardless of the gaps. If there are more than 3 valid days, only the last 3 days will be used. If there are only 1 or 2 valid days, the average of these days will be used.
- Change from TV/OV1 (baseline) in PDQ-39 sub-scores (mobility score, activities of daily living, bodily discomfort score, emotional wellbeing score, social support score, communication score, cognitive impairment score, and stigma score) and summary index score. The questionnaire provides scores on eight dimensions as outlined below:
  - o mobility (10 items, #1 to 10)
  - o activities of daily living (6 items, #11 to 16)
  - o emotional well-being (6 items, #17 to 22)
  - o stigma (4 items, #23 to 26)
  - o social support (3 items, #27 to 29)
  - o cognitions (4 items, #30 to 33)
  - o communication (3 items, #34 to 36)
  - o bodily discomfort (3 items, #37 to 39)

Items are scored from 0 (never) to 4 (always). Dimension scores are obtained by dividing the sum of the item scores by the maximum possible score for any given dimension and expressing this as a percentage. For example:

- o mobility = (sum of scores of #1 to 10)/(4 x 10) x 100
- o activities of daily living = (sum of scores of #11 to 16)/(4 x 6) x 100

For social support, if the response indicates that a patient does not have a spouse or partner for #28, social support can be calculated as [(sum of scores of #27 and 29)/(4 x 2) x 100].

A summary index is then calculated as the sum of the total score of the dimensions divided by the number of dimensions, i.e. (sum of dimension scores / 8). If any item score is missing, the relevant dimension score and the summary index will be missing.



## Statistical Analysis Plan

- The PGI-C score. The non-missing values will be categorized as improvements (much improved, improved, a little improved) or non-improvements (no change, a little worse, worse, much worse).
- Change from TV/OV1 (baseline) Schwab and England (S&E) Activities of Daily Living (ADL). No further derivation will be done for the S&E scores.
- Change from TV/OV1 (baseline) in the UPDRS Part 2 score. The UPDRS Part 2 score will be calculated as the sum of the individual items of the UPDRS Part 2 questionnaire (UPDRS items 5-17). Missing individual items will not be imputed and the sum score will be missing in case of 1 or more missing items.




### Statistical Analysis Plan

### 5. ANALYSIS SETS

### 5.1. ALL AVAILABLE POPULATION (AAP)

The AAP will include all patients who have consented for the study, including screening failures. Unless specified otherwise, the AAP will be used for patient listings and for the summary of patient disposition.

#### 5.2. SAFETY POPULATION

The Safety Population will include all randomized patients who received at least 1 dose of inhaled CVT-301 and patients from the Observational Cohort. Patients will be analyzed according to study treatment that they received. The Safety Population will be used for all analyses of safety endpoints and summaries of patient demographics and baseline characteristics.

### 5.3. INTENT-TO-TREAT POPULATION (ITT)

The ITT population will include all patients from the safety population. Patients will be analyzed according to randomized treatment. The ITT Population will be used for all analyses of exploratory efficacy endpoints.

### 5.4. PROTOCOL DEVIATIONS

A protocol deviation is any significant finding indicating that the study investigator or patient failed to adhere to the protocol requirements (e.g., drug noncompliance, failure to return for defined number of visits or within an acceptable visit window for completion of study assessments). The deviation may necessitate premature termination of the patient from the visit assessments, or from the study.

The deviations will be classified during a review process with the Sponsor and other study personnel (as appropriate) before database lock. The deviations will be classified as minor or major with/without impact on pulmonary assessments during the review process. All decisions regarding major deviations will also be discussed between the Sponsor, other study personnel (as appropriate), and the study statistician prior to commencing the final analysis on the locked database. The following deviations will be identified, but do not necessarily represent a complete list of potential deviations:

- Administration of PD medications after the usual morning dose of PD medication and before study drug administration
- Incorrect study drug administered at a visit
- Drug non-compliance including but not limited to unapproved dose modification



## Statistical Analysis Plan

• Failure to return for defined study visits or within an acceptable visit window for completion of study assessments

The number of subjects with minor, major with/without impact on pulmonary assessments protocol deviations will be summarized by treatment groups and overall. All protocol deviations will be listed.



### Statistical Analysis Plan

### 6. GENERAL ASPECTS FOR STATISTICAL ANALYSIS

#### 6.1. GENERAL METHODS

All patient data will be included in listings. All patients entered into the database will be included in patient data listings. The listings will be generally sorted by Patient ID (and by visit and by time point, if applicable), unless specified otherwise.

All applicable data will be summarized by treatment group (Observational Cohort or CVT-301) and overall in tables, unless specified otherwise. The CVT-301 group will be broken down into CVT-301-naïve patients and patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies. Where appropriate, data will be summarized by visit and/or time point in addition to treatment group. Unscheduled or repeat assessments will not be included in summary tables, but will be included in listings.

For the Observational Cohort, the "start of treatment" will be defined as attendance of TV/OV1, unless specified otherwise. Baseline will be defined as the assessments performed at TV/OV1. In case of missing data, the last non-missing screening assessment will be used as the baseline value.

Continuous variables will be summarized using the number of observations (n), mean, SD, median, minimum, and maximum. Standard error of the mean (SEM) will also be provided for summaries of UPDRS and other exploratory efficacy endpoints, if relevant. The same number of decimal places as in the raw data will be presented when reporting minimum and maximum, 1 more decimal place than in the raw data will be presented when reporting mean and median, and 2 more decimal places than in the raw data will be presented when reporting SD and SEM.

Descriptive statistics for categorical/qualitative data will include frequency counts and percents. The total number of patients in the treatment group overall (N) will be used as the denominator for percent calculations, unless stated otherwise in the table shell. All percents will be presented with one decimal point, unless specified otherwise. Percents equal to 100 will be presented as 100% and percents will not be presented for zero frequencies.

Significance testing will be 2-tailed using  $\alpha$  = 0.05, unless otherwise specified. All analyses and summaries will be produced using SAS® version 9.3 (or higher).

Deviations from the statistical plan will be reported in the clinical study report, including the rationale for use.

Acorda Therapeutics, Inc. CVT-301-005




### Statistical Analysis Plan

#### 6.2. KEY DEFINITIONS

#### <u>Age</u>

Age, as an integer, will be calculated using the date of birth and the date of informed consent.

Age = int ((date of informed consent- date of birth)/365.25)

### **Body Mass Index (BMI)**

BMI will be calculated as follows and rounded to 1 decimal place:

BMI  $(kg/m^2)$  = weight (kg) /  $[height (m)]^2$ 

### Parkinson's Disease History

The following parameters will be calculated for the PD history:

Time since diagnosis of PD (months) = Date of Screening Visit 1 (M/Y) - Date of diagnosis (M/Y)

Duration of levodopa treatment (months) = Date of Screening Visit 1 (M/Y) - Start date of levodopa treatment (M/Y)

Time since onset of wearing off episodes (months) = Date of Screening Visit 1 (M/Y) - Date of onset of wearing off episodes (M/Y)

If the month is missing, the first month of the year will be used.

### Change from pre-dose to post-dose

The change from pre-dose to post-dose within each visit will be calculated for each post-dose assessment as:

Change from Pre-dose to Post-dose = Post-dose value - Pre-dose value

### Percent change from pre-dose to post-dose

The percent change from pre-dose to post-dose within each visit will be calculated for each post-dose assessment as:

Percent Change from Pre-dose to Post-dose =



### Statistical Analysis Plan

(Post-dose value - Pre-dose value)\*100/Pre-dose value

#### Baseline

For CVT-301 patients, baseline is defined as the last non-missing assessment before the first dose of study drug, unless specified otherwise. For the Observational Cohort, baseline is defined as TV/OV1, or, in the case of missing data, the last non-missing assessment before TV/OV1, unless specified otherwise. However, for all patients who were included in the CVT 301-002 or CVT-301-003 studies, TV/OV1 of the CVT-301-005 study will be used as baseline.

### Change from baseline

The change from baseline will be calculated for each post-baseline assessment as:

Change from Baseline = Post-baseline value - Baseline value

#### Percent change from baseline

The percent change from baseline will be calculated for specified post-baseline assessments as:

Percent Change from Baseline = (Post-baseline value - Baseline value)\*100/Baseline value

DLCO predicted and DLCO predicted, adjusted for hemoglobin (Hb)

#### **DLCO** predicted

DLCO predicted will be calculated by Miller equation. (Miller A, Thornton JC, Warshaw R, Anderson H, Teirstein AS, Selikoff IJ. Single breath diffusing capacity in a representative of Michigan, a large industrial state. Am Rev Resp Dis 1983; 127: 270-277).

- Men predicted DLCO = 12.9113 (0.229 x age) + (0.418 x height in)
- Women predicted DLCO = 2.2382 (0.1111 x age) + (0.4068 x height in)

Where age is the age at the time of assessment taken, height is measured in inches.

### DLCO Predicted, adjusted for Hb

DLCO predicted adjusted for Hb is calculated using the Cotes method, according to the 2005 ATS/ERS guidelines for DLco.



- DLCO predicted, adjusted for Hb in <u>adult men</u>:
   DLCO predicted for Hb = DLCO predicted 1.7\* Hb / (10.22 + Hb)
- DLCO predicted, adjusted for Hb in <u>adult women</u>:

  DLCO predicted for Hb = DLCO predicted 1.7 \*Hb / (9.38 + Hb)

Where DLCO<sub>predicted</sub> is the DLCO calculated from Miller equation; Hb = hemoglobin, measured in g/dL. The Hb closest to the date/time of DLCO taken will be used.

### Percent predicted of FEV1 and FVC

The percent predicted of FEV1 and FVC will be calculated using the following equation.

Percent Predicted = 100 \* (Observed) / Predicted

where observed value is the value provided by TechEd, and the predicted value is the predicted value that provided by BMS and is the values closest to the date of observed value taken. The details are listed in table below.

| DLCO <sub>predicted</sub> , percent predicted of FEV1 and FVC | Value selection for Hb, predicted FEV1 and FVC |
|---|---|
| Screening (prior to randomization) | From TV/OV1 or the value closest to the date of DLCO |
| | assessment if the value at TV/OV1 is missing |
| TV/OV3, within 2 weeks prior to 3 | From TV/OV3 or the value closest to the date of DLCO |
| | assessment if the value at TV/OV3 is missing |
| TV/OV4, within 2 weeks prior to 6 | From TV/OV4 or the value closest to the date of DLCO |
| | assessment if the value at TV/OV4 is missing |
| TV/OV5, within 2 weeks prior to 9 | From TV/OV5 or the value closest to the date of DLCO |
| | assessment if the value at TV/OV5 is missing |
| TV/OV6, within 2 weeks prior to 12 | From TV/OV6 or the value closest to the date of DLCO |
| | assessment if the value at TV/OV6 is missing |
| 4 to 5 weeks after TV/OV6 | The latest non-missing Hb that closest to the date of |
| | DLCO assessment taken. |

#### 6.3. MISSING DATA

Several different methods to handle the missing data will be used.

 For calculation of the UPDRS part 3 scores, the missing single UPDRS items will be imputed as described in Section 4.3.



### Statistical Analysis Plan

- For the primary analysis of spirometry and selected explorative efficacy endpoints, likelihood-based modeling approach will be used to handle incomplete data. For this purpose, Mixed Model for Repeated Measures (MMRM) will be applied, see Section 8.1.
- Sensitivity analysis for spirometry and selected explorative efficacy endpoints will be conducted using the Multiple Imputation (MI) approach, i.e. by replacing each missing value with a set of plausible values that represent the uncertainty about the right value to impute, see Section 8.1.
- For the binary explorative efficacy endpoints, sensitivity analyses will be conducted using worst case imputation, where visits with missing data are counted as non-resolved (primary method), see Section 9.1.
- For AEs, the overall incidence of TEAEs, normalized for duration of exposure will be calculated to account for the shorter follow-up time in patients who discontinue the study prematurely, see Section 8.4.

The Safety and ITT populations will be used for the analysis of the primary, secondary and exploratory endpoints. The patients with no post-baseline data will not contribute to the analyses performed with the MMRM approach, but they do contribute to the sensitivity analyses using the MI approach. Due to this, no additional population, like a modified ITT population including only the patients with post-baseline will be defined.

#### 6.4. VISIT WINDOWS

The visits recorded in database will be used for all analyses. There is no plan to re-assign visits based on actual visit dates.

For the patients who discontinue the study prematurely, a set of assessments is scheduled to be performed at the Early Termination (ET) visit (PDQ-39, UPDRS Part 2, UPDRS Part 4, S&E ADL score and safety assessments). CVT 301 treated patients will also perform the UPDRS Part 3 assessments at 10, 20, 30, and 60 minutes post dose as well as the PGI-C. The following rules will be used to analyze the data collected at the ET visit:

- For the PDQ-39, PGI-C, UPDRS Part 2, UPDRS Part 3, UPDRS Part 4 and S&E ADL score, the data from the ET visit will be re-assigned to TV/OV6 in case there is no TV/OV6 assessment.
- In case there are PD diary assessments performed during the three days before the ET visit, these assessments will be re-assigned to the first visit at which the PD diary assessments were scheduled but are missing due to the premature withdrawal.



- The safety assessment assessments performed at the ET visit will be re-assigned to the first time point at which the corresponding safety assessments were scheduled but are missing due to the premature withdrawal.
- Any other data collected at the ET visit will not be used.

#### 6.5. POOLING OF SITES

Not applicable.

#### 6.6. SUBGROUPS

At least the following subgroup analyses have been pre-planned. The subgroup analyses will be performed for selected efficacy endpoints (at least the Change from pre-dose in UPDRS Part 3 motor score at 30 minutes post-dose and the mean daily OFF time). Selected baseline data will be presented for the subgroups as well.

- Patients with baseline PD severity < 2.5 points on the Hoehn & Yahr scale versus patients with baseline PD severity ≥ 2.5 points on the Hoehn & Yahr scale
- Patients who are dyskinetic before TV/OV1 versus non-dyskinetic patients. The classification will be done based on the Parkinson's disease diary data. The patients who have recorded at least 1 hour of dyskinesia (either ON with nontroublesome dyskinesia or ON with troublesome dyskinesia) on at least 2 days before TV/OV1 will be classified as dyskinetic
- Patient with the baseline daily levodopa dose less than or equal to the median versus the patients with the baseline daily levodopa dose higher than the median
- Patients who have less than 4.5 hours of PD diary mean daily OFF time before TV/OV1 versus patients who have 4.5 hours or more of OFF time
- Patients with FEV1 <60% of predicted or FEV1/FVC ratio <70% at baseline versus patients with FEV1 ≥60% of predicted and FEV1/FVC ratio ≥70%
- Non-elderly (<65 years) versus elderly (≥65 years) patients
- Female versus male patients.




### Statistical Analysis Plan

# 7. DEMOGRAPHIC, OTHER BASELINE CHARACTERISTICS AND MEDICATION

### 7.1. PATIENT DISPOSITION AND WITHDRAWALS

The patient disposition table will summarize the following and will be presented for each treatment group, as applicable, and overall. The percentages will be calculated based on the number of randomized patients, unless otherwise specified). The randomized set will include all randomized patients as well as those from CVT-301-002 and CVT-301-003 studies who were assigned to the CVT 301 treatment group.

- The number of patients screened (i.e. the number of patients in the AAP population)
- The number of patients who failed screening
- The number (%) of patients randomized into the study (% calculated from the AAP population)
- The number (%) of patients in the different study populations (Safety and ITT populations)
- The number (%) of patients who completed the study (based on end-of-study case record page)
- The number (%) of patients who withdrew from the study and associated reasons (% calculated from the Safety population)

### 7.2. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Demographics and baseline characteristics will be summarized descriptively for the Safety population by treatment group and overall. The following variables will be summarized:

- Demographics (age (continuous), age categorized as <65 years versus ≥65 years, gender, ethnicity, race, height, weight, BMI, country)
- Smoking history (current, former, never, Number of Years Smoked and Number of Cigarettes/Day)
- Cognitive status (MMSE)
- Average number of daily OFF episodes experienced from the Screening ON/OFF Log. The screening ON/OFF log data collected on 3 days prior to TV/OV1 will be used as baseline. If the data are only available on 1 or 2 days prior to TV/OV1, the available data will be used as baseline. If there is no data prior to TV/OV1, the data collected on 3 days prior to SV2 will be used as baseline.



### Statistical Analysis Plan

- Proportion of patients who changed the timing of their usual levodopa medication and proportion of patients who took an extra dose of levodopa or other PD medication from the Screening ON/OFF Log. The screening ON/OFF log data collected on 3 days prior to TV/OV1 will be used as baseline. If the data are only available on 1 or 2 days prior to TV/OV1, the available data will be used as baseline. If there is no data prior to TV/OV1, the data collected on 3 days prior to SV2 will be used as baseline.
- Average daily OFF time, ON time Without Dyskinesia, ON time with troublesome and non-troublesome dyskinesia (from PD diary before TV/OV1)
- Proportion of patients with total daily OFF time <4.5 hours or ≥4.5 hours (from PD diary before TV/OV1)
- Distribution of average daily OFF time in 30-minute intervals (00:00 00:30, 00:30 01:00, ...). The percentage based on the total daily OFF time will also be presented and is calculated as the average of total OFF time collected three days prior to TV1 and is normalized to 16 awake hours per day.
- PD history (time since diagnosis of PD, duration of levodopa treatment, time since onset of wearing off episodes)
- Total daily levodopa dose, number of levodopa doses per day
- PD disease severity (Modified Hoehn and Yahr Staging in "ON" State)
- UPDRS Part 3 Motor score in ON/OFF (from screening assessment); the change from OFF to ON state in UPDRS part 3 Motor score at the Screening will also be classified as ≥6 points, or ≥11 points reduction.
- Baseline Dyskinesia (Dyskinetic before TV/OV1, Non-dyskinetic before TV/OV1).
   The classification will be done based on the Parkinson's disease diary data. The patients who have recorded at least 1 hour of dyskinesia (either ON with non-troublesome dyskinesia or ON with troublesome dyskinesia) on at least 2 days before TV will be classified as dyskinetic.
- Proportion of patients with FEV1 <60% of predicted or FEV1/FVC ratio <70% at baseline versus FEV1 ≥60% of predicted and FEV1/FVC ratio ≥70% (based on the randomization strata).
- Screening spirometry data: FEV1, FVC, and FEV1/FVC ratio, presented for each motor status, ON or OFF, separately.

Demographics and PD disease data will also be summarized by subgroups (Patients with baseline PD severity < 2.5 points on the Hoehn & Yahr scale versus  $\geq$  2.5 points; Patients who are dyskinetic before TV/OV1 versus non-dyskinetic; Patient with the baseline less than or equal to the median versus above median; Patients who have less than 4.5 hours of PD diary mean daily OFF time before TV/OV1 versus 4.5 hours or more; Patients with FEV1 <60% of predicted or FEV1/FVC ratio <70% at baseline versus FEV1  $\geq$ 60% of predicted and FEV1/FVC ratio  $\geq$ 70%, Non-elderly (<65 years) versus elderly ( $\geq$ 65 years) patients, Female versus Male patients).



### Statistical Analysis Plan

### 7.3. MEDICAL HISTORY

Medical history data will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 17.0. The medical history data will be summarized with frequencies and percentages of patients with at least one medical history item, and patient frequencies and percentages on the system organ class (SOC) and preferred term (PT) levels. The events will also be summarized. The table, using the Safety population, will be sorted by overall descending frequency of SOC and then, within a SOC, by overall descending frequency of PT.

#### 7.4. MEDICATION

All medications will be classified using the Anatomical Therapeutic Chemical (ATC) classification codes and preferred drug names from the World Health Organization Drug Dictionary (WHO-DD), Q1March2014.

For the medications recorded on CRF page "Prior and Concomitant Medications", medications with a stop date before the first date of study drug dosing or TV/OV1 for the observational cohort will be considered prior medications. Medications with start date or stop date on or after the first date of study drug dosing will be considered concomitant medications.

Tables will be generated for the Safety Population. Summaries of baseline PD treatment medications (medications which start with ATC code NO4) will be presented in tabular form using the ATC Level 4 and preferred term. Other prior medications and concomitant medications will be presented in tabular form using the ATC Level 1, ATC Level 2, and PT. Frequencies and percentages will be presented by treatment group and overall. The counts of medications will also be summarized. The tables will be sorted by overall descending frequency of ATC Level(s) and then, within an ATC Level, by overall descending frequency of PT.

If the medication start date is incomplete, then it will be imputed as follows for the purpose of determining concomitance only:

- If the start date is completely missing, the start date will be equal to the first dose date. However, if the stop date is not missing and is before the first dose date, then the stop date will be used instead.
- If the start day is missing, the first day of the month will be used.
- If the start day and month are missing, then the first day of the first month (January) will be used.

If the medication stop date is partial, then it will be imputed as follows for the purpose of determining concomitance only:



## Statistical Analysis Plan

- If the stop date is completely missing and the medication is not ongoing, the stop date will be equal to the last dose date or date of completion/withdrawal, whichever is the latest.
- If the stop day is missing, the last day of the month will be used.
- If the stop day and month are missing, then the last day of the last month (December) will be used.


## Statistical Analysis Plan

### 8. SAFETY

The population used for safety analyses will be the Safety Population. The analyses are outlined below.

#### 8.1. SPIROMETRY

Spirometry will be performed by trained and qualified staff at each study site. Spirometry data obtained in the study site will reviewed by a central spirometry laboratory (Biomedical Systems, Inc.) which will provide a quality over read of all evaluations based on acceptability and repeatability metrics in accordance with ATS criteria. FEV1, FVC and FEV1/FVC ratio will be recorded from the single "best test" (based on effort with highest summed FEV1 and FVC). Variables will include the absolute FEV1, FVC, and FEV1/FVC ratio and FEV1 and FVC expressed as % of predicted value.

FEV1, FVC, FEV1/FVC ratio and DLco will be summarized descriptively by treatment group and overall. For screening data, the summary will be presented for each motor status, ON or OFF, separately. For other visits, data in ON or OFF state will be combined for summary. The following will be summarized:

- Change from baseline to other visits Arrival values for each parameter. The baseline is defined as the TV/OV1 Arrival value. If the TV/OV1 Arrival value is missing, the last available value in ON state before the first dose of study drug will be used.
- Number and percentage of patients with FEV1/FVC < 60% and <70% by Visit</li>
- Spirometry data will also be provided to indicate whether specific determinations met American Thoracic Society (ATS) quality criteria. The proportion of spirometry data measurements meeting or not meeting ATS quality criteria will be summarized by treatment group and overall. The summary will also be performed for ON state measurements, OFF state measurements, and all measurements, separately. The reasons for not meeting ATS quality criteria will be classified as not meeting the criteria for acceptability, not meeting the criteria for repeatability or as other/unknown and summarized.

The spirometry analyses will be repeated for the subset of assessments meeting the ATS quality criteria.

Another subset analysis will be performed by excluding the spirometry data from patients with a very high intra-individual variability. For the purpose of this analysis, all patients who have a co-efficient of variation (CV) value >7.5% for FEV1 will be excluded. The CV will be calculated for each patient as standard deviation divided by the mean.



# Statistical Analysis Plan

The screening visit FEV1 data (assessed in ON state) and arrival values at subsequent visits will be used for the calculation.

In addition to the descriptive statistics, the changes in the spirometry values within each treatment group and differences between the treatment groups will be estimated with MMRM. The model will include the treatment group (CVT-301 or observational cohort), visit (visits at 1, 3, 6, 9, and 12 months), the stratification variables (Hoehn and Yahr stage and screening FEV1 and/or FEV1/FVC) and the interaction between the treatment group and visit as fixed factors. The baseline spirometry value will be included as a covariate. An unstructured covariance structure will be applied for MMRM. In case the model will not converge with the unstructured covariance structure, the heterogeneous compound symmetry (CSH) or the heterogeneous Toeplitz structure (TOEPH) will be used instead. If the unstructured covariance structure will be used, the denominator degrees of freedom will be computed using the Kenward-Roger method. In case of other covariance structures, the BETWITHIN option will be used for the denominator degrees of freedom. The least square (LS) mean, standard error, and LS mean difference between CVT-301 and observational cohort at each visit; along with the 95% confidence interval (CI) will be provided in a table. Treatment difference will be assessed with a 2-sided alpha level of 0.05, unless specified otherwise.

The SAS code planned for the analysis is outlined below.

```
proc mixed data=&data;
class pdsevbl fev1bl trta avisit usubjid;
model chg=base pdsevbl fev1bl trta avisit trta*avisit / ddfm=kr;
repeated avisit / subject=usubjid(trtp) type=un;
lsmeans trtp*avisit / cl;
estimate 'CVT vs OBS Month 1'
       trta 1 -1 trta*avisit 1 0 0 0 0 -1 0 0 0 0 / cl;
estimate 'CVT vs OBS Month 3'
        trta 1 -1 trta*avisit 0 1 0 0 0 0 -1 0 0 0 / cl;
estimate 'CVT vs OBS Month 6'
       trta 1 -1 trta*avisit 0 0 1 0 0 0 0 -1 0 0 / cl;
estimate 'CVT vs OBS Month 9'
       trta 1 -1 trta*avisit 0 0 0 1 0 0 0 0 -1 0 / cl;
estimate 'CVT vs OBS Month 12'
       trta 1 -1 trta*avisit 0 0 0 0 1 0 0 0 0 -1 / cl;
run;
```

The Safety population will be used for the primary analysis.

### Sensitivity analyses of the spirometry data

The following sensitivity analysis will be performed for the primary endpoint.



## Statistical Analysis Plan

MI analysis: MI techniques based on Pattern Mixture Models (PMM) will be applied (Ratitch et al., 2011) as a further sensitivity analysis in the Safety population. This methodology will structure data based on missing data patterns. The method will be based on a missingness pattern having a monotone structure, i.e. if among the observations over time one data value is missing, all other values after this missing value will also be treated as missing. For patients with intermittent missing values, before performing MI based on the PMM, it will be necessary to create a monotone missingness pattern. Intermittent missing values will be imputed using the Markov Chain Monte Carlo (MCMC) methodology which assumes a multivariate normal distribution over all variables included in the imputation model. The MI procedure in SAS will be used for this purpose and this first MI step is planned to be repeated 100 times, creating several different datasets with a monotone missing data structure. Seed value of 201508 will be used in the MI procedure. The imputation is based on the missing at random (MAR) assumption, i.e. the missing data are assumed to follow the same model as the other patients in their respective treatment arm that have complete data.

After this, the remaining missing data can be imputed using a method for monotone missingness, also based on the MAR assumption. Thus, for each of the created datasets with a monotone missing data pattern, the MI procedure in SAS will used to impute missing values based on a sequential procedure reflecting the monotone missing data pattern. Patients with the first missing value occurring at visit at Month 1 will have their missing Month 1 value replaced by an imputed value from a regression model with treatment group, baseline spirometry value and the stratification factors as explanatory variables. In the next step, patients with their Month 3 value missing will have their missing Month 3 value replaced by an imputed value from a regression model with treatment group, baseline spirometry value, stratification factors and the Month 1 value as explanatory variables. Similar procedure will be used to replace the missing values at Month 6, 9 and 12.

The imputed datasets generated with the approach described above do contain only non-missing values and are used as input in the model for the primary endpoint. MMRM models similar as described above will thus be run on each of the generated imputed datasets and the difference between the treatment groups will be estimated. The MMRM model will be similar to the primary analysis. Finally, the MIANALYZE procedure in SAS will be applied to combine the results from these several datasets to derive an overall estimate of the within-group changes and treatment differences. Estimates and corresponding 95% confidence intervals will be calculated.

#### 8.2. EXTENT OF EXPOSURE

The following information will be summarized for CVT-301 treated subjects:




## Statistical Analysis Plan

- The number of patients with dose change
- Duration of exposure (days)
- Total exposure to study treatment, expressed as person years (sum of exposure to study treatment over all CVT - 301 treated patients)
- Total number of doses and capsules taken, by visit and overall. Average number of daily doses and number of capsules, by visit and overall
- Proportion of days with 5, 4, 3, 2, 1 or 0 doses administered
- Proportion of patients using 5, 4, 3, 2, 1 or 0 doses/day at least once

In addition, these in-clinic data will be summarized by treatment group and visit:

- Standard morning dose of LD-containing medications to in-clinic OFF (mins)
- In-clinic OFF to start of study drug inhalation (mins)
- Standard morning dose of LD-containing medications to start of study drug inhalation (mins)
- Duration of study drug inhalation (mins), calculated as (Completion time of last inhalation Time of start of first capsule inhalation).

Furthermore, the distribution of time of intake of study medication (00:00 - 00:30, 00:30 - 01:00, ...) as percentage of the total number of study medication intakes will be displayed during the whole treatment period. This data will be collected on the Inhaled Dosing Log.

All study drug data will be listed. A listing will also be provided to show how many times each patient will take study drug and the capsules taken for each day.

#### 8.3. TREATMENT COMPLIANCE

Patients will be instructed to administer inhaled study drug up to 5 times each day during the treatment period. In-clinic administration of study drug will be supervised by study personnel, and at-home diary data will be reviewed to ensure patient compliance. Since there are no fixed scheduled doses for each day, compliance will not be calculated for this study; alternatively, study drug use will be evaluated based on the inhaled medication treatment log by summarizing the proportion of days with >5, 5, 4, 3, 2, 1 or 0 doses administered.

### 8.4. ADVERSE EVENTS

All AEs will be coded using the MedDRA version 17.0.

Treatment-emergent adverse events (TEAEs) are defined as all AEs that start after the patient receives the first dose of study drug. For the observational cohort, TEAE will



# Statistical Analysis Plan

be defined as events that occur during/after TV/OV1. Events will be classified as drug-related if the AE is classified as possibly, probably, or definitely related to study drug.

Events with a missing start time, but with a start date equal to the date of first dose of study drug will be considered treatment-emergent. If the AE start date is incomplete, then it will be imputed as follows for the purpose of determining TEAE:

- If the start date is completely missing, the start date will be equal to the first dose date. However, if the stop date is not missing and is before the first dose date, then the stop date will be used instead.
- If the start day is missing, the first day of the month will be used.
- If the start day and month are missing, then the first day of the first month (January) will be used.

The original date and time will be shown on all listings of AEs. Listings will be provided for all AEs, serious AEs, AEs leading to study drug discontinuation, AEs leading to dose reduction, and deaths.

TEAEs will be summarized by SOC and PT for each treatment group and overall total. TEAEs with onset after the treatment period are attributed to the treatment group and dose level during the treatment period. Both event and patient counts, where applicable, will be summarized. The counts will be complemented by percentages will be calculated for the patient counts unless otherwise specified. In addition, the incidence of TEAEs, normalized for duration of exposure will be presented (number of TEAEs divided by the total exposure to CVT 301 or observation, measured as patient years).

- An overall summary of the number and percentage of patients reporting TEAEs and the number of TEAE events, drug-related TEAEs, severe TEAEs, serious TEAEs, TEAEs leading to dose interruption, TEAEs leading to study drug discontinuation, TEAEs leading to dose reduction and TEAEs leading to death
- TEAEs by SOC and PT, both as event and patient counts
- TEAEs by PT, both as event and patient counts
- Drug-related TEAEs by SOC and PT, both as event and patient counts
- Severe TEAEs by SOC and PT, both as event and patient counts
- Drug-related TEAEs by SOC, PT and severity, as event counts; percentages will be calculated for the event count out of total number of events
- Drug-related TEAEs by SOC, PT and relationship, as event counts; percentages will be calculated for the event count out of total number of events
- Serious TEAEs by SOC and PT, both as event and patient counts
- TEAEs leading to study drug interruption, both as event and patient counts
- TEAEs leading to study drug withdrawal, both as event and patient counts



# Statistical Analysis Plan

- TEAEs leading to dose reduction, both as event and patient counts
- Most common AEs, both as event and patient counts, most common TEAEs is defined any AE preferred term occurred in greater than 10% total patients.
- Time to first onset of most common AEs, classified as 0-1 months, >1-3 months, >3-6 months, >6-9 months and after 9 months, where the date of TEAE onset will be used as the time point for classification.

The tables will be sorted by overall descending frequency of SOC and then, within a SOC, by overall descending frequency of PT based on the patient count for the Total column. If only event count is presented, the sorting will be done based on the event count.

#### 8.5. LABORATORY EVALUATIONS

Laboratory samples for hematology and clinical chemistry will be analyzed by a central laboratory (located in the United Kingdom for EU sites and the United States for US sites) to ensure consistent interpretation of results. In the event of an unexplained clinically significant abnormal laboratory test value, the test should be repeated immediately and followed up until it has returned to the normal range and/or an adequate explanation of the abnormality is found.

All parameters will be converted to consistent units according to the International System of Units (SI) before summarization. The following will be summarized by treatment group and overall:

- Actual values and change from baseline, if applicable, at each visit for each parameter (for handling of data from the ET visit, see Section 6.4)
- Number and percentage of patients with normal or "abnormal" (i.e., out of reference range) labs at each visit for each parameter
- Number and percentage of patients with potentially clinically significant (PCS) lab values at each visit for each parameter
- Number and percentage of patients with potentially clinically significant changes (PCSC) in lab values at each post-baseline visit for each parameter

PCS and PCSC will be identified for specific laboratory parameters as outlined in the following table.

| Laboratory | Units | Criteria for PCS Values (Actual | | Criteria for PCSC values | |
|---|---|---|---|---|---|
| Parameter | | values) | | (Changes from baseline values) | |
| | | | Ι. | | , |
| | | High | Low | % increase | % decrease |
| Hemoglobin | g/L | > 10 above ULN | >20 below LLN | NA | 25% |
| Hematocrit | 1 | >0.04 above ULN | >0.05 below LLN | NA | 25% |
| WBC | GI/L | >5 above ULN | >1 below LLN | 100% | 50% |




## Statistical Analysis Plan

| Neutrophils | GI/L | NA | <0.5xLLN | 100% | 50% |
|--------------------|--------|---------------|----------------|------|-----|
| Neutrophils | % | NA | <0.5xLLN | 100% | 50% |
| Lymphocytes | GI/L | NA | <0.5xLLN | 100% | 50% |
| Lymphocytes | % | NA | <0.5xLLN | 100% | 50% |
| Total bilirubin | µmol/L | >1.5xULN | NA | 300% | NA |
| Total protein | g/L | >15 above ULN | >15 below LLN | 200% | 60% |
| Albumin | g/L | >5 above ULN | >5 below LLN | NA | 60% |
| AST | U/L | >3xULN | NA | 300% | NA |
| ALT | U/L | >3xULN | NA | 300% | NA |
| Alkaline | U/L | >3xULN | NA | 300% | NA |
| Phosphatase | | | | | |
| GGT | U/L | >3xULN | NA | 300% | NA |
| Creatinine | µmol/L | >1.5xULN | NA | 200% | NA |
| Urea | mmol/L | >2.5xULN | NA | 300% | NA |
| Uric Acid | µmol/L | >3xULN | NA | 300% | NA |
| Sodium | mmol/L | >5 above ULN | >5 below LLN | 10% | 10% |
| Potassium | mmol/L | >1 above ULN | >0.5 below LLN | 25% | 20% |
| Carbon dioxide | mmol/L | >40 | <16 | 25% | 25% |
| Calcium | mmol/L | >2.99 | <1.78 | 30% | 30% |
| Glucose (fasting)* | mmol/L | >11.1 | <2.8 | 300% | 40% |

ULN = Upper limit of normal range, LLN = Lower limit of normal range

Baseline is defined as the visit 3 assessment. If the visit 3 assessment is missing, the last non-missing screening assessment will be used as baseline. \* fasting defined as ≥4 hr from prior meal

The tables showing the normal/abnormal values, PCS values and PCSCs will be done both as summaries of all data and as shift tables (i.e., classified by the baseline status).

Values which fall outside the central laboratory normal range will be flagged as "L" - below normal range, or "H" - above normal range, on the data listings. PCS and PCSC values will also be flagged. All repeated values will be presented on the data listings but not included in the summaries showing data by visit.

### 8.6. VITAL SIGNS

Standard vital sign measurements will include RR, systolic and diastolic BP (SBP, DBP), and HR. At SV1 (or SV2) and each of the subsequent study visits, and in the event of a clinically significant finding that could be suggestive of symptomatic orthostatic hypotension (e.g., dizziness, lightheadedness, or other AE), orthostatic vital signs will be performed. Orthostatic vital sign measurements will include SBP, DBP, and HR.

The following will be summarized:

• Change from baseline to other visit for each parameter. The baseline is defined as the TV/OV1. If TV/OV1, the last non-missing screening assessment will be used as baseline.



# Statistical Analysis Plan

- Actual values and change from pre-dose to post-dose time points at TV/OV1 by time point for each parameter for CVT-301 treated patients
- Number and percentage of patients with PCS values at each applicable visit and time point for each standard vital sign parameter
- Number and percentage of patients with PCSC values at each applicable visit and time point for each standard vital sign parameter
- Number and percentage of patients with Orthostatic hypotension at each applicable visit

PCS and PCSC for standard vital sign will be identified as outlined in the following table.

| Vital Sign | Units | Criteria for PCS Values<br>(Actual values) | | Criteria for PCSC values<br>(Change from Baseline or<br>pre-dose values *) | |
|---|---|---|---|---|---|
| | | High | Low | increase | decrease |
| Pulse rate | bpm | >120 | <40 | 2x | 0.5x |
| Respiration Rate | brpm | >32 | <8 | 1.5x | NA |
| Systolic Blood | mmHg | >200 | <85 | 1.6x | 0.2x |
| Pressure (supine) | | | | | |
| Diastolic Blood | mmHg | >120 | <40 | | 0.2x |
| pressure (supine) | | | | | |

\*Pre-dose values will be used for corresponding post-dose values assessment at TV/OV1. Otherwise baseline values are used.

Orthostatic hypotension will be defined as a reduction in SBP of 20 mmHg or more, and/or a reduction in DBP of 10 mmHg or more, for the standing measurement compared to the supine/semi-supine measurement.

#### 8.7. ELECTROCARDIOGRAM

Standard 12-lead ECGs will be obtained after the patient has rested in a supine position for at least 5 minutes. Electrocardiograms will be measured using an ECG machine that automatically calculates the HR and measures PR, QRS, QT, QT interval corrected using Bazett's formula (QTcB) and QT interval corrected using Fridericia's formula (QTcF).

The following will be summarized:

- Change from baseline to other visit for each parameter. The baseline is defined as the TV/OV1 value. If TV/OV1 value is missing, the last non-missing screening assessment will be used as baseline.
- Number and percentage of patients with PCS values at each applicable visit for each parameter



# Statistical Analysis Plan

 Number and percentage of patients with PCSC values at each applicable visit for each parameter

PCS and PCSC will be identified as outlined in the following table.

| ECG | Units | Criteria for PCS Values<br>(Actual values) | | Criteria for PCSC values (Change from Baseline) | |
|---|---|---|---|---|---|
| | | High | Low | increase | decrease |
| PR interval | msec | >300 | NA | >25% for baseline ≥200<br>>50% for baseline <200 | NA |
| QRS interval | msec | >200 | NA | >25% for baseline ≥100<br>>50% for baseline <100 | NA |
| QTcB | msec | >500 | NA | >15% for baseline ≥440<br>>30% for baseline <440<br>>30 msec increase<br>>60 msec increase<br>Change>30 and value>500<br>Change>60 and value>500 | NA |
| QTcF | msec | >500 | NA | >15% for baseline ≥440<br>>30% for baseline <440<br>>30 msec increase<br>>60 msec increase<br>>Change>30 and value>500<br>Change>60 and value>500 | NA |
| Heart Rate | bpm | >120 | <35 | NA | NA |

## 8.8. PHYSICAL EXAMINATION

A complete physical examination (head, eyes, ears, nose, and throat [HEENT], heart, lungs, abdomen, skin, cervical and axillary lymph nodes, neurological, and musculoskeletal systems) will be performed at screening. Genital, rectal, and breast examination may be excluded if not clinically indicated.

The following will be summarized:

 Total number and percentage of patients reporting abnormal clinically significant physical examination results

## 8.9. COLUMBIA-SUICIDALITY SEVERITY RATING SCALE

The C-SSRS is a measure of suicidal ideation and behavior. The rating scale has 4 general categories: suicidal ideation, intensity of ideation, suicidal behavior, and actual attempts. All C-SSRS data will be listed. The frequency and percentage of patients



# Statistical Analysis Plan

with each response for suicidal ideation, intensity of ideation, and suicidal behavior items will be summarized as appropriate by treatment group and overall.

A shift from baseline table will be constructed to assess any changes in the subjects' suicidal ideation and behavior during the treatment period.

### 8.10. EPWORTH SLEEPINESS SCALE

The Epworth Sleepiness Scale is used to determine the level of daytime sleepiness. There are 8 situations listed for which patients rate their likelihood of dozing or sleeping (0=would never doze or sleep, 1=slight chance of dozing or sleeping, 2=moderate chance of dozing or sleeping, and 3=high chance of dozing or sleeping). The total score is the sum of 8 item scores and can range between 0 and 24. In case of missing item scores, the missing value will be replaced by the average of non-missing scores at the same visit from the same patient. In case all item scores are missing, the total score will be set as missing. The higher total score indicates the higher level of daytime sleepiness. A score of 10 or more is considered sleepy, and a score of 18 or more is very sleepy.

All Epworth Sleepiness Scale data will be listed. The total score and change from baseline will be summarized by treatment group and overall (for handling of data from the ET visit, see Section 6.4).

# 8.11. QUESTIONNAIRE FOR IMPULSIVE-COMPULSIVE DISORDERS IN PARKINSON'S DISEASE

The QUIP is an instrument used to measure the extent of impulsive and compulsive behaviors in PD patients. The QUIP has 3 sections: Section 1 assesses any impulsive control disorder (gambling, sexual, buying, and eating disorders); Section 2 assesses other compulsive behaviors (punding, hobbyism, and walkabout); and Section 3 assesses compulsive medication use.

The frequency and percentage of patients with positive response for each of the item within each section will be summarized by visit treatment group and overall. The assessment of positive response for each item will be based on the table below.

| Section and Item | Number of items with positive response |
|-------------------------------|----------------------------------------|
| A. Impulse Control Disorders | |
| Compulsive gambling | any 2 of the 5 gambling items |
| Compulsive sexual behavior | any 1 of the 5 sexual behavior items |
| Compulsive buying | any 1 of the 5 buying items |
| Compulsive eating | any 2 of the 5 eating items |
| B. Other Compulsive Behaviors | |

1003805 Acorda Therapeutics, Inc. CVT-301-005




# Statistical Analysis Plan

| Hobbyism | item #1A |
|------------------------------|-----------------|
| Punding | item #1B |
| Walkabout | item #1C |
| C. Compulsive Medication Use | items #1 and #4 |

### **8.12. UPDRS PART 4**

Changes from baseline to the subsequent visits in UPDRS Part 4 sum scores (dyskinesia sum score, wearing-off sum score) will be analyzed using a similar MMRM as for the UPDRS Part 3 scores (described below) to estimate the within-group changes. Otherwise, the data will be presented with descriptive statistics only classified by visit for CVT treated patients. The observed cases will be used in the analysis and summaries.

### 8.13. EXAMINER-RATED DYSKINESIA

The occurrence and severity will be tabulated by treatment group and visit. The observed cases will be used in the summaries. No formal statistical methods will be used.



## Statistical Analysis Plan

### 9. EXPLORATORY EFFICACY

#### 9.1. EXPLORATORY EFFICACY ENDPOINT AND ANALYSIS

The ITT population will be used for the exploratory efficacy analysis. Patients will be analyzed according to randomized treatment. The within group changes from baseline in continuous efficacy variables will be estimated using an MMRM. No between group differences will be calculated, unless otherwise specified. The model will include visit and the stratification variables (Hoehn and Yahr stage and screening FEV1 and/or FEV1/FVC) as fixed factors. The baseline value will be used as a covariate. For variables which do not have a pretreatment baseline assessment, OFF-state baseline UPDRS Part 3 score will be used as the baseline covariate. An unstructured covariance structure will be applied for the MMRM. In case the model will not converge with the unstructured covariance structure, compound symmetry will be used instead. For all patients, categorical data will be evaluated descriptively. Each visit will be evaluated separately for the categorical endpoints. The exploratory efficacy endpoints and associated analyses are as follows. For the detailed definition of the endpoints, see Section 4.3.

- Change from pre-dose in UPDRS Part 3 motor score at 10, 20, 30, and 60 minutes and the average of the motor score at 10-60 following treatment of patients experiencing an OFF episode in the clinic. Change from pre-dose in the average UPDRS Part 3 score at 10 to 60 minutes is calculated as the mean of change of UPDRS Part III total score from pre-dose to each time point post-dose if UPDRS Part III total score is available for at least 2 time points post-dose. The scheduled post-dose UPDRS Part III assessments are at 10, 20, 30, 60 minutes post-dose, respectively. If there is more than 2 time points post-dose with missing UPDRS Part III total score, the change of UPDRS Part III total score from pre-dose to 10 to 60 minutes post-dose will be missing. A MMRM model as defined above will be used.
- Time curve of the UPDRS response shown as change from pre-dose in UPDRS Part 3 motor score to 10, 20, 30 and 60 minutes following treatment of patients experiencing an OFF episode in the clinic. A separate MMRM model will be fitted for each of the time points.
- A ≥3, ≥6, and ≥11 point reduction in the UPDRS Part 3 motor score from pre-dose to post-dose, at 10 to 60 minutes following treatment in the clinic (cumulative and non-cumulative). For the non-cumulative analysis, the proportions of patients with a reduction will be tabulated by treatment group, visit and time point. For the cumulative analysis, the cumulative proportions of patients who achieved the first reduction before or at the time point in question will be tabulated by visit and time point.



# Statistical Analysis Plan

- Resolution of an OFF to an ON state within 60 minutes after study drug is administered in the clinic and maintaining the ON at 60 minutes after study drug administration (per the examiner's subjective assessment). This endpoint will be based on the examiner's subjective assessment. The proportions of patients will be summarized descriptively for each CVT-301 treated patients. The missing values will be counted as non-resolved.
- Change from baseline (3 consecutive days prior to TV/OV1) in patient-recorded total daily OFF time, assessed by the patient and recorded in the PD Diary for 3 consecutive days prior to the visit. Similar methods as for primary endpoint will be used. However, the baseline daily OFF time will be used as a covariate in the MMRM model instead of the OFF-state baseline UPDRS part 3 score. Only valid diary days will be included in the diary summarizations. In addition, change from baseline in total daily ON time without dyskinesia, total daily ON time with non-troublesome dyskinesia, and total daily ON time with troublesome dyskinesia.
- The PGI-C score. The proportions of patients who improved (much improved, improved or a little improved) will be tabulated by visit for CVT-301 treated patients. This summary will be complemented by the distribution of each response category (much improved, improved, a little improved, no change, a little worse, worse, much worse) tabulated by the treatment group.
- Changes from TV/OV1 in endpoints based on S&E ADL score, UPDRS Part 2 score, and PDQ-39 sub-scores. An ANCOVA model with the treatment group and stratification variables as fixed factors and the TV/OV1 value as a covariate will be used to estimate the treatment differences. Otherwise, the data will be presented with descriptive statistics only classified by treatment group and visit. The observed cases will be used in the analysis and summaries.

### Sensitivity analyses of the exploratory efficacy data

The following sensitivity analysis will be performed for the UPDRS Part 3 motor scores at 30 minutes post-dose and daily OFF time exploratory efficacy endpoints.

• MI analysis: MI techniques based on Pattern Mixture Models (PMM) will be applied (Ratitch et al., 2011) as a further sensitivity analysis in the ITT population. This methodology will structure data based on missing data patterns. The method will be based on a missingness pattern having a monotone structure, i.e. if among the observations over time one data value is missing, all other values after this missing value will also be treated as missing. For patients with intermittent missing values, before performing MI based on the PMM, it will be necessary to create a monotone missingness pattern. Intermittent missing values will be imputed using the Markov Chain Monte Carlo (MCMC) methodology which assumes a multivariate normal



# Statistical Analysis Plan

distribution over all variables included in the imputation model. The MI procedure in SAS will be used for this purpose and this first MI step is planned to be repeated 100 times, creating several different datasets with a monotone missing data structure. Seed value of 201508 will be used in the MI procedure. The imputation is based on the missing at random (MAR) assumption, i.e. the missing data are assumed to follow the same model as the other patients in their respective treatment arm that have complete data.

After this, the remaining missing data can be imputed using a method for monotone missingness, also based on the MAR assumption. Thus, for each of the created datasets with a monotone missing data pattern, the MI procedure in SAS will used to impute missing values based on a sequential procedure reflecting the monotone missing data pattern. Patients with the first missing value occurring at visit at Month 1 will have their missing Month 1 value replaced by an imputed value from a regression model with baseline value and the stratification factors as explanatory variables. In the next step, patients with their Month 3 value missing will have their missing Month 3 value replaced by an imputed value from a regression mode with baseline spirometry value, stratification factors and the Month 1 value as explanatory variables. Similar procedure will be used to replace the missing values at Month 6, 9 and 12.

The imputed datasets generated with the approach described above do contain only non-missing values and are used as input in the model for the exploratory efficacy endpoint. MMRM models similar as described above will thus be run on each of the generated imputed datasets. Finally, the MIANALYZE procedure in SAS will be applied to combine the results from these several datasets to derive an overall estimate of the within-group changes.



## Statistical Analysis Plan

### 10. INTERIM ANALYSES

Safety data will be reviewed by a Data Safety Monitoring Committee (DSMC) that will include relevant medical experts (including a neurologist and pulmonologist), an independent statistician, and additional representatives (as will be defined in the DSMC Charter). Safety data, including but not limited to AEs, spirometry, vital signs, and ECG data will be reviewed. The safety review will be documented in a DSMC Charter prior to the start of the study. In the event that potential safety issues are identified, the committee may recommend modification of the study design or study termination, which will be communicated promptly with investigators, IRBs, IECs, and regulatory agencies, in accordance with legal and regulatory requirements. There will be no prospective interim evaluation of efficacy endpoint data.

Data summary, which will not affect study conduct, may be prepared to support regulatory submission. These analyses will be described in the Interim Analysis Charter.



# Statistical Analysis Plan

# 11. CHANGE FROM ANALYSIS PLANNED IN PROTOCOL

There are no changes from the analyses planned in the protocol.




## Statistical Analysis Plan

## 12. PROGRAMMING CONSIDERATIONS

All tables, listings, figures (TLFs), and statistical analyses will be generated using SAS® for Windows, Release 9.3 (SAS® Institute Inc., Cary, NC, USA) or higher. Computergenerated table, listing and figure output produced by INC Research will adhere to the following specifications.

#### 12.1. GENERAL CONSIDERATIONS

- One SAS program can create several outputs.
- One output file can contain several outputs.
- Output files will be delivered in Word format.
- Numbering of TFLs will follow ICH E3 guidance

## 12.2. TABLE, LISTING, AND FIGURE FORMAT

#### 12.2.1. General

- All TLFs will be produced in landscape format, unless otherwise specified.
- All TLFs will be produced using the Courier New font, size 8
- The data displays for all TLFs will have a 1.5-inch binding margin on top of a landscape oriented page and a minimum 1-inch margin on the other 3 sides.
- Headers and footers for figures will be in Courier New font, size 8.
- Legends will be used for all figures with more than 1 variable, group, or item displayed.
- TLFs will be in black and white (no color), unless otherwise specified. For spirometry graphs, separate colors will be used for ON (red circles) and OFF (blue triangles) State data.
- Specialized text styles, such as bolding, italics, borders, shading, and superscripted and subscripted text, will not be used in the TLFs, unless otherwise specified.
- Only standard keyboard characters will be used in the TLFs. Special characters, such as non-printable control characters, printer-specific, or font-specific characters, will not be used.
- Mixed case will be used for all titles, column headers, and programmer-supplied formats, as appropriate.

## 12.2.2. Headers

All output should have the following header at the top left of each page:




# Statistical Analysis Plan

Civitas Therapeutics, Inc.

- All output should have Page n of N at the top or bottom right corner of each page. TLFs should be internally paginated in relation to the total length (i.e., the page number should appear sequentially as page n of N, where N is the total number of pages in the table).
- The date and time (date and time output was generated) should appear along with program name and location as the last footer on each page.

### 12.2.3. Display Titles

• Each TLF should be identified by the designation and a numeral. (i.e., Table 14.1.1). The title is centered. The title and table designation are single spaced. A solid line spanning the margins will separate the display titles from the column headers. There will be 1 blank line between the last title and the solid line.

### 12.2.4. Column Headers

- Column headings should be displayed immediately below the solid line described above.
- Analysis set sizes will be presented for each treatment group in the column heading as (N=xx) (or in the row headings if applicable). This is distinct from the 'n' used for the descriptive statistics representing the number of patients in the analysis set.
- The order of treatments in the tables will be Placebo first, followed by CVT-301 and a total column (if applicable in tables).

## 12.2.5. Body of the Data Display

### 12.2.5.1. General Conventions

Data in columns of a table or listing should be formatted as follows:

- alphanumeric values are left-justified;
- whole numbers (e.g., counts) are right-justified; and
- · numbers containing fractional portions are decimal aligned.

### 12.2.5.2. Table Conventions

- Units will be included where available
- Unless otherwise specified, the estimated mean and median for a set of values should be printed out to 1 more significant digit than the original values, and

Acorda Therapeutics, Inc. CVT-301-005




## Statistical Analysis Plan

standard deviations should be printed out to 2 more significant digits than the original values. The minimum and maximum should report the same significant digits as the original values. For example, for systolic blood pressure:

| N | XX |
|---------|-------|
| Mean | XXX.X |
| Std Dev | X.XX |
| Median | XXX.X |
| Minimum | XXX, |
| Maximum | XXX |

- P-values should be output in the format: "0.xxx", where xxx is the value rounded to 3 decimal places. Any p-value less than 0.001 will be presented as <0.001. If the p-value is returned as >0.999 then present as >0.999.
- Percentage values should be printed to one decimal place, in parentheses with no spaces, one space after the count, e.g., 7 (12.8%), 13 (5.4%). For a value that rounds down to 0.0, display it as "<0.1". Unless otherwise noted, for all percentages, the number of patients in the analysis set for the treatment group who have an observation will be the denominator. Percentages after zero counts should not be displayed and percentages equating to 100% should be presented as 100%, without any decimal places.

## 12.2.5.3. Listing Conventions

- Listings will be sorted for presentation in order of patient number, visit/collection day, and visit/collection time.
- Dates should be printed in SAS® DATE9.format ("ddMMMyyyy": 01JUL2000). Missing portions of dates should be represented on patient listings as dashes (--JUL2000).
- All observed time values must be presented using a 24-hour clock HH:MM or HH:MM:SS format (e.g., 11:26:45, or 11:26).

#### 12.2.6. Footnotes

- A solid line spanning the margins will separate the body of the data display from the footnotes.
- All footnotes will be left justified with single-line spacing immediately below the solid line underneath the data display.



# Statistical Analysis Plan

• The last line of the footnote section will be a standard source line that indicates the name of the program used to produce the data display, date and time the program was run.



# Statistical Analysis Plan

## 13. QUALITY CONTROL

SAS programs are developed to produce clinical trial output such as analysis data sets, summary tables, data listings, figures or statistical analyses. INC Research SOP 03.010.00 and 03.013.00 provide an overview of the development of such SAS programs.

INC Research SOP 03.009.00 describes the quality control procedures that are performed for all SAS programs and output. Quality control is defined here as the operational techniques and activities undertaken to verify that the SAS programs produce the proper clinical trial output by checking for their logic, efficiency and commenting and by review of the produced output.



# Statistical Analysis Plan

# 14. INDEX OF TABLES

| Table 14.1.1.2Number of Subjects in Each Population by Study Center All SubjectsTable 14.1.2.1Summary of Protocol Deviation Randomized SetTable 14.1.3.1.1Demographic and Baseline Characteristics (Safety Population)Table 14.1.3.1.2Demographic and Baseline Characteristics (ITT Population)Table 14.1.3.1.3Demographic and Baseline Characteristics by Baseline PD Severity (ITT Population)Table 14.1.3.1.4Demographic and Baseline Characteristics by Baseline Dyskinesia (ITT Population)Table 14.1.3.1.5Demographic and Baseline Characteristics by Baseline Daily Levodopa Dose (ITT |
|---|
| Table 14.1.3.1.1 Demographic and Baseline Characteristics (Safety Population) Table 14.1.3.1.2 Demographic and Baseline Characteristics (ITT Population) Table 14.1.3.1.3 Demographic and Baseline Characteristics by Baseline PD Severity (ITT Population) Table 14.1.3.1.4 Demographic and Baseline Characteristics by Baseline Dyskinesia (ITT Population) |
| Table 14.1.3.1.2 Demographic and Baseline Characteristics (ITT Population) Table 14.1.3.1.3 Demographic and Baseline Characteristics by Baseline PD Severity (ITT Population) Table 14.1.3.1.4 Demographic and Baseline Characteristics by Baseline Dyskinesia (ITT Population) |
| Table 14.1.3.1.3 Demographic and Baseline Characteristics by Baseline PD Severity (ITT Population) Table 14.1.3.1.4 Demographic and Baseline Characteristics by Baseline Dyskinesia (ITT Population) |
| Population) Table 14.1.3.1.4 Demographic and Baseline Characteristics by Baseline Dyskinesia (ITT Population) |
| Table 14.1.3.1.4 Demographic and Baseline Characteristics by Baseline Dyskinesia (ITT Population) |
| Population) |
| Table 14.1.3.1.5 Demographic and Baseline Characteristics by Baseline Daily Levodopa Dose (ITT |
| Population) |
| Table 14.1.3.1.6 Demographic and Baseline Characteristics by PD Diary Mean Daily OFF Time during Screening (ITT Population) |
| Table 14.1.3.1.7 Demographic and Baseline Characteristics by Screening Spirometry (ITT Population) |
| Table 14.1.3.1.8 Demographic and Baseline Characteristics by Age Group (ITT Population) |
| Table 14.1.3.1.9 Demographic and Baseline Characteristics by Gender (ITT Population) |
| Table 14.1.3.2.1 Parkinson's Disease History (Safety Population) |
| Table 14.1.3.2.2 Parkinson's Disease History (ITT Population) |
| Table 14.1.3.2.3 Parkinson's Disease History by Baseline PD Severity (ITT Population) |
| Table 14.1.3.2.4 Parkinson's Disease History by Baseline Dyskinesia (ITT Population) |
| Table 14.1.3.2.5 Parkinson's Disease History by Baseline Daily Levodopa Dose (ITT Population) |
| Table 14.1.3.2.6 Parkinson's Disease History by PD Diary Mean Daily OFF Time during Screening (ITT Population) |
| Table 14.1.3.2.7 Parkinson's Disease History by Screening Spirometry (ITT Population) |
| Table 14.1.3.2.8 Parkinson's Disease History by Age Group (ITT Population) |
| Table 14.1.3.2.9 Parkinson's Disease History by Gender (ITT Population) |
| Table 14.1.3.2.10 Modified Hoehn and Yahr Staging in "ON" State (Safety Population) |
| Table 14.1.3.2.11 Modified Hoehn and Yahr Staging in "ON" State (ITT Population) |
| Table 14.1.3.2.12 Distribution of Average Daily OFF Time (Safety Population) |
| Table 14.1.3.2.13 Distribution of cumulative Average Daily OFF Time (Safety Population) |
| Table 14.1.3.3 Medical History (Safety Population) |
| Table 14.1.4.1 Prior Medications (Safety Population) |
| Table 14.1.4.2 Concomitant Medications (Safety Population) |
| Table 14.1.4.3 Parkinson's disease Treatment Medications at Baseline (ITT Population) |
| Table 14.2.1.1 Exploratory Efficacy Analysis: Change from Pre-dose in the UPDRS Part 3 Score |
| at 10 Minutes Post-dose by Visit (ITT Population) |
| Table 14.2.1.2 Exploratory Efficacy Analysis: Change from Pre-dose in the UPDRS Part 3 Score |
| at 20 Minutes Post-dose by Visit (ITT Population) |
| Table 14.2.1.3.1 Exploratory Efficacy Analysis: Change from Pre-dose in the UPDRS Part 3 Score |
| at 30 Minutes Post-dose by Visit (ITT Population) |
| Table 14.2.1.3.2 Sensitivity Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 30 |
| Minutes Post-dose by Visit (ITT Population) |



| Table 14.2.1.3.3 | Exploratory Efficacy Subgroup Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 30 Minutes Post-dose by Visit by Baseline PD Severity (ITT Population) |
|---|---|
| Table 14.2.1.3.4 | Exploratory Efficacy Subgroup Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 30 Minutes Post-dose by Visit by Baseline Dyskinesia (ITT Population) |
| Table 14.2.1.3.5 | Exploratory Efficacy Subgroup Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 30 Minutes Post-dose by Visit by Baseline Daily Levodopa Dose (ITT Population) |
| Table 14.2.1.3.6 | Exploratory Efficacy Subgroup Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 30 Minutes Post-dose by Visit by PD Diary Mean Daily OFF Time during Screening (ITT Population) |
| Table 14.2.1.3.7 | Exploratory Efficacy Exploratory Efficacy Subgroup Analysis: Change from Predose in the UPDRS Part 3 Score at 30 Minutes Post-dose by Visit by Screening Spirometry (ITT Population) |
| Table 14.2.1.3.8 | Exploratory Efficacy Exploratory Efficacy Subgroup Analysis: Mean Change from Pre-dose in the UPDRS Part 3 Score at 30 Minutes Post-dose by Visit by Age Group (ITT Population) |
| Table 14.2.1.3.9 | Exploratory Efficacy Exploratory Efficacy Subgroup Analysis: Mean Change from Pre-dose in the UPDRS Part 3 Score at 30 Minutes Post-dose by Visit by Gender (ITT Population) |
| Table 14.2.1.4 | Exploratory Efficacy Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 60 Minutes Post-dose by Visit (ITT Population) |
| Table 14.2.1.5 | Exploratory Efficacy Analysis: Change from Pre-dose in the Average UPDRS Part 3 Score at 10 to 60 Minutes Post-dose by Visit (ITT Population) |
| Table 14.2.2.1 | Exploratory Efficacy Analysis: Change from Pre-dose in UPDRS Part 3 Score to 10, 20, 30, 60 minutes Post-dose by Visit (ITT Population) |
| Table 14.2.2.2 | Exploratory Efficacy Analysis: Change from Pre-Dose to 10, 20, 30, 60 minutes Post-dose in UPDRS Part 3 Score by Visit and Timepoint (ITT Population) |
| Table 14.2.2.3 | Exploratory Efficacy Analysis: Change from Pre-Dose to 10, 20, 30, 60 minutes Post-dose in UPDRS Part 3 Score by Timepoint and Visit (ITT Population) |
| Table 14.2.3.1 | Exploratory Efficacy Analysis Subjects with a >= 3 Reduction from Pre-dose to Post-dose in the UPDRS Part 3 Score by Visit (ITT Population) |
| Table 14.2.3.2 | Exploratory Efficacy Analysis Subjects with a >= 3 Reduction from Pre-dose to Post-dose in the UPDRS Part 3 Score by Visit With Percentages Based on N (ITT Population) |
| Table 14.2.3.3 | Exploratory Efficacy Analysis Subjects with a >=6 Reduction from Pre-dose to Post-dose in the UPDRS Part 3 Score by Visit (ITT Population) |
| Table 14.2.3.4 | Exploratory Efficacy Analysis Subjects with a >=6 Reduction from Pre-dose to Post-dose in the UPDRS Part 3 Score by Visit With Percentages Based on N (ITT Population) |
| Table 14.2.3.5 | Exploratory Efficacy Analysis Subjects with a >=11 Reduction from Pre-dose to Post-dose in the UPDRS Part 3 Score by Visit (ITT Population) |
| Table 14.2.3.6 | Exploratory Efficacy Analysis Subjects with a >=11 Reduction from Pre-dose to Post-dose in the UPDRS Part 3 Score by Visit With Percentages Based on N (ITT Population) |
| Table 14.2.4.1 | Exploratory Efficacy Analysis: Subjects Achieving Resolution of an OFF to an ON |



| | State within 60 Minutes by Visit Worst Case Imputation [a] (ITT Population) |
|---|---|
| Table 14.2.5.1.1 | Exploratory Efficacy Analysis: Mean of Total Daily OFF Time by Visit (ITT |
| Table 14.2.5.1.1 | Population) |
| Table 14.2.5.1.2 | Sensitivity Analysis: Mean of Total Daily OFF Time by Visit MI analysis with |
| | Missing At Random Assumption (ITT Population |
| Table 14.2.5.1.3 | Exploratory Efficacy Subgroup Analysis: Mean of Total Daily OFF Time by Visit by |
| | Baseline PD Severity (ITT Population) |
| Table 14.2.5.1.4 | Exploratory Efficacy Subgroup Analysis: Mean of Total Daily OFF Time by Visit by |
| | Baseline Dyskinesia (ITT Population) |
| Table 14.2.5.1.5 | Exploratory Efficacy Subgroup Analysis: Mean of Total Daily OFF Time by Visit by |
| | Baseline Daily Levodopa Dose (ITT Population) |
| Table 14.2.5.1.6 | Exploratory Efficacy Subgroup Analysis: Mean of Total Daily OFF Time by Visit by |
| | PD Diary Mean Daily OFF Time during Screening (ITT Population) |
| Table 14.2.5.1.7 | Exploratory Efficacy Subgroup Analysis: Mean of Total Daily OFF Time by Visit by |
| | Screening Spirometry (ITT Population) |
| Table 14.2.5.1.8 | Exploratory Efficacy Subgroup Analysis: Mean of Total Daily OFF Time by Visit by |
| | Age Group (ITT Population) |
| Table 14.2.5.1.9 | Exploratory Efficacy Subgroup Analysis: Mean of Total Daily OFF Time by Visit by |
| | Gender (ITT Population) |
| Table 14.2.5.2 | Exploratory Efficacy Analysis: Mean of Total Daily ON Time without Dyskinesia |
| | by Visit (ITT Population) |
| Table 14.2.5.3 | Exploratory Efficacy Analysis: Mean of Total Daily ON Time with non- |
| | Troublesome Dyskinesia by Visit (ITT Population) |
| Table 14.2.5.4 | Exploratory Efficacy Analysis: Mean of Total Daily ON Time with Troublesome |
| | Dyskinesia by Visit (ITT Population) |
| Table 14.2.6.1 | Exploratory Efficacy Analysis: Subjects Global Impression of Change (PGI-C) by |
| | Visit Worst Case Imputation [a] (ITT Population) |
| Table 14.2.7.1 | Exploratory Efficacy Analysis: UPDRS Part 2 Score at TV4/OV4 (ITT Population) |
| Table 14.2.7.2 | Exploratory Efficacy Analysis: UPDRS Part 2 Score at TV6/OV6 (ITT Population) |
| Table 14.2.8.1 | Exploratory Efficacy Analysis: Schwab and England (S&E) Activities of Daily |
| | Living (ADL) Score at TV4/OV4 (ITT Population) |
| Table 14.2.8.2 | Exploratory Efficacy Analysis: Schwab and England (S&E) Activities of Daily |
| | Living (ADL) Score at TV6/OV6 (ITT Population) |
| Table 14.2.9.1 | Exploratory Efficacy Analysis: 39 Item Parkinson's disease Questionnaire (PDQ- |
| | 39) Sub-scores and Summary Index Score at TV4/OV4 (ITT Population) |
| Table 14.2.9.2 | Exploratory Efficacy Analysis: 39 Item Parkinson's disease Questionnaire (PDQ- |
| | 39) Sub-scores and Summary Index Score at TV6/OV6 (ITT Population) |
| Table 14.3.1.1 | Extent of Exposure: Overall (Safety Population) |
| Table 14.3.1.2 | In-Clinic Study Drug Administration (Safety Population) |
| Table 14.3.1.3 | Distribution of Time of Study Drug Administration (Safety Population) |
| Table 14.3.2.1 | Treatment-emergent adverse events -Overall Summary (Safety Population) |
| Table 14.3.2.2.1 | Treatment-emergent adverse events by System Organ Class and Preferred Term |
| | (Safety Population) |
| Table 14.3.2.2.2 | Treatment-emergent adverse events by Preferred Term (Safety Population) |
| Table 14.3.2.3 | Drug-Related Treatment-emergent adverse events by System Organ Class, |
| | Preferred Term and Severity (Safety Population) |
| | , |



| Table 14.3.2.4 | Drug -Related Treatment-emergent adverse events by System Organ Class, Preferred Term and Relationship (Safety Population) |
|---|---|
| Table 14.3.2.5 | Drug-related Treatment-emergent adverse events by System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.2.6 | Serious Treatment-emergent adverse events by System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.2.7 | Listing of Serious Adverse Events |
| Table 14.3.2.8 | Listing of Adverse Events Leading to Death |
| Table 14.3.2.9 | Severe Treatment-emergent adverse events by System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.2.10 | Listing of Severe Treatment-Emergent Adverse Events |
| Table 14.3.2.11 | Treatment-emergent adverse events Leading to Study Drug Interruption by System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.2.12 | Listing of Adverse Events Leading to Study Drug Interruption |
| Table 14.3.2.13 | Treatment-emergent adverse events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.2.14 | Listing of Adverse Events Leading to Study Drug Discontinuation |
| Table 14.3.2.15 | Treatment-emergent adverse events Leading to Dose Reduction by System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.2.16 | Listing of Adverse Events Leading to Dose Reduction |
| Table 14.3.2.17 | Most Common Treatment-Emergent Adverse Events (Preferred Term Occurred in >10% of Over Patients) by System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.2.18 | Listing of Most Common Treatment-Emergent Adverse Events |
| Table 14.3.2.19 | Time to first Onset of most Common Treatment-Emergent Adverse Events (Preferred Term Occurred in >10% of Over Patients) (Safety Population) |
| Table 14.3.4.1 | Clinical Laboratory Results: PCS and PCSC Criteria |
| Table 14.3.4.1.1.1 | Summary of Clinical Laboratory Results: Hematology (Safety Population) |
| Table 14.3.4.1.1.2 | Summary of Clinical Laboratory Results: Hematology Abnormal Values (Safety Population) |
| Table 14.3.4.1.1.3 | Summary of Clinical Laboratory Results: Hematology Abnormal Values -Shift from Baseline (Safety Population) |
| Table 14.3.4.1.1.4 | Summary of Clinical Laboratory Results: Hematology PCS Values -Shift from Baseline (Safety Population) |
| Table 14.3.4.1.1.5 | Summary of Clinical Laboratory Results: Hematology PCSC Values -Shift from Baseline (Safety Population) |
| Table 14.3.4.1.1.6 | Clinical Laboratory Results - Hematology PCS and PCSC Values (Safety Population) |
| Table 14.3.4.1.2.1 | Summary of Clinical Laboratory Results: Chemistry (Safety Population) |
| Table 14.3.4.1.2.2 | Summary of Clinical Laboratory Results: Chemistry Abnormal Values (Safety Population) |
| Table 14.3.4.1.2.3 | Summary of Clinical Laboratory Results: Chemistry Abnormal Values -Shift from Baseline (Safety Population) |
| Table 14.3.4.1.2.4 | Summary of Clinical Laboratory Results: Chemistry PCS Values -Shift from Baseline (Safety Population) |
| Table 14.3.4.1.2.5 | Summary of Clinical Laboratory Results: Chemistry PCSC Values -Shift from |



| | Baseline (Safety Population) |
|---|---|
| Table 14.3.4.1.2.6 | Clinical Laboratory Results - Chemistry PCS and PCSC Values (Safety Population) |
| Table 14.3.4.1.2.0 | Ctiffical Laboratory Results - Chemistry PCs and PCsC values (safety Population) |
| Table 14.3.4.2 | Vital Signs: PCS and PCSC Criteria |
| Table 14.3.4.2.1 | Summary of Vital Signs: Actual Values and Change from Baseline across Visits |
| | (Safety Population) |
| Table 14.3.4.2.2 | Summary of Vital Signs: Actual Values and Change from Pre-dose at TV1 (Safety |
| | Population) |
| Table 14.3.4.2.3 | Summary of Standard Vital Signs: PCS and PCSC Values by Visit (Safety |
| | Population) |
| Table 14.3.4.2.4 | Summary of Standard Vital Signs: PCS and PCSC Values by Scheduled Timepoint |
| | at TV1 (Safety Population) |
| Table 14.3.4.2.5 | Standard Vital Signs: PCS and PCSC Values |
| Table 14.3.4.2.6 | Summary of Vital Signs: Orthostatic Hypotension by Visit (Safety Population) |
| Table 14.3.4.2.7 | Summary of Vital Signs: Orthostatic Hypotension by Scheduled Timepoint at TV1 |
| | (Safety Population) |
| Table 14.3.4.2.8 | Orthostatic Vital Signs |
| Table 14.3.4.3 | 12-Lead ECG:PCS and PCSC Criteria |
| Table 14.3.4.3.1 | Summary of 12-Lead ECG: Actual Values and Change across Visits (Safety |
| | Population) |
| Table 14.3.4.3.2 | Summary of 12-Lead ECG: PCS and PCSC Values (Safety Population) |
| Table 14.3.4.3.3 | 12-Lead Electrocardiogram (ECG): PCS and PCSC Values |
| Table 14.3.4.4 | Physical Examination (Safety Population) |
| Table 14.3.4.5.1.1 | Summary of Spirometry(Neurology Office): Actual Values and Change from Baseline for FEV1 and FVC by Visit (Safety Population) |
| Table 14.3.4.5.1.2 | Summary of Spirometry(Neurology Office): Actual Values and Change from |
| | Baseline for FEV1 and FVC by Visit Using Subset of Assessments Meeting the ATS |
| | Quality Criteria (Safety Population) |
| Table 14.3.4.5.1.3 | Summary of Spirometry(Neurology Office): Actual Values and Change from |
| | Baseline for FEV1 and FVC by Visit Excluding Patients with Co-efficient of |
| | Variation (CV) of FEV1 >7.5% (Safety Population) |
| Table 14.3.4.5.1.4 | MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for |
| T:11: 44 2 4 5 4 5 | FEV1 by Visit (Safety Population) |
| Table 14.3.4.5.1.5 | MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for |
| | FEV1 by Visit Using Subset of Assessments Meeting the ATS Quality Criteria |
| Table 14.3.4.5.1.6 | (Safety Population) MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for |
| Table 14.3.4.3.1.6 | FEV1 by Visit Excluding Patients with Co-efficient of Variation (CV) of FEV1 |
| | >7.5% (Safety Population) |
| Table 14.3.4.5.1.7 | Sensitivity Analysis Using MMRM: Change from Baseline for FEV1 by Visit MI |
| | analysis with Missing At Random Assumption (ITT Population) |
| Table 14.3.4.5.1.8 | MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for |
| | Percentage Predicted FEV1 by Visit (Safety Population) |
| Table 14.3.4.5.1.9 | MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for |
| | Percentage Predicted FEV1 by Visit Using Subset of Assessments Meeting the ATS |
| | Quality Criteria (Safety Population) |



| Table 14.3.4.5.1.10 | MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for Percentage Predicted FEV1 by Visit Excluding Patients with Co-efficient of Variation (CV) of FEV1 >7.5% (Safety Population) |
|---|---|
| Table 14.3.4.5.1.11 | Sensitivity Analysis Using MMRM: Change from Baseline for Percentage Predicted FEV1 by Visit MI analysis with Missing At Random Assumption (ITT Population) |
| Table 14.3.4.5.1.12 | MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for FVC by Visit (Safety Population) |
| Table 14.3.4.5.1.13 | MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for FVC by Visit Using Subset of Assessments Meeting the ATS Quality Criteria (Safety Population) |
| Table 14.3.4.5.1.14 | MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for FVC by Visit Excluding Patients with Co-efficient of Variation (CV) of FEV1 >7.5% (Safety Population) |
| Table 14.3.4.5.1.15 | Sensitivity Analysis Using MMRM: Change from Baseline for FVC by Visit MI analysis with Missing At Random Assumption (ITT Population) |
| Table 14.3.4.5.1.16 | MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for Percentage Predicted FVC by Visit (Safety Population) |
| Table 14.3.4.5.1.17 | MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for Percentage Predicted FVC by Visit Using Subset of Assessments Meeting the ATS Quality Criteria (Safety Population) |
| Table 14.3.4.5.1.18 | MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for Percentage Predicted FVC by Visit Excluding Patients with Co-efficient of Variation (CV) of FEV1 >7.5% (Safety Population) |
| Table 14.3.4.5.1.19 | Sensitivity Analysis Using MMRM: Change from Baseline for Percentage Predicted FVC by Visit MI analysis with Missing At Random Assumption (ITT Population) |
| Table 14.3.4.5.2.1 | Summary of Spirometry: (Neurology Office): Actual Values and Change from Baseline for FEV1/FVC by Visit (Safety Population) |
| Table 14.3.4.5.2.2 | Summary of Spirometry: (Neurology Office): Actual Values and Change from Baseline for FEV1/FVC by Visit Using Subset of Assessments Meeting the ATS Quality Criteria (Safety Population) |
| Table 14.3.4.5.2.3 | Summary of Spirometry: (Neurology Office): Actual Values and Change from Baseline for FEV1/FVC by Visit Excluding Patients with Co-efficient of Variation (CV) of FEV1 >7.5% (Safety Population) |
| Table 14.3.4.5.2.4 | MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for FEV1/FVC by Visit (Safety Population) |
| Table 14.3.4.5.2.5 | MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for FEV1/FVC by Visit Using Subset of Assessments Meeting the ATS Quality Criteria (Safety Population) |
| Table 14.3.4.5.2.6 | MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for FEV1/FVC by Visit Excluding Patients with Co-efficient of Variation (CV) of FEV1 >7.5% (Safety Population) |
| Table 14.3.4.5.2.7 | Sensitivity Analysis Using MMRM: Change from Baseline for FEV1/FVC by Visit MI analysis with Missing At Random Assumption (ITT Population) |
| Table 14.3.4.5.3.1 | Summary of Spirometry (Neurology Office): Summary of FEV1/FVC < 60% and <70% by Visit (Safety Population) |
| Table 14.3.4.5.3.2 | Summary of Spirometry (Neurology Office): Summary of FEV1/FVC < 60% and |



| | 700/ b Maria Harris C. basel of Assessment Maria and baseling the ATC C. 199 C. 199 |
|---|---|
| | <70% by Visit Using Subset of Assessments Meeting the ATS Quality Criteria (Safety Population) |
| Table 14.3.4.5.3.3 | Summary of Spirometry (Neurology Office): Summary of FEV1/FVC < 60% and |
| ומטוכ וד.ט.ד.ט.ט | <70% by Visit Excluding Patients with Co-efficient of Variation (CV) of FEV1 |
| | >7.5% (Safety Population) |
| Table 14.3.4.5.4 | Spirometry(Neurology Office): 70% or Smaller FEV1/FVC Values and >=200 |
| 14566 1 1.5. 1.5. 1 | Reduction from Pre-dose |
| Table 14.3.4.5.5 | Summary of Spirometry (Neurology Office): Measurements Meeting ATS Quality |
| | Criteria (Safety Population) |
| Table 14.3.4.5.6 | Summary of Spirometry(Pulmonary Function Facility): Actual Values and Change |
| | from Baseline for Calculated DLco Parameters by Visit (Safety Population) |
| Table 14.3.4.5.7 | Summary of Spirometry(Pulmonary Function Facility): Actual Values and Change |
| | from Baseline for FEV1 and FVC by Visit (Safety Population) |
| Table 14.3.4.5.8 | Summary of Spirometry(Pulmonary Function Facility): Actual Values and Change |
| <del></del> | from Baseline for FEV1/FVC by Visit (Safety Population) |
| Table 14.3.4.5.9 | Summary of Spirometry (Pulmonary Function Facility): Summary of FEV1/FVC < |
| Table 44.2.4.5.40 | 60% and <70%by Visit (Safety Population) Spirometry(Pulmonary Function Facility):70% or Smaller FEV1/FVC Values by |
| Table 14.3.4.5.10 | Visit |
| Table 14.3.4.5.11 | Summary of Spirometry(Pulmonary Function Facility): Measurements Meeting |
| 14.5.4.5.11 | ATS Quality Criteria (Safety Population) |
| Table 14.3.4.6.1 | Summary of Columbia-Suicide Severity Rating Scale (C-SSRS) (Safety Population) |
| | ballinary or columnia ballone covering reality (caree) reparationly |
| Table 14.3.4.6.2 | Shift from Baseline in Columbia-Suicide Severity Rating Scale (C-SSRS) (Safety |
| | Population) |
| Table 14.3.4.7 | Summary of Epworth Sleepiness Scale Total Score: Actual Values and Change |
| | from Baseline by Visit (Safety Population) |
| Table 14.3.4.8 | Summary of Questionnaire for Impulsive-Compulsive Disorders in Parkinson's |
| | (QUIP) by Visit (Safety Population) |
| Table 14.3.4.9.1 | MMRM Analysis of UPDRS Part 4: Change from Baseline in the UPDRS Part 4 Score |
| | at TV4 (Safety Population) |
| Table 14.3.4.9.2 | MMRM Analysis of UPDRS Part 4 Dyskinesias Score: Change from Baseline in the |
| Table 14.3.4.9.3 | UPDRS Part 4 Score at TV4 (Safety Population) MMRM Analysis of UPDRS Part 4 Fluctuations Score: Change from Baseline in the |
| Table 14.3.4.9.3 | LIDDES Part 4 Score at TV4 (Safety Population) |
| Table 14.3.4.9.4 | UPDRS Part 4 Score at TV4 (Safety Population) Summary of UPDRS Part 4: Actual Values and Change from Baseline by Visit |
| 14.3.4.7.4 | (Safety Population) |
| Table 14.3.4.9.5 | Summary of UPDRS Part 4 Dyskinesias Score: Actual Values and Change from |
| | Baseline by Visit (Safety Population) |
| Table 14.3.4.9.6 | Summary of UPDRS Part 4 Fluctuations Score: Actual Values and Change from |
| 1 | Baseline by Visit (Safety Population) |
| Table 14.3.4.10 | Dyskinesia: Occurrence and Severity (In-clinic) by Visit (ITT Population) |

1003805 Acorda Therapeutics, Inc. CVT-301-005




# Statistical Analysis Plan

# 15. INDEX OF LISTINGS

| Listing 16.2.1 | Patient Disposition |
|---|---|
| Listing 16.2.2.1 | Protocol Deviations |
| Listing 16.2.3.1 | Inclusion Criteria not Met at Screening |
| Listing 16.2.3.2 | Exclusion Criteria Met at Screening |
| Listing 16.2.3.3 | Analysis Populations |
| Listing 16.2.4.1 | Demographics |
| Listing 16.2.4.2 | Medical History |
| Listing 16.2.4.3 | Parkinson's Disease History |
| Listing 16.2.4.4 | Smoking History |
| Listing 16.2.4.5 | ON and OFF Concordance Testing at Screening |
| Listing 16.2.4.6 | Modified Hoehn and Yahr Staging in "ON" State at Screening |
| Listing 16.2.4.7 | Mini Mental State Examination (MMSE) at Screening |
| Listing 16.2.4.8 | Parkinson's Disease Diary Data at Screening: Derived Time |
| Listing 16.2.4.9 | Screening ON/OFF Log |
| Listing 16.2.4.10 | Randomization |
| Listing 16.2.4.11.1 | Prior and Concomitant Medications |
| Listing 16.2.4.11.2 | Parkinson's disease Treatment Medications at Baseline |
| Listing 16.2.4.12 | Baseline Pulmonary Assessment Part 2 - Pulmonary History |
| Listing 16.2.4.13 | Baseline Pulmonary Assessment Part 3 - Assessments of Symptoms |
| Listing 16.2.5.1.1 | Study Drug Administration: in Clinic and at Home |
| Listing 16.2.5.1.2 | Study Drug Administration: Derived Variables (in Clinic) |
| Listing 16.2.5.1.3 | Study Drug Administration: Derived Variables (Overall) |
| Listing 16.2.5.1.4 | Study Drug Administration: Derived Variables (Overall by Visit) |
| Listing 16.2.5.1.5 | Listing of Study Drug Dose Change |
| Listing 16.2.5.2 | Study Drug Kit Dispensation |
| Listing 16.2.5.3 | Daily Levodopa Dose |
| Listing 16.2.6.1.1 | Unified Parkinson's Disease Rating Scale (UPDRS) Part 3 |
| Listing 16.2.6.1.2 | Unified Parkinson's Disease Rating Scale (UPDRS) Part 3: Derived |
| | Variables |
| Listing 16.2.6.2.1 | Clinic Assessment |
| Listing 16.2.6.2.2 | Parkinson's Disease Diary Data |
| Listing 16.2.6.2.3.1 | Parkinson's Disease Diary Data - Derived Variable by Dairy Date |
| Listing 16.2.6.2.3.2 | Parkinson's Disease Diary Data - Derived Variable by Visit |
| Listing 16.2.6.2.4 | Patient's Global Impression of Change (PGI-C) |
| Listing 16.2.6.2.5 | Impact of Parkinson's OFF Episodes |
| Listing 16.2.6.3.1 | Unified Parkinson's Disease Rating Scale (UPDRS) Part 2 |
| Listing 16.2.6.3.2 | Listing of S&E Activities of Daily Living |
| Listing 16.2.6.3.3 | 39 Item Parkinson's Disease Questionnaire (PDQ-39) |
| Listing 16.2.7.1 | Adverse Events |
| Listing 16.2.8.1.1 | Clinical Laboratory Results - Hematology |
| Listing 16.2.8.1.2 | Clinical Laboratory Results - Chemistry |
| Listing 16.2.8.1.3 | Serum Pregnancy Test - Positive Only |
| Listing 16.2.8.2.1 | Vital Signs |



| Listing 16.2.8.2.2 | 12-Lead Electrocardiogram (ECG) |
|---|---|
| Listing 16.2.8.2.3 | Physical Examination |
| Listing 16.2.8.2.4.1 | Spirometry( Neurology Office) |
| Listing 16.2.8.2.4.2 | Spirometry( Neurology Office) Measurements Not Meeting ATS Quality |
| | Criteria |
| Listing 16.2.8.2.4.3 | Spirometry(Pulmonary Function Facility): DLco Parameters |
| Listing 16.2.8.2.4.4 | Spirometry(Pulmonary Function Facility): Spirometry/DLco Measurements |
| | Not Meeting ATS Quality Criteria |
| Listing 16.2.8.2.5 | Columbia-Suicide Severity Rating Scale (C-SSRS) |
| Listing 16.2.8.2.6 | Epworth Sleepiness Scale |
| Listing 16.2.8.2.7 | Questionnaire for Impulsive-Compulsive Disorders in Parkinson's (QUIP) |
| Listing 16.2.8.2.8.1 | Unified Parkinson's Disease Rating Scale (UPDRS) Part 4 |
| Listing 16.2.8.2.8.2 | Unified Parkinson's Disease Rating Scale (UPDRS) Part 4: Derived |
| | Variables |
| Listing 16.2.8.2.9.1 | Telephone Contact |
| Listing 16.2.8.2.9.2 | Telephone Contact: Challenges with Inhaler or Capsules Data |

1003805 Acorda Therapeutics, Inc. CVT-301-005



# Statistical Analysis Plan

# 16. INDEX OF FIGURES

Not Applicable.


#### Attachment 1 Table Mock-ups

#### Table of Contents

| Table 14.1.1.1 Number of Subjects Enforced and Study Termination (All Available Population) |
|---|
| Table 14.1.1.2 Number of Subjects in Each Population by Study Center All Subjects |
| Table 14.1.2.1 Summary of Protocol Deviation Randomized Set |
| Table 14.1.3.1.1 Demographic and Baseline Characteristics (Safety Population) |
| Table 14.1.3.1.2 Demographic and Baseline Characteristics (ITT Population) |
| Table 14.1.3.1.3 Demographic and Baseline Characteristics by Baseline PD Severity (ITT Population) |
| Table 14.1.3.1.4 Demographic and Baseline Characteristics by Baseline Dyskinesia (ITT Population) |
| Table 14.1.3.1.5 Demographic and Baseline Characteristics by Baseline Daily Levodopa Dose (ITT Population) |
| Table 14.1.3.1.6 Demographic and Baseline Characteristics by PD Diary Mean Daily OFF Time during Screening (ITT Population) |
| Table 14.1.3.1.7 Demographic and Baseline Characteristics by Screening Spirometry (ITT Population) |
| Table 14.1.3.1.8 Demographic and Baseline Characteristics by Age Group (ITT Population) |
| Table 14.1.3.1.9 Demographic and Baseline Characteristics by Gender (ITT Population) |
| Table 14.1.3.2.1 Parkinson's Disease History (Safety Population) |
| Table 14.1.3.2.2 Parkinson's Disease History (ITT Population) |
| Table 14.1.3.2.3 Parkinson's Disease History by Baseline PD Severity (ITT Population) |
| Table 14.1.3.2.4 Parkinson's Disease History by Baseline Dyskinesia (ITT Population) |
| Table 14.1.3.2.5 Parkinson's Disease History by Baseline Daily Levodopa Dose (ITT Population) |
| Table 14.1.3.2.6 Parkinson's Disease History by PD Diary Mean Daily OFF Time during Screening (ITT Population) |
| Table 14.1.3.2.7 Parkinson's Disease History by Screening Spirometry (ITT Population) |
| Table 14.1.3.2.8 Parkinson's Disease History by Age Group (ITT Population) |
| Table 14.1.3.2.9 Parkinson's Disease History by Gender (ITT Population) |
| Table 14.1.3.2.10 Modified Hoehn and Yahr Staging in "ON" State (Safety Population) |
| Table 14.1.3.2.11 Modified Hoehn and Yahr Staging in "ON" State (ITT Population) |
| Table 14.1.3.2.12 Distribution of Average Daily OFF Time at Baseline (Safety Population) |
| Table 14.1.3.2.13 Distribution of Cumulative Average Daily OFF Time at Baseline (Safety Population) |
| Table 14.1.3.3 Medical History (Safety Population) |
| Table 14.1.4.1 Prior Medications (Safety Population) |
| Table 14.1.4.2 Concomitant Medications (Safety Population) |
| Table 14.1.4.3 Parkinson's disease Treatment Medications at Baseline (ITT Population) |
| Table 14.2.1.1 Exploratory Efficacy Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 10 Minutes Post-dose by Visit (ITT |
| Population) |
| Table 14.2.1.2 Exploratory Efficacy Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 20 Minutes Post-dose by Visit (ITT |
| Population) |
| Table 14.2.1.3.1 Exploratory Efficacy Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 30 Minutes Post-dose by Visit |
| (ITT Population) |
| Table 14.2.1.3.2 Sensitivity Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 30 Minutes Post-dose by Visit MI analysis |
| with Missing At Random Assumption (ITT Population)2 |
| Table 14.2.1.3.3 Subgroup Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 30 Minutes Post-dose by Visit by Baseline PD |
| Severity (ITT Population) |
| Table 14.2.1.3.4 Exploratory Efficacy Subgroup Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 30 Minutes Post-dose by |
| Visit by Baseline Dyskinesia (ITT Population) |
| Table 14.2.1.3.5 Exploratory Efficacy Subgroup Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 30 Minutes Post-dose |
| by Visit by Baseline Daily Levodopa Dose (ITT Population) |
| Table 14.2.1.3.6 Exploratory Efficacy Subgroup Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 30 Minutes Post-dose by |
| Visit by PD Diary Mean Daily OFF Time during Screening (ITT Population) |
| Table 14.2.1.3.7 Exploratory Efficacy Subgroup Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 30 Minutes Post-dose by |
| Visit by Screening Spirometry (ITT Population) |

| Table 14.2.1.3.8 Exploratory Efficacy Subgroup Analysis: Mean Change from Pre-dose in the UPDRS Part 3 Score at 30 Minutes |
|---|
| Post-dose by Visit by Age Group (ITT Population) |
| Table 14.2.1.3.9 Exploratory Efficacy Subgroup Analysis: Mean Change from Pre-dose in the UPDRS Part 3 Score at 30 Minutes Post-dose by Visit by Gender (ITT Population) |
| Table 14.2.1.4 Exploratory Efficacy Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 60 Minutes Post-dose by Visit (ITT |
| Population) |
| Table 14.2.1.5 Exploratory Efficacy Analysis: Change from Pre-dose in the Average UPDRS Part 3 Score at 10 to 60 Minutes Post-dose |
| by Visit (ITT Population) |
| Table 14.2.2.1 Exploratory Efficacy Analysis: Change from Pre-dose in UPDRS Part 3 Score to 10, 20, 30, 60 minutes Post-dose by Visit (ITT Population) |
| Table 14.2.2.2 Exploratory Efficacy Analysis: Change from Pre-Dose to 10, 20, 30, 60 minutes Post-dose in UPDRS Part 3 Score by |
| Visit and Timepoint (ITT Population) |
| Table 14.2.2.3 Exploratory Efficacy Analysis: Change from Pre-Dose to 10, 20, 30, 60 minutes Post-dose in UPDRS Part 3 Score by |
| Timepoint and Visit (ITT Population) |
| Table 14.2.3.1 Exploratory Efficacy Analysis: Subjects with a >=3 Reduction from Pre-dose to Post-dose in the UPDRS Part 3 Score by |
| Visit (ITT Population) |
| 3 Score by Visit With Percentages Based on N (ITT Population) |
| Table 14.2.3.3 Exploratory Efficacy Analysis: Subjects with a >=6 Reduction from Pre-dose to Post-dose in the UPDRS Part 3 Score |
| by Visit (ITT Population) |
| Table 14.2.3.4 Exploratory Efficacy Analysis: Subjects with a >=6 Reduction from Pre-dose to Post-dose in the UPDRS Part 3 Score by |
| Visit With Percentages Based on N (ITT Population) |
| Table 14.2.3.5 Exploratory Efficacy Analysis: Subjects with a >=11 Reduction from Pre-dose to Post-dose in the UPDRS Part 3 Score by Visit (ITT Population) |
| Table 14.2.3.6 Exploratory Efficacy Analysis: Subjects with a >=11 Reduction from Pre-dose to Post-dose in the UPDRS Part 3 |
| Score by Visit With Percentages Based on N (ITT Population) |
| Table 14.2.4.1 Exploratory Efficacy Analysis: Subjects Achieving Resolution of an OFF to an ON State within 60 Minutes by Visit |
| Worst Case Imputation [a] (ITT Population) |
| Table 14.2.5.1.1 Exploratory Efficacy Analysis: Mean of Total Daily OFF Time by Visit (ITT Population) |
| Table 14.2.5.1.2 Sensitivity Analysis: Mean of Total Daily OFF Time by Visit MI analysis with Missing At Random Assumption (ITT |
| Population) |
| Population) |
| Table 14.2.5.1.4 Exploratory Efficacy Subgroup Analysis: Mean of Total Daily OFF Time by Visit by Baseline Dyskinesia (ITT |
| Population) |
| Table 14.2.5.1.5 Exploratory Efficacy Subgroup Analysis: Mean of Total Daily OFF Time by Visit by Baseline Daily Levodopa Dose |
| (ITT Population) |
| Table 14.2.5.1.6 Exploratory Efficacy Subgroup Analysis: Mean of Total Daily OFF Time by Visit by PD Diary Mean Daily OFF Time during Screening (ITT Population) |
| Table 14.2.5.1.7 Exploratory Efficacy Subgroup Analysis: Mean of Total Daily OFF Time by Visit by Screening Spirometry (ITT |
| Population) |
| Table 14.2.5.1.8 Exploratory Efficacy Subgroup Analysis: Mean of Total Daily OFF Time by Visit by Age Group (ITT Population) 44 |
| Table 14.2.5.1.9 Exploratory Efficacy Subgroup Analysis: Mean of Total Daily OFF Time by Visit by Gender (ITT Population) 44 |
| Table 14.2.5.2 Exploratory Efficacy Analysis: Mean of Total Daily ON Time without Dyskinesia by Visit (ITT Population) |
| Table 14.2.5.3 Exploratory Efficacy Analysis: Mean of Total Daily ON Time with non-Troublesome Dyskinesia by Visit (ITT Population) |
| Table 14.2.5.4 Exploratory Efficacy Analysis: Mean of Total Daily ON Time with Troublesome Dyskinesia by Visit (ITT Population) 45 |
| Table 14.2.6.1 Exploratory Efficacy Analysis: Subjects Global Impression of Change (PGI-C) by Visit Worst Case Imputation [a] (ITT |
| Population) |
| Table 14.2.7.1 Exploratory Efficacy Analysis: UPDRS Part 2 Score at TV4/OV4 (ITT Population) |
| Table 14.2.7.2 Exploratory Efficacy Analysis: UPDRS Part 2 Score at TV6/OV6 (ITT Population) |

Page x of y

| Table 14.2.8.1 Exploratory Efficacy Analysis: Schwab and England (S&E) Activities of Daily Living (ADL) Score at TV4/OV4 (ITT |
|---|
| Population) |
| Table 14.2.8.2 Exploratory Efficacy Analysis: Schwab and England (S&E) Activities of Daily Living (ADL) Score at TV6/OV6 (ITT |
| Population) |
| Table 14.2.9.1 Exploratory Efficacy Analysis: 39 Item Parkinson's disease Questionnaire (PDQ-39) Sub-scores and Summary Index Score |
| at TV4/OV4 (ITT Population) |
| Table 14.2.9.2 Exploratory Efficacy Analysis: 39 Item Parkinson's disease Questionnaire (PDQ-39) Sub-scores and Summary Index |
| Score at TV6/OV6 (ITT Population) |
| Table 14.3.1.1 Extent of Exposure: Overall for CVT-301 Group Only (Safety Population) |
| Table 14.3.1.2 In-Clinic Study Drug Administration (Safety Population) |
| Table 14.3.1.3 Distribution of Time of Study Drug Administration for CVT-301 Group Only (Safety Population) |
| Table 14.3.2.1 Treatment-Emergent Adverse Events -Overall Summary (Safety Population) |
| Table 14.3.2.2.2 Treatment-Emergent Adverse Events by Preferred Term (Safety Population) |
| Table 14.3.2.3 Drug-Related Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and Severity (Safety Population) |
| Table 14.3.2.4 Drug -Related Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and Relationship (Safety |
| Population) |
| Table 14.3.2.5 Drug-related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.2.6 Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.2.6 Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.2.8 Listing of Adverse Events Leading to Death |
| Table 14.3.2.0 Easting of Adverse Events Leading to Death |
| Table 14.3.2.10 Listing of Severe Treatment-Emergent Adverse Events |
| Table 14.3.2.10 Disting of Severe freatment-Emergent Adverse Events. Table 14.3.2.11 Treatment-Emergent Adverse Events Leading to Study Drug Interruption by System Organ Class and Preferred Term |
| (Safety Population) |
| Table 14.3.2.12 Listing of Adverse Events Leading to Study Drug Interruption |
| Table 14.3.2.13 Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term |
| (Safety Population) |
| Table 14.3.2.14 Listing of Adverse Events Leading to Study Drug Discontinuation |
| Table 14.3.2.15 Treatment-Emergent Adverse Events Leading to Dose Reduction by System Organ Class and Preferred Term (Safety |
| Population) |
| Table 14.3.2.16 Listing of Adverse Events Leading to Dose Reduction. |
| Table 14.3.2.17 Most Common Treatment-Emergent Adverse Events (Preferred Term Occurred in >10% of Over Patients) by System Organ |
| Class and Preferred Term (Safety Population) |
| Table 14.3.2.18 Listing of Most Common Treatment-Emergent Adverse Events |
| Table 14.3.2.19 Time to first Onset of Most Common Treatment-Emergent Adverse Events (Preferred Term Occurred in >10% of Over |
| Patients) (Safety Population) |
| Table 14.3.4.1 Clinical Laboratory Results: PCS and PCSC Criteria |
| Table 14.3.4.1.1.1 Summary of Clinical Laboratory Results: Hematology (Safety Population) |
| Table 14.3.4.1.1.2 Summary of Clinical Laboratory Results: Hematology Abnormal Values (Safety Population) |
| Table 14.3.4.1.1.3 Summary of Clinical Laboratory Results: Hematology Abnormal Values -Shift from Baseline (Safety Population) |
| Table 14.3.4.1.1.4 Summary of Clinical Laboratory Results: Hematology PCS Values -Shift from Baseline (Safety Population) 68 |
| Table 14.3.4.1.1.5 Summary of Clinical Laboratory Results: Hematology PCSC Values -Shift from Baseline (Safety Population) |
| Table 14.3.4.1.1.6 Clinical Laboratory Results - Hematology PCS and PCSC Values (Safety Population) |
| Table 14.3.4.1.2.1 Summary of Clinical Laboratory Results: Chemistry (Safety Population) |
| Table 14.3.4.1.2.2 Summary of Clinical Laboratory Results: Chemistry Abnormal Values (Safety Population) |
| Table 14.3.4.1.2.3 Summary of Clinical Laboratory Results: Chemistry Abnormal Values -Shift from Baseline (Safety Population)71 |
| Table 14.3.4.1.2.4 Summary of Clinical Laboratory Results: Chemistry PCS Values -Shift from Baseline (Safety Population) |
| Table 14.3.4.1.2.5 Summary of Clinical Laboratory Results: Chemistry PCSC Values -Shift from Baseline (Safety Population) |
| Table 14.3.4.1.2.6 Clinical Laboratory Results - Chemistry PCS and PCSC Values (Safety Population) |

| Table 14.3.4.2 Vital Signs: PCS and PCSC Criteria |
|---|
| Table 14.3.4.2.1 Summary of Vital Signs: Actual Values and Change from Baseline across Visits (Safety Population) |
| Table 14.3.4.2.2 Summary of Vital Signs: Actual Values and Change from Pre-dose at dose at TV1 (Safety Population) |
| Table 14.3.4.2.3 Summary of Standard Vital Signs: PCS and PCSC Values by Visit (Safety Population) |
| Table 14.3.4.2.4 Summary of Standard Vital Signs: PCS and PCSC Values by Scheduled Timepoint at TV1 (Safety Population) |
| Table 14.3.4.2.5 Standard Vital Signs: PCS and PCSC Values |
| Table 14.3.4.2.6 Summary of Vital Signs: Orthostatic Hypotension by Visit (Safety Population) |
| Table 14.3.4.2.7 Summary of Vital Signs: Orthostatic Hypotension by Scheduled Timepoint at TV1 (Safety Population) |
| Table 14.3.4.2.8 Orthostatic Vital Signs |
| Table 14.3.4.3 12-Lead ECG:PCS and PCSC Criteria |
| Table 14.3.4.3.1 Summary of 12-Lead ECG: Actual Values and Change across Visits (Safety Population) |
| Table 14.3.4.3.2 Summary of 12-Lead ECG: PCS and PCSC Values (Safety Population) |
| Table 14.3.4.3.3 12-Lead Electrocardiogram (ECG): PCS and PCSC Values |
| Table 14.3.4.4 Physical Examination (Safety Population) |
| Table 14.3.4.5.1.1 Summary of Spirometry (Neurology Office): Actual Values and Change from Baseline for FEV1 and FVC by Visit |
| (Safety Population) |
| Table 14.3.4.5.1.2 Summary of Spirometry (Neurology Office): Actual Values and Change from Baseline for FEV1 and FVC by Visit |
| Using Subset of Assessments Meeting the ATS Quality Criteria (Safety Population) |
| Table 14.3.4.5.1.3 Summary of Spirometry (Neurology Office): Actual Values and Change from Baseline for FEV1 and FVC by Visit |
| Excluding Patients with Co-efficient of Variation (CV) of FEV1 >7.5% (Safety Population) |
| Table 14.3.4.5.1.4 MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for FEV1 by Visit (Safety Population) 89 |
| Table 14.3.4.5.1.5 MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for FEV1 by Visit Using Subset of |
| Assessments Meeting the ATS Quality Criteria (Safety Population) |
| Table 14.3.4.5.1.6 MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for FEV1 by Visit Excluding Patients |
| with Co-efficient of Variation (CV) of FEV1 >7.5% (Safety Population) |
| Table 14.3.4.5.1.7 Sensitivity Analysis Using MMRM: Change from Baseline for FEV1 by Visit MI analysis with Missing At Random |
| Assumption (Safety Population)91 |
| Table 14.3.4.5.1.8 MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for Percentage Predicted FEV1 by Visit |
| (Safety Population)92 |
| Table 14.3.4.5.1.9 MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for Percentage Predicted FEV1 by Visit |
| Using Subset of Assessments Meeting the ATS Quality Criteria (Safety Population) |
| Table 14.3.4.5.1.10 MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for Percentage Predicted FEV1 by |
| Visit Excluding Patients with Co-efficient of Variation (CV) of FEV1 >7.5% (Safety Population) |
| Table 14.3.4.5.1.11 Sensitivity Analysis Using MMRM: Change from Baseline for Percentage Predicted FEV1 by Visit MI analysis with |
| Missing At Random Assumption (Safety Population) |
| Table 14.3.4.5.1.12 MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for FVC by Visit (Safety Population) 93 |
| Table 14.3.4.5.1.13 MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for FVC by Visit Using Subset of |
| Assessments Meeting the ATS Quality Criteria (Safety Population) |
| Table 14.3.4.5.1.14 MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for FVC by Visit Excluding Patients |
| with Co-efficient of Variation (CV) of FEV1 >7.5% (Safety Population) |
| Table 14.3.4.5.1.15 Sensitivity Analysis Using MMRM: Change from Baseline for FVC by Visit MI analysis with Missing At Random |
| Assumption (Safety Population)94 |
| Table 14.3.4.5.1.16 MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for Percentage Predicted FVC by Visit |
| (Safety Population)94 |
| Table 14.3.4.5.1.17 MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for Percentage Predicted FVC by Visit |
| Using Subset of Assessments Meeting the ATS Quality Criteria (Safety Population) |
| Table 14.3.4.5.1.18 MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for Percentage Predicted FVC by Visit |
| Excluding Patients with Co-efficient of Variation (CV) of FEV1 >7.5% (Safety Population) |
| Table 14.3.4.5.1.19 Sensitivity Analysis Using MMRM: Change from Baseline for Percentage Predicted FVC by Visit MI analysis with |
| Missing At Random Assumption (Safety Population) |

| Table 14.3.4.5.2.1 Summary of Spirometry : ( Neurology Office): Actual Values and Change from Baseline for FEV1/FVC by Visit |
|---|
| (Safety Population) |
| Table 14.3.4.5.2.3 Summary of Spirometry : ( Neurology Office): Actual Values and Change from Baseline for FEV1/FVC by Visit Excluding Patients with Co-efficient of Variation (CV) of FEV1 >7.5% (Safety Population) |
| Table 14.3.4.5.2.4 MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for FEV1/FVC by Visit (Safety Population) |
| Table 14.3.4.5.2.5 MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for FEV1/FVC by Visit Using Subset of Assessments Meeting the ATS Quality Criteria (Safety Population) |
| Table 14.3.4.5.2.6 MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for FEV1/FVC by Visit Excluding Patients with Co-efficient of Variation (CV) of FEV1 >7.5% (Safety Population) |
| Table 14.3.4.5.2.7 Sensitivity Analysis Using MMRM: Change from Baseline for FEV1/FVC by Visit MI analysis with Missing At Random Assumption (Safety Population) |
| Table 14.3.4.5.3.1 Summary of Spirometry (Neurology Office): Summary of FEV1/FVC < 60% and <70% by Visit (Safety Population) |
| Assessments Meeting the ATS Quality Criteria (Safety Population) |
| Table 14.3.4.5.4 Spirometry (Neurology Office): 70% or Smaller FEV1/FVC Values |
| Table 14.3.4.5.6 Summary of Spirometry (Pulmonary Function Facility): Actual Values and Change from Baseline for Calculated DLco Parameters by Visit (Safety Population) |
| Table 14.3.4.5.7 Summary of Spirometry (Pulmonary Function Facility): Actual Values and Change from Baseline for FEV1 and FVC by Visit (Safety Population) |
| Table 14.3.4.5.8 Summary of Spirometry (Pulmonary Function Facility): Actual Values and Change from Baseline for FEV1/FVC by Visit (Safety Population) |
| Table 14.3.4.5.9 Summary of Spirometry (Pulmonary Function Facility): Summary of FEV1/FVC < 60% and <70% by Visit (Safety Population) |
| Table 14.3.4.5.10 Spirometry (Pulmonary Function Facility):70% or Smaller FEV1/FVC Values by Visit |
| Population) |
| Table 14.3.4.7 Summary of Epworth Sleepiness Scale Total Score: Actual Values and Change from Baseline by Visit (Safety Population) 111 Table 14.3.4.8 Summary of Questionnaire for Impulsive-Compulsive Disorders in Parkinson's (QUIP) by Visit (Safety Population) 112 |
| Table 14.3.4.9.1 MMRM Analysis of UPDRS Part 4: Change from Baseline in the UPDRS Part 4 Score by Visit (Safety Population) |
| (Safety Population) |
| (Safety Population) |
| Population) |
Civitas Therapeutics, Inc.

Page x of y

Protocol No. CVT-301-005


Table 14.1.1.1

Number of Subjects Enrolled and Study Termination
(All Available Population)

| | CVT-301 | | | | |
|---|---|---|---|---|---|
| | O.C. | 002/003 | Naive | Total | Overall |
| | n (%) | n (%) | n (%) | n (%) | n (%) |
| Screened | | | | | XX |
| Failed Screening [a] | | | | | xx (xx.x) |
| Randomized [a] | xx | xx | XX | XX | xx (xx.x) |
| Safety Population [b] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ITT Population [b] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Completed Study [b] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Withdrawn from Study [b] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reason for Withdrawal from Study [c] | | | | | |
| Adverse Event | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lack of Efficacy | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subject Withdrew Consent | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Protocol Violation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lost to Follow-up | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients.

<sup>[</sup>a] Percentages are based on the number of screened subjects.

<sup>[</sup>b] Percentages are based on the number of randomized subjects.

<sup>[</sup>c] Percentages are based on the number of randomized and dosed subjects withdrawn from study.

<sup>[</sup>d] Percentages are based on the number of subjects in safety population.

Cross-reference: Listing 16.2.1, 16.2.3.3

Table 14.1.1.2 Number of Subjects in Each Population by Study Center All Subjects

| | | O.C. | | | 002/003 | | | Naive | |
|---|---|---|---|---|---|---|---|---|---|
| | Randomized | Safety | ITT | Randomized | Safety | ITT | Randomized | Safety | ITT |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Overall | xxx | xxx | xxx | XXX | xxx | xxx | XXX | xxx | xxx |
| Site 1 | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) |
| Site 2 | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) |
| Site 3 | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) |
| | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) |

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. PP=Per-protocol; Percentages are based on the number of subjects in each population for each treatment group.

Cross-reference: Listing 16.2.1, 16.2.3.3

Table 14.1.1.2 Number of Subjects in Each Population by Study Center All Subjects

| | CVT-301 Total | | | Overall | | |
|---|---|---|---|---|---|---|
| | Randomized | Safety | ITT | Randomized | Safety | ITT |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Overall | xxx | xxx | xxx | xxx | xxx | xxx |
| Site 1 | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) |
| ite 2 | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) |
| Site 3 | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) |
| | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) |

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. PP=Per-protocol; Percentages are based on the number of subjects in each population for each treatment group.

Cross-reference: Listing 16.2.1, 16.2.3.3

Table 14.1.2.1 Summary of Protocol Deviation Randomized Set

| | | | CVT-301 | | |
|---|---|---|---|---|---|
| | O. C.<br>N=xxx | 002/003 | Naive | Total | Overall |
| | | N=xxx | N=xxx | N=xxx | N=xxx |
| | n (%) | n (%) | n (%) | n (%) | n (%) |
| Any Protocol Deviation | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Any Minor Protocol Deviation | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Any Major Protocol Deviation | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Without Impact on Pulmonary Assessments | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| With Pulmonary Impact on Assessments | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Percentages are based on the number of subjects in each treatment group.

Cross-reference: Appendix 16.2.2.1

Program Name: Lxxxxx.sas Table Generation: ddmonyyyy hh:mm

Table 14.1.3.1.1 Demographic and Baseline Characteristics (Safety Population)

| | | | CVT-301 | | | _ |
|---|---|---|---|---|---|---|
| | | O. C. | 002/003 | Naïve | Total | Overall |
| Characteristic | Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Age (years) | n | XX | xx | XX | XX | XX |
| 1190 (10010) | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Age (years) | | | | | | |
| <65 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >=65 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gender | | | | | | |
| Male | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Female | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ethnicity | | | | | | |
| Hispanic or Latino | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Hispanic or Latino | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Race | | | | | | |
| American Indian or Alaska Native | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Asian | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Black or African American | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Native Hawaiian or other | | | | | | |
| Pacific Islander | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| White | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Height (cm) | n | XX | XX | xx | xx | xx |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Weight (kg) BMI ((kg/m^2) [a] | • • • • | | | | | |

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients.

<sup>[</sup>a] BMI was calculated as weight (kg) / [height (m)]^2.

Cross-reference: Listing 16.2.4.1, 16.2.4.4, 16.2.4.7, 16.2.4.10

Table 14.1.3.1.1 Demographic and Baseline Characteristics (Safety Population)

| - | | | | CVT-301 | | |
|---|---|---|---|---|---|---|
| Characteristic | Statistic | O. C.<br>(N=xx) | 002/003<br>(N=xx) | Naïve<br>(N=xx) | Total<br>(N=xx) | Overall (N=xx) |
| Country | | | | | | |
| United States | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Canada | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ••• | ( - / | , | , , | , , | , | , , |
| Smoking History | | | | | | |
| Never | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Former | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Current | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of Years Smoked | n | XX | xx | xx | xx | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Number of Cigarettes/Day | n | XX | xx | xx | xx | xx |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| MMSE Total Score | n | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| Screening Spirometry | ••• | | | | | |
| FEV1 <60% or FEV1/FVC ratio <70% | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| FEV1 >=60% and FEV1/FVC ratio >=70% | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1211 / 000 and 1211,110 14010 / 700 | 11 (0) | 1111 (111111) | (, | (, | 1111 (1111 • 111) | (1111) |
| Baseline PD Severity | | | | | | |
| Hoehn & Yahr scale < 2.5 points | n (응) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Hoehn & Yahr scale>= 2.5 points | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Randomization Strata | | | | | | |
| Hoehn & Yahr scale < 2.5 points AND FEV1 <60% or FEV1/FVC ratio <70% | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Hoehn & Yahr scale < 2.5 points AND FEV1 >=60% and FEV1/FVC ratio >=70% | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Hoehn & Yahr scale>= 2.5 points AND FEV1 <60% or FEV1/FVC ratio <70% | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Hoehn & Yahr scale>= 2.5 points AND FEV1 >=60% and FEV1/FVC ratio >=70% | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients.

<sup>[</sup>a] BMI was calculated as weight (kg) / [height (m)]^2.

Cross-reference: Listing 16.2.4.1, 16.2.4.4, 16.2.4.7, 16.2.4.10


Table 14.1.3.1.2

Demographic and Baseline Characteristics

(ITT Population)

Table 14.1.3.1.3

Demographic and Baseline Characteristics

by Baseline PD Severity

(ITT Population)

will have similar format as Table 14.1.2.1. Summarize for "Hoehn & Yahr scale < 2.5 points" and "Hoehn & Yahr scale >= 2.5 points" respectively.

Table 14.1.3.1.4

Demographic and Baseline Characteristics

by Baseline Dyskinesia

(ITT Population)

will have similar format as Table 14.1.2.1. Summarize for "Dyskinetic before TV1" and "Non-dyskinetic before TV1" respectively.

Table 14.1.3.1.5

 ${\tt Demographic\ and\ Baseline\ Characteristics}$ 

by Baseline Daily Levodopa Dose

(ITT Population)

Table 14.1.3.1.6

Demographic and Baseline Characteristics

by PD Diary Mean Daily OFF Time during Screening

(ITT Population)

will have similar format as Table 14.1.2.1. Summarize for "PD Diary Mean Daily OFF Time during Screening < 4.5 Hours" and "PD Diary Mean Daily OFF Time during Screening >=4.5 Hours" respectively.

Table 14.1.3.1.7

Demographic and Baseline Characteristics

by Screening Spirometry

(ITT Population)

will have similar format as Table 14.1.2.1. Summarize for "FEV1 <60% or FEV1/FVC ratio <70%" and "FEV1  $\geq$ 60% and FEV1/FVC ratio  $\geq$ 70%" respectively.

Table 14.1.3.1.8

Demographic and Baseline Characteristics

by Age Group

(ITT Population)

will have similar format as Table 14.1.3.1.1 Summarize for "Non-elderly (<65 years)" and "Elderly (≥65 years) patients" respectively.

Table 14.1.3.1.9

Demographic and Baseline Characteristics
by Gender
(ITT Population)

will have similar format as Table 14.1.3.1.1 Summarize for "Female" and "Male" respectively.

Table 14.1.3.2.1 Parkinson's Disease History (Safety Population)

| | | | | CVT-301 | | |
|---|---|---|---|---|---|---|
| | Statistic | O. C.<br>(N=xx) | 002/003<br>(N=xx) | Naïve<br>(N=xx) | Total<br>(N=xx) | Overall (N=xx) |
| | 504015010 | (21 2227) | (11 1111) | (11 1111) | (11 1111) | (11 1111) |
| Time Since Diagnosis of Parkinson's Disease (months) | n | XX | XX | XX | xx | XX |
| | Mean | xx.x | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | XX, XX | xx, xx | XX, XX |
| Duration of Levodopa Treatment (months) | | | | | | |
| Duration since Onset of Fluctuation (Wearing Off) Episodes (months) | ••• | | | | | |
| Baseline Average Daily Levodopa Dose (mg) | n | XX | XX | xx | xx | xx |
| | mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| Baseline Average # of Daily Levodopa Doses | n | XX | XX | XX | XX | XX |
| | mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| Screening UPDRS III Total Score (ON State) | n | XX | XX | XX | XX | xx |
| | mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| Screening UPDRS III Total Score (OFF State) | n | XX | XX | XX | XX | XX |
| · · · · · · | mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| Difference from OFF to ON State in Screening | n | | | | | |
| UPDRS III Total Score | | XX | XX | XX | XX | XX |
| | mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| Percent Difference from OFF to ON in Screening | n | | | | | |
| UPDRS III Total Score (%)[a] | | XX | XX | XX | XX | XX |
| | mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| Average Number of Daily OFF Episodes Experienced | n | XX | XX | XX | XX | XX |
| | mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| Patients who Changed the Timing of Their Usual<br>Levodopa Medication | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Patients who Took an Extra Dose of Levodopa or other PD Medication | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients.

<sup>[</sup>a] % was calculated as OFF-ON/OFF \* 100%'.

<sup>[</sup>b] The patients who have recorded at least 1 hour of dyskinesia (either ON with non-troublesome dyskinesia or ON with troublesome Cross-reference: Listing 16.2.4.3, 16.2.4.8, 16.2.4.9, 16.2.5.3, 16.2.6.1.1, 16.2.8.2.4.1

Table 14.1.3.2.1 Parkinson's Disease History (Safety Population)

| | | | | CVT-301 | | |
|---|---|---|---|---|---|---|
| | | O. C. | 002/003 | Naïve | Total | Overall |
| | Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Screening PD Diary | | | | | | |
| Mean Daily OFF Time (hours) | n | XX | XX | XX | XX | xx |
| nean barry off fime (notio) | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | 222.2 | 7171 • 21 | 2121 • 21 | 7171 • 71 | 2121 • 21 |
| Mean Daily OFF Time during Screening< 4.5 Hours | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Mean Daily OFF Time during Screening>= 4.5 Hours | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| noun burly off fime during beforening, 1.0 hours | 11 (0) | 7171 (2121 • 21) | 7171 (2121 • 21) | 111 (111·11) | 1121 (2121 • 21) | 2121 (2121 • 21) |
| Mean Daily ON Time Without Dyskinesia (hours) | n | XX | XX | XX | XX | XX |
| | mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| Mean Daily ON Time With | | | | | | |
| Non-troublesome Dyskinesia (hours) | n | XX | XX | XX | XX | XX |
| | mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| Mean Daily ON Time With | | | | | | |
| Troublesome Dyskinesia (hours) | n | XX | XX | XX | XX | XX |
| | mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| Baseline Dyskinesia | | | | | | |
| Dyskinetic before TV1/OV1[b] | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Non-dyskinetic before TV1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Canada Carina Carina Carina Carina (ON) | | | | | | |
| Screening Spirometry data (ON) FEV1 | n | xx | xx | xx | xx | xx |
| LEVI | mean | | XX.X | | XX<br>XX.X | |
| | | XX.X | AA.A | XX.X | **** | XX.X |
| FVC | n | XX | xx | XX | XX | XX |
| r v C | mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| FEV1/FVC | n | XX | XX | XX | XX | XX |
| T T A T \ T A C | mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| Screening Spirometry data (OFF) | IIICa11 | ^^.^ | ^^.^ | ^^.^ | ^^.^ | ^^.^ |
| FEV1 | | | | | | |
| FVC | | | | | | |
| FEV1/FVC | | | | | | |

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients.

Cross-reference: Listing 16.2.4.3, 16.2.4.8, 16.2.4.9, 16.2.5.3, 16.2.6.1.1, 16.2.8.2.4.1

<sup>[</sup>a] % was calculated as OFF-ON/OFF \* 100%.

<sup>[</sup>b] The patients who have recorded at least 1 hour of dyskinesia (either ON with non-troublesome dyskinesia or ON with troublesome dyskinesia) on at least 2 days before TV1/OV1 will be classified as dyskinetic.

Table 14.1.3.2.2 Parkinson's Disease History (ITT Population)

will have similar format as Table 14.1.3.2.1.

Table 14.1.3.2.3 Parkinson's Disease History by Baseline PD Severity (ITT Population)

will have similar format as Table 14.1.3.2.1, but to summarize for "Hoehn & Yahr scale < 2.5 points" and "Hoehn & Yahr scale >= 2.5 points" respectively. No need to summarize "Baseline PD Severity".

> Table 14.1.3.2.4 Parkinson's Disease History by Baseline Dyskinesia (ITT Population)

will have similar format as Table 14.1.3.2.1, but to summarize for "Dyskinetic before Visit 3" and "Non-dyskinetic before Visit 3" respectively. No need to summarize "Baseline Dyskinesia".

> Table 14.1.3.2.5 Parkinson's Disease History by Baseline Daily Levodopa Dose (ITT Population)

will have similar format as Table 14.1.3.2.1. Summarize for "Baseline Daily Levodopa Dose< = Median of Baseline Daily Levodopa Dose" and "Baseline Daily Levodopa Dose >= Median of Baseline Daily Levodopa Dose " respectively.

> Table 14.1.3.2.6 Parkinson's Disease History by PD Diary Mean Daily OFF Time during Screening (ITT Population)

will have similar format as Table 14.1.3.2.11, but to summarize for "PD Diary Mean Daily OFF Time during Screening <4.5 Hours" and "PD Diary Mean Daily OFF Time during Screening >=4.5 Hours".


Table 14.1.3.2.7
Parkinson's Disease History
by Screening Spirometry
(ITT Population)

will have similar format as Table 14.1.3.2.1. Summarize for "FEV1 <60% or FEV1/FVC ratio <70%" and "FEV1  $\geq$ 60% and FEV1/FVC ratio  $\geq$ 70%" respectively.

Table 14.1.3.2.8
Parkinson's Disease History
by Age Group
(ITT Population)

will have similar format as Table 14.1.3.2.1. Summarize for "Non-elderly (<65 years)" and "Elderly (≥65 years) patients" respectively.

Table 14.1.3.2.9
Parkinson's Disease History
by Gender
(ITT Population)

will have similar format as Table 14.1.3.2.1. Summarize for "Female" and "Male" respectively.

Table 14.1.3.2.10

Modified Hoehn and Yahr Staging in "ON" State (Safety Population)

| | CVT-301 | | | | |
|---|---|---|---|---|---|
| | O. C.<br>(N=xx)<br>n (%) | 002/003<br>(N=xx)<br>n (%) | Naive<br>(N=xx)<br>n (%) | Total<br>(N=xx)<br>n (%) | Overall<br>(N=xx)<br>n (%) |
| odified Hoehn and Yahr | | | | | |
| Stage 0 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Stage 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Stage 1.5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| Stage 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Stage 2.5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Stage 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Stage 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Stage 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients.

Cross-reference: Listing 16.2.4.6

Table 14.1.3.2.11
Modified Hoehn and Yahr Staging in "ON" State
(ITT Population)

will have similar format as Table 14.1.3.2.11.

# Table 14.1.3.2.12 Distribution of Average Daily OFF Time at Baseline (Safety Population)

| | _ | | _ | | |
|---|---|---|---|---|---|
| Time Interval/OFF Hours (%) | O. C.<br>(N=xx) | 002/003<br>(N=xx) | Naive<br>(N=xx) | Total<br>(N=xx) | Overall<br>(N=xx) |
| Average Total Daily OFF Time (Hours) | xx.x | xx.x | xx.x | xx.x | XX.X |
| Average Daily OFF Hours (%) | | | | | |
| 00:00 -< 00:30 | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| 00:30 -< 01:00 | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| 01:00 -< 01:30 | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| 01:30 -< 02:00 | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |

Continue with 30 mins interval until 23:30 -< 24:00

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients.

Total daily OFF time is calculated as the average of total OFF time collected three days prior to TV1/OVland is normalized to 16 awake hours per day. Average daily OFF Hours at each interval will be calculated similarly. The percentage is based on Total Daily OFF Time. Cross-reference: Listing 16.2.6.2.2

# Table 14.1.3.2.13 Distribution of Cumulative Average Daily OFF Time at Baseline (Safety Population)

| | | | _ | | |
|---|---|---|---|---|---|
| Time Interval/OFF Hours (%) | O. C.<br>(N=xx) | 002/003<br>(N=xx) | Naive<br>(N=xx) | Total<br>(N=xx) | Overall<br>(N=xx) |
| Average Total Daily OFF Time (Hours) | xx.x | XX.X | XX.X | XX.X | XX.X |
| Cumulative Average Daily OFF Hours (%) | | | | | |
| 00:00 -< 00:30 | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| 00:00 -< 01:00 | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| 00:00 -< 01:30 | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| 00:00 -< 02:00 | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |

Continue with 30 mins interval until 00:00 -< 24:00

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients.

Total daily OFF time is calculated as the average of total OFF time collected three days prior to TV1/OVland is normalized to 16 awake hours per day. Cumulative Average daily OFF Hours are calculated similarly. The percentage is based on Total Daily OFF Time. Cross-reference: Listing 16.2.6.2.2

Table 14.1.3.3
Medical History
(Safety Population)

| | | | CVT-301 | | |
|---|---|---|---|---|---|
| | O. C. | 002/003 | Naïve | Total | Overall |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| System Organ Class | Subjects Events | Subjects Events | Subjects Events | Subjects Events | Subjects Events |
| Preferred Term [a] | n (%) n | n (%) n | n (%) n | n (%) n | n (%) n |
| Any Medical History | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| System Organ Class 1 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term 1 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term 2 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| ••• | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| System Organ Class 2 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term 1 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term 2 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| ••• | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients.

Cross-reference: Listing 16.2.4.2

Programming note: The table will be sorted by total descending frequency of SOC and then, within a SOC, by total descending frequency of PT.

<sup>[</sup>a] Medical history data were coded into system organ class and preferred term by using MedDRA version 17.0.

Table 14.1.4.1 Prior Medications (Safety Population)

| | | | CVT-301 | | |
|---|---|---|---|---|---|
| ATC Level 1 | O. C. | 002/003 | Naive | Total | Overall |
| ATC Level 2 | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Preferred Term | Subjects Meds | Subjects Meds | Subjects Meds | Subjects Medi | Subjects Meds |
| [a] | n (%) n | n (%) n | n (%) n | n (%) n | n (%) n |
| Any Medications | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| ATC Level 1 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| ATC Level 2 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| ATC Level 2 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| ••• | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| ATC Level 1 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| ATC Level 2 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| • • • | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| ATC Level 2 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |

Note: Meds = Medications; O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Data from "Prior and Concomitant Medications" CRF page were summarized in this table. The medications with a stop date before the first date of study drug dosing will be considered prior medications.

[a] Medications were coded into ATC and preferred term using the WHO Drug Dictionary,Q1March2014.

Cross-reference: Listing 16.2.4.11.1

Programming note: The table will be sorted by total descending frequency of ATC1 and ATC2 and then, within a ATC2, by total descending frequency of PT.

Table 14.1.4.2
Concomitant Medications
(Safety Population)

Will have same format as Table 14.1.4.1

Note: Meds = Medications; O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients.

Data from "Prior and Concomitant Medications" CRF page were summarized in this table. The medications with start date or stop date on or after the first date of study drug dosing will be considered concomitant medications.

[a] Medications were coded into ATC and preferred term using the WHO Drug Dictionary, Q1March2014.

Cross-reference: Listing 16.2.4.11.2

Table 14.1.4.3 Parkinson's disease Treatment Medications at Baseline (ITT Population)

| | | | CVT-301 | | |
|---|---|---|---|---|---|
| | o. c. | 002/003 | Naive | Total | Overall |
| ATC Level 4 | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Preferred Term | Subjects Meds | Subjects Meds | Subjects Meds | Subjects Meds | Subjects Meds |
| [a] | n (%) n | n (%) n | n (%) n | n (%) n | n (%) n |
| Any Medications | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| ATC Level 4 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| ATC Level 4 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| ••• | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| ATC Level 4 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| ATC Level 4 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |

Programming note: The table will be sorted by total descending frequency of ATC and then, within a ATC, by total descending frequency of PT.

Note: Meds = Medications; O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients.

<sup>[</sup>a] Medications were coded into ATC and preferred term using the WHO Drug Dictionary, Q1March2014. The medications which start with ATC code N04 are considered as baseline PD treatment medications. Cross-reference: Listing 16.2.4.11.2

Civitas Therapeutics, Inc.

Page x of y


Table 14.2.1.1

Exploratory Efficacy Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 10 Minutes Post-dose by Visit (ITT Population)

| | | CVT-301 | |
|--------|-------------------------------|--------------|---------|
| /isit | Statistic | (N=xx) | p-value |
| verall | Overall p-value | | |
| | Baseline Hoehn and Yahr stage | | 0.xxx |
| | Screening Spirometry | | 0.xxx |
| | Visit | | 0.xxx |
| | Baseline UPDRS Part 3 Score | | 0.xxx |
| V2 | n | xx | |
| | LS Mean | XX.X | |
| | SE (LS Mean) | XX.XX | |
| | 95% CI (LS Mean) | (xx.x, xx.x) | |
| V3 | | | |
| V4 | | | |
| V5 | | | |
| V6 | | | |

Note: TV = Treatment Visit;

MMRM model uses the change from pre-dose in UPDRS Part 3 total scores at 10 minutes at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes visit (TV2, TV3, TV4, TV5 or TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus  $\geq$ 2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1  $\geq$ 60% and FEV1/FVC ratio  $\geq$ 70%)) as fixed factors; the baseline UPDRS part 3 score will be included as a covariate, assuming an unstructured covariance matrix.

Cross-reference: Listing 16.2.6.1.2

Civitas Therapeutics, Inc. Page x of y Protocol No. CVT-301-005


Table 14.2.1.2

Exploratory Efficacy Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 20 Minutes Post-dose by Visit (ITT Population)

Note: TV = Treatment Visit;

MMRM model uses the change from pre-dose in UPDRS Part 3 total scores at 20 minutes at each post-baseline visit (TV2, TV3,TV4, TV5 or TV6) as the dependent variable, and includes visit ((TV2, TV3,TV4, TV5 or TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus ≥2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1 ≥60% and FEV1/FVC ratio ≥70%)) as fixed factors; the baseline UPDRS part 3 score will be included as a covariate, assuming an unstructured covariance matrix.

Cross-reference: Listing 16.2.6.1.2

Table 14.2.1.3.1

Exploratory Efficacy Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 30 Minutes Post-dose by Visit (ITT Population)

Note: TV = Treatment Visit;

MMRM model uses the change from pre-dose in UPDRS Part 3 total scores at 30 minutes at each post-baseline visit (TV2, TV3,TV4, TV5 or TV6) as the dependent variable, and includes visit (TV2, TV3,TV4, TV5 or TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus ≥2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1 ≥60% and FEV1/FVC ratio ≥70%)) as fixed factors; the baseline UPDRS part 3 score will be included as a covariate, assuming an unstructured covariance matrix.

Cross-reference: Listing 16.2.6.1.2

will have similar format as Table 14.2.1.1.1.

Civitas Therapeutics, Inc.

Page x of y


### Table 14.2.1.3.2

Sensitivity Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 30 Minutes Post-dose by Visit
MI analysis with Missing At Random Assumption
(ITT Population)

| <pre>Visit/Statistic((Number of Datasets = 100)</pre> | CVT-301<br>(N=xx) |
|-------------------------------------------------------|-------------------|
| TV2 | |
| MI Mean (SE) | xx.x(xx.xx) |
| MI Median | XX.X |
| MI Minimum, MI Maximum | XX, XX |
| TV3 | |
| TV4 | |
| TV5 | |
| TV6 | |
| TV3 | |

Note: TV = Treatment Visit;

The non-monotone missing values will be imputed using the Markov Chain Monte Carlo (MCMC) methodology which assumes a multivariate normal distribution over all variables included in the imputation model. The monotone missing values are imputed using pattern mixture model assuming missing at random. MMRM model uses the change from pre-dose in UPDRS Part 3 total scores at 30 minutes at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus  $\ge 2.5$ ) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1  $\ge 60$ % and FEV1/FVC ratio  $\ge 70$ %)) as fixed factors; the Baseline UPDRS part 3 score will be included as a covariate, assuming an unstructured covariance matrix. The MIANALYZE procedure in SAS will be applied to combine the results from these datasets to derive an overall estimate at each visi

Cross-reference: Listing 16.2.6.1.2

Table 14.2.1.3.3 Subgroup Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 30 Minutes Post-dose by Visit by Baseline PD Severity (ITT Population)

# Hoehn & Yahr scale < 2.5 points

| Visit | Statistic | CVT-301<br>(N=xx) | p-value |
|---------|-----------------------------|-------------------|---------|
| Overall | Overall p-value | | |
| 0.01011 | Screening Spirometry | | 0.xxx |
| | Visit | | 0.xxx |
| | Baseline UPDRS Part 3 Score | | 0.xxx |
| TV2 | n | xx | |
| | LS Mean | XX.X | |
| | SE (LS Mean) | XX.XX | |
| | 95% CI (LS Mean) | (xx.x, xx.x) | |
| TV3 | | | |
| TV4 | | | |
| TV5 | | | |
| TV6 | | | |

Note: TV = Treatment Visit;

MMRM model uses the change from pre-dose in UPDRS Part 3 total scores at 30 minutes at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes visit (TV2, TV3, TV4, TV5, TV6), the stratification variable (screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1 ≥60% and FEV1/FVC ratio ≥70%)) as fixed factors; the baseline UPDRS part 3 score will be included as a covariate, assuming an unstructured covariance matrix. Cross-reference: Listing 16.2.6.1.2

Programming Note: Do separate analysis for "Hoehn & Yahr scale < 2.5 points" and "Hoehn & Yahr scale >= 2.5 points", and do not include baseline PD severity in MMRM model.

Table 14.2.1.3.4 Exploratory Efficacy Subgroup Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 30 Minutes Post-dose by Visit by Baseline

> Dyskinesia (ITT Population)

Dyskinetic before TV1

| | | CVT-301 | |
|---------|-------------------------------|--------------|---------|
| Visit | Statistic | (N=xx) | p-value |
| Overall | Overall p-value | | |
| | Baseline Hoehn and Yahr stage | | 0.xxx |
| | Screening Spirometry | | 0.xxx |
| | Visit | | 0.xxx |
| | Baseline UPDRS Part 3 Score | | 0.xxx |
| TV2 | n | xx | |
| | LS Mean | XX.X | |
| | SE (LS Mean) | XX.XX | |
| | 95% CI (LS Mean) | (xx.x, xx.x) | |
| TV3 | | | |
| TV4 | | | |
| TV5 | | | |
| TV6 | | | |

Note: TV = Treatment Visit;

MMRM model uses the change from pre-dose in UPDRS Part 3 total scores at 30 minutes at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus ≥2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1 ≥60% and FEV1/FVC ratio ≥70%)) and the interaction between the treatment group and visit as fixed factors; the Baseline UPDRS part 3 score will be included as a covariate, assuming an unstructured covariance matrix. Cross-reference: Listing 16.2.6.1.2

Programming Note: Do separate analysis for Dyskinetic before TV1/OV1versus Non-Dyskinetic before TV1


# Table 14.2.1.3.5

Exploratory Efficacy Subgroup Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 30 Minutes Post-dose by Visit by Baseline Daily Levodopa Dose (ITT Population)

### Baseline Daily Levodopa Dose <= Median of Baseline Daily Levodopa Dose

| | | CVT-301 | |
|---------|-------------------------------|--------------|---------|
| Visit | Statistic | (N=xx) | p-value |
| Overall | Overall p-value | | |
| | Baseline Hoehn and Yahr stage | | 0.xxx |
| | Screening Spirometry | | 0.xxx |
| | Visit | | 0.xxx |
| | Baseline UPDRS Part 3 Score | | 0.xxx |
| TV2 | n | xx | |
| | LS Mean | XX.X | |
| | SE (LS Mean) | XX.XX | |
| | 95% CI (LS Mean) | (xx.x, xx.x) | |
| TV3 | | | |
| TV4 | | | |
| TV5 | | | |
| TV6 | | | |

Note: TV = Treatment Visit;

MMRM model uses the change from pre-dose in UPDRS Part 3 total scores at 30 minutes at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus ≥2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1 ≥60% and FEV1/FVC ratio ≥70%)) and the interaction between the treatment group and visit as fixed factors; the Baseline UPDRS part 3 score will be included as a covariate, assuming an unstructured covariance matrix. Cross-reference: Listing 16.2.6.1.2

Programming Note: Do separate analysis for "Baseline Daily Levodopa Dose< = Median of Baseline Daily Levodopa Dose" and "Baseline Daily Levodopa Dose>=Median of Baseline Daily Levodopa Dose" respectively.

Table 14.2.1.3.6 Exploratory Efficacy Subgroup Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 30 Minutes Post-dose by Visit by PD Diary Mean Daily OFF Time during Screening (ITT Population)

PD Diary Mean Daily OFF Time during Screening <4.5 Hours

| Statistic | (27 | |
|---|---|---|
| | (N=xx) | p-value |
| Overall p-value | | |
| | | 0.xxx |
| | | 0.xxx |
| Visit | | 0.xxx |
| Baseline UPDRS Part 3 Score | | 0.xxx |
| n | xx | |
| LS Mean | XX.X | |
| SE (LS Mean) | xx.xx | |
| 95% CI (LS Mean) | (xx.x, xx.x) | |
| | Baseline UPDRS Part 3 Score n LS Mean SE (LS Mean) | Baseline Hoehn and Yahr stage Screening Spirometry Visit Baseline UPDRS Part 3 Score n LS Mean xx SE (LS Mean) xx.xx |

Note: TV = Treatment Visit;

MMRM model uses the change from pre-dose in UPDRS Part 3 total scores at 30 minutes at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus ≥2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1 ≥60% and FEV1/FVC ratio ≥70%)) and the interaction between the treatment group and visit as fixed factors; the Baseline UPDRS part 3 score will be included as a covariate, assuming an unstructured covariance matrix. Cross-reference: Listing 16.2.6.1.2

Programming Note: Do separate analysis for "PD Diary Mean Daily OFF Time during Screening<4.5 Hours" and "PD Diary Mean Daily OFF Time during Screening>=4.5 Hours".


# Table 14.2.1.3.7

Exploratory Efficacy Subgroup Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 30 Minutes Post-dose by Visit by Screening Spirometry

(ITT Population)

# FEV1 <60% or FEV1/FVC ratio <70%

| | | CVT-301 | |
|---------------|-------------------------------|--------------|---------|
| <i>J</i> isit | Statistic | (N=xx) | p-value |
| Overall | Overall p-value | | |
| | Baseline Hoehn and Yahr stage | | 0.xxx |
| | Visit | | 0.xxx |
| | Baseline UPDRS Part 3 Score | | 0.xxx |
| rv2 | n | xx | |
| | LS Mean | XX.X | |
| | SE (LS Mean) | xx.xx | |
| | 95% CI (LS Mean) | (xx.x, xx.x) | |
| rv3 | | | |
| rv4 | | | |
| rv5 | | | |
| rv6 | | | |

Note: TV = Treatment Visit;

MMRM model uses the change from pre-dose in UPDRS Part 3 total scores at 30 minutes at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus  $\ge 2.5$ )) and the interaction between the treatment group and visit as fixed factors; the Baseline UPDRS part 3 score will be included as a covariate, assuming an unstructured covariance matrix. Cross-reference: Listing 16.2.6.1.2

Programming Note: Do separate analysis for FEV1 <60% or FEV1/FVC ratio <70% and FEV1 ≥60% and FEV1/FVC ratio ≥70%

Table 14.2.1.3.8

Exploratory Efficacy Subgroup Analysis: Mean Change from Pre-dose in the UPDRS Part 3 Score at 30 Minutes Post-dose by Visit by Age
Group
(ITT Population)

# Non-elderly (<65 years)

| | CVT-301 | |
|---|---|---|
| Statistic | (N=xx) | p-value |
| Overall p-value | | |
| | | 0.xxx |
| <del>-</del> | | 0.xxx |
| | | 0.xxx |
| Baseline UPDRS Part 3 Score | | 0.xxx |
| n | xx | |
| LS Mean | xx.x | |
| SE (LS Mean) | xx.xx | |
| 95% CI (LS Mean) | (xx.x, xx.x) | |
| | Overall p-value Baseline Hoehn and Yahr stage Screening Spirometry Visit Baseline UPDRS Part 3 Score n LS Mean SE (LS Mean) | Overall p-value Baseline Hoehn and Yahr stage Screening Spirometry Visit Baseline UPDRS Part 3 Score n LS Mean SE (LS Mean) (N=xx) xx xx xx |

Note: TV = Treatment Visit;

MMRM model uses the change from pre-dose in UPDRS Part 3 total scores at 30 minutes at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus >2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1 >60% and FEV1/FVC ratio >70%)) and the interaction between the treatment group and visit as fixed factors; the Baseline UPDRS part 3 score will be included as a covariate, assuming an unstructured covariance matrix. Cross-reference: Listing 16.2.6.1.2

Programming Note: Do separate analysis for 'Non-elderly (<65 years)' and 'Elderly (>=65 years)' respectively.


Table 14.2.1.3.9

Exploratory Efficacy Subgroup Analysis: Mean Change from Pre-dose in the UPDRS Part 3 Score at 30 Minutes Post-dose by Visit by Gender

(ITT Population)

| | | CVT-301 | |
|---------|-------------------------------|--------------|---------|
| Visit | Statistic | (N=xx) | p-value |
| Overall | Overall p-value | | |
| | Baseline Hoehn and Yahr stage | | 0.xxx |
| | Screening Spirometry | | 0.xxx |
| | Visit | | 0.xxx |
| | Baseline UPDRS Part 3 Score | | 0.xxx |
| rv2 | n | xx | |
| | LS Mean | XX.X | |
| | SE (LS Mean) | XX.XX | |
| | 95% CI (LS Mean) | (xx.x, xx.x) | |
| TV3 | | | |
| TV4 | | | |
| rv5 | | | |
| rv6 | | | |

Note: TV = Treatment Visit;

MMRM model uses the change from pre-dose in UPDRS Part 3 total scores at 30 minutes at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus  $\ge2.5$ ) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1  $\ge60\%$  and FEV1/FVC ratio  $\ge70\%$ )) and the interaction between the treatment group and visit as fixed factors; the Baseline UPDRS part 3 score will be included as a covariate, assuming an unstructured covariance matrix. Cross-reference: Listing 16.2.6.1.2

Programming Note: Do separate analysis for 'Male' and 'Female' respectively.

Table 14.2.1.4

Exploratory Efficacy Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 60 Minutes Post-dose by Visit (ITT Population)

Note: TV = Treatment Visit;

MMRM model uses the change from pre-dose in UPDRS Part 3 total scores at 60 minutes at each post-baseline visit (TV2, TV3, TV4, TV5 or TV6) as the dependent variable, and includes visit (TV2, TV3, TV4, TV5 or TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus >2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1 >60% and FEV1/FVC ratio >70%)) as fixed factors; the baseline UPDRS part 3 score will be included as a covariate, assuming an unstructured covariance matrix.

Cross-reference: Listing 16.2.6.1.2

Table 14.2.1.5

Exploratory Efficacy Analysis: Change from Pre-dose in the Average UPDRS Part 3 Score at 10 to 60 Minutes Post-dose by Visit (ITT Population)

Note: TV = Treatment Visit;

MMRM model uses the change from pre-dose to the average of the 4 post-dose UPDRS Part 3 total scores (10,20,30 and 60 minutes) at each post-baseline visit (TV2, TV3,TV4, TV5 or TV6) as the dependent variable, and includes visit (TV2, TV3,TV4, TV5 or TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus  $\geq$ 2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1  $\geq$ 60% and FEV1/FVC ratio  $\geq$ 70%)) as fixed factors; the baseline UPDRS part 3 score will be included as a covariate, assuming an unstructured covariance matrix.

Cross-reference: Listing 16.2.6.1.2

will have similar format as Table 14.2.1.1.1.

Table 14.2.2.1 Exploratory Efficacy Analysis: Change from Pre-dose in UPDRS Part 3 Score to 10, 20, 30, 60 minutes Post-dose by Visit (ITT Population)

| Timeponit | Visit | Statistic | CVT-301<br>(N=xx) | p-value |
|---|---|---|---|---|
| 0 mins Post-dose | Overall | Overall p-value | | |
| .o mino robe dobe | OVCIUII | Baseline Hoehn and Yahr stage | | 0.xxx |
| | | Screening Spirometry | | 0.xxx |
| | | Treatment | | 0.xxx |
| | | Visit | | 0.xxx |
| | | Baseline UPDRS Part 3 Score | | 0.xxx |
| | TV2 | n | xx | |
| | | LS Mean | XX.X | |
| | | SE (LS Mean) | XX.XX | |
| | | 95% CI (LS Mean) | (xx.x, xx.x) | |
| | TV3 | | | |
| | TV4 | ••• | | |
| | TV5 | | | |
| | TV6 | | | |
| 0 mins Post-dose | | | | |
| 30 mins Post-dose | | | | |
| 60 mins Post-dose | | | | |

Note: TV = Treatment Visit;

MMRM model uses the change from pre-dose in UPDRS Part 3 score to 10, 20, 30, or 60 minutes at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes visit (TV2, TV3, TV4, TV5, TV6) the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus ≥2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1 ≥60% and FEV1/FVC ratio ≥70%)) as fixed factors; baseline UPDRS part 3 score will be included as a covariate, assuming an unstructured covariance matrix. A separate MMRM model will be fitted for each of the time points.

Cross-reference: Listing 16.2.6.1.2

Table 14.2.2.2

Exploratory Efficacy Analysis: Change from Pre-Dose to 10, 20, 30, 60 minutes Post-dose in UPDRS Part 3 Score by Visit and Timepoint (ITT Population)

| Timepoint | Visit | Statistic | CVT-301<br>(N=xx) |
|-------------------|---------|--------------|-------------------|
| Pre-dose | TV2 | Actual value | |
| | | n | XX |
| | | Mean | xx.x |
| | | SD | XX.XX |
| | | SEM | xx.x |
| | | Median | XX.X |
| | | Min, Max | XX, XX |
| | TV3 | | |
| | TV4 | ••• | |
| 10 mins post-dose | <br>TV2 | Actual value | |
| | | n | XX |
| | | Mean | XX.X |
| | | SD | XX.XX |
| | | SEM | XX.X |
| | | Median | XX.X |
| | | Min, Max | XX, XX |
| | | n | XX |
| | | Mean | XX.X |
| | | SD | XX.XX |
| | | SEM | XX.X |
| | | Median | XX.X |
| | | Min, Max | XX, XX |
| | TV3 | ••• | |
| | TV4 | | |
| 20 mins Post-dose | | | |
| 30 mins Post-dose | | | |
| 60 mins Post-dose | | | |

Note: TV = Treatment Visit; Cross-reference: Listing 16.2.6.1.2

Table 14.2.2.3

Exploratory Efficacy Analysis: Change from Pre-Dose to 10, 20, 30, 60 minutes Post-dose in UPDRS Part 3 Score by Timepoint and Visit (ITT Population)

| Visit | Timepoint | Statistic | CVT-301<br>(N=xx) |
|---|---|---|---|
| TV2 | Pre-dose | Actual value | |
| | | n | XX |
| | | Mean | XX.X |
| | | SD | xx.xx |
| | | SEM | xx.x |
| | | Median | xx.x |
| | | Min, Max | xx, xx |
| | 10 mins Post-dose | Actual value | |
| | | n | XX |
| | | Mean | XX.X |
| | | SD | XX.XX |
| | | SEM | XX.X |
| | | Median | XX.X |
| | | Min, Max | XX, XX |
| | | Change from Pre-dose | |
| | | n | XX |
| | | Mean | XX.X |
| | | SD | XX.XX |
| | | SEM | XX.X |
| | | Median | XX.X |
| | | Min, Max | XX, XX |
| | 20 mins Post-dose | | |
| | 30 mins Post-dose | | |
| | 60 mins Post-dose | | |
| Continue with TV3, TV4, TV5, | , TV6 | | |

Note: TV = Treatment Visit;

Cross-reference: Listing 16.2.6.1.2

Civitas Therapeutics, Inc. Page x of y Protocol No. CVT-301-005


Table 14.2.3.1 Exploratory Efficacy Analysis: Subjects with a >= 3 Reduction from Pre-dose to Post-dose in the UPDRS Part 3 Score by Visit (ITT Population)

| | CVT-30<br>(N=xx) |
|---|---|
| risit/Time Point | n (%) |
| V2 | |
| Any Time Post-dose | |
| n* | XX |
| Cumulative number of subjects having achieved the response | xx (xx. |
| 10 mins Post-dose | |
| n* | XX |
| Number of subjects achieving the first response | xx (xx. |
| 20 mins Post-dose | xx (xx. |
| n* | XX |
| Number of subjects achieving the first response | xx (xx. |
| Cumulative number of subjects having achieved the response[a] | xx (xx. |
| 30 mins Post-dose | xx (xx. |
| n* | XX |
| Number of subjects achieving the first response | xx (xx. |
| Cumulative number of subjects having achieved the response | xx (xx. |
| 60 mins Post-dose | xx (xx. |
| n* | XX |
| Number of subjects achieving the first response | xx (xx. |
| Cumulative number of subjects having achieved the response | xx (xx. |
| V3 | |
| vs<br>V4 | |
| 75 | |
| V6 | |

Note: TV = Treatment Visit;; Percentages are based on n\*, the number of subjects with UPDRS Part 3 performed at any time post-dose and pre-dose.

[a] Cumulative numbers of subjects refer to the subjects who achieved the first reduction before or at the time point.

Cross-reference: Listing 16.2.6.1.2

Civitas Therapeutics, Inc.

Page x of y


Table below will use the table 14.2.3.1 template except that percentages are based on N

Table 14.2.3.2

Additional Exploratory Efficacy Analysis: Subjects with a >=3 Reduction from Pre-dose to Post-dose in the UPDRS Part 3 Score by Visit

With Percentages Based on N

(ITT Population)

Note: Percentages are based on the header count N. Cross-reference: Listing 16.2.6.1.2

Table 14.2.3.3

Exploratory Efficacy Analysis: Subjects with a >= 6 Reduction from Pre-dose to Post-dose in the UPDRS Part 3 Score by Visit (ITT Population)

Table 14.2.3.4

Exploratory Efficacy Analysis: Subjects with a >=6 Reduction from Pre-dose to Post-dose in the UPDRS Part 3 Score by Visit
With Percentages Based on N

(ITT Population)

Note: TV = Treatment Visit; Percentages are based on the header count N. Cross-reference: Listing 16.2.6.1.2

Table 14.2.3.5

Exploratory Efficacy Analysis: Subjects with a >=11 Reduction from Pre-dose to Post-dose in the UPDRS Part 3 Score by Visit (ITT Population)

Table 14.2.3.6

Exploratory Efficacy Analysis: Subjects with a >=11 Reduction from Pre-dose to Post-dose in the UPDRS Part 3 Score by Visit
With Percentages Based on N
(ITT Population)

Note: TV = Treatment Visit; Percentages are based on the header count N. Cross-reference: Listing 16.2.6.1.2

Table 14.2.4.1

Exploratory Efficacy Analysis: Subjects Achieving Resolution of an OFF to an ON State within 60 Minutes by Visit

Worst Case Imputation [a]

(ITT Population)

| Visit/ | | CVT-301<br>(N=xx) |
|--------------------------------|-----------|-------------------|
| Category | Statistic | |
| TV2 | | |
| Turned ON within 60 Minutes | | |
| Yes | n (%) | xx (xx.x) |
| No | n (%) | xx (xx.x) |
| Turned ON within 60 Minutes (C | Observed) | |
| Yes | n (%) | xx (xx.x) |
| No | n (%) | xx (xx.x) |
| Missing | n (%) | xx (xx.x) |
| rv3 | | |
| rv4 | | |
| rv5 | | |
| rv6 | | |

Note: TV = Treatment Visit;

[a] The patient who achieved resolution of an OFF to an ON state within 60 minutes after study drug is administered in the clinic and maintaining the ON at 60 minutes after study drug administration will be counted as Yes. The missing values will be counted as non-resolved.

Cross-reference: Listing 16.2.6.2.1
Table 14.2.5.1.1 Exploratory Efficacy Analysis: Mean of Total Daily OFF Time by Visit (ITT Population)

| Visit | Statistic | O.C.<br>(N=xx) | CVT-301<br>(N=xx) | p-value |
|---|---|---|---|---|
| VISIC | Statistic | (IV-XX) | (N-XX) | p-varue |
| Overall | Overall p-value | | | |
| | Baseline Hoehn and Yahr stage | | | 0.xxx |
| | Screening Spirometry | | | 0.xxx |
| | Treatment | | | 0.xxx |
| | Visit | | | 0.xxx |
| | Treatment-by-Visit Interaction | | | 0.xxx |
| | Baseline Daily OFF time | | | 0.xxx |
| TV2/OV2 | n | xx | xx | |
| | LS Mean | XX.X | XX.X | |
| | SE (LS Mean) | XX.XX | xx.xx | |
| | 95% CI (LS Mean) | (xx.x, xx.x) | (xx.x, xx.x) | |
| | LS Mean Difference (CVT-301 - O.C.) | | XX.X | |
| | 95% CI (LS Mean Difference) | | (xx.x, xx.x) | |
| | p-value (LS Mean Difference) | | 0.xxx | |
| TV3/OV3 | <del>-</del> | | | |

Note: TV = Treatment Visit; OV = Observational Visit; MMRM model uses the total daily OFF time at each post-baseline visit (TV2, TV3, TV4, TV5 or TV6) as the dependent variable, and includes the treatment group (CVT-301 or O.C.), visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus  $\ge$ 2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1  $\ge$ 60% and FEV1/FVC ratio  $\ge$ 70%)) and the interaction between the treatment group and visit as fixed factors. The total daily OFF time at baseline will be included as a covariate, assuming an unstructured covariance matrix.

Cross-reference: Listing 16.2.6.2.3.2


Table below will use format Table 14.2.1.3.2 except for two treatment group.

Table 14.2.5.1.2

Sensitivity Analysis: Mean of Total Daily OFF Time by Visit

MI analysis with Missing At Random Assumption

(ITT Population)

Note: TV = Treatment Visit; OV = Observational Visit;

The non-monotone missing values will be imputed using the Markov Chain Monte Carlo (MCMC) methodology which assumes a multivariate normal distribution over all variables included in the imputation model. The monotone missing values are imputed using pattern mixture model assuming missing at random. MMRM model uses the total daily OFF time at each post-baseline visit (TV2, TV3, TV4, TV5 or TV6) as the dependent variable, and includes the treatment group (CVT-301 or O.C.), visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus >2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1 >60% and FEV1/FVC ratio >70%)) and the interaction between the treatment group and visit as fixed factors. The total daily OFF time at baseline will be included as a covariate, assuming an unstructured covariance matrix. The MIANALYZE procedure in SAS will be applied to combine the results from these datasets to derive an overall estimate at each visit.

Cross-reference: Listing 16.2.6.2.3.2

Table below will use the table 14.2.5.1.1 template except will be performed for "Hoehn & Yahr scale < 2.5 points" and "Hoehn & Yahr scale >= 2.5 points" and removed 'baseline Hoehn and Yahr stage (<2.5 versus  $\ge 2.5$ )' in the model. Footnote revised.

Table 14.2.5.1.3

Exploratory Efficacy Subgroup Analysis: Mean of Total Daily OFF Time by Visit by Baseline PD Severity (ITT Population)

Note: TV = Treatment Visit; OV = Observational Visit; MMRM model uses the total daily OFF time at each post-baseline visit (TV2, TV3, TV4, TV5 or TV6) as the dependent variable, and includes the treatment group (CVT-301 or O.C.), visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1  $\geq$ 60% and FEV1/FVC ratio  $\geq$ 70%)) and the interaction between the treatment group and visit as fixed factors. The total daily OFF time at baseline will be included as a covariate, assuming an unstructured covariance matrix.

Cross-reference: Listing 16.2.6.2.3.2

Table below will use the table 14.2.5.1.1 template and footnote except will be performed for "Dyskinetic before TV1" and "Non-dyskinetic before TV1"

Table 14.2.5.1.4

Exploratory Efficacy Subgroup Analysis: Mean of Total Daily OFF Time by Visit by Baseline Dyskinesia (ITT Population)

Table below will use the table 14.2.5.1.1 template and footnote except will be performed for "Baseline Daily Levodopa Dose<=Median of Baseline Daily Levodopa Dose" and "Baseline Daily Levodopa Dose".

Table 14.2.5.1.5

Exploratory Efficacy Subgroup Analysis: Mean of Total Daily OFF Time by Visit by Baseline Daily Levodopa Dose (ITT Population)

Table below will use the table 14.2.5.1.1 template and footnote except will be performed for "PD Diary Mean Daily OFF Time during Screening < 4.5 Hours" and "PD Diary Mean Daily OFF Time during Screening >=4.5 Hours".

Table 14.2.5.1.6

Exploratory Efficacy Subgroup Analysis: Mean of Total Daily OFF Time by Visit by PD Diary Mean Daily OFF Time during Screening (ITT Population)

Table below will use the table 14.2.5.1.1 template and footnote except will be performed for "FEV1 <60% or FEV1/FVC ratio <70%" and "FEV1  $\geq$ 60% and FEV1/FVC ratio  $\geq$ 70%" removed 'screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1  $\geq$ 60% and FEV1/FVC ratio  $\geq$ 70%' in the model. Footnote revised.

Table 14.2.5.1.7

Exploratory Efficacy Subgroup Analysis: Mean of Total Daily OFF Time by Visit by Screening Spirometry (ITT Population)

Note: TV = Treatment Visit; OV = Observational Visit; MMRM model uses the total daily OFF time at each post-baseline visit (TV2, TV3, TV4, TV5 or TV6) as the dependent variable, and includes the treatment group (CVT-301 or O.C.), visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus  $\geq$ 2.5)) and the interaction between the treatment group and visit as fixed factors. The total daily OFF time at baseline will be included as a covariate, assuming an unstructured covariance matrix.

Cross-reference: Listing 16.2.6.2.3.2

Table below will use the table 14.2.5.1.1 template and footnote except will be performed for "Non-elderly (<65 years)" and "Elderly ( $\geq$ 65 years) patients".

Table 14.2.5.1.8

Exploratory Efficacy Subgroup Analysis: Mean of Total Daily OFF Time by Visit by Age Group (ITT Population)

Table below will use the table 14.2.5.1.1 template and footnote except will be performed for "Female" and "Male".

Table 14.2.5.1.9

Exploratory Efficacy Subgroup Analysis: Mean of Total Daily OFF Time by Visit by Gender (ITT Population)

Table below will use the table 14.2.5.1.1 template.


Table 14.2.5.2

Exploratory Efficacy Analysis: Mean of Total Daily ON Time without Dyskinesia by Visit (ITT Population)

Note: TV = Treatment Visit; OV = Observational Visit; MMRM model uses the total daily ON time without dyskinesia at each postbaseline visit (TV2, TV3, TV4, TV5 or TV6) as the dependent variable, and includes visit (TV2, TV3, TV4, TV5 or TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus ≥2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1 ≥60% and FEV1/FVC ratio ≥70%)) as fixed factors; the total daily ON time without dyskinesia at baseline will be included as a covariate, assuming an unstructured covariance matrix.

Cross-reference: Listing 16.2.6.2.3.2

Table 14.2.5.3

Exploratory Efficacy Analysis: Mean of Total Daily ON Time with non-Troublesome Dyskinesia by Visit (ITT Population)

Note: TV = Treatment Visit; OV = Observational Visit; MMRM model uses the total daily ON time with non-troublesome dyskinesia at each post-baseline visit (TV2, TV3, TV4, TV5 or TV6) as the dependent variable, and includes visit (TV2, TV3, TV4, TV5 or TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus ≥2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1 ≥60% and FEV1/FVC ratio ≥70%)) as fixed factors; the total daily ON time with non-troublesome dyskinesia at baseline will be included as a covariate, assuming an unstructured covariance matrix.

Cross-reference: Listing 16.2.6.2.3.2

Table 14.2.5.4

Exploratory Efficacy Analysis: Mean of Total Daily ON Time with Troublesome Dyskinesia by Visit (ITT Population)

Note: TV = Treatment Visit; OV = Observational Visit; MMRM model uses the total daily ON time with troublesome dyskinesia at each post-baseline visit (TV2, TV3, TV4, TV5 or TV6) as the dependent variable, and includes visit (TV2, TV3, TV4, TV5 or TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus ≥2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1 ≥60% and FEV1/FVC ratio ≥70%)) as fixed factors; the total daily ON time with troublesome dyskinesia at baseline will be included as a covariate, assuming an unstructured covariance matrix.

Cross-reference: Listing 16.2.6.2.3.2

will have similar format as Table 14.2.5.1.1.


Table 14.2.6.1
Exploratory Efficacy Analysis: Subjects Global Impression of Change (PGI-C) by Visit
Worst Case Imputation [a]
(ITT Population)

| | CVT-301 |
|---------------------|-----------|
| | (N=xx) |
| /isit/Statistic | n (%) |
| V4/0V4 | |
| n | XX |
| Much Improved | xx (xx.x) |
| Improved | xx (xx.x) |
| A little Improved | xx (xx.x) |
| No Change | xx (xx.x) |
| A Little Worse | xx (xx.x) |
| Worse | xx (xx.x) |
| Much Worse | xx (xx.x) |
| Improved [b] | |
| Yes | xx (xx.x) |
| No | xx (xx.x) |
| Improved (Observed) | |
| Yes | xx (xx.x) |
| No | xx (xx.x) |
| Missing | xx (xx.x) |

Note: TV = Treatment Visit; OV = Observational Visit; Percentages are based on n, the number of subjects with PGI-C performed at each visit.

Cross-reference: Listing 16.2.6.2.4

<sup>[</sup>a] The missing values will be counted as No.

<sup>[</sup>b] The patient who had PGI-C response of much improved, improved or a little improved will be counted as Yes.


Table 14.2.7.1 Exploratory Efficacy Analysis: UPDRS Part 2 Score at TV4/OV4 (ITT Population)

| | | O. C. | CVT-301 |
|---|---|---|---|
| /isit | Statistic | (N=xx) | (N=xx) |
| Baseline | Actual Value | | |
| | n | xx | XX |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min, Max | xx, xx | XX, XX |
| TV4/OV4 | Actual value | | |
| | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min, Max | xx, xx | XX, XX |
| | Change from Baseline | | |
| | n | xx | xx |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min, Max | xx, xx | XX, XX |
| | LS Mean | xx.xx | XX.XX |
| | SE (LS Mean) | xx.xxx | xx.xxx |
| | 95% CI (LS Mean) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| | LS Mean Difference (CVT-301 - O. C.) | | xx.xx |
| | 95% CI (LS Mean Difference) | | (xx.xx, xx.xx) |
| | p-value (LS Mean Difference) | | 0.xxx |

Note: TV = Treatment Visit; OV = Observational Visit; Baseline is defined as the assessments performed at TV1/OV1. If the TV1/OV1 assessment is missing, the last non-missing screening assessment will be used as baseline. An ANCOVA model with the treatment group and stratification variables (baseline Hoehn and Yahr stage (<2.5 versus ≥2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1 ≥60% and FEV1/FVC ratio ≥70%)) as fixed factors and the baseline value as a covariate will be used to estimate the treatment differences.

Cross-reference: Listing 16.2.6.3.1

Table below s will use the table 14.2.7.1 template.

Table 14.2.7.2

Page x of y

Exploratory Efficacy Analysis: UPDRS Part 2 Score at TV6/OV6 (ITT Population)

Table below s will use the table 14.2.7.1 template with revised cross-reference

Table 14.2.8.1

Exploratory Efficacy Analysis: Schwab and England (S&E) Activities of Daily Living (ADL) Score at TV4/OV4 (ITT Population)

Table 14.2.8.2

Exploratory Efficacy Analysis: Schwab and England (S&E) Activities of Daily Living (ADL) Score at TV6/OV6 (ITT Population)

Note: TV = Treatment Visit; OV = Observational Visit; Baseline is defined as the assessments performed at TV1/OV1. If the TV1/OV1 assessment is missing, the last non-missing screening assessment will be used as baseline. An ANCOVA model with the treatment group and stratification variables (baseline Hoehn and Yahr stage (<2.5 versus  $\geq$ 2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1  $\geq$ 60% and FEV1/FVC ratio  $\geq$ 70%)) as fixed factors and the baseline value as a covariate will be used to estimate the treatment differences.

Cross-reference: Listing 16.2.6.3.2

Table below s will use the table 14.2.7.1 template with revised cross-reference

Table 14.2.9.1

Exploratory Efficacy Analysis: 39 Item Parkinson's disease Questionnaire (PDQ-39) Sub-scores and Summary Index Score at TV4/OV4 (ITT Population)

Table 14.2.9.2

Exploratory Efficacy Analysis: 39 Item Parkinson's disease Questionnaire (PDQ-39) Sub-scores and Summary Index Score at TV6/OV6 (ITT Population)

Note: TV = Treatment Visit; OV = Observational Visit; Baseline is defined as the assessments performed at TV1/OV1. If the TV1/OV1 assessment is missing, the last non-missing screening assessment will be used as baseline. An ANCOVA model with the treatment group and stratification variables (baseline Hoehn and Yahr stage (<2.5 versus  $\geq$ 2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1  $\geq$ 60% and FEV1/FVC ratio  $\geq$ 70%)) as fixed factors and the baseline value as a covariate will be used to estimate the treatment differences.

Cross-reference: Listing 16.2.6.3.2

Table 14.3.1.1
Extent of Exposure: Overall for CVT-301 Group Only (Safety Population)

| N | | | 002/003 | Naive | Total |
|---|---|---|---|---|---|
| Dicease | | | (N=xx) | (N=xx) | (N=xx) |
| Dicease | Subjects with Dose Change | n (§) | vv (vv v) | vv (vv v) | vv (vv v) |
| Decrease n (%) | | | | | |
| Number of Exposure (days) [a] | | | | | |
| Mean | Decrease | 11 (0) | AA (AA.A) | AA (AA•A) | AA (AA.A) |
| SD | Duration of Exposure (days) [a] | | XX | XX | XX |
| Median XX. X XX. | | | XX.X | XX.X | XX.X |
| Min, Max | | | XX.XX | XX.XX | XX.XX |
| Summed Total XXX | | | XX.X | XX.X | XX.X |
| Number of Capsules Taken (Overall) | | Min, Max | xx, xx | xx, xx | XX, XX |
| TV1- <tv2 (overall)="" doses="" number="" of="" taken="" td="" total="" tv1-<tv3="" tv2-<tv3="" tv2-ctv3="" tv3-<tv4="" tv3-ctv4="" tv4-ctv5="" tv4-tv5="" tv5-tv6="" tv5-tv7="" tv7-c<="" tv7-ctv7=""><td></td><td>Summed Total</td><td>XXX</td><td>XXX</td><td>XXX</td></tv2> | | Summed Total | XXX | XXX | XXX |
| TV1- <tv2 (overall)="" doses="" number="" of="" taken="" td="" total="" tv1-<tv3="" tv2-<tv3="" tv2-ctv3="" tv3-<tv4="" tv3-ctv4="" tv4-ctv5="" tv4-tv5="" tv5-tv6="" tv5-tv7="" tv7-c<="" tv7-ctv7=""><td>Total Number of Capsules Taken (Overall)</td><td>n</td><td>XX</td><td>XX</td><td>xx</td></tv2> | Total Number of Capsules Taken (Overall) | n | XX | XX | xx |
| TV1- <tv2 10="" 1<="" td=""><td>, , , , , , , , , , , , , , , , , , ,</td><td></td><td></td><td></td><td></td></tv2> | , | | | | |
| TV1- <tv2 rean<="" td=""><td></td><td></td><td></td><td></td><td></td></tv2> | | | | | |
| TV2- <tv3 (overall)="" average="" capsules="" daily="" doses="" number="" of="" potal="" taken="" td="" tv1-<tv2="" tv2-<tv3="" tv2-tv3="" tv3-<tv4="" tv3-ctv4="" tv3-tv4="" tv4-ctv5="" tv4-tv5="" tv5-tv6="" tv5-tv6<=""><td>TV1-<tv2< td=""><td></td><td>XX</td><td>xx</td><td>XX</td></tv2<></td></tv3> | TV1- <tv2< td=""><td></td><td>XX</td><td>xx</td><td>XX</td></tv2<> | | XX | xx | XX |
| TV2- <tv3 (overall)="" **<="" **cotal="" **potal="" doses="" number="" of="" taken="" td="" tv3-<tv4="" tv4-<tv5="" tv5-tv6=""><td></td><td></td><td></td><td></td><td></td></tv3> | | | | | |
| TV2- <tv3 (overall)="" average="" daily="" doses="" n="" number="" of="" potal="" taken="" td="" tv1-<tv2="" tv2-ctv3="" tv3-ctv4="" tv3-tv4="" tv4-ctv5="" tv5-tv6="" xx="" xx<=""><td></td><td></td><td></td><td></td><td></td></tv3> | | | | | |
| TV3- <tv4 (overall)="" doses="" n<="" number="" octal="" of="" taken="" td="" tv4-<tv5="" tv5-tv6=""><td>TV2-<tv3< td=""><td></td><td></td><td></td><td></td></tv3<></td></tv4> | TV2- <tv3< td=""><td></td><td></td><td></td><td></td></tv3<> | | | | |
| TV5-TV6 TV5-TV6 TV5-TV6 TV5-TV6 TV5-TV6 TV5-TV6 TV5-TV6 TV7-TV2 TV1- <tv2 (overall)="" average="" daily="" doses="" td="" tv1-<tv2="" tv2-<tv3="" tv3-<tv4="" tv4-tv5="" tv5-tv6="" tv5-tv7="" tv7-tv7="" tv7-tv7<=""><td></td><td></td><td></td><td></td><td></td></tv2> | | | | | |
| TV5-TV6 Potal Number of Doses Taken (Overall) n | | | | | |
| Number of Doses Taken (Overall) Number of Doses Taken (Overall) Number of Doses Taken (Overall) Number of Capsules ( | | | | | |
| Mean | | | vv | vv | VV |
| TV1- <tv2 (overall)="" average="" daily="" doses="" mean="" n="" td="" tv2-ctv3="" tv3-ctv4="" tv4-ctv5="" tv5-tv6="" xx="" xx<=""><td>rotal Nambel of Boses Taken (overall)</td><td></td><td></td><td></td><td></td></tv2> | rotal Nambel of Boses Taken (overall) | | | | |
| TV1- <tv2 (overall)="" average="" daily="" doses="" n="" td="" tv2-tv3="" tv3-<tv4="" tv4-ctv5="" tv5-tv6="" xx="" xx<=""><td></td><td></td><td>AA • A</td><td>AA · A</td><td>AA·A</td></tv2> | | | AA • A | AA · A | AA·A |
| TV2- <tv3 (overall)="" average="" daily="" doses="" n<="" td="" tv3-<tv4="" tv4-<tv5="" tv5-tv6=""><td>TV1 - &lt; TV2</td><td></td><td></td><td></td><td></td></tv3> | TV1 - < TV2 | | | | |
| TV3- <tv4 (overall)="" average="" daily="" doses="" n<="" td="" tv4-<tv5="" tv5-tv6=""><td></td><td></td><td></td><td></td><td></td></tv4> | | | | | |
| TV4- <tv5 (overall)="" average="" daily="" doses="" n<="" td="" tv5-tv6=""><td></td><td></td><td></td><td></td><td></td></tv5> | | | | | |
| TV5-TV6 Average Daily Doses (Overall) n xx xx xx Mean xx.x | | ••• | | | |
| Mean xx.x xx.x xx.x TV1- <tv2 (overall)="" average="" capsules="" daily="" mean="" n="" number="" of="" td="" tv2-<tv3="" tv3-<tv4="" tv4-<tv5="" tv5-tv6="" xx="" xx.x="" xx.x<=""><td></td><td></td><td></td><td></td><td></td></tv2> | | | | | |
| Mean xx.x xx.x xx.x TV1- <tv2 (overall)="" average="" capsules="" daily="" mean="" n="" number="" of="" td="" tv2-<tv3="" tv3-<tv4="" tv4-<tv5="" tv5-tv6="" xx="" xx.x="" xx.x<=""><td>Average Daily Deces (Overall)</td><td>_</td><td></td><td></td><td></td></tv2> | Average Daily Deces (Overall) | _ | | | |
| TV1- <tv2 (overall)="" average="" capsules="" daily="" n="" number="" of="" td="" tv2-<tv3="" tv3-<tv4="" tv4-<tv5="" tv5-tv6="" xx="" xx<=""><td>average Daily Doses (Overall)</td><td></td><td></td><td></td><td></td></tv2> | average Daily Doses (Overall) | | | | |
| TV1- <tv2 (overall)="" average="" capsules="" daily="" n="" number="" of="" td="" tv2-<tv3="" tv3-<tv4="" tv4-<tv5="" tv5-tv6="" xx="" xx.x<=""><td></td><td></td><td>xx.x</td><td>xx.x</td><td>XX.X</td></tv2> | | | xx.x | xx.x | XX.X |
| TV2- <tv3 (overall)="" average="" capsules="" daily="" mean="" n="" number="" of="" td="" tv3-<tv4="" tv4-<tv5="" tv5-tv6="" xx="" xx.x="" xx.x<=""><td>mt/1 /mt/0</td><td></td><td></td><td></td><td></td></tv3> | mt/1 /mt/0 | | | | |
| TV3- <tv4 (overall)="" average="" capsules="" daily="" n="" number="" of="" td="" tv4-<tv5="" tv5-tv6="" xx="" xx<=""><td></td><td></td><td></td><td></td><td></td></tv4> | | | | | |
| TV4- <tv5 (overall)="" average="" capsules="" daily="" n="" number="" of="" td="" tv5-tv6="" xx="" xx<=""><td></td><td></td><td></td><td></td><td></td></tv5> | | | | | |
| TV5-TV6 Average Daily Number of Capsules (Overall) n xx xx xx xx Mean xx.x xx.x xx.x | | • • • | | | |
| verage Daily Number of Capsules (Overall) n xx xx xx xx xx xx.x xx.x | | | | | |
| Mean xx.x xx.x xx.x | TV5-TV6 | | | | |
| Mean xx.x xx.x xx.x | Average Daily Number of Capaules (Overall) | _ | | | |
| ••• | Average parry number or capsures (Overall) | | | | |
| | | | XX.X | XX.X | XX.X |
| | | • • • | | | |

TV2-<TV3
TV3-<TV4
TV4-<TV5
TV5-TV6

Note: TV = Treatment Visit; Total column is for all CVT-301 treated patients, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Data presented is self-reported by study participants and is subject to limitations of self-report measures.

[a] Duration of exposure (days) is calculated as documented last dose date-first dose date +1. Cross-reference: Listing 16.2.5.1.3, 16.2.5.1.4, 16.2.5.1.5

Table 14.3.1.1
Extent of Exposure: Overall for CVT-301 Group Only (Safety Population)

| | | 002/003<br>(N=xx) | Naive<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|
| Proportion of Days with >5 Doses per Day | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | ••• | | | |
| Proportion of Days with 5 Doses per Day | n | XX | XX | XX |
| | Mean | xx.x | XX.X | XX.X |
| | • • • | | | |
| Proportion of Days with 4 Doses per Day | n | xx | XX | XX |
| | Mean | xx.x | XX.X | XX.X |
| | ••• | | | |
| Proportion of Days with 3 Doses per Day | n | xx | XX | XX |
| | Mean | xx.x | XX.X | XX.X |
| | ••• | | | |
| Proportion of Days with 2 Doses per Day | n | xx | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | ••• | | | |
| Proportion of Days with 1 Dose per Day | n | xx | XX | XX |
| | Mean | xx.x | XX.X | XX.X |
| | • • • | | | |
| Proportion of Days with 0 Dose per Day | n | xx | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| Proportion of Patients using >5 Doses/day at least once | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | • • • | | | |
| Proportion of Patients using 5 Doses/day at least once | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | • • • | | | |
| Proportion of Patients using 4 Doses/day at least once | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | • • • | | | |
| Proportion of Patients using 3 Doses/day at least once | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | • • • | | | |
| Proportion of Patients using 2 Doses/day at least once | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | • • • | | | |
| Proportion of Patients using 1 Dose/day at least once | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| Proportion of Patients using 0 Dose/day at least once | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |

Note: TV = Treatment Visit; Total column is for all CVT-301 treated patients, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients.

Data presented is self-reported by study participants and is subject to limitations of self-report measures.

<sup>[</sup>b] Duration of exposure (days) is calculated as documented last dose date-first dose date +1. Cross-reference: Listing 16.2.5.1.1, 16.2.5.1.3


Table 14.3.1.2 In-Clinic Study Drug Administration (Safety Population)

| Visit | Parameter | Statistic | 002/003<br>(N=xx) | Naive<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|---|
| TV1 | Standard Morning Dose of LD-containing Medications | | | | |
| IVI | to in-clinic OFF (mins) | n | xx | XX | XX |
| | to in time of (mins) | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.XX | XX.XX | XX.XX |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | xx, xx | xx, xx | xx, xx |
| | <= 180 mins | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | > 180 to <= 210 mins | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | > 210 to <= 240 mins | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | > 240 to <= 270 mins | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | > 270 mins | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | In-clinic OFF to Start of Study Drug Inhalation (mins) | n | xx | XX | xx |
| | | Mean | XX.X | XX.X | XX.X |
| | | • • • | | | |
| | <= 10 mins | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | > 10 to <= 15 mins | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | > 15 to <= 20 mins | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | > 20 to <= 25 mins | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | > 25 to <= 30 mins | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | > 30 mins | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Standard Morning Dose of LD-containing Medications | | | | |
| | to Start of Study Drug Inhalation (mins) | n | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | Duration of Study Drug Inhalation (mins) | n | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X |
| TV2 | ••• | | | | |
| TV3 | ••• | | | | |

Note: TV = Treatment Visit; Total column is for all CVT-301 treated patients, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients.

Percentages are based on the number of subjects with results for each parameter at each treatment visit within each treatment group or Overall.

Cross-reference: Listing 16.2.5.1.2

Table 14.3.1.3

Distribution of Time of Study Drug Administration for CVT-301 Group Only (Safety Population)

| Time Interval | Statistic | 002/003<br>(N=xx) | Naive<br>(N=xx) | Total (N=xx) |
|---|---|---|---|---|
| Total Study Medication Intakes | n | xx | xx | xx |
| 00:00 -< 00:30 | n (%) | xx (%) | xx (%) | xx (%) |
| 00:30 -< 01:00 | n (%) | xx (%) | xx (%) | xx (%) |
| 01:00 -< 01:30 | n (%) | xx (%) | xx (%) | xx (%) |
| 01:30 -< 02:00 | n (%) | xx (%) | xx (%) | xx (%) |

Continue with 30 mins interval until 23:30 -< 24:00

Note: Total column is for all CVT-301 treated patients, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. The percentage is based on the total # of study medication intakes.

Cross-reference: Listing 16.2.5.1.1

Table 14.3.2.1
Treatment-Emergent Adverse Events -Overall Summary (Safety Population)

| | | | CVT- 301 | | |
|---|---|---|---|---|---|
| | O. C. | 002/003 | Naive | Total | Overall |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| | Subjects Events | Subjects Events | Subjects Events | Subjects Events | Subjects Events |
| | n (%) n | n (%) n | n (%) n | n (%) n | n (%) n |
| Any TEAEs | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) |
| Drug-related TEAEs [a] | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) |
| Severe TEAEs | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) |
| Serious TEAEs | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) |
| TEAEs Leading to Study Drug Interruption | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) |
| TEAEs Leading to Study<br>Drug Discontinuation | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) |
| TEAEs Leading to Dose<br>Reduction | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) |
| TEAEs Leading to Death | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) |

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Treatment-emergent adverse events (TEAEs) are defined as all AEs that start after the patient receives the first dose of study drug.

Cross-reference: Listing 16.2.7.1

<sup>[</sup>a] Adverse events are considered drug-related if the event is classified as possibly, probably, or definitely related to study drug.

## ${\tt Table~14.3.2.2.1}$ Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population)

| | O. C.<br>(N=xx) | 002/003<br>(N=xx) | Naive<br>(N=xx) | Total<br>(N=xx) | Overall (N=xx) |
|---|---|---|---|---|---|
| System Organ Class | Subjects Events | Subjects Events | Subjects Events | Subjects Events | Subjects Events |
| Preferred Term [a] | n (%) n | n (%) n | n (%) n | n (%) n | n (%) n |
| Any TEAEs | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| System Organ Class | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| • • • | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| System Organ Class | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| • • • | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Treatment-Emergent Adverse Events (TEAEs) are defined as all AEs that start after the patient receives the first dose of study drug.

[a] Adverse events were coded into system organ class and preferred term using MedDRA version 17.0.

Cross-reference: Listing 16.2.7.1

Programming note: The table will be sorted by total descending frequency of SOC and then, within a SOC, by total descending frequency of PT.

# Table 14.3.2.2.2 Treatment-Emergent Adverse Events by Preferred Term (Safety Population)

| | | CVT- 301 | | | |
|---|---|---|---|---|---|
| | O. C. | 002/003 | Naive | Total | Overall |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| | Subjects Events | Subjects Events | Subjects Events | Subjects Events | Subjects Events |
| Preferred Term [a] | n (%) n | n (%) n | n (%) n | n (%) n | n (%) n |
| Any TEAEs | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term 1 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term 2 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term 3 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term 4 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| • • • | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Na $\"{\text{ave}}$  is for the CVT-301 na $\acute{\text{naive}}$  patients. Treatment-Emergent Adverse Events (TEAEs) are defined as all AEs that start after the patient receives the first dose of study drug

[a] Adverse events were coded into system organ class and preferred term using MedDRA version 17.0.

Cross-reference: Listing 16.2.7.1

Programming note: The table will be sorted by total descending frequency of PT.

Table 14.3.2.3

Drug-Related Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and Severity (Safety Population)

| | | | | CVT- 301 | | |
|---|---|---|---|---|---|---|
| | | o. c. | 002/003 | Naive | Total | Overall |
| System Organ Class | | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Preferred Term [a] | Severity | n (%) | n (%) | n (%) | n (%) | n (%) |
| All TEAEs | Total | XX | XX | XX | XX | XX |
| | Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class | Total | XX | XX | XX | XX | XX |
| | Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term<br>Preferred Term | ••• | | | | | |
| System Organ Class Preferred Term Preferred Term | | | | | | |
| • • • | | | | | | |

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Treatment-Emergent Adverse Events (TEAEs) are defined as all AEs that start after the patient receives the first dose of study drug. Adverse events are considered drug-related if the event is classified as possibly, probably, or definitely related to study drug. The percentages are calculated based on the total number of TEAEs.

[a] Adverse events were coded into system organ class and preferred term using MedDRA version 17.0.

Cross-reference: Listing 16.2.7.1

Programming note: The table will be sorted by total descending frequency of SOC then PT in total row, total column.

Table 14.3.2.4

Drug -Related Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and Relationship (Safety Population)

| | | | CVT- 301 | | |
|---|---|---|---|---|---|
| Maximal<br>Severity [b] | O. C.<br>(N=xx)<br>n (%) | 002/003<br>(N=xx)<br>n (%) | Naive<br>(N=xx)<br>n (%) | Total<br>(N=xx)<br>n (%) | Overall<br>(N=xx)<br>n (%) |
| <u>-</u> | | | | | |
| Total | XX | XX | xx | XX | XX |
| Possibly Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Probably Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Definitely Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total | XX | xx | xx | xx | xx |
| Possibly Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Probably Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Definitely Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Total Possibly Related Probably Related Definitely Related Total Possibly Related Probably Related Probably Related Definitely Related | Maximal (N=xx) Severity [b] n (%) Total xx Possibly Related xx (xx.x) Probably Related xx (xx.x) Definitely Related xx (xx.x) Total xx Possibly Related xx (xx.x) Probably Related xx (xx.x) Probably Related xx (xx.x) Definitely Related xx (xx.x) | Maximal Severity [b] (N=xx) n (%) (N=xx) n (%) Total XX XX XX XX (XX.X) XX (XX.X) Probably Related XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) Definitely Related XX (XX.X) XX (XX.X) XX XX XX Possibly Related XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) Probably Related XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) Definitely Related XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | Maximal O. C. (N=xx) 002/003 Naive (N=xx) Severity [b] n (%) n (%) n (%) Total xx xx xx Possibly Related xx (xx.x) xx (xx.x) xx (xx.x) Probably Related xx (xx.x) xx (xx.x) xx (xx.x) Total xx xx (xx.x) xx (xx.x) Total xx xx xx Possibly Related xx (xx.x) xx (xx.x) xx (xx.x) Probably Related xx (xx.x) xx (xx.x) xx (xx.x) Definitely Related xx (xx.x) xx (xx.x) xx (xx.x) | Maximal O. C. (N=xx) 002/003 Naive (N=xx) Total (N=xx) Severity [b] n (%) n (%) n (%) n (%) Total xx xx xx xx Possibly Related xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) Probably Related xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) Total xx xx xx xx xx Possibly Related xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) Probably Related xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) Definitely Related xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) |

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Treatment-Emergent Adverse Events (TEAEs) are defined as all AEs that start after the patient receives the first dose of study drug. Adverse events are considered drug-related if the event is classified as possibly, probably, or definitely related to study drug. The percentages are calculated based on the total number of TEAEs.

[a] Adverse events were coded into system organ class and preferred term using MedDRA version 17.0.

Cross-reference: Listing 16.2.7.1

Programming note: The table will be sorted by Definitely Not Related descending frequency of SOC then PT in total row, total column.

Table below s will have same format as T14.3.2.4.1 and note:

Table below s will have same format as 14.3.2.2.1 and note:

Table 14.3.2.5

Drug-related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population)

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Treatment-Emergent Adverse Events (TEAEs) are defined as all AEs that start after the patient receives the first dose of study drug Adverse events are considered drug-related if the event is classified as possibly, probably, or definitely related to study drug.

[a] Adverse events were coded into system organ class and preferred term using MedDRA version 17.0.

Cross-reference: Listing 16.2.7.1

Table 14.3.2.6

Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population)

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Treatment-Emergent Adverse Events (TEAEs) are defined as all AEs that start after the patient receives the first dose of study drug

[a] Adverse events were coded into system organ class and preferred term using MedDRA version 17.0.

Cross-reference: Listing 16.2.7.1, Table 14.3.2.7


### Table 14.3.2.7 Listing of Serious Adverse Events

| Treatment Group: 0. C. | | AE Start<br>Date | | <pre>I: Intensity R: Relationship</pre> | | |
|---|---|---|---|---|---|---|
| Su<br>bject | System Organ Class/<br>Preferred Term/ | and Time/<br>Study Day | | to Study<br>Medication | | |
| ID | Verbatim Term [a] | [b] | AE Stop Date and Time | A: Action Taken | Outcome | SAE? If Yes, Specify [c] |
| | xxxxxxxxx/ | ddmonyyyy | | I: xxxxxxxx | | |
| | xxxxxxxx/ | hh:mm/ | ddmonyyyy | R: xxxxxxxx | | |
| xxx-xxx | xxxxxxxx | -XX | Hh:mm | A: xxxxxxxxx | Resolved | Yes: 1 |
| | xxxxxxxxx/ | ddmonyyyy | | I: xxxxxxxx | | |
| | xxxxxxxx/ | hh:mm/ | | R: xxxxxxxx | | |
| | xxxxxxxx | xx# | Ongoing | A: xxxxxxxxx | Unknown | No |
| | xxxxxxxxx/ | ddmonyyyy | | I: xxxxxxxx | | |
| | xxxxxxxx/ | hh:mm/ | ddmonyyyy | R: xxxxxxxx | | |
| xxxx-xxx | xxxxxxxxx | -xx | Hh:mm | A: xxxxxxxxx | Resolved | Yes: 2 |

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. TEAE=Treatment-emergent AE. SAE=Serious AE.

- [a] Adverse events were coded into system organ class and preferred term using MedDRA version 17.0.
- [b] TEAEs were flagged with a #. The AEs occurred on the clinic visit were flagged with \*. Study day is relative to date of first study medication (date of first dose = Day 1).
- [c] 1 = The event is fatal or life-threatening, 2 = The event is permanently disabling (incapacitating or interfering with the ability to resume usual life patterns), 3 = The event results in unplanned in subject hospitalization or prolongation of existing hospitalization, 4 = The event is a congenital anomaly, 5 = The event requires medical intervention of any kind in order to prevent any of the aforementioned outcomes.

Cross-reference: Listing 16.2.7.1

Table below s will have same format as T14.3.2.7

Table 14.3.2.8

Listing of Adverse Events Leading to Death

Table below s will have same format as T14.3.2.2.1and revised Cross-reference

Table 14.3.2.9

Severe Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population)

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Treatment-Emergent Adverse Events (TEAEs) are defined as all AEs that start after the patient receives the first dose of study drug Adverse events are considered drug-related if the event is classified as possibly, probably, or definitely related to study drug.

[a] Adverse events were coded into system organ class and preferred term using MedDRA version 17.0.

Cross-reference: Listing 16.2.7.1, table 14.3.2.10

Table below s will have same format as T14.3.2.7

Table 14.3.2.10

Listing of Severe Treatment-Emergent Adverse Events

(Safety Population)

Table below s will have same format as T14.3.2.2.1and revised Cross-reference

Table 14.3.2.11

Treatment-Emergent Adverse Events Leading to Study Drug Interruption by System Organ Class and Preferred Term (Safety Population)

Cross-reference: Listing 16.2.7.1, table 14.3.2.12

Table below s will have same format as T14.3.2.7

Table 14.3.2.12

Listing of Adverse Events Leading to Study Drug Interruption

Table below s will have same format as T14.3.2.2.1and revised Cross-reference

Table 14.3.2.13

Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term (Safety Population)

Cross-reference: Listing 16.2.7.1, table 14.3.2.14


Table below will have same format as T14.3.2.7

Table 14.3.2.14

Listing of Adverse Events Leading to Study Drug Discontinuation

Table below will have same format as T14.3.2.2.1and revised Cross-reference

Table 14.3.2.15

Treatment-Emergent Adverse Events Leading to Dose Reduction by System Organ Class and Preferred Term (Safety Population)

Cross-reference: Listing 16.2.7.1, table 14.3.2.16

Table below will have same format as T14.3.2.7

Table 14.3.2.16

Listing of Adverse Events Leading to Dose Reduction

Table 14.3.2.17

Most Common Treatment-Emergent Adverse Events (Preferred Term Occurred in >10% of Over Patients) by System Organ Class and Preferred

(Safety Population)

Cross-reference: Listing 16.2.7.1, table 14.3.2.18

Table 14.3.2.18

Listing of Most Common Treatment-Emergent Adverse Events

Table 14.3.2.19 Time to first Onset of Most Common Treatment-Emergent Adverse Events (Preferred Term Occurred in >10% of Over Patients) (Safety Population)

| | | CTV-301 | | | |
|---|---|---|---|---|---|
| Parameter | O.C.<br>(N=xx) | 002/003<br>(N=xx) | Naive<br>(N=xx) | Total<br>(N=xx) | Overall (N=xx) |
| 0 -< 30 Days | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 30 -< 90 Days | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 90 -< 180 Days | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 180 -< 270 Days | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >= 270 Days | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. TEAE=Treatment-emergent AE. Percentages are based on the number of subjects at each treatment group or Overall. Most common TEAEs is defined any AE preferred term occurred in greater than 10% of overall patients. Time to first onset of most common TEAE is calculated as onset of first common TEAE-first dose date (or date of OV1) +1).

Cross-reference: Listing 16.2.7.1


Table 14.3.4.1 Clinical Laboratory Results: PCS and PCSC Criteria

| Laboratory Parameter (Units) | Criteria for PCS V | alues (Actual values) | Criteria for PCSC v | values (Changes from baseline values) |
|---|---|---|---|---|
| | High | Low | % Increase | % Decrease |
| Hemoglobin (g/L) | > 10 above ULN | >20 below LLN | NA | 25% |
| Hematocrit (1) | >0.04 above ULN | >0.05 below LLN | NA | 25% |
| WBC (GI/L) | >5 above ULN | >1 below LLN | 100% | 50% |
| Neutrophils (GI/L) | NA | <0.5xLLN | 100% | 50% |
| Neutrophils (% ) | NA | <0.5xLLN | 100% | 50% |
| Lymphocytes (GI/L) | NA | <0.5xLLN | 100% | 50% |
| Lymphocytes (% ) | NA | <0.5xLLN | 100% | 50% |
| Total bilirubin (µmol/L) | >1.5xULN | NA | 300% | NA |
| Total protein (g/L) | >15 above ULN | >15 below LLN | 200% | 60% |
| Albumin (g/L) | >5 above ULN | >5 below LLN | NA | 60% |
| AST (U/L) | >3xULN | NA | 300% | NA |
| ALT (U/L) | >3xULN | NA | 300% | NA |
| Alkaline Phosphatase (U/L) | >3xULN | NA | 300% | NA |
| GGT (U/L) | >3xULN | NA | 300% | NA |
| Creatinine (µmol/L) | >1.5xULN | NA | 200% | NA |
| Urea (mmol/L) | >2.5xULN | NA | 300% | NA |
| Uric Acid (µmol/L) | >3xULN | NA | 300% | NA |
| Sodium (mmol/L) | >5 above ULN | >5 below LLN | 10% | 10% |
| Potassium (mmol/L) | >1 above ULN | >0.5 below LLN | 25% | 20% |
| Carbon dioxide (mmol/L) | >40 | <16 | 25% | 25% |
| Calcium (mmol/L) | >2.99 | <1.78 | 30% | 30% |
| Glucose (fasting)* (mmol/L) | >11.1 | <2.8 | 300% | 40% |

Note: ALT = alanine aminotransferase; AST = aspartate aminotransferase; GGT = gamma glutamyl transferase; LLN = lower limit of normal range; NA = not applicable; PCS = potentially clinically significant; PCSC = potentially clinically significant changes; Baseline is defined as the assessments performed at TV1/OV1. If the TV1/OV1 assessment is missing, the last non-missing screening assessment will be used as baseline. \* fasting defined as >=4 hr from prior meal.


Table 14.3.4.1.1.1 Summary of Clinical Laboratory Results: Hematology (Safety Population)

| | | | | | CVT- 301 | | |
|---|---|---|---|---|---|---|---|
| Test (unit) | Visit | Visit Statistic | O. C.<br>(N=xx) | 002/003<br>(N=xx) | Naive<br>(N=xx) | Total<br>(N=xx) | Overall (N=xx) |
| Test 1 (unit) | Baseline | Actual value | | | | | |
| | | n | XX | xx | XX | xx | xx |
| | | Mean | XX.X | XX.X | XX.X | XX.X | xx.x |
| | | SD | XX.XX | xx.xx | XX.XX | XX.XX | xx.xx |
| | | Median | XX.X | XX.X | XX.X | XX.X | xx.x |
| | | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX |
| | TV3/OV3 | Actual value | | | | | |
| | | n | XX | XX | xx | XX | xx |
| | | Mean | xx.x | XX.X | xx.x | XX.X | XX.X |
| | | SD | XX.XX | XX.XX | xx.xx | XX.XX | XX.XX |
| | | Median | XX.X | XX.X | xx.x | XX.X | xx.x |
| | | Min, Max | XX, XX | XX, XX | xx, xx | xx, xx | XX, X |
| | | Change from Baseline | | | | | |
| | | n | XX | XX | xx | XX | XX |
| | | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.XX | xx.xx | xx.xx | XX.XX | XX.XX |
| | | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | Min, Max | xx, xx | xx, xx | xx, xx | XX, XX | XX, X |
| | TV4/OV4 | | | | | | |
| Test 2 (unit) | Baseline | | | | | | |

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Baseline is defined as the TV1/OV1 assessment. If the TV1/OV1 assessment is missing, the last non-missing screening assessment will be used as baseline.

Cross-reference: Listing 16.2.8.1.1

Table 14.3.4.1.1.2

Summary of Clinical Laboratory Results: Hematology Abnormal Values (Safety Population)

| | | | | CVT- 301 | | |
|---|---|---|---|---|---|---|
| Test (unit) | Visit<br>Assessment | O. C.<br>(N=xx)<br>n (%) | 002/003<br>(N=xx)<br>n (%) | Naive<br>(N=xx)<br>n (%) | Total<br>(N=xx)<br>n (%) | Overall (N=xx) n (%) |
| Test 1 (unit) | SV1 | | | | | |
| rest i (unitt) | n | XX | XX | XX | XX | XX |
| | Normal | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | Abnormal: Low | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | Abnormal: High | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | PCS Low | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | PCS High | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | PCSC Low | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | PCSC High | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | SV2 | | | | | |
| | n | xx | xx | XX | xx | XX |
| | Normal | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | Abnormal: Low | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | Abnormal: High | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | • • • | | | | | |
| | TV3/OV3 | | | | | |
| | ••• | | | | | |
| | Followup | | | | | |
| Test 2 (unit) | | | | | | |

Note: SV = Screening Visit; TV = Treatment Visit; O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Percentages are based on n, the number of subjects with the test performed at each visit.

PCS = potentially clinically significant values. PCSC = potentially clinically significant changes.

Cross-reference: Listing 16.2.8.1.1, Table 14.3.4.1.1.6

Table 14.3.4.1.1.3

Summary of Clinical Laboratory Results: Hematology Abnormal Values -Shift from Baseline (Safety Population)

Test 1

| | | | Base | eline | |
|---|---|---|---|---|---|
| | Visit | Normal | Abnormal: Low | Abnormal: High | Total |
| Treatment | Assessment | n (%) | n (%) | n (%) | n (%) |
| o. c. | TV3/OV3 | | | | |
| | Normal | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | Abnormal: Low | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Abnormal: High | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | Total | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | <br>Followup | | | | |
| CVT-301 (002/003)<br>CVT-301 (Naïve)<br>CVT-301 Total<br>Overall | | | | | |
| Continue with other tests | | | | | |

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Percentages are based on the number of subjects with the test performed at both baseline and the visit.

Cross-reference: Listing 16.2.8.1.1, Table 14.3.4.1.1.6

Test 1

| | Visit | | Base | eline | |
|---|---|---|---|---|---|
| | | Not PCS | PCS: Low | PCS: High | Total |
| Treatment | Assessment | n (%) | n (%) | n (%) | n (%) |
| o. c. | TV3/OV3 | | | | |
| | Not PCS | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | PCS: Low | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | PCS: High | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Total | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Followup | | | | |
| | ••• | | | | |
| CVT-301 (002/003) | | | | | |
| CVT-301 (Naïve) | | | | | |
| CVT-301 Total | | | | | |
| Overall | | | | | |
| Continue with other | | | | | |
| tests | | | | | |

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Percentages are based on the number of subjects with the test performed at both baseline and the visit.

Cross-reference: Listing 16.2.8.1.1, Table 14.3.4.1.1.6

PCS = potentially clinically significant values.

Table 14.3.4.1.1.5 Summary of Clinical Laboratory Results: Hematology PCSC Values -Shift from Baseline (Safety Population)

Test 1

| Treatment | Visit<br>Assessment | Normal<br>(N=xx)<br>n (%) | Abnormal: Low (N=xx) n (%) | Abnormal: High (N=xx) n (%) | Total<br>(N=xx)<br>n (%) |
|---|---|---|---|---|---|
| o. c. | TV4 | | | | |
| | Normal | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Abnormal: Low | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Abnormal: High<br>Total | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Followup | | | | |
| CVT-301 (002/003)<br>CVT-301(Naïve)<br>CVT-301 Total<br>Overall | | | | | |
| Continue with other tests | | | | | |

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Percentages are based on the number of subjects with the test performed at both baseline and the visit.

Cross-reference: Listing 16.2.8.1.1, Table 14.3.4.1.1.6

PCSC = potentially clinically significant changes.


Table 14.3.4.1.1.6

Clinical Laboratory Results - Hematology PCS and PCSC Values (Safety Population)

Treatment Group: O. C.

| Patient<br>ID | Visit | Date and Time<br>of Sample | Test Name<br>(unit) | Normal<br>Range | Result<br>[a] |
|---|---|---|---|---|---|
| xxxx-xxx | Screening | ddmonyyyy hh:mm | xxxxxxx (xxx) | xxxx-xxx | Xx H** |
| | | | xxxxxxx (xxx) | xxxx-xxx | xx L* |
| | | | • • • | | |
| | TV3 | ddmonyyyy hh:mm | xxxxxxx (xxx) | xxxx-xxx | Xx L** |
| | | | xxxxxxx (xxx) | xxxx-xxx | xx H* |
| | OV3 | | | | |
| | Followup | | | | |

xxxx-xxx

. . .

Programmer note: Please display all values for the parameter if there is at least one PCS or PCSC for the parameter  $\alpha$ 

Continue with CVT-301 (002/003), CVT-301 (Naïve)

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Na $\"{\text{Na}}$ ve is for the CVT-301 naive patients.

 $L^*$  = potentially clinically significant (PCS) low value,  $H^*$  = PCS high value,

 $L^{**}$  = potentially clinically significant change (PCSC) low,  $H^{**}$  = PCSC high.

Cross-reference: Listing 16.2.8.1.1

Table below will have same format as T14.3.4.1.1.1

Table 14.3.4.1.2.1 Summary of Clinical Laboratory Results: Chemistry (Safety Population)

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Baseline is defined as the TV1/OV1 assessment. If the TV1/OV1 assessment is missing, the last non-missing screening assessment will be used as baseline.

Cross-reference: Listing 16.2.8.1.2

Table below will have same format as T14.3.4.1.1.2 with revised cross reference

Table 14.3.4.1.2.2

Summary of Clinical Laboratory Results: Chemistry Abnormal Values (Safety Population)

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Percentages are based on n, the number of subjects with the test performed at each visit.

Cross-reference: Listing 16.2.8.1.2, Table 14.3.4.1.2.6

Table below will have same format as T14.3.4.1.1.3 with revised cross reference

Table 14.3.4.1.2.3

Summary of Clinical Laboratory Results: Chemistry Abnormal Values -Shift from Baseline (Safety Population)

Cross-reference: Listing 16.2.8.1.2, Table 14.3.4.1.2.6

Table below will have same format as T14.3.4.1.1.4with revised cross reference

Table 14.3.4.1.2.4

Summary of Clinical Laboratory Results: Chemistry PCS Values -Shift from Baseline (Safety Population)

Cross-reference: Listing 16.2.8.1.2, Table 14.3.4.1.2.6

Table below will have same format as T14.3.4.1.1.5with revised cross reference

Table 14.3.4.1.2.5

Summary of Clinical Laboratory Results: Chemistry PCSC Values -Shift from Baseline (Safety Population)

Cross-reference: Listing 16.2.8.1.2, Table 14.3.4.1.2.6

Table below will have same format as T14.3.4.1.1.6 with revised cross reference

Table 14.3.4.1.2.6

Clinical Laboratory Results - Chemistry PCS and PCSC Values (Safety Population)

Cross-reference: Listing 16.2.8.1.2

Table 14.3.4.2

Vital Signs: PCS and PCSC Criteria

| Vital Sign Parameters (Units) | Criteria for I | PCS Values (Actual | : (Actual Criteria for PCSC values (Change from Base values *) | |
|---|---|---|---|---|
| | High | Low | Increase | Decrease |
| Pulse rate(bpm) | >120 | <40 | 2x | 0.5x |
| Respiration Rate (brpm) | >32 | <8 | 1.5x | NA |
| SBP (Supine) (mmHg) | >200 | <85 | 1.6x | 0.2x |
| DBP (Supine) (mmHg) | >120 | <40 | 1.2x | 0.2x |

Note: bpm = beats per minute; brpm = breaths per minute; NA = not applicable; SBP = Systolic Blood Pressure; DBP = Diastolic Blood pressure; PCS = potentially clinically significant; PCSC = potentially clinically significant change.

<sup>\*</sup> Baseline values will be used for pre-dose and pre-dose values assessment at each treatment visits. Pre-dose values will be used for corresponding post-dose values assessment.

| | | | | | CVT- 301 | | |
|---|---|---|---|---|---|---|---|
| Parameter (unit) | Visit | Statistic | O. C.<br>(N=xx) | 002/003<br>(N=xx) | Naive<br>(N=xx) | Total<br>(N=xx) | Overal<br>(N=xx) |
| Standard Systolic | | | | | | | |
| Blood Pressure (unit) | Baseline | Actual value | | | | | |
| proce from the came, | 200011110 | n | XX | XX | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X | XX.X | xx.x |
| | | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX |
| | TV2/OV2 Pre-dose | Actual value | | | | | |
| | | n | XX | XX | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X | XX.X | xx.x |
| | | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | Min, Max | xx, xx | XX, XX | xx, xx | xx, xx | XX, X |
| | | Change from Baseli | ne | | | | |
| | | n | XX | XX | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | Min, Max | xx, xx | xx, xx | XX, XX | xx, xx | XX, X |
| | TV3/OV3 Pre-dose | | | | | | |
| | Followup | • • • | | | | | |

Standard Diastolic Blood Pressure (unit)

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naïve patients. The baseline is defined as the TV1/OV1 pre-dose value. If TV1/OV1 pre-dose value is missing, the last non-missing screening assessment will be used as baseline.

Cross-reference: Listing 16.2.8.2.1

Programming Note: Repeat for Standard Diastolic Blood Pressure, Standard Heart Rate, Standard Respiratory Rate, Upright Systolic Blood Pressure, Upright Diastolic Blood Pressure, Upright Heart Rate, Respiration Rate


| Parameter (unit) | Time Point | Statistic | CVT-301<br>(N=xx) |
|---|---|---|---|
| Standard Systolic | | | |
| Blood Pressure (unit) | Pre-dose | Actual value | |
| biood flessure (unit) | ile dose | n | XX |
| | | Mean | XX.X |
| | | SD | XX.XX |
| | | Median | XX.X |
| | | Min, Max | XX, XX |
| | | MIN, MAX | AA, AA |
| | 10 mins Post-dose | Actual value | |
| | | n | XX |
| | | Mean | XX.X |
| | | SD | XX.XX |
| | | Median | XX.X |
| | | Min, Max | XX, XX |
| | | Change from Pre-dose | |
| | | n | XX |
| | | Mean | XX.X |
| | | SD | XX.XX |
| | | Median | XX.X |
| | | Min, Max | XX, XX |
| | ••• | | |
| Standard Diastolic | | | |
| Standard Diastolic<br>Blood Pressure (unit) | | | |
| •• | | | |

Cross-reference: Listing 16.2.8.2.1

Programming Note: Repeat for Standard Diastolic Blood Pressure, Standard Heart Rate, Standard Respiratory Rate, Upright Systolic Blood Pressure, Upright Diastolic Blood Pressure, Upright Heart Rate, Respiration Rate

> Table 14.3.4.2.3 Summary of Standard Vital Signs: PCS and PCSC Values by Visit (Safety Population)

| | | | CVT- 301 | | | |
|---|---|---|---|---|---|---|
| | | O. C. | 002/003 | Naive | Total | Overall |
| | Visit | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Parameter (unit) | Assessment | n (%) | n (%) | n (%) | n (%) | n (%) |
| Standard Systolic | SV1 | | | | | |
| Blood Pressure (unit) | n | XX | xx | xx | XX | XX |
| | PCS Low | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | PCS High | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | PCSC Low | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | PCSC High | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | SV2 | | | | | |
| | n | XX | XX | xx | XX | XX |
| | PCS Low | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | PCS High | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | PCSC Low | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | PCSC High | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | TV1/OV1 Pre-dose | | | | | |
| | n | XX | XX | XX | XX | XX |
| | TV2/OV2 Pre-dose | | | | | |
| | <br>TV3/OV3 Pre-dose | | | | | |
| | ••• | | | | | |
| | Followup | | | | | |
| Standard Diastolic<br>Blood Pressure (unit) | ••• | | | | | |
| Blood Pressure (unit) | | | | | | |

Note: SV = Screening Visit; TV = Treatment Visit; O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Percentages are based on n, the number of subjects with the test performed at each visit. PCS = potentially clinically significant values, PCSC = potentially clinically significant changes.

Cross-reference: Listing 16.2.8.2.1, Table 14.3.4.2.5

Programming Note: Repeat for Standard Diastolic Blood Pressure, Standard Heart Rate, Standard Respiratory Rate. Only visits with any PCS or PCSC values are included.

Table 14.3.4.2.4

Summary of Standard Vital Signs: PCS and PCSC Values by Scheduled Timepoint at TV1 (Safety Population)

| | | CVT- 301 |
|------------------------|-------------------|-----------|
| | Timepoint | (N=xx) |
| Parameter (unit) | Assessment | n (%) |
| Standard Systolic | Pre-dose | |
| Blood Pressure (unit) | n | xx |
| siood flessale (diffe) | PCS Low | xx (xx.x) |
| | PCS High | xx (xx.x) |
| | PCSC Low | xx (xx.x) |
| | PCSC High | xx (xx.x) |
| | 10 mins post-dose | |
| | n | XX |
| | PCS Low | xx (xx.x) |
| | PCS High | xx (xx.x) |
| | PCSC Low | xx (xx.x) |
| | PCSC High | xx (xx.x) |
| | 20 mins post-dose | |
| | n | XX |
| | | **** |
| | 30 mins post-dose | |
| | ••• | |
| | 60 mins post-dose | |
| | ••• | |
| Standard Diastolic | | |
| Blood Pressure (unit) | | |
| •• | | |

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients.

Percentages are based on n, the number of subjects with the test performed at each visit.

PCS = potentially clinically significant values, PCSC = potentially clinically significant changes.

Cross-reference: Listing 16.2.8.2.1, Table 14.3.4.2.5

Programming Note: Repeat for Standard Diastolic Blood Pressure, Standard Heart Rate, Standard Respiratory Rate. Only visits with any PCS or PCSC values are included.
Table 14.3.4.2.5 Standard Vital Signs: PCS and PCSC Values

Treatment Group: O. C.

| | | | | | | Blood P<br>(mm | | | |
|---|---|---|---|---|---|---|---|---|---|
| Patient<br>ID | Visit | Time Point | Date<br>Performed | Time<br>Performed | Position | SBP | BBP DBP | Heart Rate<br>(Beats/Min) | Respiratory Rate<br>(Breaths/Min) |
| | | | | hh:mm | SUPINE/SEMI- | xx | | | |
| XXXX-XXX | Screening | | ddmonyyyy | | SUPINE | | XX | XX | xx |
| | | | | hh:mm | STANDING | XX | Xx H | XX | XX |
| | | Pre-dose | | hh:mm | SUPINE/SEMI- | xx L** | | | |
| | TV3/OV3 | | ddmonyyyy | | SUPINE | | XX | XX | XX |
| | | | | hh:mm | STANDING | xx L* | XX | XX | XX |

. . .

xxxx-xxx

CVT-301 (002/003) CVT-301(Naïve) CVT-301 Total

Programmer note: Please display all related values if there is one Orthostatic Hypertension Data

Note: SV = Screening Visit; TV = Treatment Visit; O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. L\* = potentially clinically significant (PCS) low value,  $H^* = PCS$  high value,  $L^{**}$  = potentially clinically significant change (PCSC) low,  $H^{**}$  = PCSC high.

Table 14.3.4.2.6

Summary of Vital Signs: Orthostatic Hypotension by Visit (Safety Population)

| | | | CVT- 301 | | |
|------------------|-----------|-----------|-----------|-----------|-----------|
| | O. C. | 002/003 | Naive | Total | Overall |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Visit | n (%) | n (%) | n (%) | n (%) | n (%) |
| SV1 | | | | | |
| n | XX | xx | XX | xx | XX |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SV2 | | | | | |
| n | XX | xx | XX | XX | XX |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TV1/OV1 Pre-dose | | | | | |
| n | XX | xx | XX | XX | XX |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TV2/OV2 Pre-dose | | | | | |
| TV3/OV3 Pre-dose | | | | | |
| ••• | | | | | |
| <br>Pallanna | | | | | |
| Followup | | | | | |
| • • • | | | | | |

Note: SV = Screening Visit; TV = Treatment Visit; O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Percentages are based on n, the number of subjects with the test performed at each visit.

Orthostatic hypotension is defined as a reduction in SBP of 20 mmHg or more, and/or a reduction in DBP of 10 mmHg or more, for the standing measurement compared to the semi-supine measurement.

Cross-reference: Listing 16.2.8.2.1 and Table 14.3.4.2.8

# Table 14.3.4.2.7 Summary of Vital Signs: Orthostatic Hypotension by Scheduled Timepoint at TV1 (Safety Population)

| | CVT- 301 |
|-------------------|-----------|
| | (N=xx) |
| Timepoint | n (%) |
| Pre-dose | |
| n | xx |
| Yes | xx (xx.x) |
| No | xx (xx.x) |
| 10 mins post-dose | |
| n | XX |
| Yes | xx (xx.x) |
| No | xx (xx.x) |
| 20 mins post-dose | |
| n | XX |
| Yes | xx (xx.x) |
| No | xx (xx.x) |
| 30 mins post-dose | |
| • | |
| 60 mins post-dose | |

Percentages are based on n, the number of subjects with the test performed at each visit. Orthostatic hypotension is defined as a reduction in SBP of 20 mmHg or more, and/or a reduction in DBP of 10 mmHg or more, for the standing measurement compared to the semi-supine measurement.

Cross-reference: Listing 16.2.8.2.1 and Table 14.3.4.2.8

Table 14.3.4.2.8 Orthostatic Vital Signs

Treatment Group: O. C.

| | | | | | | Blood Pressure<br>(mmHg) | | | |
|---|---|---|---|---|---|---|---|---|---|
| Patient<br>ID | Visit | Time Point | Date<br>Performed | Time<br>Performed | Position | SBP | DBP | Heart Rate<br>(Beats/Min) | Respiratory Rate (Breaths/Min) |
| | | | | hh:mm | SUPINE/SEMI- | xx | | | |
| xxxx-xxx | Screening | | ddmonyyyy | | SUPINE | | XX | XX | XX |
| | | | | hh:mm | STANDING * | XX | XX | XX | XX |
| | | Pre-dose | | hh:mm | SUPINE/SEMI- | XX | | | |
| | Visit 3 | | ddmonyyyy | | SUPINE | | XX | XX | XX |
| | | | | hh:mm | STANDING * | XX | XX | XX | XX |

. . .

xxxx-xxx

CVT-301 (002/003)

CVT-301(Naïve)

CVT-301 Total

Programmer note: Please display all related values if there is one Orthostatic Hypertension Data

Note: SV = Screening Visit; TV=Treatment Visit; FU= Follow-up; UNS= unscheduled; O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients.

<sup>\*</sup> denotes orthostatic hypotension that is defined as a reduction in SBP of 20 mmHg or more, and/or a reduction in DBP of 10 mmHg or more, for the standing measurement compared to the Semi-supine measurement. Cross-reference: Listing 16.2.8.2.1

# Table 14.3.4.3 12-Lead ECG:PCS and PCSC Criteria

| ECG Parameters(Units) | Criteria for PCS Values (Actual values) | | Criteria for PCSC values (Change from 1 | Baseline or pre-dose values *) |
|---|---|---|---|---|
| | High | Low | Increase | Decrease |
| PR interval (msec) | >300 | NA | >25% for baseline >=200 | NA |
| | | | >50% for baseline <200 | |
| QRS interval (msec) | >200 | NA | >25% for baseline >=100 | NA |
| | | | >50% for baseline <100 | |
| QTcB (msec) | >500 | NA | >15% for baseline >=440 | NA |
| | | | >30% for baseline <440 | |
| QTcF (msec) | >500 | NA | >15% for baseline >=440 | NA |
| | | | >30% for baseline <440 | |
| Heart Rate (bpm) | >120 | <35 | NA | NA |

Note: bpm = beats per minute; msec = Micro Second; NA = not applicable; SBP = Systolic Blood Pressure; DBP = Diastolic Blood Pressure; PCS = potentially clinically significant; PCSC = potentially clinically significant change.

<sup>\*</sup> Baseline values will be used for pre-dose and pre-dose values assessment at each treatment visits. Pre-dose values will be used for corresponding post-dose values assessment.

Table 14.3.4.3.1 Summary of 12-Lead ECG: Actual Values and Change across Visits (Safety Population)

| | | | | | CVT- 301 | | |
|---|---|---|---|---|---|---|---|
| Parameter (unit) | Visit | Statistic | O. C.<br>(N=xx) | 002/003<br>(N=xx) | Naive<br>(N=xx) | Total<br>(N=xx) | Overall<br>(N=xx) |
| PR Interval (unit) | Baseline | Actual value | | | | | |
| , | | n | XX | XX | XX | XX | XX |
| | | Mean | XX.X | xx.x | xx.x | XX.X | XX.X |
| | | SD | XX.XX | xx.xx | XX.XX | XX.XX | xx.xx |
| | | Median | XX.X | xx.x | xx.x | XX.X | XX.X |
| | | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX |
| | TV1/OV1 | Actual value | | | | | |
| | | n | XX | XX | XX | XX | xx |
| | | Mean | XX.X | xx.x | xx.x | XX.X | xx.x |
| | | SD | XX.XX | xx.xx | XX.XX | XX.XX | xx.xx |
| | | Median | XX.X | xx.x | xx.x | XX.X | xx.x |
| | | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX |
| | | Change from Baseline | | | | | |
| | | n | XX | XX | XX | XX | xx |
| | | Mean | XX.X | xx.x | xx.x | XX.X | XX.X |
| | | SD | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx |
| | | Median | XX.X | XX.X | XX.X | XX.X | xx.x |
| | | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX |
| | TV3/OV3 | ••• | | | | | |
| | ••• | | | | | | |

. . .

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. The baseline is defined as the TV1/OV1 pre-dose value. If TV1/OV1 pre-dose value is missing, the last non-missing screening assessment will be used as baseline.

Cross-reference: Listing 16.2.8.2.2

Programming Note: Repeat for other ECG parameters.

# Table 14.3.4.3.2 Summary of 12-Lead ECG: PCS and PCSC Values (Safety Population)

| | | | | CVT- 301 | | |
|---|---|---|---|---|---|---|
| | Visit | O. C.<br>(N=xx) | 002/003<br>(N=xx) | Naive<br>(N=xx) | Total<br>(N=xx) | Overall (N=xx) |
| Parameter (unit) | Assessment | n (%) | n (%) | n (응) | n (%) | n (%) |
| PR Interval (unit) | TV1/OV1 | | | | | |
| | n | xx | xx | XX | xx | XX |
| | PCS High | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | PCSC High | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | ••• | | | | | |
| | TV3/OV3 | | | | | |

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Percentages are based on n, the number of subjects with the test performed at each visit.

PCS = potentially clinically significant values, PCSC = potentially clinically significant changes.

Cross-reference: Listing 16.2.8.2.2, Table 14.3.4.3.3

Programming Note: For PCS repeat for other applicable ECG parameters (QRS Interval, QTcB, QTcF, Heart Rate). For Heart Rate, both PCS Low and PCS High will be assessed.

For PCSC repeat for other applicable ECG parameters (QRS Interval, QTcB, QTcF). PCSC Low values will not be assessed. Only visits with any PCS or PCSC values are included.

# Protocol No. CVT-301-005 Confidential

Table 14.3.4.3.3
12-Lead Electrocardiogram (ECG): PCS and PCSC Values

Treatment Group: O. C.

| Patient<br>ID | Visit | Time Point | Date and Time<br>Of Assessment | Test (Unit) | Result |
|---|---|---|---|---|---|
| xxxx-xxx | SV1<br>OV3 | Pre-dose<br>+5mins<br>+20mins<br>+30mins | ddmonyyyy hh:mm<br>ddmonyyyy hh:mm | xxx (xxx) | xx H*<br>xx L** |
| | | ••• | | | |

xxxx-xxx

. . .

CVT-301 (002/003)

CVT-301(Naïve)

CVT-301 Total

Programmer note: Please display all values for the parameter if there is at least one PCS or PCSC for the parameter

Note: SV = Screening Visit; TV = Treatment Visit; OV = Observational Cohort; O.C. column is for the patients in Observational Cohort, 002/003 is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients.

Note:  $L^*$  = potentially clinically significant (PCS) low value,  $H^*$  = PCS high value,  $L^{**}$  = potentially clinically significant change (PCSC) low,  $H^{**}$  = PCSC high.


Table 14.3.4.4
Physical Examination
(Safety Population)

| | | | | CVT- 301 | | |
|---|---|---|---|---|---|---|
| | | O. C.<br>(N=xx) | 002/003<br>(N=xx) | Naive<br>(N=xx) | Total<br>(N=xx) | Overall (N=xx) |
| Visit | Assessment | n (%) | n (응) | n (%) | n (%) | n (%) |
| Screening | Any Clinically Significant Abnormal Findings | | | | | |
| <u> </u> | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TV1/OV1 | Any Clinically Significant Abnormal Findings That Are New or Have Worsened | | | | | |
| | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TV2/OV2<br>TV3/OV3 | | | | | | |

Note: SV = Screening Visit; TV = Treatment Visit; OV = Observational Cohort; O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients.

Table 14.3.4.5.1.1 Summary of Spirometry (Neurology Office): Actual Values and Change from Baseline for FEV1 and FVC by Visit (Safety Population)

| | | | <u>_</u> | | CVT- 301 | | <u> </u> |
|---|---|---|---|---|---|---|---|
| Parameter (unit) | Visit | Statistic | O. C.<br>(N=xx) | 002/003<br>(N=xx) | Naive<br>(N=xx) | Total<br>(N=xx) | Overall<br>(N=xx) |
| FEV1 (unit) | Screening (ON state) | Actual value | | | | | |
| | Screening (OFF state) | Actual value | | | | | |
| | TV1/OV1 Arrival | Actual value | | | | | |
| | Baseline | Actual value | | | | | |
| | TV2/OV2 Arrival | Actual value n Mean SD Median Min, Max Change from Baseline Percent Change from Baseline (%) | xx<br>xx.x<br>xx.xx<br>xx.x<br>xx.x | xx<br>xx.x<br>xx.xx<br>xx.x<br>xx.x | xx<br>xx.x<br>xx.xx<br>xx.x<br>xx.x | xx<br>xx.x<br>xx.xx<br>xx.x<br>xx.x | xx<br>xx.x<br>xx.xx<br>xx.x |
| | TV3/OV3 Arrival<br>TV4/OV4 Arrival<br>TV5/OV5 Arrival<br>TV6/OV6 Arrival | ::: | | | | | |

Percentage Predicted FVC

Note: SV = Screening Visit; TV = Treatment Visit; OV = Observational Visit; O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Screening is the latest assessment during screening period. Baseline is defined as the TV1/OV1 arrival value. If the TV1/OV1 arrival value is missing, the last available value in ON state before the first dose of study drug is used.

Cross-reference: Listing 16.2.8.2.4.1

Programming Note: Repeat for Percentage predicted FEV1, FVC, Percentage predicted FVC. No need to summarize percent change for Predicted FEV1 and Predicted FVC.

Table 14.3.4.5.1.2

Summary of Spirometry (Neurology Office): Actual Values and Change from Baseline for FEV1 and FVC by Visit Using Subset of Assessments Meeting the ATS Quality Criteria (Safety Population)

Table 14.3.4.5.1.3

Summary of Spirometry (Neurology Office): Actual Values and Change from Baseline for FEV1 and FVC by Visit Excluding Patients with Co-efficient of Variation (CV) of FEV1 >7.5% (Safety Population)

Note: SV = Screening Visit; TV = Treatment Visit; OV = Observational Visit; O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Screening is the latest assessment during screening period. Baseline is defined as the TV1/OV1 arrival value. If the TV1/OV1 arrival value is missing, the last available value in ON state before the first dose of study drug is used. The CV will be calculated for each patient as standard deviation divided by the mean. The screening visit FEV1 data (assessed in ON state) and arrival values at subsequent visits will be used for the calculation.

Cross-reference: Listing 16.2.8.2.4.1

Programming Note: Repeat for Percentage predicted FEV1, FVC, Percentage predicted FVC. No need to summarize percent change for Predicted FEV1 and Predicted FVC.

Table 14.3.4.5.1.4 MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for FEV1 by Visit (Safety Population)

| Visit | Statistic | O. C.<br>(N=xx) | CVT-301<br>(N=xx) | n-walue |
|---|---|---|---|---|
| VISIL | Statistic | (IV-XX) | (N-XX) | p-value |
| Overall | Overall p-value | | | |
| | Baseline Hoehn and Yahr stage | | | 0.xxx |
| | Screening Spirometry | | | 0.xxx |
| | Treatment | | | 0.xxx |
| | Visit | | | 0.xxx |
| | Treatment-by-Visit Interaction | | | 0.xxx |
| | Baseline Spirometry | | | 0.xxx |
| TV2/OV2 | n | xx | XX | |
| | LS Mean | XX.X | xx.x | |
| | SE (LS Mean) | XX.XX | xx.xx | |
| | 95% CI (LS Mean) | (xx.x, xx.x) | (xx.x, xx.x) | |
| | LS Mean Difference (CVT-301 - O. C.) | | XX.X | |
| | 95% CI (LS Mean Difference) | | (xx.x, xx.x) | |
| | p-value (LS Mean Difference) | | 0.xxx | |
| TV3/OV3 | | | | |
| TV4/OV4 | | | | |
| TV5/OV5 | | | | |
| TV6/OV6 | | | | |

Note: TV = Treatment Visit; OV = Observational Visit. O.C. column is for the patients in Observational Cohort. MMRM model uses the Change from baseline for FEV1 at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes the treatment group (CVT-301 or O.C.), visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus ≥2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1 ≥60% and FEV1/FVC ratio ≥70%)) and the interaction between the treatment group and visit as fixed factors. Baseline FEV1 will be included as a covariate, assuming an unstructured covariance matrix. Cross-reference: Listing 16.2.8.2.4.1


#### Table 14.3.4.5.1.5

MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for FEV1 by Visit
Using Subset of Assessments Meeting the ATS Quality Criteria
(Safety Population)

### Table 14.3.4.5.1.6

MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for FEV1 by Visit Excluding Patients with Co-efficient of Variation (CV) of FEV1 >7.5% (Safety Population)

Note: TV = Treatment Visit; OV = Observational Visit. O.C. column is for the patients in Observational Cohort. The CV will be calculated for each patient as standard deviation divided by the mean. The screening visit FEV1 data (assessed in ON state) and arrival values at subsequent visits will be used for the calculation.

MMRM model uses the Change from baseline for FEV1 at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes the treatment group (CVT-301 or O.C.), visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus  $\geq$ 2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1  $\geq$ 60% and FEV1/FVC ratio  $\geq$ 70%)) and the interaction between the treatment group and visit as fixed factors. Baseline FEV1 will be included as a covariate, assuming an unstructured covariance matrix.

Table 14.3.4.5.1.7 Sensitivity Analysis Using MMRM: Change from Baseline for FEV1 by Visit MI analysis with Missing At Random Assumption (Safety Population)

| Visit/Statistic | O. C.<br>(N=xx) | CVT-301<br>(N=xx) |
|---|---|---|
| TV2/OV2 | | |
| MI mean (SE) | xx.xx(x.xxx) | xx.xx(x.xxx) |
| MI Treatment Difference in Mean Change from Baseline (SE) | | xx.xx(x.xxx) |
| 95% CI (MI Treatment Difference) | | (xx.xx, xx.xx) |
| P-Value | | 0.xxx |
| TV3/OV3 | | |
| TV4/OV4 | | |
| TV5/OV5 | | |
| TV6/OV6 | | |

Note: TV = Treatment Visit; OV = Observational Visit. O.C. column is for the patients in Observational Cohort. The non-monotone missing values will be imputed using the Markov Chain Monte Carlo (MCMC) methodology which assumes a multivariate normal distribution over all variables included in the imputation model. The monotone missing values are imputed using pattern mixture model assuming missing At Random. MMRM model uses the Change from baseline for FEV1 at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes the treatment group (CVT-301 or O.C.), visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus ≥2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1 ≥60% and FEV1/FVC ratio ≥70%)) and the interaction between the treatment group and visit as fixed factors. Baseline FEV1 will be included as a covariate, assuming an unstructured covariance matrix. The MIANALYZE procedure in SAS will be applied to combine the results from these datasets to derive an overall estimate of the treatment difference at each visit.


Table 14.3.4.5.1.8

MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for Percentage Predicted FEV1 by Visit (Safety Population)

Note: TV = Treatment Visit; OV = Observational Visit. O.C. column is for the patients in Observational Cohort. MMRM model uses the Change from baseline for percentage predicted FEV1 at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes the treatment group (CVT-301 or O.C.), visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus ≥2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1 ≥60% and FEV1/FVC ratio ≥70%)) and the interaction between the treatment group and visit as fixed factors; Baseline Percentage predicted FEV1 will be included as a covariate, assuming an unstructured covariance matrix. Cross-reference: Listing 16.2.8.2.4.1

Table 14.3.4.5.1.9

MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for Percentage Predicted FEV1 by Visit Using Subset of Assessments Meeting the ATS Quality Criteria (Safety Population)

Note: TV = Treatment Visit; OV = Observational Visit. O.C. column is for the patients in Observational Cohort. MMRM model uses the Change from baseline for percentage predicted FEV1 at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes the treatment group (CVT-301 or O.C.), visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus ≥2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1 ≥60% and FEV1/FVC ratio ≥70%)) and the interaction between the treatment group and visit as fixed factors; Baseline Percentage predicted FEV1 will be included as a covariate, assuming an unstructured covariance matrix. Cross-reference: Listing 16.2.8.2.4.1

Table 14.3.4.5.1.10

MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for Percentage Predicted FEV1 by Visit Excluding Patients with Co-efficient of Variation (CV) of FEV1 >7.5% (Safety Population)

Note: TV = Treatment Visit; OV = Observational Visit. O.C. column is for the patients in Observational Cohort. The CV will be calculated for each patient as standard deviation divided by the mean. The screening visit FEV1 data (assessed in ON state) and arrival values at subsequent visits will be used for the calculation.

MMRM model uses the Change from baseline for percentage predicted FEV1 at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes the treatment group (CVT-301 or O.C.), visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus ≥2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1 ≥60% and FEV1/FVC ratio ≥70%)) and the interaction between the treatment group and visit as fixed factors; Baseline Percentage predicted FEV1 will be included as a covariate, assuming an unstructured covariance matrix. Cross-reference: Listing 16.2.8.2.4.1

Table 14.3.4.5.1.11

Sensitivity Analysis Using MMRM: Change from Baseline for Percentage Predicted FEV1 by Visit MI analysis with Missing At Random Assumption (Safety Population)

Note: TV = Treatment Visit; OV = Observational Visit. O.C. column is for the patients in Observational Cohort. The non-monotone missing values will be imputed using the Markov Chain Monte Carlo (MCMC) methodology which assumes a multivariate normal distribution over all variables included in the imputation model. The monotone missing values are imputed using pattern mixture model assuming missing At Random. MMRM model uses the change from baseline for percentage predicted FEV1 at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes the treatment group (CVT-301 or O.C.), visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus ≥2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1 ≥60% and FEV1/FVC ratio ≥70%)) and the interaction between the treatment group and visit as fixed factors. Baseline percentage predicted FEV1 will be included as a covariate, assuming an unstructured covariance matrix. The MIANALYZE procedure in SAS will be applied to combine the results from these datasets to derive an overall estimate of the treatment difference at each visit.

Cross-reference: Listing 16.2.8.2.4.1

Table 14.3.4.5.1.12 MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for FVC by Visit (Safety Population)

Note: TV = Treatment Visit; OV = Observational Visit. O.C. column is for the patients in Observational Cohort. MMRM model uses the Change from Baseline for FVC at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes the treatment group (CVT-301 or O.C.), visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus ≥2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1 ≥60% and FEV1/FVC ratio ≥70%)) and the interaction between the treatment group and visit as fixed factors; Baseline FVC will be included as a covariate, assuming an unstructured covariance matrix. Cross-reference: Listing 16.2.8.2.4.1

Table 14.3.4.5.1.13

MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for FVC by Visit Using Subset of Assessments Meeting the ATS Quality Criteria (Safety Population)

Note: TV = Treatment Visit; OV = Observational Visit. O.C. column is for the patients in Observational Cohort. MMRM model uses the Change from Baseline for FVC at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes the treatment group (CVT-301 or O.C.), visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus ≥2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1 ≥60% and FEV1/FVC ratio ≥70%)) and the interaction between the treatment group and visit as fixed factors; Baseline FVC will be included as a covariate, assuming an unstructured covariance matrix. Cross-reference: Listing 16.2.8.2.4.1

Table 14.3.4.5.1.14

MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for FVC by Visit Excluding Patients with Co-efficient of Variation (CV) of FEV1 >7.5% (Safety Population)


Note: TV = Treatment Visit; OV = Observational Visit. O.C. column is for the patients in Observational Cohort. The CV will be calculated for each patient as standard deviation divided by the mean. The screening visit FEV1 data (assessed in ON state) and arrival values at subsequent visits will be used for the calculation.

MMRM model uses the Change from Baseline for FVC at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes the treatment group (CVT-301 or O.C.), visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus ≥2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1 ≥60% and FEV1/FVC ratio ≥70%)) and the interaction between the treatment group and visit as fixed factors; Baseline FVC will be included as a covariate, assuming an unstructured covariance matrix.

Page x of y

Cross-reference: Listing 16.2.8.2.4.1

Table 14.3.4.5.1.15

Sensitivity Analysis Using MMRM: Change from Baseline for FVC by Visit MI analysis with Missing At Random Assumption (Safety Population)

Note: TV = Treatment Visit; OV = Observational Visit. O.C. column is for the patients in Observational Cohort. The non-monotone missing values will be imputed using the Markov Chain Monte Carlo (MCMC) methodology which assumes a multivariate normal distribution over all variables included in the imputation model. The monotone missing values are imputed using pattern mixture model assuming missing At Random. MMRM model uses the change from baseline for FVC at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes the treatment group (CVT-301 or O.C.), visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus ≥2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1 ≥60% and FEV1/FVC ratio ≥70%)) and the interaction between the treatment group and visit as fixed factors. Baseline FVC will be included as a covariate, assuming an unstructured covariance matrix. The MIANALYZE procedure in SAS will be applied to combine the results from these datasets to derive an overall estimate of the treatment difference at each visit.

Cross-reference: Listing 16.2.8.2.4.1

Table 14.3.4.5.1.16

MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for Percentage Predicted FVC by Visit (Safety Population)

Note: TV = Treatment Visit; OV = Observational Visit. O.C. column is for the patients in Observational Cohort. MMRM model uses the change from baseline for percentage predicted FVC at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes the treatment group (CVT-301 or O.C.), visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus ≥2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1 ≥60% and FEV1/FVC ratio ≥70%)) and the interaction between the treatment group and visit as fixed factors; Baseline percentage predicted FVC will be included as a covariate, assuming an unstructured covariance matrix. Cross-reference: Listing 16.2.8.2.4.1

Will use format for 14.3.4.5.1.2

Table 14.3.4.5.1.17

MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for Percentage Predicted FVC by Visit Using Subset of Assessments Meeting the ATS Quality Criteria (Safety Population)

Note: TV = Treatment Visit; OV = Observational Visit. O.C. column is for the patients in Observational Cohort. MMRM model uses the change from baseline for percentage predicted FVC at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes the treatment group (CVT-301 or O.C.), visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus ≥2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70%


versus FEV1  $\geq$ 60% and FEV1/FVC ratio  $\geq$ 70%)) and the interaction between the treatment group and visit as fixed factors; Baseline percentage predicted FVC will be included as a covariate, assuming an unstructured covariance matrix. Cross-reference: Listing 16.2.8.2.4.1 Will use format for 14.3.4.5.1.2

Table 14.3.4.5.1.18

MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for Percentage Predicted FVC by Visit

Excluding Patients with Co-efficient of Variation (CV) of FEV1 >7.5%

(Safety Population)

Note: TV = Treatment Visit; OV = Observational Visit. O.C. column is for the patients in Observational Cohort. The CV will be calculated for each patient as standard deviation divided by the mean. The screening visit FEV1 data (assessed in ON state) and arrival values at subsequent visits will be used for the calculation.

MMRM model uses the change from baseline for percentage predicted FVC at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes the treatment group (CVT-301 or 0.C.), visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus  $\ge$ 2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1  $\ge$ 60% and FEV1/FVC ratio  $\ge$ 70%)) and the interaction between the treatment group and visit as fixed factors; Baseline percentage predicted FVC will be included as a covariate, assuming an unstructured covariance matrix.

Cross-reference: Listing 16.2.8.2.4.1 Will use format for 14.3.4.5.1.2

Table 14.3.4.5.1.19

Sensitivity Analysis Using MMRM: Change from Baseline for Percentage Predicted FVC by Visit
MI analysis with Missing At Random Assumption
(Safety Population)

Note: TV = Treatment Visit; OV = Observational Visit. O.C. column is for the patients in Observational Cohort. The non-monotone missing values will be imputed using the Markov Chain Monte Carlo (MCMC) methodology which assumes a multivariate normal distribution over all variables included in the imputation model. The monotone missing values are imputed using pattern mixture model assuming missing At Random. MMRM model uses the change from Baseline for percentage predicted FVC at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes the treatment group (CVT-301 or 0.C.), visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus <2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1 <60% and FEV1/FVC ratio <70%)) and the interaction between the treatment group and visit as fixed factors. Baseline percentage predicted FVC will be included as a covariate, assuming an unstructured covariance matrix. The MIANALYZE procedure in SAS will be applied to combine the results from these datasets to derive an overall estimate of the treatment difference at each visit.

Cross-reference: Listing 16.2.8.2.4.1

Will use format for Table 14.3.4.5.1.2 and Table 14.3.4.5.1.3 respectively.

Table 14.3.4.5.2.1

Summary of Spirometry : ( Neurology Office): Actual Values and Change from Baseline for FEV1/FVC by Visit (Safety Population)

| | | | | CVT- 301 | | |
|---|---|---|---|---|---|---|
| Visit | Statistic | O. C.<br>(N=xx) | 002/003<br>(N=xx) | Naive<br>(N=xx) | Total<br>(N=xx) | Overall<br>(N=xx) |
| Screening (ON state) | Actual value | | | | | |
| soluting (on souse, | n | xx | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx |
| Screening (OFF state) | | | | | | |
| TV1/OV1 Arrival | | | | | | |
| Baseline | | | | | | |
| TV2/OV2 Arrival | Actual value | | | | | |
| | n | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX |
| | Change from Baseline | | | | | |
| | Percent Change from Baseline | | | | | |
| TV3/OV3 Arrival<br>TV4/OV4 Arrival<br>TV5/OV5 Arrival<br>TV6/OV6 Arrival | | | | | | |

SV = Screening Visit; TV = Treatment Visit; OV = Observational Cohort; O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Screening is the latest assessment during screening period. Baseline is defined as the TV1/OV1 arrival value. If the TV1/OV1 arrival value is missing, the last available value in ON state before the first dose of study drug is used.

Civitas Therapeutics, Inc.

Page x of y


Table 14.3.4.5.2.2

Summary of Spirometry : ( Neurology Office): Actual Values and Change from Baseline for FEV1/FVC by Visit
Using Subset of Assessments Meeting the ATS Quality Criteria
(Safety Population)

Table 14.3.4.5.2.3

Summary of Spirometry : ( Neurology Office): Actual Values and Change from Baseline for FEV1/FVC by Visit Excluding Patients with Co-efficient of Variation (CV) of FEV1 >7.5% (Safety Population)

Table 14.3.4.5.2.4

MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for FEV1/FVC by Visit (Safety Population)

Note: TV = Treatment Visit; OV = Observational Visit. O.C. column is for the patients in Observational Cohort. MMRM model uses the change from baseline for FEV1/FVC at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes the treatment group (CVT-301 or O.C.), visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus  $\geq$ 2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1  $\geq$ 60% and FEV1/FVC ratio  $\geq$ 70%)) and the interaction between the treatment group and visit as fixed factors; Baseline FEV1/FVC will be included as a covariate, assuming an unstructured covariance matrix.

#### Will use format for table 14.3.4.5.1.2

Table 14.3.4.5.2.5

MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for FEV1/FVC by Visit
Using Subset of Assessments Meeting the ATS Quality Criteria
(Safety Population)

Note: TV = Treatment Visit; OV = Observational Visit. O.C. column is for the patients in Observational Cohort.

MMRM model uses the change from baseline for FEV1/FVC at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes the treatment group (CVT-301 or O.C.), visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus  $\ge$ 2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1  $\ge$ 60% and FEV1/FVC ratio  $\ge$ 70%)) and the interaction between the treatment group and visit as fixed factors; Baseline FEV1/FVC will be included as a covariate, assuming an unstructured covariance matrix.

#### Will use format for table 14.3.4.5.1.2

Table 14.3.4.5.2.6

MMRM Analysis of Spirometry Data (Neurology Office): Change from Baseline for FEV1/FVC by Visit Excluding Patients with Co-efficient of Variation (CV) of FEV1 >7.5% (Safety Population)

Note: TV = Treatment Visit; OV = Observational Visit. O.C. column is for the patients in Observational Cohort. The CV will be calculated for each patient as standard deviation divided by the mean. The screening visit FEV1 data (assessed in ON state) and arrival values at subsequent visits will be used for the calculation.

MMRM model uses the change from baseline for FEV1/FVC at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes the treatment group (CVT-301 or 0.C.), visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus  $\geq$ 2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1  $\geq$ 60% and FEV1/FVC ratio  $\geq$ 70%)) and the interaction between the treatment group and visit as fixed factors; Baseline FEV1/FVC will be included as a covariate, assuming an unstructured covariance matrix.

Will use format for table 14.3.4.5.1.2

Table 14.3.4.5.2.7

Sensitivity Analysis Using MMRM: Change from Baseline for FEV1/FVC by Visit

MI analysis with Missing At Random Assumption

(Safety Population)

Note: TV = Treatment Visit; OV = Observational Visit

The non-monotone missing values will be imputed using the Markov Chain Monte Carlo (MCMC) methodology which assumes a multivariate normal distribution over all variables included in the imputation model. The monotone missing values are imputed using pattern mixture model assuming missing At Random. MMRM model uses the change from baseline for **FEV1/FVC** at each post-baseline visit (TV2, TV3, TV4, TV5, TV6) as the dependent variable, and includes the treatment group (CVT-301 or 0.C.), visit (TV2, TV3, TV4, TV5, TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus  $\ge2.5$ ) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1  $\ge60\%$  and FEV1/FVC ratio  $\ge70\%$ )) and the interaction between the treatment group and visit as fixed factors. Baseline FEV1/FVC will be included as a covariate, assuming an unstructured covariance matrix. The MIANALYZE procedure in SAS will be applied to combine the results from these datasets to derive an overall estimate of the treatment difference at each visit.

Cross-reference: Listing 16.2.8.2.4.1

Will use format for table 14.3.4.5.1.3

Table 14.3.4.5.3.1 Summary of Spirometry (Neurology Office): Summary of FEV1/FVC < 60% and <70% by Visit (Safety Population)

| | | | | CVT- 301 | | |
|---|---|---|---|---|---|---|
| Category/Visit | Statistic | O. C.<br>(N=xx) | 002/003<br>(N=xx) | Naive<br>(N=xx) | Total<br>(N=xx) | Overall (N=xx) |
| FEV1/FVC < 60% | | | | | | |
| Screening (ON state) | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Screening (OFF state) | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TV1/OV1 Arrival | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Baseline | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TV2/OV2 Arrival | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| • • • | | | | | | |
| FEV1/FVC < 70% | | | | | | |
| Screening (ON state) | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Screening (OFF state) | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TV1/OV1 Arrival | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Baseline | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TV2/OV2 Arrival | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: SV = Screening Visit; TV = Treatment Visit; OV = Observational Visit; O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Screening is the latest assessment during screening period. Baseline is defined as the TV1/OV1 arrival value. If the TV1/OV1 arrival value is missing, the last available value in ON state before the first dose of study drug is used.

Cross-reference: Listing 16.2.8.2.4.1, Table 14.3.4.5.8

Table 14.3.4.5.3.2

Summary of Spirometry (Neurology Office): Summary of FEV1/FVC < 60% and <70% by Visit Using Subset of Assessments Meeting the ATS Quality Criteria (Safety Population)

Table 14.3.4.5.3.3

Summary of Spirometry (Neurology Office): Summary of FEV1/FVC < 60% and <70% by Visit Excluding Patients with Co-efficient of Variation (CV) of FEV1 >7.5% (Safety Population)

Note: SV = Screening Visit; TV = Treatment Visit; OV = Observational Visit; O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Screening is the latest assessment during screening period. Baseline is defined as the TV1/OV1 arrival value. If the TV1/OV1 arrival value is missing, the last available value in ON state before the first dose of study drug is used. The CV will be calculated for each patient as standard deviation divided by the mean. The screening visit FEV1 data (assessed in ON state) and arrival values at subsequent visits will be used for the calculation. Cross-reference: Listing 16.2.8.2.4.1, Table 14.3.4.5.8


# 

Treatment Group: CVT-301 (002/003)

| Patient<br>ID | Visit | Time<br>Point | Motor<br>State | Date and Time<br>of Assessment | Test (Unit) | Result |
|---|---|---|---|---|---|---|
| xxxx-xxx@ | TV2 | Pre-dose<br>Pre-dose | ON<br>ON | ddmonyyyy hh:mm ddmonyyyy hh:mm # | xxx (xxx) | Xx*<br>Xx \$ |
| | TV3 | rie-dose | ON | danonyyyy mi:nun # | xxx (xxx) | XX Ş |

#### XXXX-XXX

Programmer note: please display all FEV1, FVC and FEV1/FVC from all timepoint if any criteria meet.

# Continue with CVT-301 (Naïve)

Note: TV = Treatment Visit;

# indicates spirometry measurement not meeting ATS quality criteria. \* indicates imputed values. \$ indicates manual data @ indicates patients with Co-efficient of Variation (CV) of FEV1 >7.5%

Data with 70% or smaller FEV1/FVC Values at each timepoint/visit are included.

| | | | | _ | | |
|---|---|---|---|---|---|---|
| State | Statistic | O. C.<br>(N=xx) | 002/003<br>(N=xx) | Naive<br>(N=xx) | Total<br>(N=xx) | Overall<br>(N=xx) |
| State | Statistic | (IV-XX) | (IN-XX) | (IV-XX) | (N-XX) | (N-XX) |
| Overall | | | | | | |
| Total Number of Spirometry Measurements | n | XX | XXX | XXX | XXX | XX |
| Total Number (Percent) of Measurements | | | | | | |
| Meeting ATS Quality Criteria [a] | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| Total Number (Percent) of Measurements | | | | | | |
| Not Meeting ATS Quality Criteria [a] | n (%) | xx (xx.x) | xx (xx.x | xx (xx.x | xx (xx.x | xx (xx.x |
| Reason for Not Meeting ATS Quality Criteria [b] | | | | | | |
| Acceptable Effort of ANY and Repeatable Effort of O | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| Acceptable Effort of 3 and Repeatable Effort of 0 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| Acceptable Effort of 2 and Repeatable Effort of 0 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Acceptable Effort of 1 and Repeatable Effort of 0 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| Acceptable Effort of 0 and Repeatable Effort of 0 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Acceptable Effort of 2 and Repeatable Effort of 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Proportion of Measurements Meeting ATS | | | | | | |
| Quality Criteria at Subject Level[c] | n | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

. . .

OFF State

. . .

Note: O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients.

<sup>[</sup>a] Percent is based on the total number of spirometry measurements.

<sup>[</sup>b] Percent is based on the total number of spirometry measurements not meeting ATS quality criteria.

<sup>[</sup>c] For each subject, the proportion is calculated as spirometry measurements meeting ATS criteria divided by total the count of records with unique assessment date/time and non-missing ATS Quality Criteria Flag.

Cross-reference: Listing 16.2.8.2.4.1, Listing 16.2.8.2.4.3

Table 14.3.4.5.6

Summary of Spirometry (Pulmonary Function Facility): Actual Values and Change from Baseline for Calculated DLco Parameters by Visit (Safety Population)

| | | | _ | | CVT-301 | | |
|---|---|---|---|---|---|---|---|
| Parameter (unit) | Visit | Statistic | O. C.<br>(N=xx) | 002/003<br>(N=xx) | Naive<br>(N=xx) | Total<br>(N=xx) | Overall (N=xx) |
| Discount distant (solt) | D 1 / | Patrick and the second | | | | | |
| DLco predicted (unit) | Baseline | Actual value | | | | | |
| | | n | XX | XX | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| | TV2/OV2 | Actual value | | | | | |
| | | n | XX | XX | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | Median | xx.x | XX.X | XX.X | xx.x | xx.x |
| | | Min, Max | xx, xx | xx, xx | xx, xx | XX, XX | xx, xx |
| | | Change from Baseline | | | | | |
| | | Percent Change from Baseline (%) | | | | | |
| | TV4/OV4<br>TV5/OV5<br>TV6/OV6 | | | | | | |

# Continue with all Applicable Calculated Parameters

Note: TV = Treatment Visit; OV = Observational Visit. O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. The baseline is defined as the DLco results taken after SV2 and before randomization.

Table 14.3.4.5.7

Summary of Spirometry (Pulmonary Function Facility): Actual Values and Change from Baseline for FEV1 and FVC by Visit (Safety Population)

| | | | | | CVT- 301 | | |
|---|---|---|---|---|---|---|---|
| Parameter (unit) | Visit | Statistic | O. C.<br>(N=xx) | 002/003<br>(N=xx) | Naive<br>(N=xx) | Total<br>(N=xx) | Overall (N=xx) |
| FEV1 (unit) | Baseline | Actual value | | | | | |
| | | n | XX | XX | XX | XX | XX |
| | | Mean | xx.x | XX.X | XX.X | XX.X | xx.x |
| | | SD | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx |
| | | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| | TV2/OV2 | Actual value | | | | | |
| | | n | XX | XX | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | Min, Max | XX, XX | XX, XX | XX, XX | xx, xx | xx, xx |
| | | Change from Baseline | | | | | |
| | | Percent Change from Baseline (%) | | | | | |
| | TV4/OV4 | | | | | | |
| | TV5/OV5 | | | | | | |
| | TV6/OV6 | | | | | | |

# Continue with all Applicable Parameters

Note: TV = Treatment Visit; OV = Observational Visit. O.C. column is for the patients in Observational Cohort, OOZ/OO3 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients.

The baseline is defined as the DLco results taken after SV2 and before randomization.

Table 14.3.4.5.8

Summary of Spirometry (Pulmonary Function Facility): Actual Values and Change from Baseline for FEV1/FVC by Visit (Safety Population)

| Parameter (unit) | Visit | Statistic | O. C.<br>(N=xx) | 002/003<br>(N=xx) | Naive<br>(N=xx) | Total<br>(N=xx) | Overall<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| FEV1/FVC(unit) | Baseline | Actual value | | | | | |
| , | | n | XX | XX | XX | XX | XX |
| | | Mean | xx.x | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | Min, Max | xx, xx | xx, xx | XX, XX | XX, XX | XX, XX |
| | TV2/OV2 Actual value | Actual value | | | | | |
| | | n | XX | XX | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | Min, Max | xx, xx | xx, xx | XX, XX | XX, XX | xx, xx |
| | | Change from Baseline | | | | | |
| | | Percent Change from Baseline (%) | | | | | |
| | TV4/OV4 | | | | | | |
| | TV5/OV5 | | | | | | |
| | TV6/OV6 | | | | | | |

Note: TV = Treatment Visit; OV = Observational Visit; O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. The baseline is defined as the DLco results taken after SV2 and before randomization.

| | | | | CVT- 301 | | |
|---|---|---|---|---|---|---|
| Category/Visit | Statistic | O. C.<br>Statistic (N=xx) | 002/003<br>(N=xx) | Naive<br>(N=xx) | Total<br>(N=xx) | Overall (N=xx) |
| FEV1/FVC < 60% | | | | | | |
| Baseline | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TV2/OV2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TV4/OV4 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TV5/OV5 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TV6/OV6 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| • • • | | | | | | |
| FEV1/FVC < 70% | | | | | | |
| Baseline | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TV2/OV2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TV4/OV4 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TV5/OV5 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TV6/OV6 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: TV = Treatment Visit; OV = Observational Visit. O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. The baseline is defined as the DLco results taken after SV2 and before randomization.

Cross-reference: Listing 16.2.8.2.4.4, Table 14.3.4.5.19

Table 14.3.4.5.10 Spirometry (Pulmonary Function Facility):70% or Smaller FEV1/FVC Values by Visit

Treatment Group: Observational Cohort

| Patient<br>ID | Visit | Time<br>Point | Motor<br>State | Date and Time<br>of Assessment | Test (Unit) | Result | Change from<br>Baseline |
|---|---|---|---|---|---|---|---|
| xxxx-xxx | TV2/OV2<br>TV3/OV3 | Pre-dose<br>Pre-dose | ON<br>ON | ddmonyyyy hh:mm<br>ddmonyyyy hh:mm # | xxx (xxx) | xx<br>Xx \$ | |

#### xxxx-xxx

Programmer note: please display all FEV1, FVC and FEV1/FVC from all timepoint if any criteria meet.

# Continue with CVT-301 (002/003), CVT-301 (Naïve)

Note: TV = Treatment Visit; OV = Observational Visit;

# indicates spirometry measurement not meeting ATS quality criteria. \* indicates imputed values. \$ indicates manual data. Data with 70% or smaller FEV1/FVC Values are included.

Table 14.3.4.5.11
Summary of Spirometry (Pulmonary Function Facility): Measurements Meeting ATS Quality Criteria (Safety Population)

| | | | | CVT-301 | | |
|---|---|---|---|---|---|---|
| State | Statistio | O.C.<br>(N=5) | 002/003<br>(N=7) | Naive<br>(N=8) | Total (N=20) | Overall (N=xx) |
| <u> </u> | Deacibeic | (11 0) | (14 / / | (14 0) | (11 20) | (11 2121) |
| Overall | | | | | | |
| Total Number of Spirometry/DLCO Measurements | n | xx | xx | XX | XX | |
| Total Number (Percent) of Spirometry Measurements | | | | | | |
| Meeting ATS Quality Criteria [a] | n (%) | xx (xx) | xx (xx) | xx (xx) | xx ( xx) | xx (xx) |
| Total Number (Percent) of Spirometry Measurements | | | | | | |
| Not Meeting ATS Quality Criteria [b] | n (%) | xx ( xx) | xx (xx) | xx (xx) | xx (xx) | xx ( xx) |
| Total Number (Percent) of DLCO Measurements | | | | | | |
| Meeting ATS Quality Criteria [a] | n (%) | xx (xx) | xx (xx) | xx (xx) | xx ( xx) | xx (xx) |
| Total Number (Percent) of DLCO Measurements | | | | | | |
| Not Meeting ATS Quality Criteria [b] | n (%) | xx ( xx) | xx (xx) | xx ( xx) | xx (xx) | xx (xx) |
| Proportion of Spirometry Measurements Meeting | | | | | | |
| ATS Quality Criteria at Subject Level[c] | n | XX | XX | XX | XX | XX |
| | Mean | 0.xxxx | 0.xxxx | 0.xxxx | 0.xxxx | 0.xxxx |
| | SD | 0.xxxxx | 0.xxxxx | 0.xxxxx | 0.xxxxx | 0.xxxxx |
| | Median | 0.xxxx | 0.xxxx | 0.xxxx | 0.xxxx | 0.xxxx |
| | Min, Max | 0.xxx, x.xxx | 0.xxx, x.xxx | 0.xxx, x.xxx | 0.xxx, x.xxx | 0.xxx, x.xxx |
| Proportion of DLCO Measurements Meeting | | | | | | |
| ATS Quality Criteria at Subject Level[c] | n | XX | XX | XX | XX | |
| | Mean | 0.xxxx | 0.xxxx | 0.xxxx | 0.xxxx | |

Note: TV = Treatment Visit; OV = Observational Visit; O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients.

<sup>[</sup>a] Percent is based on the total number of DLco measurements.

<sup>[</sup>b] Percent is based on the total number of DLco measurements not meeting ATS quality criteria.

<sup>[</sup>c] For each subject, the proportion is calculated as Dlco measurements meeting ATS criteria divided by total the count of records with unique assessment date/time and non-missing ATS Quality Criteria Flag.

Cross-reference: Listing 16.2.8.2.4.4, Listing 16.2.8.2.4.6

Table 14.3.4.6.1
Summary of Columbia-Suicide Severity Rating Scale (C-SSRS)
(Safety Population)

| | | | | CVT- 301 | | |
|---|---|---|---|---|---|---|
| | | O. C. | 002/003 | Naive | Total | Overall |
| Section | Visit | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Item | Assessment | n (%) | n (응) | n (%) | n (%) | n (%) |
| Baseline (TV1/OV1) | | | | | | |
| Any Suicidal Ideation or Behavior | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Suicidal Ideation | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Suicidal Behavior | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| Post Baseline | | | | | | |
| Any Suicidal Ideation or Behavior | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Suicidal Ideation | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Suicidal Behavior | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Suicidal Ideation | | | | | | |
| Wish to be Dead | TV1/OV1 | | | | | |
| | n | XX | XX | xx | XX | XX |
| | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | TV2/OV2 | | | | | |
| | n | XX | XX | XX | XX | XX |
| | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | TV3/OV3 | | | | | |
| | TV4/OV4 | | | | | |
| | TV5/OV5 | | | | | |
| | TV6/OV6 | | | | | |

Non-Specific Active Suicidal Thoughts

. . .

Intensity of Ideation

Suicidal Behavior

TV2/OV2...

. . .

Note: TV = Treatment Visit; OV = Observational Cohort; O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Percentages are based on n, the number of subjects assessed at each visit.

Table 14.3.4.6.2
Shift from Baseline in Columbia-Suicide Severity Rating Scale (C-SSRS) (Safety Population)

| | | TV1/OV1 n (%) | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| В | Baseline | No Suicidal Behavior or Ideation | | Suicidal Ideation | | Suicidal Behavior | | Missing | | Total | |
| | No Suicidal Ideation or Behavior | xx | (xx.x) | xx | (xx.x) | xx | (xx.%) | xx | (xx.%) | xx | (xx.x) |
| S¹ | uicidal Ideation | XX | (xx.x) | XX | (xx.x) | XX | (xx.%) | XX | (xx.%) | XX | (xx.x) |
| S <sup>1</sup> | uicidal Behavior | XX | (xx.x) | XX | (xx.x) | XX | (xx.%) | XX | (xx.%) | XX | (xx.x) |
| M: | Missing | xx | (xx.x) | XX | (xx.x) | XX | (xx.%) | XX | (xx.%) | XX | (xx.x) |
| (002/003) | To Suicidal Ideation<br>or Behavior | xxx | (xx.x) | XXX | (xx.x) | XXX | (xx.%) | xx | (xx.%) | xx | (xx.x) |
| S <sup>,</sup> | uicidal Ideation | XX | (xx.x) | XX | (xx.x) | XX | (xx.%) | XX | (xx.%) | XX | (xx.x) |
| S, | Suicidal Behavior | XX | (xx.x) | XX | (xx.x) | XX | (xx.%) | XX | (xx.%) | XX | (xx.x) |
| | Missing | XX | (xx.x) | vv | (xx.x) | XX | (xx.%) | XX | (xx.%) | XX | (xx.x) |

Note: O.C. rows is for the patients in Observational Cohort, 002/003 rows is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients.

Percentages are based on N, the number of subjects in each treatment group.

Table 14.3.4.7 Summary of Epworth Sleepiness Scale Total Score: Actual Values and Change from Baseline by Visit (Safety Population)

| Visit | Statistic | | | | | |
|---|---|---|---|---|---|---|
| | | O. C.<br>(N=xx) | 002/003<br>(N=xx) | Naive<br>(N=xx) | Total<br>(N=xx) | Overall (N=xx) |
| Baseline | Actual value | | | | | |
| | n | xx | XX | xx | xx | XX |
| | Mean | XX.X | xx.x | xx.x | xx.x | XX.X |
| | SD | XX.XX | xx.xx | xx.xx | xx.xx | XX.XX |
| | Median | XX.X | XX.X | xx.x | xx.x | XX.X |
| | Min, Max | XX, XX | xx, xx | XX, XX | xx, xx | xx, xx |
| TV4/OV4 | Actual value | | | | | |
| | n | XX | XX | xx | xx | XX |
| | Mean | XX.X | XX.X | XX.X | xx.x | XX.X |
| | SD | xx.xx | XX.XX | xx.xx | xx.xx | XX.XX |
| | Median | XX.X | XX.X | XX.X | xx.x | XX.X |
| | Min, Max | XX, XX | xx, xx | XX, XX | xx, xx | xx, xx |
| | Change from Baseline | | | | | |
| | n | XX | XX | XX | xx | XX |
| | Mean | xx.x | XX.X | xx.x | xx.x | XX.X |
| | SD | XX.XX | xx.xx | xx.xx | xx.xx | XX.XX |
| | Median | XX.X | XX.X | xx.x | xx.x | XX.X |
| | Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx |
| TV6/OV6 | • • • | | | | | |

Note: TV = Treatment Visit; OV = Observational Cohort; O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Baseline is the last non-missing assessment before the first dose of study drug.

Table 14.3.4.8

Summary of Questionnaire for Impulsive-Compulsive Disorders in Parkinson's (QUIP) by Visit (Safety Population)

| | | | CVT-301 | | | |
|---|---|---|---|---|---|---|
| | | O. C. | 002/003 | Naive | Total<br>(N=xx) | Overall (N=xx) |
| Section | Visit | (N=xx) | (N=xx) | (N=xx) | | |
| Item | Assessment | n (%) | n (응) | n (%) | n (%) | n (응) |
| Any Impulse or Other Compulsive Behaviors | TV1/OV1 | | | | | |
| | n | XX | XX | XX | XX | XX |
| | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx. |
| | TV4/OV4 | | | | | |
| | n | XX | XX | XX | XX | XX |
| | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx. |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx. |
| | TV6/OV6 | | | | | |
| | n | XX | XX | XX | XX | XX |
| | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx. |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx. |
| Any Impulse Behaviors | TV1/OV1 | | | | | |
| | n | XX | XX | XX | XX | XX |
| | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx. |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx. |
| | TV4/OV4 | | | | | |
| | n | XX | XX | XX | XX | XX |
| | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx. |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx. |
| | TV6/OV6 | | | | | |
| | n | XX | XX | XX | XX | XX |
| | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx. |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx. |
| Any Other Compulsive Behaviors | TV1/OV1 | | | | | |
| | n | XX | xx | XX | xx | XX |
| | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx. |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx. |
| | TV4/OV4 | | | | | |

| Civitas Therapeutics, Inc. | Page x of y |
|----------------------------|-------------|

| | n | XX | XX | XX | XX | XX |
|---|---|---|---|---|---|---|
| | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | TV6/OV6 | | | | | |
| | n | XX | XX | XX | XX | XX |
| | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Impulse Control Disorders | | | | | | |
| _ | TV1/OV1 | | | | | |
| Compulsive Gambling | n | XX | XX | XX | XX | XX |
| | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | TV4/OV4 | | | | | |
| | n | XX | XX | XX | XX | XX |
| | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | • • • | | | | | |
| Compulsive Sexual Behavior | | | | | | |

Compulsive Sexual Behavior Compulsive Buying Compulsive Eating

Other Compulsive Behaviors Hobbyism Punding Walkabout

Compulsive Medication Use

Note: TV = Treatment Visit; OV = Observational Cohort; O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Percentages are based on n, the number of subjects assessed at each visit.
Table 14.3.4.9.1

MMRM Analysis of UPDRS Part 4: Change from Baseline in the UPDRS Part 4 Score by Visit

(Safety Population)

| Visit | Statistic | CVT-301<br>(N=xx) | p-value |
|---------|-------------------------------|-------------------|---------|
| Overall | Overall p-value | | |
| | Baseline Hoehn and Yahr stage | | 0.xxx |
| | Screening Spirometry | | 0.xxx |
| | Visit | | 0.xxx |
| | Baseline UPDRS Part 3 Score | | 0.xxx |
| :V4 | n | xx | |
| | LS Mean | XX.X | |
| | SE (LS Mean) | XX.XX | |
| | 95% CI (LS Mean) | (xx.x, xx.x) | |
| ľV6 | | | |

Note: TV = Treatment Visit;

MMRM model uses the change from baseline in UPDRS Part 4 total scores at each post-baseline visit (TV4, TV6) as the dependent variable, and includes visit (TV4 or TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus  $\geq$ 2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1  $\geq$ 60% and FEV1/FVC ratio  $\geq$ 70%)) as fixed factors; The baseline UPDRS part 4 score will be included as a covariate, assuming an unstructured covariance matrix.

Cross-reference: Listing 16.2.8.2.8.2

Tables below will have similar format as Table 14.3.4.9.1

Table 14.3.4.9.2

MMRM Analysis of UPDRS Part 4 Dyskinesias Score: Change from Baseline in the UPDRS Part 4 Score by Visit (Safety Population)

Note: TV = Treatment Visit;

MMRM model uses the change from baseline in UPDRS Part 4 **D**yskinesias scores at each post-baseline visit (TV4, TV6) as the dependent variable, and includes visit (TV4 or TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus  $\ge$ 2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1  $\ge$ 60% and FEV1/FVC ratio  $\ge$ 70%)) as fixed factors; The baseline UPDRS part 4 score will be included as a covariate, assuming an unstructured covariance matrix.

Cross-reference: Listing 16.2.8.2.8.2

Table 14.3.4.9.3

MMRM Analysis of UPDRS Part 4 **Fluctuations Score:** Change from Baseline in the UPDRS Part 4 Score by Visit (Safety Population)

Note: TV = Treatment Visit;

MMRM model uses the change from baseline in UPDRS Part 4 Fluctuations scores at each post-baseline visit (TV4, TV6) as the dependent variable, and includes visit (TV4 or TV6), the stratification variables (baseline Hoehn and Yahr stage (<2.5 versus  $\ge$ 2.5) and screening spirometry ([FEV1] <60% or FEV1/forced vital capacity [FVC] ratio <70% versus FEV1  $\ge$ 60% and FEV1/FVC ratio  $\ge$ 70%)) as fixed factors; The baseline UPDRS part 4 score will be included as a covariate, assuming an unstructured covariance matrix.

Cross-reference: Listing 16.2.8.2.8.2

Table 14.3.4.9.4

Summary of UPDRS Part 4: Actual Values and Change from Baseline by Visit (Safety Population)

| Visit | Statistic | 002/003<br>(N=xx) | Naive<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|
| ATSTC | SCACISCIC | (IV-XX) | (1v-XX) | (N-XX) |
| Baseline | Actual value | | | |
| | n | XX | xx | xx |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | xx.xx |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | XX, XX |
| TV4/OV4 | Actual value | | | |
| | n | xx | XX | xx |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | xx.xx |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | XX, XX |
| | Change from Baseline | | | |
| | n | XX | XX | xx |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | xx.xx |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | XX, XX |
| TV6/OV6 | | | | |

Note: TV = Treatment Visit; OV = Observational Cohort; Total column is for all CVT-301 treated patients, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. Baseline is the last non-missing assessment before the first dose of study drug.

Cross-reference: Listing 16.2.8.2.6

Table below will have similar format as Table 14.3.4.9.4

Table 14.3.4.9.5

Summary of UPDRS Part 4 Dyskinesias Score: Actual Values and Change from Baseline by Visit (Safety Population)

Table 14.3.4.9.6

Summary of UPDRS Part 4 Fluctuations Score: Actual Values and Change from Baseline by Visit (Safety Population)

Table 14.3.4.10 Dyskinesia: Occurrence and Severity (In-clinic) by Visit (ITT Population)

| Visit | Statistic | O. C.<br>(N=xx) | 002/003<br>(N=xx) | Naive<br>(N=xx) | Total<br>(N=xx) | Overall<br>(N=xx) |
|---|---|---|---|---|---|---|
| TV2/OV2 | Dyskinesia | | | | | |
| | Yes (Percentages based on N) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | No (Percentages based on N) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Severity of Dyskinesia | | | | | |
| | Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Unknown | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TV3/OV3 | ••• | | | | | |

Note: TV = Treatment Visit; OV = Observational Cohort; O.C. column is for the patients in Observational Cohort, 002/003 column is for the patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies and Naïve is for the CVT-301 naive patients. [a] The data for which a subject was dyskinetic already before the study drug administration was excluded from summary.

Cross-reference: Listing 16.2.6.2.1

## Attachment 2 Listing Mock-ups

Page x of y

### Table of Contents

| Listing | 16.2.1 | Patient Disposition | . 3 |
|---|---|---|---|
| | | Protocol Deviations | |
| Listing | 16.2.3.1 | Inclusion Criteria not Met at Screening | . 5 |
| Listing | 16.2.3.2 | Exclusion Criteria Met at Screening | . 7 |
| Listing | 16.2.4.1 | Demographics | 10 |
| Listing | 16.2.4.2 | Medical History | 11 |
| Listing | 16.2.4.3 | Parkinson's Disease History | 12 |
| Listing | 16.2.4.4 | Smoking History | 13 |
| Listing | 16.2.4.5 | | |
| Listing | 16.2.4.6 | Modified Hoehn and Yahr Staging in "ON" State at Screening | 15 |
| Listing | 16.2.4.7 | | |
| Listing | 16.2.4.8 | | |
| Listing | | | 18 |
| Listing | 16.2.4.1 | 0 Randomization | 19 |
| | | 1.1 Prior and Concomitant Medications. | |
| Listing | 16.2.4.1 | 1.2 Parkinson's disease Treatment Medications at Baseline | 21 |
| Listina | 16.2.4.1 | 2 Baseline Pulmonary Assessment Part 2 - Pulmonary History | 22 |
| | | 3 Baseline Pulmonary Assessment Part 3 - Assessments of Symptoms | |
| | | .1 Study Drug Administration: in Clinic and at Home | |
| Listing | 16.2.5.1 | .2 Study Drug Administration: Derived Variables (in Clinic) | 26 |
| | | .3 Study Drug Administration: Derived Variables (Overall) | |
| | | .4 Study Drug Administration: Derived Variables (Overall by Visit) | |
| | | .5 Listing of Study Drug Dose Change | |
| | | Study Drug Kit Dispensation. | |
| | | Daily Levodopa Dose. | |
| | | .1 Unified Parkinson's Disease Rating Scale (UPDRS) Part 3 | |
| | | .2 Unified Parkinson's Disease Rating Scale (UPDRS) Part 3: Derived Variables | |
| | | 1 Clinic Assessment. | |
| | | 2 Parkinson's Disease Diary Data. | |
| | | .3.1 Parkinson's Disease Diary Data - Derived Variable by Dairy Date | |
| | | .3.2 Parkinson's Disease Diary Data - Derived Variable by Visit | |
| | | 4 Patient's Global Impression of Change (PGI-C) | |
| | | .5 Impact of Parkinson's OFF Episodes. | |
| | | .1 Unified Parkinson's Disease Rating Scale (UPDRS) Part 2 | |
| | | .2 Listing of S&E Activities of Daily Living | |
| | | 3 39 Item Parkinson's Disease Questionnaire (PDO-39). | |
| | | Adverse Events. | |
| | | .1 Clinical Laboratory Results - Hematology | |
| | | 2 Clinical Laboratory Results - Chemistry | |
| | | .3 Serum Pregnancy Test - Positive Only | |
| | | .1 Vital Signs | |
| | | 2 12-Lead Electrocardiogram (ECG). | |
| | | .3 Physical Examination | |
| | | .4.1 Spirometry( Neurology Office) | |
| | | .4.2 Spirometry (Neurology Office) Measurements Not Meeting ATS Quality Criteria | |
| | | .4.2 Spirometry (Pulmonary Function Facility): DLco Parameters | |
| Listing | | | |
| | | transmill (- almonal) randolon radiffely, optionodily, blood head atometres not needling into Quartely Cliteria | |

Civitas Therapeutics, Inc.

Page x of y


| Listing 16.2.8.2.5 Columbia-Suicide Severity Rating Scale (C-SSRS) | 60 |
|---|---|
| Listing 16.2.8.2.6 Epworth Sleepiness Scale | 64 |
| Listing 16.2.8.2.7 Questionnaire for Impulsive-Compulsive Disorders in Parkinson's (QUIP) | |
| Listing 16.2.8.2.8.1 Unified Parkinson's Disease Rating Scale (UPDRS) Part 4 | 68 |
| Listing 16.2.8.2.8.1 Unified Parkinson's Disease Rating Scale (UPDRS) Part 4 | 68 |
| Listing 16.2.8.2.8.2 Unified Parkinson's Disease Rating Scale (UPDRS) Part 4: Derived Variables | 69 |
| Listing 16.2.8.2.9.1 Telephone Contact | 70 |
| Listing 16.2.8.2.9.2 Telephone Contact: Challenges with Inhaler or Capsules Data | 71 |


Listing 16.2.1 Patient Disposition

Treatment Group: Observational Cohort

| | | | Date of Completion/ | | | |
|---|---|---|---|---|---|---|
| Patient | Date of First | Date of | Withdrawal (Study Day) | Completed | Primary Reason | Screen |
| ID | Dose | Last Dose | [a] | Study? | for Withdrawal | Failure/Date |
| XXXX-XXX | ddmonyyyy | ddmonyyyy | ddmonyyyy | Yes | | |
| XXXX-XXX | ddmonyyyy | ddmonyyyy | ddmonyyyy | No | Adverse Event: AE #x | Yes |
| XXXX-XXX | ddmonyyyy | ddmonyyyy | ddmonyyyy | No | Lack of Efficacy | |
| XXXX-XXX | ddmonyyyy | ddmonyyyy | ddmonyyyy | No | Patient Withdrew Consent | No |
| | | | | | Protocol Violation: | |
| xxxx-xxx | ddmonyyyy | ddmonyyyy | ddmonyyyy | No | XXXXXXXXX | |

. . .

Continue with CVT-301 (002/003), CVT-301 (Naïve)

Note: [a] Study Day = Date of Completion/Withdrawal - Date of first Dose + 1.

# Listing 16.2.2.1 Protocol Deviations

Treatment Group: Observational Cohort

| Patient ID | Deviation Type | Deviation Description | Created Date | Major<br>Deviation | Affect Pulmonary<br>Assessments |
|---|---|---|---|---|---|
| xxxx-xxx | xxxxxxxxxx | xxxxxxxxxxxxxxx | ddmonyyyy | | |
| | | xxxxxxxxxxxxxx | ddmonyyyy | | |
| xxxx-xxx | xxxxxxxxxx | xxxxxxxxxxxxxxx | ddmonyyyy | Yes | Yes |
| | xxxxxxxxxx | xxxxxxxxxxxxxxx | ddmonyyyy | | |

# Listing 16.2.3.1 Inclusion Criteria not Met at Screening

### Inclusion Criteria:

- 1. Has signed and dated an IRB/IEC-approved informed consent form before any protocol-specific screening procedures are performed.
- 2. Is a male or female aged 30 to 80 years, inclusive. Women of child-bearing potential must use protocol-defined contraceptive measures (see Section 11.1.5) and must have a negative serum human chorionic gonadotropin (hCG) test at screening. These patients must be willing to remain on their current form of contraception for the duration of the study.
- 3. Patients who have idiopathic PD (i.e., not induced by drugs or other diseases) as defined by fulfilling Steps 1 and 2 of the United Kingdom (UK) Brain Bank criteria, diagnosed after the age of 30 years.
- 4. Patients who are classified as Stage 1 to 3 (in the ON state) on the modified Hoehn and Yahr scale for staging of PD severity.
- 5. Patients who have experienced motor fluctuations for a minimum of 2 hours of average daily OFF time per waking day (excluding early morning OFF time) by self-report and confirmed by the PD Diary (on 3 consecutive days) during the screening period.
- 6. Patients must be stable on oral LD-containing therapy for at least 2 weeks prior to SV1 with a LD/DDI-containing regimen, which must include doses at least 4 times during the waking day and a total daily LD dose of ≤1600 mg (exclusive of PRN LD-containing medications).
- 7. Patients should be stable on other PD medications for at least 4 weeks prior to SV1.
- 8. Patients must have a ≥25% difference between UPDRS Part 3 scores recorded in their ON and OFF states at screening.
- 9. Patients must understand (with or without caregiver assistance) their daily medication regimen and must agree that they will not change their daily medication doses during the study.
- 10. Patients must have normal cognition as confirmed by a score of ≥25 on the Mini Mental State Examination (MMSE).
- 11. Patients must be able to perform a spirometry maneuver in the ON and OFF states and must have a screening FEV1 ≥50% of predicted, and a FEV1/FVC ratio >60% of predicted in the ON state at screening. (A pulmonologist will review the spirometry tracings/morphology of any patient with FEV1 <60% or FEV1/FVC <70% in order to determine eligibility. Patients with an FEV1/FVC <70% will complete spirometry before and after the administration of a bronchodilator in a pulmonary function laboratory. Testing will be performed in accordance with the 2005 ATS/European Respiratory Society (ERS) criteria prior to randomization. The results of the bronchodilator challenge will be reviewed by a pulmonologist prior to potential randomization.)

Listing 16.2.3.1
Inclusion Criteria not Met at Screening

Treatment Group: Observational Cohort

| | Any Criterion | Criterion Not Met at SV1 | | Patient Has >= 2 Hours of OFF - | Criterion Not Met at SV2 | |
|---|---|---|---|---|---|---|
| Patient<br>ID | Violation<br>at SV1 | Criterion Number | Comment | Time during the Waking Day<br>Confirmed by Diary. | Criterion Number | Comment |
| xxxx-xxx | Yes | Х | xxxxxxx | x | х | xxxxxx |
| | | X | XXXXXXX | X | X | XXXXXXX |
| xxxx-xxx | | Х | XXXXXX | х | Х | xxxxxx |
| • • • | | | | | | |
| Continue w | ith CVT-301 (002/00 | 3), CVT-301 (Naïve) | | | | |

Civitas Therapeutics, Inc.

Page x of y


# Listing 16.2.3.2 Exclusion Criteria Met at Screening

### Exclusion Criteria

- 1. Patients who have dyskinesia of a severity that would significantly interfere with their ability to participate or perform study procedures.
- 2. Pregnant or lactating females or females wishing to become pregnant.
- 3. Patients who have any known contraindication to the use of LD, including a history of malignant melanoma or a history of narrow-angle glaucoma.
- 4. Patients who have had previous surgery for PD (including but not limited to deep brain stimulation or cell transplantation) or plan to have stereotactic surgery during the study period.
- 5. Patients with a history of psychotic symptoms requiring treatment, or suicidal ideation or attempt within the prior 12 months (stable regimens [for at least 4 weeks prior to SV1] of anti-depressant medications and certain low-dose atypical antipsychotic medications are permitted).
- 6. Patients who have cancer with the exception of the following: basal cell carcinoma or successfully treated squamous cell carcinoma of the skin; cervical carcinoma in situ; prostatic carcinoma in situ; or other malignancies curatively treated and with no evidence of disease recurrence for at least 3 years.
- 7. Patients taking certain prohibited medications (see Section 9.4.2).
- 8. Patients with a history of drug or alcohol abuse within the prior 12 months.
- 9. Patients with chronic obstructive pulmonary disease (COPD), asthma, or other chronic respiratory disease within the last 5 years (or if a patient is receiving treatment for any of these conditions).
- 10. Patients with any contraindication to performing routine spirometry or who are unable to perform a spirometry maneuver (see Appendix 14 for a list of contraindications).
- 11. Patients with a current history of symptomatic orthostatic hypotension despite adequate treatment.
- 12. Patients with any condition that in the investigator's opinion would make patients unable to comply with study procedures or make them unsuitable for participation in the study.
- 13. Patients who have any clinically significant abnormality or finding from examination, tests, or history that may compromise patient safety. Potential issues of concern should be raised to the medical monitor during eligibility review.
- 14. Patients who have participated in any prior CVT-301 study, regardless of treatment group assignment.

# Listing 16.2.3.2 Exclusion Criteria Met at Screening

Treatment Group: Observational Cohort

| Any Criterion | Criterion Met at SV1 | | — Patient Has >= 2 Hours of | Criterion Met at SV2 | |
|---|---|---|---|---|---|
| Violation<br>at SV1 | Criterion Number | Comment | OFF time during the Waking<br>Day Confirmed by Diary. | Criterion Number | Comment |
| Yes | Х | xxxxxxx | х | х | xxxxxx |
| | X | XXXXXXX | X | x | XXXXXXX |
| | X | XXXXXXX | X | X | XXXXXXX |
| | Violation<br>at SV1 | Violation at SV1 Criterion Number Yes x x | Violation at SV1 Criterion Number Comment Yes x xxxxxxx x xxxxxxxxxxxxxxxxxxxxxxxx | Violation at SV1 Criterion Number Comment Day Confirmed by Diary. Yes x xxxxxxx x x xxxxxxx x | Violation at SV1 Criterion Number Comment Day Confirmed by Diary. Criterion Number Yes x xxxxxxx x x x x x x x x x x x x x x |

# Listing 16.2.3.3 Analysis Populations

Treatment Group: Observational Cohort

| | Safety | ITT | | | | Compl | eted Visit | |
|---|---|---|---|---|---|---|---|---|
| Patient ID | Population | Population | TV1/OV1 | TV2/OV2 | TV3/OV3 | TV4/OV4 | TV5/OV5 | TV6/OV6 |
| xxxx-xxx | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes |
| xxxx-xxx | No | No | Yes | Yes | Yes | Yes | Yes | Yes |

Program Name: xxxx.sas Page 194 of 335 Listing Generation: ddmomyyyy

Listing 16.2.4.1

Demographics

| Patient ID | Date of<br>Informed<br>Consent | Date of<br>Birth | Age<br>(years)<br>[a] | Sex | Race | Ethnicity | Height<br>(cm) | Weight<br>(kg) | BMI<br>(kg/m^2)<br>[b] |
|---|---|---|---|---|---|---|---|---|---|
| xxxx-xxx | ddmonyyyy | ddmonyyyy | XX | Male | White | Hispanic or Latino | XXX.X | xx.x | xx.x |
| xxxx-xxx | ddmonyyyy | ddmonyyyy | xx | Male | Black or African<br>American | Not Hispanic or<br>Latino | xxx.x | XX.X | XX.X |
| xxx-xxx | ddmonyyyy | ddmonyyyy | xx | Female | Other: xxxxx | Hispanic or Latino | xxx.x | xx.x | xx.x |
| xxx-xxx | ddmonyyyy | ddmonyyyy | XX | Female | Asian | Unknown | xxx.x | XX.X | xx.x |
| Continue wi | th CVT-301 (00 | 2/003), CVT-301 | (Naïve) | | | | | | |

<sup>[</sup>a] Age was calculated as the difference between date of birth and date of Informed Consent, in years.

<sup>[</sup>b] BMI was calculated as weight (kg) / [height (m)]^2.


Listing 16.2.4.2 Medical History

Treatment Group: Observational Cohort

| Patient<br>ID | Body System | Description | System Organ Class/<br>Preferred Term [a] | Start Date | Stop Date |
|---|---|---|---|---|---|
| xxxx-xxx | HEENT | xxxxxxxxxx | xxxxxxxxxxx/<br>xxxxxxxxx | ddmonyyyy | ddmonyyyy |
| | Dermatological | xxxxxxxxxx | ************************************** | ddmonyyyy | Ongoing |
| | Psychiatric | xxxxxxxxxx | xxxxxxxxxxxxx/<br>xxxxxxxxx | ddmonyyyy | Ongoing |
| | Neurological | xxxxxxxxxx | xxxxxxxxxxxx/<br>xxxxxxxxx | ddmonyyyy | Ongoing |
| | Other: xxxxxx | | | ddmonyyyy<br>Unknown | Ongoing<br>Unknown |
| xxx-xxx | | | | | |
| Continue wit | th CVT-301 (002/003), CVT | -301 (Naïve) | | | |

<sup>[</sup>a] Medical history data were coded into system organ class and preferred term by using MedDRA version 17.0.

# Listing 16.2.4.3 Parkinson's Disease History

| Treatment Group | : Observational Cohor | t | |
|---|---|---|---|
| Patient<br>ID | Date of<br>Diagnosis | Start Date<br>of Levodopa<br>Treatment | Date of Onset of<br>Motor Fluctuation<br>(Wearing Off) Episodes |
| xxxx-xxx | monyyyy | monyyyy | топуууу |
| xxxx-xxx | monyyyy | топуууу | топуууу |
| xxxx-xxx | monyyyy | monyyyy | топуууу |
| xxxx-xxx | monyyyy | monyyyy | топуууу |
| Continue with C | VT-301 (002/003), CVT | -301 (Naïve) | |

Listing 16.2.4.4 Smoking History

Treatment Group: Observational Cohort

| | _ , , , | _ | | - 11 | _ | If Former or Curren | · |
|---|---|---|---|---|---|---|---|
| Patient | Ever Smoked | Age | Current | Smoking | Age | Average Number of Cigarettes | Number of Years |
| ID | Cigarettes | Started | Smoker | Status | Quitted | per Day | Smoked |
| XXX-XXX | Yes | 25 | No | Former | XX | XX | XX |
| XXX-XXX | Yes | 26 | Yes | Current | XX | XX | XX |
| xxx-xxx | No | | | Never | | | |
| XXX-XXX | | | | | | | |

Number of Years Smoked = (Age-Age Started+1)(Current Smoker) OR = (Age Quitted-Age Started+1)(Former Smoker).

## 

Treatment Group: Observational Cobort

| Patient<br>ID | Visit | Date of<br>Assessment | Has the Patient Been Tested for Competence in self-rating with at least 75% concordance with the ratings of the examiner? |
|---|---|---|---|
| xxxx- | SV1<br>SV2 | ddmonyyyy<br>Not Done | Yes |
| xxxx-<br>xxx | UNS<br>SV1 | ddmonyyyy<br>ddmonyyyy | No<br>Yes |

Note: SV = Screening Visit; UNS = Unscheduled;

### Listing 16.2.4.6 Modified Hoehn and Yahr Staging in "ON" State at Screening

Treatment Group: Observational Cohort

| Patient<br>ID | Date of<br>Assessment | Stage in "ON"<br>State [a] |
|---|---|---|
| xxxx-xxx | ddmonyyyy | 0 = No signs of disease |
| xxxx-xxx | ddmonyyyy | 1 = Unilateral disease |
| xxxx-xxx<br>••• | Not Done, xxxxxx | |
| Continue with CV | 7T-301 (002/003), CVT-301 (Naïve) | |

<sup>[</sup>a] 0 = No signs of disease, 1 = Unilateral disease, 1.5 = Unilateral plus axial involvement,

<sup>2 =</sup> Bilateral disease, without impairment of balance, 2.5 = Mild bilateral disease, with recovery on pull test,

<sup>3 =</sup> Mild to moderate bilateral disease; some postural instability; physical independent,

<sup>4 =</sup> Severe disability; still able to walk or stand unassisted, 5 = Wheelchair-bound or bedridden unless aided.


Listing 16.2.4.7 Mini Mental State Examination (MMSE) at Screening

| Patient | | Date of | | | | | | | | | | | | Total |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ID | Visit | Assessment | Q1 | Q2 | Q3 | Q4 | Q5 | Q6 | Q7 | Q8 | Q9 | Q10 | Q11 | Score [a] |
| xxxx-xxx | SV1 | ddmonyyyy | Х | X | Х | Х | Х | X | х | X | Х | х | Х | XX |
| xxxx-xxx | SV2 | ddmonyyyy | Х | х | Х | Х | Х | х | Х | х | Х | Х | Х | XX |
| xxxx-xxx | | Not Done, | | | | | | | | | | | | |

Note: SV= Screening Visit; UNS=Unscheduled Visit;

<sup>[</sup>a] >=25 points = normal, 21-24 points = mild cognitive impairment, 10-20 points = moderate cognitive impairment, 0-9 points = severe cognitive impairment.

### Confidential

Listing 16.2.4.8 Parkinson's Disease Diary Data at Screening: Derived Time

Treatment Group: Observational Cohort

| | | | Mean Daily<br>ON Time With | | |
|---|---|---|---|---|---|
| Patient<br>ID | Mean OFF<br>Time<br>(hours) | Mean Daily<br>ON Time Without<br>Dyskinesia<br>(hours) | Non-<br>troublesome<br>Dyskinesia<br>(hours) | Mean Daily<br>ON Time With Troublesome<br>Dyskinesia<br>(hours) | Dyskinetic<br>Before<br>TV1 [a] |
| xxx-xxx | xx.x | xx.x | xx.x | xx.x | Yes |
| xxxx-xxx | XX.X | xx.x | xx.x | xx.x | No |
| xxxx-xxx | XX.X | xx.x | XX.X | xx.x | |
| xxx-xxx | XX.X | XX.X | XX.X | xx.x | |

Continue with CVT-301 (002/003), CVT-301 (Naïve)

Note: TV = Treatment Visit; All diary data were normalized to 16 awake hours per day.

<sup>[</sup>a] Patients who have recorded at least 1 hour of dyskinesia (either ON with non-troublesome dyskinesia or ON with troublesome dyskinesia) on at least 2 days before TV1 are classified as dyskinetic.

# Protocol No. CVT-301-005

Listing 16.2.4.9 Screening ON/OFF Log

Treatment Group: Observational Cohort

| Patient<br>ID | Date of<br>Assessment | Time of Start<br>of OFF Episode | Changed the Timing of<br>Usual LD Medication? | Take an Extra Dose of LD/<br>Other Parkinson's Medication? | Daily<br>Number of<br>OFF Episodes<br>Experienced |
|---|---|---|---|---|---|
| xxxx-xxx | ddmonyyyy | hh:mm a.m. | Yes | Yes | xx |
| | | hh:mm a.m. | No | No | |
| | ddmonyyyy | hh:mm p.m. | No | | |
| | • • • | | | | |
| xxx-xxx | | | | | |
| • • • | | | | | |
| Continue w | ith CVT-301 (002/ | '003), CVT-301 (Naïve) | | | |

Listing 16.2.4.10 Randomization

Treatment Group: Observational Cohort

| Patient<br>ID | Date of<br>Randomization | Kit Number | Baseline Disease<br>Severity [a] | Screening Spirometry | Country | Site |
|---|---|---|---|---|---|---|
| xxxx-xxx | ddmonyyyy | NA | Low | FEV1 <60% or FEV1/FVC ratio <70% | US | xx |
| xxxx-xxx | ddmonyyyy | NA | High | FEV1 ≥60% and FEV1/FVC ratio ≥70% | US | xx |
| xxxx-xxx<br>••• | ddmonyyyy | NA | High | FEV1 ≥60% and FEV1/FVC ratio ≥70% | Canada | xx |
| Continue | with CVT-301 (00 | 2/003), CVT-301 (Naïve) | | | | |

<sup>[</sup>a] Low = Hoehn and Yahr Stage < 2.5, High = Hoehn and Yahr Stage >= 2.5.

<sup>[</sup>b] Patients who have recorded at least 1 hour of dyskinesia (either ON with non-troublesome dyskinesia or ON with troublesome dyskinesia) on at least 2 days before Visit 3 are classified as dyskinetic.

# Listing 16.2.4.11.1 Prior and Concomitant Medications

| Patient | ATC Level 1/ | Preferred Term [a]/ | Start/ | P/C | Dose | | | |
|---|---|---|---|---|---|---|---|---|
| ID | ATC Level 2 [a] | Medication Name | Stop Date | [b] | (Unit) | Frequency | Route | Indication |
| | xxxxxxxx/ | xxxxxxxx/ | | | | | XXXXX | |
| xxx-xxx | xxxxxxxxxxx | xxxxxxxxxxx | Ddmonyyyy/ddmonyyyy | P | xxxxx (xxx) | XXX | | Medical History: x |
| | | xxxxxxxx/ | ddmonyyyy/ | | | | | |
| | xxxxxxxx/ | xxxxxxxxxxx | ddmonyyyy | | | | XXXXX | |
| | xxxxxxxxxxx | | | С | xxxxx (xxx) | XXX | | Adverse Event: x |
| | | xxxxxxxx/ | | | | | XXXXX | |
| | | xxxxxxxxxxx | ddmonyyyy/ Ongoing | С | xxxxx (xxx) | Other: xxx | | |
| xxx-xxx | | | | | | | | |
| Continue | with CVT-301 (002/00 | 3). CVT-301 (Naïve) | | | | | | |

<sup>[</sup>a] Medications were coded into ATC and preferred term using the WHO Drug Dictionary Q1March2014.

<sup>[</sup>b] P=Prior, C=Concomitant.

### COMPTACHETA

# Listing 16.2.4.11.2 Parkinson's disease Treatment Medications at Baseline

| Patient | ATC Level 1/ | Preferred Term [a]/ | Start/ | P/C | Dose | | | |
|---|---|---|---|---|---|---|---|---|
| ID | ATC Level 2 [a] | Medication Name | Stop Date | [b] | (Unit) | Frequency | Route | Indication |
| | xxxxxxxx/ | xxxxxxx/ | | | | | xxxxx | |
| xxxx-xxx | xxxxxxxxxx<br>xxxxxxx/ | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | ddmonyyyy/ddmonyyyy | P | xxxxx (xxx) | XXX | xxxxx | Medical History: x |
| | xxxxxxxxxx | xxxxxxxxxx<br>xxxxxxx/ | ddmonyyyy/ddmonyyyy | С | xxxxx (xxx) | XXX | xxxxx | Adverse Event: x |
| | | xxxxxxxxxx | ddmonyyyy/ Ongoing | С | xxxxx (xxx) | Other: xxx | | |
| xxx-xxx | | | | | | | | |
| <br>Continue v | with CVT-301 (002/003 | 3), CVT-301 (Naïve) | | | | | | |

<sup>[</sup>a] Medications were coded into ATC and preferred term using the WHO Drug Dictionary, Q1March2014. The medications which start with ATC code NO4 are considered as baseline PD treatment medications.


### Listing 16.2.4.12 Baseline Pulmonary Assessment Part 2 - Pulmonary History

### Part 2: Pulmonary History

- A. Asthma Questions:
- 1. Have you ever been told by an MD or other health care provider that you have asthma?/Details
- 2. If yes, how old were you when you were diagnosed with asthma?(years)
- 3. Do you still have asthma?
- 4. If no, at what age did your asthma resolve?
- 5. If yes, do you take medicine for asthma?
- 6. Which medicine(s) do you take for asthma?
- 7. What things cause your asthma to worsen or asthma attacks to occur?
- B. COPD Questions:
- 1. Have you ever been told by an MD or other health care provider that you have smoker's cough, COPD, emphysema, or chronic bronchitis?
- 2. If yes, how old were you when you were diagnosed with this condition?
- 3. What has/have been your primary occupation(s)?
- 4. Have you worked in jobs with significant dust exposure?
- 5. If yes, for how many years?
- 6. Do you currently take medicines for COPD?
- 7. If yes, which medicine(s) for COPD do you take?
- C. Other Lung or Airway Disease:
- 1. Do you have any condition that may have affected your breathing or lung health, such as congenital conditions of the chest wall or spine (for example, scoliosis) or other conditions, such as sleep apnea?
- 2. Have you ever sustained any chest or lung injuries or trauma that have had a long-term impact on your breathing?
- 3. Have you had any medical issues affecting your heart, such as a heart attack or congestive heart failure, that have caused you to have shortness of breath or limited your ability to exercise?
- 4. Have you ever needed to be put on a mechanical ventilator or respirator for any reason?/ If yes, was this needed for
  - 5. Have there been any other illnesses, chronic conditions, injuries or anything you can think of in your past, even as a child, that may have had a lasting impact on your lungs or respiratory health?

### Confidential

## Listing 16.2.4.12 Baseline Pulmonary Assessment Part 2 - Pulmonary History

| Datelant | Α. | Asthma | Ques | stion | S | | | В | . CO | PD Que | stion | S | | | C. Ot | her Lung c | r Airway | Disease | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient -<br>ID | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 1 | 2 | 3 | 4 | 5 |
| xxxx-xxx | No | | | | | | | Yes | XX | xxx | No | | No | | Yes | No | xx | Yes./xxx | XX |
| xxxx-xxx<br> | Yes/xxx | xxx | No | xx | xx | xxx | xxx | No | | | | | | | | | | | |

Programming note: The actual listing started with new page

### Listing 16.2.4.13 Baseline Pulmonary Assessment Part 3 - Assessments of Symptoms

- 1. Shortness of breath or breathlessness? / If yes, when does this seem to occur?
- 2. Chest Tightness? / If yes, when does this seem to occur?
- 3. Chest Pain? / If yes, when does this seem to occur?
- 4. Persistent Cough? / If yes, when does this seem to occur?
- 5. Sputum Production/If yes, when does this seem to occur?
- 6. Episodes of coughing up blood or blood in your sputum?/ If yes, when does this seem to occur?

## Listing 16.2.4.13 Baseline Pulmonary Assessment Part 3 - Assessments of Symptoms

Treatment Group: Observational Cohort

| | | | Assessments | of Symptoms | | |
|---|---|---|---|---|---|---|
| Patient<br>ID | 1 | 2 | 3 | 4 | 5 | 6 |
| xxxx-xxx | Yes,xxx | No | Yes,xxx | No | Yes,xxx | Yes,xxx |
| xxxx-xxx<br> | No | Yes,xxx | Yes,xxx | Yes,xxx | No | No |

Programming note: The actual listing started with new page

### Confidencial

Treatment Group: CVT-301 (002/003)

| | | | Start | End Date/Time | | | Doses/Day | Any |
|---|---|---|---|---|---|---|---|---|
| Patient | Dosing | | Date/Time | of Treatment (Time | Capsules | Time | | Reinhalations/Which |
| ID | Category | Visit | of Treatment | 0) | Administered | Intervals | | Capsules |
| | In Clinic | | | | х | 00:00 -< | х | No |
| xxxx-xxx | | TV1 | ddmonyyyyhh:mm | ddmonyyyyhh:mm | | 00:30 | | |
| | At Home | TV1- | ddmonyyyyhh:mm | ddmonyyyyhh:mm | X | 00:30 -< | X | |
| | | <tv2< td=""><td></td><td></td><td></td><td>01:00</td><td></td><td></td></tv2<> | | | | 01:00 | | |
| | | TV2- | ddmonyyyyhh:mm | ddmonyyyyhh:mm | X | 01:00 -< | X | Yes/1st |
| | | <tv2< td=""><td></td><td></td><td></td><td>01:30</td><td></td><td></td></tv2<> | | | | 01:30 | | |
| | | TV3- | ddmonyyyyhh:mm | ddmonyyyyhh:mm | X | 01:30 -< | X | No |
| | | <tv4< td=""><td></td><td></td><td></td><td>02:00</td><td></td><td></td></tv4<> | | | | 02:00 | | |
| xxxx-xxx | | | | | | | | |
| | 1.1 004 ( | | | | | | | |
| Continue w | rith CVT-301 (N | aive) | | | | | | |

Note: TV=Treatment;

## Listing 16.2.5.1.2 Study Drug Administration: Derived Variables (in Clinic)

Treatment Group: CVT-301 (002/003)

| Patient<br>ID | Visit | Standard Morning Dose of LD-<br>Containing Medications to In-<br>clinic OFF (mins) | In-clinic OFF to Start of<br>Study Drug Inhalation<br>(mins) | Standard Morning Dose of LD-containing<br>Medications to Start of Study Drug<br>Inhalation (mins) | Duration of<br>Study<br>Drug<br>Inhalation |
|---|---|---|---|---|---|
| xxxx- | | | | | |
| XXX | TV1 | XX | XX | XX | X |
| | TV2 | XX | XX | XX | X |
| | TV3 | XX | XX | XX | X |
| | TV4 | XX | XX | XX | X |
| | | | | | X |
| xxxx- | | | | | |
| XXX | | | | | |

Note: TV=Treatment Visit;

Listing 16.2.5.1.3
Study Drug Administration: Derived Variables (Overall)

Treatment Group: CVT-301 (002/003)

| Patient | Duration of | Total # of | Average Daily | Total # of | Average Daily |
|---|---|---|---|---|---|
| ID | Exposure (days) [a] | Capsules Taken | Capsules | Doses Taken | Dose(s) |
| xxxx-xxx | XX | XX | XX | XX | 2 |
| | XX | XX | XX | XX | 3 |
| | XX | XX | XX | XX | 5 |
| | XX | XX | XX | xx | 4 |
| | xx | xx | XX | xx | 5 |
| | XX | XX | XX | xx | 4 |
| | XX | XX | XX | xx | 5 |
| XXXX-XXX | | | | | |
| • • • | | | | | |
| Continue with C | VT-301 (Naïve) | | | | |

<sup>[</sup>a] Duration of exposure (days) is calculated as documented last dose date-first dose date +1.


Listing 16.2.5.1.4 Study Drug Administration: Derived Variables (Overall by Visit)

Treatment Group: CVT-301 (002/003)

| Patient | | Total # of | Average Daily | Total # of | Average Daily |
|---|---|---|---|---|---|
| ID | Visit | Capsules Taken | Capsules | Doses Taken | Dose(s) |
| xxx-xxx | TV1- <tv2< td=""><td>XX</td><td>XX</td><td>XX</td><td>2.</td></tv2<> | XX | XX | XX | 2. |
| | TV2- <tv3< td=""><td>XX</td><td>xx</td><td>xx</td><td>3</td></tv3<> | XX | xx | xx | 3 |
| | TV3- <tv4< td=""><td>xx</td><td>XX</td><td>xx</td><td>5</td></tv4<> | xx | XX | xx | 5 |
| | | XX | XX | xx | 4 |

xxxx-xxx

Continue with CVT-301 (Naïve)

Note: TV = Treatment Visit;

# Listing 16.2.5.1.5 Listing of Study Drug Dose Change

Treatment Group: CVT-301 (002/003)

| Patient<br>ID | Type of change | Reason for<br>Change | Date of Change | Old Dose Level<br>(# capsules per<br>treatment) | New Dose Level<br>(# capsules per<br>treatment) | Was Medical Monitor<br>Contacted? |
|---|---|---|---|---|---|---|
| xxxx-xxx | Increase | xxxxx | ddmmmyyyy | 1 | 2 | Yes |
| xxxx-xxx | Decrease | xxxxxxxxx | ddmmmyyyy | 2 | 1 | No |
| xxxx-xxx | Decrease | xxxxxxxxx | ddmmmyyyy | 2 | 1 | Yes |
| | ith CVT-301 (Naïve) | | | | | |

## Listing 16.2.5.2 Study Drug Kit Dispensation

| Patient | | | Kit Number | |
|---|---|---|---|---|
| ID | Visit | Treatment | Dispensed | Date Dispensed |
| xxx-xxx | TV1 | Observational Cohort | XXXX | ddmonyyyy |
| 212121 212121 | TV2 | Observational Cohort | xxxx | ddmonyyyy |
| | TV3 | Observational Cohort | xxxx | ddmonyyyy |
| | Other: xxxx | Observational Cohort | XXXX | ddmonyyyy |
| xxx-xxx | | CVT DL1 | | |
| • • • | | | | |

Note: TV=Treatment Visit; UNS= Unscheduled;

Listing 16.2.5.3
Daily Levodopa Dose

Treatment Group: Observational Cohort

| Patient ID | Visit | How many times | Total Levodopa daily dose |
|---|---|---|---|
| xxxx-xxx | SV1 | XX | |
| | TV1 | XX | XXXX |
| | TV2 | XX | XXXX |
| | TV3 | xx | XXXX |
| | | | xxxx |
| xxxx-xxx | | | |
| • • • | | | |
| | 001 (000 (000) 001 | 7 W V | |
| Continue with CVT- | 301 (002/003), CVT-301 | (Naive) | |

Note: SV = Screening Visit; TV = Treatment Visit; UNS= Unscheduled;
Listing 16.2.6.1.1
Unified Parkinson's Disease Rating Scale (UPDRS) Part 3

Treatment Group: CVT-301 (002/003)

| | | | | | | | | | | | | ion | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | | r | | | | | |
| | | | | | | | | | | | Post | ural | | | | | |
| | | | | | | T: | remoi | at | Rest | - | Tre | mor | | Rig | gidit | У | |
| Patient | | Time | Date and Time | | Facial | | | | | | | | | | | | |
| ID | Visit | Point | of Assessment | Speech | Exp. | Face | RUE | LUE | RLE | LLE | RUE | LUE | Neck | RUE | LUE | RLE | LLE |
| xxx-xxx | SV1 - OFF | | 16APR2013 14:10 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 1 | 1 | 1 |
| | SV1 - ON | | 16APR2013 16:20 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 |
| xxx-xxx | SV1 - OFF | | 16APR2013 15:35 | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 0 |
| | SV1 - ON | | 16APR2013 14:10 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 0 |
| | SV2 | | Not Done, not applicable | | | | | | | | | | | | | | |
| | TV1 | Pre-dose | 14MAY2013 11:20 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 0 |
| | | +10 mins | 14MAY2013 11:37 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 |
| | | +20 mins | 14MAY2013 11:47 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 |
| | | +30 mins | 14MAY2013 11:57 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 |
| | | +60 mins | 14MAY2013 12:27 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 |
| | TV2 | Pre-dose | 21MAY2013 11:43 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0 |

Continue with CVT-301 (Naïve)

Note: SV = Screening Visit; TV = Treatment Visit; ET = Early Termination; UNS = Unscheduled;
\*indicates imputed item score. 18=Speech, 19=Facial Expression, 20=Tremor at Rest, 21=Action or Postural Tremor of hands, 22=Rigidity,
23=Finger Taps, 24=Hand Movements, 25=Rapid Alternating Movements of Hands, 26=Leg Agility, 27=Arising from Chair, 28=Posture,
29=Gait, 30=Postural Stability, 31=Body Bradykinesia and Hypokinesia.

Listing 16.2.6.1.1 Unified Parkinson's Disease Rating Scale (UPDRS) Part 3

Treatment Group: CVT-301 (002/003)

| | | | | Finger | Taps | Ha<br>Moven | | Rap<br>Altern<br>Movem<br>of H | ating<br>ents | Leg Ag | gility | Arising |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient | | Time | Date and Time | | | | | | | | | from |
| ID | Visit | Point | of Assessment | Right | Left | Right | Left | Right | Left | Right | Left | Chair |
| | 0111 000 | | 167770010 14 10 | 4 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | |
| XXX-XXX | SV1 - OFF | | 16APR2013 14:10 | 4 | 2 | 2 | 2 | 3 | 2<br>1 | 1 | 1 | 4 |
| | SV1 - ON | | 16APR2013 16:20 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 |
| xxx-xxx | SV1 - OFF | | 16APR2013 15:35 | 2 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 |
| | SV1 - ON | | 16APR2013 14:10 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| | SV2 | | Not Done, not applicable | | | | | | | | | |
| | TV1 | Pre-dose | 14MAY2013 11:20 | 2 | 2 | 2 | 1 | 1 | 1 | 0 | 1 | 0 |
| | | +10 mins | 14MAY2013 11:37 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 |
| | | +20 mins | 14MAY2013 11:47 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 |
| | | +30 mins | 14MAY2013 11:57 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 |
| | | +60 mins | 14MAY2013 12:27 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 2 | 0 |
| | | | | _ | _ | _ | - | = | _ | - | _ | Ü |
| | TV2 | Pre-dose | 21MAY2013 11:43 | 1 | 2 | 1 | 1 | 0 | 1 | 1 | 2 | 0 |
| G | : + b | 1 (31-") | | | | | | | | | | |

Continue with CVT-301 (Naïve)

Note: SV = Screening Visit; TV = Treatment Visit; ET = Early Termination; UNS = Unscheduled; \*indicates imputed item score. 18=Speech, 19=Facial Expression, 20=Tremor at Rest, 21=Action or Postural Tremor of hands, 22=Rigidity, 23=Finger Taps, 24=Hand Movements, 25=Rapid Alternating Movements of Hands, 26=Leg Agility, 27=Arising from Chair, 28=Posture, 29=Gait, 30=Postural Stability, 31=Body Bradykinesia and Hypokinesia.

Listing 16.2.6.1.1 Unified Parkinson's Disease Rating Scale (UPDRS) Part 3

Treatment Group: CVT-301 (002/003)

| Patient | | Time | Date and Time | | | Postural | Bradykinesia/ | UPDRS III |
|---|---|---|---|---|---|---|---|---|
| ID | Visit | Point | of Assessment | Posture | Gait | Stability | Hypokinesia | Total Score |
| xxxx-xxx | SV1 - OFF | | 16APR2013 14:10 | 1 | 2 | 0 | 3 | 38 |
| | SV1 - ON | | 16APR2013 16:20 | 1 | 1 | 0 | 2 | 16 |
| xxx-xxx | SV1 - OFF | | 16APR2013 15:35 | 2 | 1 | 1 | 2 | 24* |
| | SV1 - ON | | 16APR2013 14:10 | 2 | 1 | 0 | 1 | 15 |
| | SV2 | | Not Done, not applicable | | | | | |
| | TV1 | Pre-dose | 14MAY2013 11:20 | 1 | 1 | 0 | 2 | 24 |
| | | +10 mins | 14MAY2013 11:37 | 1 | 1 | 0 | 1 | 11 |
| | | +20 mins | 14MAY2013 11:47 | 1 | 1 | 0 | 1 | 10 |
| | | +30 mins | 14MAY2013 11:57 | 1 | 1 | 0 | 1 | 9 |
| | | +60 mins | 14MAY2013 12:27 | 2 | 1 | 0 | 1 | 21 |
| | TV2 | Pre-dose | 21MAY2013 11:43 | 2 | 1 | 0 | 2 | 22 |

Continue with CVT-301 (Naïve)

<sup>\*</sup>indicates imputed item score. 18=Speech, 19=Facial Expression, 20=Tremor at Rest, 21=Action or Postural Tremor of hands, 22=Rigidity, 23=Finger Taps, 24=Hand Movements, 25=Rapid Alternating Movements of Hands, 26=Leg Agility, 27=Arising from Chair, 28=Posture, 29=Gait, 30=Postural Stability, 31=Body Bradykinesia and Hypokinesia.

Listing 16.2.6.1.2 Unified Parkinson's Disease Rating Scale (UPDRS) Part 3: Derived Variables

Treatment Group: CVT-301 (002/003)

| | | | | | Mean Change | | | |
|---|---|---|---|---|---|---|---|---|
| | | | UPDRS III | | from Pre-dose<br>at 10 to 60 | | | >=11<br>Reduction |
| Patient | | Time | Total | Change from | mins | >=3 Reduction | >=6 Reduction | from Pre- |
| ID | Visit | Point | Score | Pre-dose | Post-dose | from Pre-dose | from Pre-dose | dose |
| xxxx-xxx | TV2 | Pre-dose | XX | | XX | | | |
| | | +10mins | XX | XX | | | | |
| | | +20mins | XX | XX | | | Y | |
| | | +30mins | XX | XX | | Y | | Y |
| | | +60mins | XX | XX | | Y | | |
| | TV3 | Pre-dose | XX | | XX | | | |
| | | +10mins | XX | XX | | | | |
| | | +20mins | XX | XX | | | | |
| | | +30mins | XX | XX | | | | |
| | | +60mins | XX | XX | | | | |
| | TV4 | Pre-dose | XX | | XX | | | |
| | | +10mins | XX | XX | | | | |
| | | +20mins | XX | XX | | | | |
| | | +30mins | XX | XX | | | | |
| | | +60mins | XX | XX | | | | |
| XXXX-XXX | | | | | | | | |
| • • • | | | | | | | | |

Continue with CVT-301 (Naïve)

Note: TV = Treatment Visit; ET = Early Termination;

## Listing 16.2.6.2.1 Clinic Assessment

Treatment Group: Observational Cohort

| Patient<br>ID | Visit | Date of<br>Assessment | Time of Standard<br>Morning Dose of LD-<br>Containing<br>Medications | Motor<br>State at<br>Arrival | Time<br>Patient<br>Turned OFF | Turned ON within the 60-min Post Dose Period? | Was Patient ON at<br>60-min Post<br>Inhaled<br>Treatment? | Experience<br>Dyskinesia | Maximum<br>Severity |
|---|---|---|---|---|---|---|---|---|---|
| | 0111 | | | | | | | | |
| XXXX- | SV1 | 1.1 | 1. 1 | | | | | | |
| XXX | 27.70 | ddmonyyyy | hh:mm | | | | | | |
| | SV2 | Not Done,<br>xxxx | | | | | | | |
| | TV1 | ddmonyyyy | hh:mm | OFF | hh:mm | Yes | No | Yes | XXX |
| | | ddmonyyyy | hh:mm | OFF | hh:mm | Yes | Yes | No | |
| xxxx- | | | | | | | | | |
| XXX | | | | | | | | | |

Continue with CVT-301 (002/003), CVT-301 (Naïve)

Listing 16.2.6.2.2 Parkinson's Disease Diary Data

Treatment Group: Observational Cohort

| | | | | | ON without | ON with Non-troublesome | ON with Troublesome |
|---|---|---|---|---|---|---|---|
| Week | Date of Assessment | Assessment | Asleep | OFF | Dyskinesia | Dyskinesia | Dyskinesia |
| SV<br>TV3 | ddmonyyyy<br>Not Done, xxxx | hh:mm | | | | | |
| TV4 | ddmonyyyy | hh:mm | 1 | 0 | 0 | 0 | 0 |
| | ddmonyyyy | hh:mm | 1 | 0 | 0 | 0 | 0 |
| S<br>T | V<br>V3<br>V4 | V ddmonyyyy<br>V3 Not Done, xxxx<br>V4 ddmonyyyy | V ddmonyyyy hh:mm<br>V3 Not Done, xxxx<br>V4 ddmonyyyy hh:mm | V ddmonyyyy hh:mm V3 Not Done, xxxx V4 ddmonyyyy hh:mm 1 | V ddmonyyyy hh:mm<br>V3 Not Done, xxxx<br>V4 ddmonyyyy hh:mm 1 0 | V ddmonyyyy hh:mm<br>V3 Not Done, xxxx<br>V4 ddmonyyyy hh:mm 1 0 0 | V ddmonyyyy hh:mm<br>V3 Not Done, xxxx<br>V4 ddmonyyyy hh:mm 1 0 0 0 |

Continue with CVT-301 (002/003), CVT-301 (Naïve)

## Listing 16.2.6.2.3.1 Parkinson's Disease Diary Data - Derived Variable by Dairy Date

Treatment Group: Observational Cohort

| Patient<br>ID | Visit | Date of<br>Assessment | Daily Awake<br>Time (Hrs) | Daily OFF Time (Hrs)/<br>% of OFF time | Daily<br>ON Time<br>Without<br>Dyskinesia<br>(hours) | Daily ON Time With Non- troublesome Dyskinesia (hours) | Daily<br>ON Time With<br>Troublesome Dyskinesia<br>(hours) |
|---|---|---|---|---|---|---|---|
| xxxx- | SV | ddmonyyyy | х.х | x.x | х.х | x.x | x.x |
| XXX | TV2<br>TV3 | ddmonyyyy<br>ddmonyyyy | x.x<br>x.x | x.x<br>x.x | x.x<br>x.x | x.x<br>x.x | x.x |
| | TV4 | ddmonyyyy | х.х | x.x | x.x | x.x | x.x |

. . .

Continue with CVT-301 (002/003), CVT-301 (Naïve)

## Listing 16.2.6.2.3.2 Parkinson's Disease Diary Data - Derived Variable by Visit

Treatment Group: Observational Cohort

| | | | | | | Mean Daily<br>ON Time | | |
|---|---|---|---|---|---|---|---|---|
| Patient<br>ID | Visit | Date of<br>Assessment | Daily<br>Awake<br>Time<br>(Hrs) | Mean Daily OFF<br>Time (Hrs)/ %<br>of OFF time | Mean Daily<br>ON Time<br>Without<br>Dyskinesia<br>(hours) | With Non- troublesome Dyskinesia (hours) | Mean Daily<br>ON Time With<br>Troublesome<br>Dyskinesia<br>(hours) | Baseline Daily OFF<br>Time/ Category at<br>Screening |
| xxxx- | SV | ddmonyyyy | х.х | x.x | х.х | х.х | х.х | x.x /<4.5 hours |
| | TV2 | ddmonyyyy | x.x | X.X | х.х | X • X | | |
| | TV3 | ddmonyyyy | x.x | X.X | X.X | x.x | X.X | |
| | TV4 | ddmonyyyy | X.X | x.x | x.x | x.x | x.x | |
| xxxx- | | | | | | | | |
| XXX | | | | | | | | |

Continue with CVT-301 (002/003), CVT-301 (Naïve)

. . .

Listing 16.2.6.2.4 Patient's Global Impression of Change (PGI-C)

Treatment Group: Observational Cohort

| Patient | | Date and Time | Response | • |
|----------|-------|----------------|----------|---|
| ID | Visit | of Assessment | [a] | |
| xxxx-xxx | TV4 | ddmonyyyyhh:mm | х | |
| xxxx-xxx | TV4 | Ddmonyyyyhh:mm | х | |
| xxxx-xxx | | | | |
| • • • | | | | |

Note: TV = Treatment Visit; [a] 1 = Much Improved, 2 = Improved, 3 = A little Improved, 4 = No change, 5 = A little worse, 6 = Worse, 7 = Much worse.

Civitas Therapeutics, Inc. Page x of y Confidential

#### Protocol No. CVT-301-005

#### Listing 16.2.6.2.5 Impact of Parkinson's OFF Episodes

#### Time Spend in OFF Time:

- 1. Over the last week, on average... how many hours in the day are you typically awake?
- 2. Over the last week, on average... how many of your awake hours are typically in an OFF state?
- 3. Over the last week, on average... how many OFF episodes do you experience in a typical day?
- 4. Over the last week, on average... what is the typical duration of each OFF episode?

#### Functional Impact of OFF time

1. Over the last week, on average, when you experience an OFF episode, did it stop you from doing things?

#### Impact of OFF Time on Activities of Daily Living

- a. Motor and Physical
- 1. Had difficulty with housework or cooking?
- 2. Had difficult with work tasks like typing?
- 3. Had difficulty getting around in public?
- 4. Been confined to the house more than you would like?
- 5. Had difficulty washing/dressing yourself?
- 6. Felt Pain?
- 7. Had difficulty walking safely?
- b. Social and Cognitive
- 1. Felt depressed?
- 2. Felt anxious?
- 3. Had problems with concentration?
- 4. Felt memory was bad?
- 5. Felt unable to communicate properly?
- 6. Had trouble mentally changing from one task to another?
- c. Any other things you would like to share about your off time

#### Impact of OFF Time on Well-being and quality of Life

1. Over the last week, on average, how do OFF periods affect your overall feeling of health and well-being?

#### Impact of OFF Time on Disability

- 1. Over the last week, on an average day when you are in an ON state, you would rate your disability:
- 2. Over the last week, on an average day when experiencing OFF time, you would rate your disability:

# Listing 16.2.6.2.5 Impact of Parkinson's OFF Episodes

Treatment Group: Observational Cohort

| | | | | | | Impa | ct of | OFF | Time | on Ac | tivit: | ies o | f Dail | ly Liv | /ing | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Date of | Tim | ne Spend | in OFF T | 'ime | | Mo | otor a | and Ph | nysica | al | | | Socia | ıl and | l Cogn | itive | |
| Visit | Assessment | 1 | 2 | 3 | 4 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 1 | 2 | 3 | 4 | 5 | 6 |
| TV1 | ddmonyyyy | х | х | х | Х | х | Х | Х | х | Х | х | Х | Х | Х | Х | Х | х | Х |
| TV1 | | Х | Х | Х | Х | Х | Х | Х | Х | Х | х | Х | Х | х | х | х | Х | Х |
| | TV1 | Visit Assessment TV1 ddmonyyyy | Visit Assessment 1 TV1 ddmonyyyy x | Visit Assessment 1 2 TV1 ddmonyyyy x x | Visit Assessment 1 2 3 TV1 ddmonyyyy x x x | Visit Assessment 1 2 3 4 TV1 ddmonyyyy x x x x x | Date of Time Spend in OFF Time | Date of Time Spend in OFF Time Mc | Date of Visit Time Spend in OFF Time Motor of | Date of Time Spend in OFF Time Motor and Provided Motor and Prov | Date of Time Spend in OFF Time Motor and Physical | Date of Time Spend in OFF Time Motor and Physical | Date of Time Spend in OFF Time Motor and Physical | Date of Time Spend in OFF Time Motor and Physical | Date of Visit Time Spend in OFF Time Motor and Physical Social Visit Assessment 1 2 3 4 1 2 3 4 5 6 7 1 2 TV1 ddmonyyyy x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x | Visit Assessment 1 2 3 4 1 2 3 4 5 6 7 1 2 3 TV1 ddmonyyyy x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x <td>Date of Visit Time Spend in OFF Time Motor and Physical Social and Cogn Visit Assessment 1 2 3 4 1 2 3 4 5 6 7 1 2 3 4 TV1 ddmonyyyy x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x <t< td=""><td>Date of Visit Time Spend in OFF Time Notor and Physical Social and Cognitive Notation Motor and Physical Social and Cognitive Notation TV1 ddmonyyyy x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x<!--</td--></td></t<></td> | Date of Visit Time Spend in OFF Time Motor and Physical Social and Cogn Visit Assessment 1 2 3 4 1 2 3 4 5 6 7 1 2 3 4 TV1 ddmonyyyy x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x <t< td=""><td>Date of Visit Time Spend in OFF Time Notor and Physical Social and Cognitive Notation Motor and Physical Social and Cognitive Notation TV1 ddmonyyyy x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x<!--</td--></td></t<> | Date of Visit Time Spend in OFF Time Notor and Physical Social and Cognitive Notation Motor and Physical Social and Cognitive Notation TV1 ddmonyyyy x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x </td |

Note: TV = Treatment Visit;

Programming note: The actual listing started with new page

# Listing 16.2.6.2.5 Impact of Parkinson's OFF Episodes

Treatment Group: Observational Cohort

| Patient<br>ID | Visit | Date of<br>Assessment | Functional Impact of OFF time | Impact of OFF Time on<br>Well-being<br>and Quality of Life | Impact of OFF T | ime on Disability | Any other things you would like to share about your OFF time |
|---|---|---|---|---|---|---|---|
| xxxx-xxx<br>xxxx-xxx | TV1<br>TV1 | ddmonyyyy | x<br>x | x<br>x | x<br>x | x<br>x | xxxx |

#### CONTIGENCIA

# Listing 16.2.6.3.1 Unified Parkinson's Disease Rating Scale (UPDRS) Part 2

Treatment Group: Observational Cohort

| Patient<br>ID | Visit | Date Of<br>Assessment | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | Total<br>Score | Change<br>from<br>Baseline |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxx- | TV1 | ddmonyyyy | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| | TV4 | Not Done,<br>xxx | | | | | | | | | | | | | | | |
| | • • • | | | | | | | | | | | | | | | | |
| xxxx- | TV1 | ddmonyyyy | Х | Х | Х | X | X | X | Х | X | X | X | X | Х | X | X | Х |
| XXX | TV4 | ddmonyyyy | х | х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |

Continue with CVT-301 (002/003), CVT-301 (Naïve)

Note: TV = Treatment Visit; ET = Early Termination;

5=Speech, 6=Salivation, 7=Swallowing, 8=Handwriting, 9=Cutting food and handling utensils, 10=Dressing, 11=Hygiene, 12=Turning in bed and adjusting bed clothes, 13=Falling(unrelated to freezing), 14=Freezing when walking, 15=Walking, 16=Tremor(Symptomatic complaint of tremor in any part of body), 17=Sensory complaints related to parkinsonism.

# Listing 16.2.6.3.2 Listing of S&E Activities of Daily Living

Treatment Group: Observational Cohort

| ID | Visit | Date of Assessment | Rating Description of ADL capability |
|----------|-------|--------------------|--------------------------------------|
| xxxx-xxx | TV1 | ddmonyyyy | х |
| | TV4 | ddmonyyyy | Х |
| xxxx-xxx | TV1 | ddmonyyyy | Х |
| | TV4 | Not Done, xxxxxxxx | |
| xxxx-xxx | | | |

Note: TV = Treatment Visit; ET = Early Termination;


Listing 16.2.6.3.3
39 Item Parkinson's Disease Questionnaire (PDQ-39)

Treatment Group: Observational Cohort

| | | Date and | | | | | | | Mobil | ity | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient<br>ID | Visit | Time of<br>Assessment | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | Dimension<br>Score |
| xxxx-xxx | TV1<br>TV4 | ddmonyyyyhh:mm<br>Not Done, xxxxx | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | х |
| xxxx-xxx | • • • | | | | | | | | | | | | |
| <br>Continue with | CVT-301 (002 | /003), CVT-301 (Naïve) | | | | | | | | | | | |

Note: SV = Screening Visit; TV = Treatment Visit; ET = Early Termination; UNS = Unscheduled; The assessments on TV1 were taken prior to study medication application.

# Listing 16.2.6.3.3 39 Item Parkinson's Disease Questionnaire (PDQ-39)

Treatment Group: Observational Cohort

| | | Date and | | Activities of Daily Living | | | | | | | | Emotional Well-being | | | | g |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient<br>ID | Visit | Time of<br>Assessment | 11 | 12 | 13 | 14 | 15 | 16 | Dimension<br>Score | 17 | 18 | 19 | 20 | 21 | 22 | Dimension<br>Score |
| xxxx-xxx | TV1<br>TV4 | ddmonyyyyhh:mm<br>Not Done, xxxxx | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| xxxx-xxx Continue wi | <br>ith CVT-30 | 1 (002/003), CVT-301 ( | Naïve) | | | | | | | | | | | | | |

Note: SV = Screening Visit; TV = Treatment Visit; ET = Early Termination; UNS = Unscheduled; The assessments on TV1 were taken prior to study medication application.

## Listing 16.2.6.3.3 39 Item Parkinson's Disease Questionnaire (PDQ-39)

Treatment Group: Observational Cohort

| | | Date and | | | S | tigma | | | Soc | cial S | upport | | | Со | gnitio | ns |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient | | Time of | | | | | Dimension | | | | Dimension | | | | | Dimension |
| ID | Visit | Assessment | 23 | 24 | 25 | 26 | Score | 27 | 28 | 29 | Score | 30 | 31 | 32 | 33 | Score |
| xxxx-xxx | TV1<br>TV4 | ddmonyyyyhh:mm<br>Not Done, xxxxx | Х | х | х | Х | х | х | х | Х | Х | Х | Х | Х | х | Х |
| xxxx-xxx | • • • | | | | | | | | | | | | | | | |
| <br>Continue w | ith CVT-3 | 301 (002/003), CVT-30 | 1 (Naï | ve) | | | | | | | | | | | | |

Note: SV = Screening Visit; TV = Treatment Visit; ET = Early Termination; UNS = Unscheduled; The assessments on TV1 were taken prior to study medication application.

# Listing 16.2.6.3.3 39 Item Parkinson's Disease Questionnaire (PDQ-39)

Treatment Group: Observational Cohort

| | | Date and | | Co | ommunic | ation | | Bodi | ly Dis | comfort | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient | | Time of | | | | Dimension | | | | Dimension | |
| ID | Visit | Assessment | 34 | 35 | 36 | Score | 37 | 38 | 39 | Score | Summary Index Score |
| xxxx-xxx | TV1<br>TV4 | ddmonyyyyhh:mm<br>Not Done, xxxxx | Х | Х | Х | Х | Х | Х | Х | х | х |
| xxxx-xxx | • • • | | | | | | | | | | |
| <br>Continue wi | th CVT-301 | 1 (002/003), CVT-301 ( | Naïve) | | | | | | | | |

Note: TV = Treatment Visit; ET = Early Termination; UNS = Unscheduled; The assessments on TV1 were taken prior to study medication application.

Listing 16.2.7.1 Adverse Events

Treatment Group: Observational Cohort

| Patient<br>ID | System Organ Class/<br>Preferred Term/<br>Verbatim Term [a] | AE Start<br>Date<br>and Time/<br>Study Day<br>[b] | AE Stop Date<br>and Time | I: Intensity R: Relationship to Study Medication A: Action Taken | Outcome | SAE? If Yes,<br>Specify [c] |
|---|---|---|---|---|---|---|
| | xxxxxxxxx/ | ddmonyyyy | | I: xxxxxxxx | | |
| | xxxxxxxx/ | hh:mm/ | ddmonyyyy | R: xxxxxxxx | | |
| XXX-XXX | xxxxxxxx | -xx | Hh:mm | A: xxxxxxxxx | Resolved | Yes: 1 |
| | xxxxxxxxx/ | ddmonyyyy | | I: xxxxxxxx | | |
| | xxxxxxxx/ | hh:mm/ | | R: xxxxxxxx | | |
| | xxxxxxxx | xx# | Ongoing | A: xxxxxxxxx | Unknown | No |
| | xxxxxxxxx/ | ddmonyyyy | | I: xxxxxxxx | | |
| | xxxxxxxx/ | hh:mm/ | ddmonyyyy | R: xxxxxxxx | | |
| | | -xx | Hh:mm | A: xxxxxxxxx | Resolved | Yes: 2 |

Continue with CVT-301 (002/003), CVT-301 (Naïve)

Notes: TEAE=Treatment-emergent AE. SAE=Serious AE.[a] Adverse events were coded into system organ class and preferred term using MedDRA version 17.0.

<sup>[</sup>b] TEAEs were flagged with a #. The AEs occurred on the clinic visit were flagged with \*.Study day is relative to date of first study medication (date of first dose = Day 1).

<sup>[</sup>c] 1 = The event is fatal or life-threatening, 2 = The event is permanently disabling (incapacitating or interfering with the ability to resume usual life patterns), 3 = The event results in unplanned inpatient hospitalization or prolongation of existing hospitalization, 4 = The event is a congenital anomaly, 5 = The event requires medical intervention of any kind in order to prevent any of the aforementioned outcomes.

# Listing 16.2.8.1.1 Clinical Laboratory Results - Hematology

Treatment Group: Observational Cohort

| Patient<br>ID | Visit | Date and Time<br>of Sample | Test1<br>unit | Test2<br>unit | Test3<br>unit | ••• |
|---|---|---|---|---|---|---|
| xxxx-xxx | SV1 | ddmonyyyyhh:mm | xx H* | xx L* | xx | |
| | TV1<br>TV4 | ddmonyyyyhh:mm<br>Not Done, xxxxx | xx<br>xx H** | xx<br>xx H** | XX<br>XX | |

XXXX-XXX

Continue with CVT-301 (002/003), CVT-301 (Naïve)

Note: SV = Screening Visit; TV=Treatment Visit; FU= Follow-up; UNS= unscheduled; L = Low, H = High,  $L^* = potentially clinically significant (PCS) low value, <math>H^* = PCS$  high value,  $L^{**}$  = potentially clinically significant change (PCSC) low,  $H^{**}$  = PCSC high.

## Below listing will has similar structure as Listing 16.2.8.1.1

Listing 16.2.8.1.2 Clinical Laboratory Results - Chemistry

Listing 16.2.8.1.3 Serum Pregnancy Test - Positive Only

Treatment Group: Observational Cohort

| Patient<br>ID | Visit | Date and Time<br>of Sample | Result |
|---|---|---|---|
| xxxx-xxx | SV1<br>TV1 | ddmonyyyyhh:mm<br>ddmonyyyyhh:mm | Positive<br>Positive |
| xxxx-xxx | SV1 | | |
| xxxx-xxx | SV1 | | |
| | • • • | | |

Continue with CVT-301 (002/003), CVT-301 (Naïve)

Note: SV = Screening Visit; TV=Treatment Visit; FU= Follow-up; UNS= unscheduled; At home pregnancy tests and an extra serum pregnancy test at TV2 visit will be performed for the CVT treated patients in Belgium and Germany.

Listing 16.2.8.2.1

Vital Signs

Treatment Group: Observational Cohort

| Patient | | | Date and Time | | | Pressure<br>mHg) | Heart Rate | Respiration Rate |
|---|---|---|---|---|---|---|---|---|
| ID | Visit | Time Point | Of Assessment | Position | SBP | DBP | (beats per minute) | (breaths per minute) |
| xxxx-xxx | SV1 | | ddmonyyyyhh:mm | Standing<br>Supine/Semi-<br>Supine | XX | xx | xx | xx |
| | TV1 | Pre-dose<br>+5mins | ddmonyyyyhh:mm | | xx<br>xx H* | xx<br>xx L** | xx<br>xx | xx<br>xx |
| | | | Not Done, xxxxx | | | | | |
| xxxx-xxx | | | | | | | | |

Note: SV = Screening Visit; TV=Treatment Visit; FU= Follow-up; UNS= unscheduled;
L\* = potentially clinically significant (PCS) low value, H\* = PCS high value,
L\*\* = potentially clinically significant change (PCSC) low, H\*\* = PCSC high.

Listing 16.2.8.2.2 12-Lead Electrocardiogram (ECG)

Treatment Group: Observational Cohort

| Patient<br>ID | Visit | Time Point | Date and Time<br>Of Assessment | Heart<br>Rate<br>(bpm) | RR<br>(ms) | PR<br>(ms) | QRS<br>(ms) | QT<br>(ms) | QTcB<br>(ms) | QTcF<br>(ms) | Result |
|---|---|---|---|---|---|---|---|---|---|---|---|
| xxx-xxx | SV1<br>TV1 | Pre-dose<br>+5mins<br>+20mins<br>+30mins | ddmonyyyyhh:mm<br>ddmonyyyyhh:mm<br>Not Done | xx<br>xx<br>xx | xx<br>xx<br>xx | XX<br>XX<br>XX L** | xx<br>xx<br>xx | XX<br>XX<br>XX H** | xx<br>xx<br>Xx | xx<br>xx<br>xx | Normal<br>Normal<br>Abnormal CS<br>Abnormal NCS |

xxxx-xxx

Continue with CVT-301 (002/003), CVT-301 (Naïve)

Note: SV = Screening Visit; TV=Treatment Visit; FU= Follow-up; UNS= unscheduled; L\* = potentially clinically significant (PCS) low value, H\* = PCS high value, For PR interval, H1= PCSC high, >25% for baseline >=200; H2= PCSC high, >25% for baseline >=200; For QRS interval, H1= PCSC high, >25% for baseline >=100; H2= PCSC high, >25% for baseline >=100; For QTcB and QTcF, H1\*\*=PCSC high, >15% for baseline >=440; H2\*\*=PCSC high, >30% for baseline <440; H3\*\*=PCSC high, Increase>30; H4\*\*=PCSC high, Increase>60, H5\*\*=PCSC high Change>30 and Value>500, H6\*\*=PCSC high, Change>60 and Value>500

Listing 16.2.8.2.3 Physical Examination

Treatment Group: Observational Cohort

| Patient | | Date of | Any Clinically Significant<br>Abnormal Findings<br>That | |
|---|---|---|---|---|
| ID | Visit | Assessment | Are New or Have Worsened? | Findings |
| xxxx-xxx | SV1<br>SV2<br>TV1 | ddmonyyyy<br>Not Done<br>ddmonyyyy | Yes | New or Worsened Clinically Significant |
| xxxx-xxx<br> | | | | |

Continue with CVT-301 (002/003), CVT-301 (Naïve)

SV = Screening Visit; TV=Treatment Visit; FU= Follow-up; UNS= unscheduled; [a] BMI was calculated as weight (kg) / [height (m)]^2.

Listing 16.2.8.2.4.1 Spirometry( Neurology Office)

Treatment Group: Observational Cohort

| Patient<br>ID | Visit | Time<br>Point | Motor<br>State | Date and Time of Assessment | FEV1<br>(Liter) | FEV1<br>(% Predicted) | FVC<br>(Liter) | FVC<br>(% Predicted) | FEV1/FVC (%) |
|---|---|---|---|---|---|---|---|---|---|
| xxxx-xxx@ | Screening | | ON | ddmonyyyyhh:mm | XX | xx | XX | XX | XX |
| | TV1 | Arrival | ON | ddmonyyyyhh:mm # | XX | XX | XX | XX | XX |
| | | Pre-dose | | ddmonyyyyhh:mm | XX | XX | XX | XX | XX |
| | | +15mins | | ddmonyyyyhh:mm | Xx * | Xx \$ | XX | XX | XX |
| | | | | Not Done, xxx | | | | | |

xxxx-xxx

Continue with CVT-301 (002/003), CVT-301 (Naïve)

Note: SV = Screening Visit; TV = Treatment Visit; # indicates spirometry measurement not meeting ATS quality criteria. \* indicates imputed values. \$ indicates manual data @ indicates patients with Co-efficient of Variation (CV) of FEV1 >7.5%

Listing 16.2.8.2.4.2 Spirometry ( Neurology Office) Measurements Not Meeting ATS Quality Criteria

Treatment Group: Observational Cohort Patient Motor Date and Time ID Visit Point State of Assessment Acceptable Efforts Repeatable Efforts ON exxx-xxxx SV ddmonyyyyhh:mm # Х Х Arrival ON ddmonyyyyhh:mm # TV1 Х Х Pre-dose ddmonyyyyhh:mm # Х Х . . .

xxxx-xxx

Continue with CVT-301 (002/003), CVT-301 (Naïve)

Note: TV = Treatment Visit; # indicates spirometry measurement not meeting ATS quality criteria. @ indicates patients with Coefficient of Variation (CV) of FEV1 >7.5%

Listing 16.2.8.2.4.3 Spirometry(Pulmonary Function Facility): DLco Parameters

Treatment Group: Observational Cohort

| Patient | | Time | Motor | Date and Time | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ID | Visit | Point | State | of Assessment | 1/20/21 | 2 | 3 | 4(13)/7(15) | 5(14)/8(16) | 6/9 | 10 | |
| xxxx-xxx@ | Screening | | ON | ddmonyyyyhh:mm | | | | XX | xx | xx | XX | XX |
| | TV1 | Arrival | ON | <pre>ddmonyyyyhh:mm #</pre> | | | | XX | XX | XX | XX | XX |
| | | Pre-<br>dose | | ddmonyyyyhh:mm | | | | XX | XX | XX | XX | XX |
| | | +15mins | | ddmonyyyyhh:mm | | | | Xx * | Xx \$ | XX | XX | XX |
| | | | | Not Done, xxx | | | | | | | | |

xxxx-xxx

Continue with CVT-301 (002/003), CVT-301 (Naïve)

Note: SV = Screening Visit; TV = Treatment Visit; # indicates spirometry measurement not meeting ATS quality criteria. \$ indicates manual data @ indicates patients with Co-efficient of Variation (CV) of FEV1 >7.5%; 1=DLCO (mL/min/mmHg), 2=IVC (L), 3=VA (L), 4=Pre Original FEV1 (L), 5=Pre Original FVC (L), 6=Pre FEV1/FVC (%),7=Post Original FEV1, 8=Post Original FVC, 9=Post FEV1/FVC (%),10=SVC (L), 13=Percentage Predicted Pre-FEV1 (%),14=Percentage Predicted Pre-FVC (%), 15=Percentage Predicted Post-FEV1 (%), 16=Percentage Predicted Post-FVC (%), 20=Percentage Predicted DLCO (%)

Listing 16.2.8.2.4.4

Spirometry(Pulmonary Function Facility): Spirometry/DLco Measurements Not Meeting ATS Quality Criteria

Will have same format as L16.2.8.2.4.3 and removed the irrelevant columns (Motor State, Repeatable Efforts and Acceptable Efforts)

# indicates DLco measurement not meeting ATS quality criteria.

Listing 16.2.8.2.5
Columbia-Suicide Severity Rating Scale (C-SSRS)

# Suicide Ideation: 1.Wish to be Dead 2.Non-Specific Suicidal Thought 3.Suicidal Ideation-No Intent 4. Ideation With Intent, No Plan 5. Ideation With Plan/Intent Intensity of Ideation: 1.Most Severe Ideation 2.Most Severe Ideation, Description 3.Most Severe Ideation, Frequency 4.Most Severe Ideation, Duration 5.Most Severe Ideation, Control 6.Most Severe Ideation, Deterrents 7.Most Severe Ideation, Reasons Suicidal Behavior: 1.Actual Attempt 2.Number of Actual Attempts 3.Non-suicidal Self-injurious Behavior 4.Interrupted Attempt 5.Number of Interrupted Attempts 6.Aborted Attempt 7.Number of Aborted Attempts 8.Preparatory Acts/Behavior 9.Suicidal Behavior 10.Completed Suicide Actual Attempts: 1.Most Recent Attempt Date 2.Most Recent Attempt Damage 3.Most Recent Attempt Potential 4.Most Lethal Attempt Date 5.Most Lethal Attempt Damage 6.Most Lethal Attempt Potential 7.First Attempt Date

8.First Attempt Damage 9.First Attempt Potential

# Listing 16.2.8.2.5 Columbia-Suicide Severity Rating Scale (C-SSRS)

Treatment Group: Observational Cohort

| Patient | | Date of | | Suicide Ideation | | | | | | | Intensity of Ideation | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ID | Visit | Assessment | 1 | 2 | 3 | 4 | 5 | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| xxxx-xxx | TV1 | ddmonyyyy | | | | | | | | | | | | |

xxxx-xxx

. . .

Continue with CVT-301 (002/003), CVT-301 (Naïve)

Note: TV = Treatment Visit;

Programming note: The actual listing started with new page

Not Done, xxxxxx

# Listing 16.2.8.2.5 Columbia-Suicide Severity Rating Scale (C-SSRS)

Treatment Group: Observational Cohort

| Patient | | Date of | Suicidal Behavior | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ID | Visit | Visit Assessment | | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | VISIC | 1155C55MC11C | ± | | | | | - | | | | |

TV1 ddmonyyyy xxx-xxx TV4 Not Done, xxxxxx

xxxx-xxx

Continue with CVT-301 (002/003), CVT-301 (Naïve)

Not Done, xxxxxx


Listing 16.2.8.2.5 Columbia-Suicide Severity Rating Scale (C-SSRS)

Treatment Group: Observational Cohort

| Patient | | Actual Attempts | | | | | | | | | |
|----------|-------|-----------------|---|---|---|---|---|---|---|---|---|
| ID | Visit | Assessment | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 |
| xxxx-xxx | TV1 | ddmonyyyy | | | | | | | | | |

xxx-xxx

Continue with CVT-301 (002/003), CVT-301 (Naïve)

TV4


Listing 16.2.8.2.6
Epworth Sleepiness Scale

Treatment Group: Observational Cohort

| Patient<br>_ID | Visit | Date of<br>Assessment | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | Total<br>Score |
|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxx-xxx | TV1<br>TV4 | ddmonyyyy<br>Not Done, xxxxxxx | xx | XX | xx | xx | xx | XX | xx | XX | xx |

xxxx-xxx

. . .

Continue with CVT-301 (002/003), CVT-301 (Naïve)

Note: TV = Treatment Visit; 1 = Sitting and reading, 2 = Watching TV, 3 = Sitting inactive in a public place, 4 = As a passenger in a car for an hour

without a break, 5 = Lying down to rest in the afternoon when circumstances permit, 6 = Sitting and talking to someone, 7 = Sitting quietly after a lunch without alcohol, 8 = In a car, while stopped for a few minutes in traffic.

Listing 16.2.8.2.7 Questionnaire for Impulsive-Compulsive Disorders in Parkinson's (QUIP)

Treatment Group: Observational Cohort

| | | | Impulse control disorders | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient | | Date of | 1. | 1. | 1. | 1. | 2. | 2. | 2. | 2. | 3. | 3. |
| ID | Visit | Assessment | Gambling | Sex | Buying | Eating | Gambling | Sex | Buying | Eating | Gambling | Sex |
| xxx-xxx | TV1<br>TV4 | ddmonyyyy Not Done, xxxxxxx | Yes | No | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes |

xxxx-xxx

Continue with CVT-301 (002/003), CVT-301 (Naïve)

Confidence

# 

Treatment Group: Observational Cohort

| | | | Impulse control disorders | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient<br>ID | Visit | Date of<br>Assessment | 3.<br>Buying | 3.<br>Eating | 4.<br>Gambling | 4.<br>Sex | 4.<br>Buying | 4.<br>Eating | 5.<br>Gambling | 5.<br>Sex | 5.<br>Buying | 5.<br>Eating |
| xxxx-xxx | TV1<br>TV4 | ddmonyyyy<br>Not Done,<br>xxxxxxx | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes |

XXXX-XXX

Continue with CVT-301 (002/003), CVT-301 (Naïve)

Listing 16.2.8.2.7 Questionnaire for Impulsive-Compulsive Disorders in Parkinson's (QUIP)

Treatment Group: Observational Cohort

| | | | | Compulsive medication use | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient<br>_ID | Visit | Date of<br>Assessment | 1A | 1B | 1C | 2 | 3 | 1 | 2 | 3 | 4 | 5 |
| xxx-xxx | TV1<br>TV4 | ddmonyyyy<br>Not Done,<br>xxxxxxx | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes |

xxxx-xxx

Continue with CVT-301 (002/003), CVT-301 (Naïve)
Civitas Therapeutics, Inc.

Page x of y


# Listing 16.2.8.2.8.1 Unified Parkinson's Disease Rating Scale (UPDRS) Part 4

#### Dyskinesias:

- 32. Duration: What proportion of the waking day are dyskinesias present?
- 33. Disability: How disabling are the dyskinesias?
- 34. Painful Dyskinesias: How painful are the dyskinesias?
- 35. Presence of Early Morning Dystonia.

#### Clinical Fluctuations:

- 36. Are "off" periods predictable?
- 37. Are "off" periods unpredictable?
- 38. Do "off" periods come on suddenly, within a few seconds?
- 39. What proportion of the waking day is the patient "off" on average?

#### Other Complications:

- 40. Does the patient have anorexia, nausea, or vomiting?
- 41. Any sleep disturbances, such as insomnia or hypersomnolence?
- 42. Does the patient have symptomatic orthostasis?

Listing 16.2.8.2.8.1

Unified Parkinson's Disease Rating Scale (UPDRS) Part 4

Treatment Group: Observational Cohort

| | | | Dyskinesias | | | Clinical Fluctuations | | | Other Complications | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient<br>ID | Visit | Date Of Assessment | 32 | 33 | 34 | 35 | 36 | 37 | 38 | 39 | 40 | 41 | 42 |
| xxxx-xxx | TV1<br>TV4 | ddmonyyyy<br>Not Done, xxx | Х | Х | Х | Х | Х | Х | Х | Х | х* | х | Х |
| xxx-xxx | TV1<br>TV4 | ddmonyyyy<br>ddmonyyyy | x<br>x | x<br>x | X<br>X | x<br>x | x<br>x | x*<br>x | x<br>x | x<br>x | x<br>x | х<br>х* | x<br>x |

Continue with CVT-301 (002/003), CVT-301 (Naïve)

Note: Note: SV = Screening Visit; TV = Treatment Visit; ET = Early Termination; UNS = Unscheduled;


Listing 16.2.8.2.8.2 Unified Parkinson's Disease Rating Scale (UPDRS) Part 4: Derived Variables

Treatment Group: Observational Cohort

| Patient ID | Score Category | Visit | Change from<br>Baseline | Percent change from<br>Baseline |
|---|---|---|---|---|
| xxxx-xxx | Total Score | TV1 | | |
| | | TV4 | xx | xx.xx |
| | Dyskinesias | TV1 | | |
| | | TV4 | xx | xx.xx |
| | Clinical Fluctuations | TV1 | | |
| | | TV4 | xx | XX.XX |
| xxxx-xxx | | | | |

Continue with CVT-301 (002/003), CVT-301 (Naïve)

Note: SV = Screening Visit; TV = Treatment Visit; ET = Early Termination; UNS = Unscheduled;

Civitas Therapeutics, Inc.

Page x of y


#### Listing 16.2.8.2.9.1 Telephone Contact

Treatment Group: Observational Cohort

| Patient<br>ID | Date of Contact | Any Changes to PD Medications? | Any Challenges with<br>Inhaler or Capsules? | Any Challenges<br>with Diary? | Any Adverse Events<br>Noted? |
|---|---|---|---|---|---|
| xxxx-xxx | ddmonyyyy | Yes | No | No | Yes |
| | ddmonyyyy | Yes | Yes, xxxxxxxxxx | Yes, xxxxxxxxxx | Yes |
| XXXX-XXX | | | | | |

# Listing 16.2.8.2.9.2 Telephone Contact: Challenges with Inhaler or Capsules Data

Treatment Group: Observational Cohort

| Patient<br>ID | Date of Contact | Any Changes to PD Medications? | Any Challenges with<br>Inhaler or Capsules? | Any Challenges with Diary? | Any Adverse Events<br>Noted? |
|---|---|---|---|---|---|
| xxx-xxx | ddmonyyyy<br>ddmonyyyy | No<br>Yes | Yes, xxxxxxxxx<br>Yes, xxxxxxxxx | No<br>Yes, xxxxxxxxxx | Yes<br>Yes |
| xxx-xxx<br>••• | ••• | | | | |
| Continue wit | h CVT-301 (002/003), CV | T-301 (Naïve) | | | |

1003805 Acorda Therapeutics, Inc. CVT-301-005

Final Version 2.0



| CVT-301-005 |
|---|
| Summary of SAP Changes From final Version 1.0 (22-Dec-2015) to Version 2.0 (13Jan2017) |
| SAP final version 2.0 (13Jan2017) |
| Cover page: |
| CVT-301-005 A Phase 3, Randomized Study Investigating the Safety of CVT-301 (Levodopa Inhalation Powder) in Parkinson's Disease Patients With Motor Response Fluctuations (OFF Phenomena) Compared to an Observational Cohort Control |
| Protocol Version and Date: Version 4.0, 07-Mar-2016 |
| SAP version and date: Final version 2.0, 13-Jan-2017 |
| 3.5 Determination of Sample Size |
| Approximately 350 CVT-301 treatment patients and 175 control patients will be enrolled in this study. |



| T1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | |
|---|---|
| The primary objective of this study will be to characterize the | |
| pulmonary safety within the CVT-301-treated patients and the | |
| differences between the groups will be estimated as a | |
| secondary objective. However, for the secondary comparison | |
| of FEV1 change between the CVT-301 treatment group and | |
| the randomized observational cohort, the standard deviation | |
| of FEV1 change from baseline is expected to be 0.281 L, | |
| based on data from Study CVT-301-003. Assuming that there | |
| is no difference in the changes from baseline between the | |
| CVT-301-treated patients and the observational cohort, the | |
| study has the following power for the comparison between | |
| the 2 groups. The upper limit of the 95% confidence interval | |
| for the difference between the 2 groups in change from | |
| baseline in FEV1 will be less than 0.121 L with 90% power, | |
| assuming 188 and 86 patients completing the study in the | |
| CVT-301 treatment group and observational cohort, | |
| respectively. The sample size calculation was performed | |
| using nQuery Advisor, Version 7.0. | |
| | 3.6 Treatment Assignment & Blinding |
| | Add sentence below: |
| | Randomization can occur before the baseline DLco has been |
| | performed. Note: Patients who were enrolled from the CVT- |
| | 301-002 and CVT-301-003 studies under an earlier version of |
| | this protocol (Version 2) were assigned only to the CVT-301 |
| | treatment group. |
| 5.2 Safety population | 5.2 Safety population |
| The Safety Population will include all randomized | The Safety Population will include all randomized |



# Statistical Analysis Plan

patients who received at least 1 dose of inhaled CVT-301 and patients from the Observational Cohort. Patients will be analyzed according to study treatment that they received. The Safety Population will be used for all analyses of safety endpoints and summaries of patient demographics and baseline characteristics.

patients who received at least 1 dose of inhaled CVT-301 and patients from the Observational <u>Cohort who came</u> <u>in for treatment visit 1.</u> Patients will be analyzed according to study treatment that they received. The Safety Population will be used for all analyses of safety endpoints and summaries of patient demographics and baseline characteristics.

#### 6.2 Key Definitions

### DLCO predicted

DLCO predicted will be calculated by Miller equation. (Miller A, Thornton JC, Warshaw R, Anderson H, Teirstein AS, Selikoff IJ. Single breath diffusing capacity in a representative of Michigan, a large industrial state. Am Rev Resp Dis 1983; 127: 270-277).

- Men predicted DLCO = 12.9113 (0.229 x age) + (0.418 x height in)
- Women predicted DLCO = 2.2382 (0.1111 x age) + (0.4068 x height in)

Where age is the age at the time of assessment taken,

### 6.2 Key Definitions

### DLCO predicted

DLCO predicted will be calculated by Miller equation. (Miller A, Thornton JC, Warshaw R, Anderson H, Teirstein AS, Selikoff IJ. Single breath diffusing capacity in a representative of Michigan, a large industrial state. Am Rev Resp Dis 1983; 127: 270-277).

- Men predicted DLCO = 12.9113 (0.229 x age) + (0.418 x height in)
- Women predicted DLCO = 2.2382 (0.1111 x age) + (0.4068 x height in)

Where age is the age <u>at baseline</u>, height is measured in



| | 1 |
|---|---|
| height is measured in inches. | inches. |
| 8.1 Spirometry | 8.1 Spirometry |
| Spirometry will be performed by trained and qualified staff at each study site. Spirometry data obtained in the study site will reviewed by a central spirometry laboratory (Biomedical Systems, Inc.) which will provide a quality over read of all evaluations based on acceptability and repeatability metrics in accordance with ATS criteria. FEV1, FVC and FEV1/FVC ratio will be recorded from the single "best test" (based on effort with highest summed FEV1 and FVC). Variables will include the absolute FEV1, FVC, and FEV1/FVC ratio and FEV1 and FVC expressed as % of predicted value. | Spirometry will be performed by trained and qualified staff at each study site. Spirometry data obtained in the study site will reviewed by a central spirometry laboratory (Biomedical Systems, Inc.) which will provide a quality over read of all evaluations based on acceptability and repeatability metrics in accordance with ATS criteria. FEV1, FVC and FEV1/FVC ratio will be recorded from the single "best test" (based on effort with highest summed FEV1 and FVC). Variables will include the absolute FEV1, FVC, and FEV1/FVC ratio and FEV1 and FVC expressed as % of predicted value. |
| FEV1, FVC, FEV1/FVC ratio and DLco will be summarized descriptively by treatment group and overall. For screening data, the summary will be presented for each motor status, ON or OFF, separately. For other visits, data in ON or OFF state will be combined for summary. The following will be summarized: | The variables from pulmonary laboratory will include the FEV1, FVC, FEV1/FVC ratio, DLCO, IVC, SVC and VA. FEV1 and FVC expressed as % of predicted value, predicted DLCO, hemoglobin (Hb) adjusted predicted DLCO, and DLCO expressed as % of these predicted values will be calculated per the method in section 6.2. The following analysis will be performed: |
| • Change from baseline to other visits Arrival values for each parameter. The baseline is defined as the | All the parameters collected at the pulmonary laboratory as well as the % of predicted DLCO and % |

1003805 Acorda Therapeutics, Inc. CVT-301-005




# Statistical Analysis Plan

TV/OV1 Arrival value. If the TV/OV1 Arrival value is missing, the last available value in ON state before the first dose of study drug will be used.

- Number and percentage of patients with FEV1/FVC < 60% and <70% by Visit</li>
- Spirometry data will also be provided to indicate whether specific determinations met American Thoracic Society (ATS) quality criteria. The proportion of spirometry data measurements meeting or not meeting ATS quality criteria will be summarized by treatment group and overall. The summary will also be performed for ON state measurements, OFF state measurements, and all measurements, separately. The reasons for not meeting ATS quality criteria will be classified as not meeting the criteria for acceptability, not meeting the criteria for other/unknown repeatability or as and summarized.

<u>The spirometry analyses</u> will be repeated for the subset of assessments meeting the ATS quality criteria.

Another subset analysis will be performed by excluding the *spirometry* data from ...

In addition to the descriptive statistics, the changes in the

of Hb adjusted predicted DLCO will be summarized descriptively by treatment group and overall.

- Change from baseline to other visits for each parameter. The summary for FEV1 will also be provided by smoker status.
- Number and percentage of patients with FEV1/FVC < 60% and <70% by Visit</li>
- <u>DLCO</u> data will also be provided to indicate whether specific determinations met American Thoracic Society (ATS) quality criteria. The proportion of <u>DLCO/</u>spirometry data measurements meeting or not meeting ATS quality criteria will be summarized by treatment group and overall.
- Categories of changes (<-50%, -50% -<-40%, -40% -</p>
  <-30%, , -30% -<-20%, , -20% -<-10%, -10% -<-10%,</p>
  10% -<20% , 20% -<30% , 30% -<40% , 40% -<50%,</p>
  >=50%) from baseline for FEV1, FEV, FEV1/FVC
  ratio and DLCO by visit. The summary for FEV1
  will also be provided by smoker status.

<u>The descriptive summaries</u> will be repeated for the subset of assessments meeting the ATS quality criteria.

Another subset analysis will be performed by excluding the *DLCO* data from ...

1003805 Acorda Therapeutics, Inc. CVT-301-005




| <u>spirometry</u> values within | In addition to the descriptive statistics, the changes in the <i>FEV1</i> , <i>FEV1/FVC ratio</i> , <i>and DLCO</i> values within |
|---|---|
| Sensitivity analyses of the spirometry data | Sensitivity analyses of the spirometry data |
| The following sensitivity analysis will be performed for the <i>primary endpoint</i> . | The following sensitivity analysis will be performed for |
| the primary enapome. | the <u>FEV1, FVC/FEV1 and DLCO assessments</u> . |
| | The following summary will be performed on the |
| | neurology sites data. |
| | • Change from baseline to other visits for each parameter. The baseline is defined as the TV/OV1 |
| | Arrival value. If the TV/OV1 Arrival value is missing, |
| | the last available value in ON state before the first dose of study drug will be used. The summary for |
| | FEV1 will also be provided by smoker status. |
| | • Number and percentage of patients with FEV1/FVC < 60% and <70% by visit |
| | <ul> <li>Spirometry data will also be provided to indicate whether specific determinations met</li> </ul> |
| | American Thoracic Society (ATS) quality criteria. The |



# Statistical Analysis Plan

proportion of DLCO/spirometry data measurements meeting or not meeting ATS quality criteria will be summarized by treatment group and overall. The summary will also be performed for ON state measurements, OFF state measurements, and all measurements, separately. The reasons for not meeting ATS quality criteria will be summarized, as data allow.

• Categories of changes (<-50%, -50% -<-40%, -40% -<-30%, , -30% -<-20%, , -20% -<-10%, -10% -<-10%, 10% -<20%, 20% -<30%, 30% -<40%, 40% -<-20%, >=50%) from baseline for FEV1, FEV, FEV1/FVC ratio and DLCO by visit. The summary for FEV1 will also be provided by smoker status.

1003805 Acorda Therapeutics, Inc. CVT-301-005




# Statistical Analysis Plan

| Document<br>Type: | Template | Document ID: |
|-------------------|-------------|-----------------------------|
| Issue Date: | 02 APR 2012 | Effective Date: 30 APR 2012 |

Sponsor Name: Civitas Therapeutics, Inc.

Protocol Number and Title: CVT-301-005

A Phase 3, Randomized Study Investigating the Safety of CVT-301 (Levodopa Inhalation Powder) in Parkinson's Disease Patients With Motor Response Fluctuations (OFF Phenomena) Compared to an Observational Cohort Control

**Protocol Version and Date:** Version 4.0, 07-Mar-2016

INC Research Project Code:

Author(s):

**SAP Version:** Final Version 2.0

SAP Version Date: 13-Jan-2017

#### Notice of Confidential and Proprietary Information:

The information contained in this document is confidential belonging to Civitas Therapeutics, Inc. Acceptance of this document constitutes agreement by the recipient that no information contained herein will be published or disclosed without prior written authorization from an official of Civitas Therapeutics, Inc. However, this document may be disclosed to appropriate Institutional Review Board and Ethics Committees or duly authorized representatives of a national regulatory authority under the condition that they are requested to keep it confidential. In the event of an actual or suspected breach of this obligation, INC Research should be notified promptly.

1003805

Acorda Therapeutics, Inc. CVT-301-005




# Statistical Analysis Plan

Version: Final Version 2.0

**Version Date:** 

13-Jan-2017

I confirm that I have reviewed this document and agree with the content.



Acorda Therapeutics, Inc. CVT-301-005





# Statistical Analysis Plan

# **TABLE OF CONTENTS**

| 1. | GLOSSARY OF ABBREVIATIONS | 14 |
|------------|------------------------------------|----|
| 2. | PURPOSE | 17 |
| 2.1. | . Responsibilities | 17 |
| 2.2. | Timings of Analyses | 17 |
| 3. | STUDY OBJECTIVES AND STUDY DESIGN | 18 |
| 3.1. | Primary Objective | 18 |
| 3.2. | Secondary Objectives | 18 |
| 3.3. | Exploratory Efficacy Objectives | 18 |
| _ | Patient Selection | 20 |
| 3.5. | Determination of Sample Size | 22 |
| 3.6. | Treatment Assignment & Blinding | 23 |
| 3.7. | Administration of Study Medication | 23 |
| 3.8. | Study Procedures and Flowchart | 24 |
| 4. | ENDPOINTS | 27 |
| 4.1. | Primary Endpoint | 27 |
| 4.2. | Secondary Endpoints | 27 |
| 4.3. | Exploratory EffiCacy Endpoints | 28 |
| <b>5</b> . | ANALYSIS SETS | 32 |
| 5.1. | . All Available Population (AAP) | 32 |






| <b>5.2.</b> | Safety Population | 32 |
|---|---|---|
| <b>5.</b> 3. | Intent-to-Treat Population (ITT) | 32 |
| 5.4. | Protocol Deviations | 32 |
| <b>6</b> . | GENERAL ASPECTS FOR STATISTICAL ANALYSIS | 34 |
| 6.1. | General Methods | 34 |
| 6.2. | Key Definitions | 35 |
| 6.3. | Missing Data | 37 |
| 6.4. | Visit Windows | 38 |
| 6.5. | Pooling of Sites | 39 |
| 6.6. | Subgroups | 39 |
| <b>7</b> . | DEMOGRAPHIC, OTHER BASELINE CHARACTERISTICS AND MEDICATION | N40 |
| • • | -, - | |
| 7.1. | · | |
| | Patient Disposition and Withdrawals | 40 |
| 7.1. | Patient Disposition and Withdrawals Demographic and Other Baseline Characteristics | 40<br>40 |
| 7.1.<br>7.2. | Patient Disposition and Withdrawals Demographic and Other Baseline Characteristics | 40<br>40<br>42 |
| 7.1.<br>7.2.<br>7.3. | Patient Disposition and Withdrawals Demographic and Other Baseline Characteristics | 40<br>40<br>42 |
| 7.1.<br>7.2.<br>7.3.<br>7.4. | Patient Disposition and Withdrawals | 40<br>40<br>42<br>42 |
| 7.1.<br>7.2.<br>7.3.<br>7.4.<br>8. | Patient Disposition and Withdrawals Demographic and Other Baseline Characteristics Medical History Medication SAFETY Spirometry | 40424244 |
| 7.1.<br>7.2.<br>7.3.<br>7.4.<br>8. | Patient Disposition and Withdrawals Demographic and Other Baseline Characteristics Medical History Medication SAFETY Spirometry Extent of Exposure | 40424444 |
| 7.1.<br>7.2.<br>7.3.<br>7.4.<br>8.<br>8.1. | Patient Disposition and Withdrawals Demographic and Other Baseline Characteristics Medical History Medication SAFETY Spirometry Extent of Exposure Treatment Compliance | 4042444447 |
| 7.1.<br>7.2.<br>7.3.<br>7.4.<br>8.<br>8.1.<br>8.2.<br>8.3. | Patient Disposition and Withdrawals Demographic and Other Baseline Characteristics Medical History Medication SAFETY Spirometry Extent of Exposure Treatment Compliance Adverse Events | 404244444748 |

Acorda Therapeutics, Inc.

CVT-301-005





| 8.7. | Electrocardiogram | 52 |
|---|---|---|
| 8.8. | Physical Examination | 53 |
| 8.9. | Columbia-Suicidality Severity Rating Scale | 54 |
| 8.10. | Epworth Sleepiness Scale | 54 |
| 8.11. | Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease | 54 |
| 8.12. | UPDRS Part 4 | 55 |
| 8.13. | examiner-rated dyskinesia | 55 |
| 9. E | XPLORATORY EFFICACY | 56 |
| 9.1. | Exploratory Efficacy Endpoint and Analysis | 56 |
| 10. | INTERIM ANALYSES | 59 |
| 11. | CHANGE FROM ANALYSIS PLANNED IN PROTOCOL | 60 |
| <b>12</b> . | PROGRAMMING CONSIDERATIONS | 61 |
| 12.1. | General Considerations | 61 |
| 12.2.<br>12.2<br>12.2<br>12.2<br>12.2<br>12.2<br>12.2 | 2.2. Headers | 61<br>62<br>62 |
| 13. | QUALITY CONTROL | 65 |
| 14. | INDEX OF TABLES | 66 |

# 1003805

Acorda Therapeutics, Inc. CVT-301-005




| <b>15</b> . | INDEX OF LISTINGS | 74 |
|-------------|-------------------|----|
| 16. | INDEX OF FIGURES | 76 |



# Statistical Analysis Plan

# 1. GLOSSARY OF ABBREVIATIONS

| Abbreviation | Description |
|--------------|--------------------------------------------|
| AAP | All Available Population |
| ADL | Activities of Daily Living |
| AE | Adverse Event |
| ANCOVA | Analysis of Covariance |
| ATC | Anatomical Therapeutic Chemical |
| ATS | American Thoracic Society |
| BMI | Body Mass Index |
| BMS | Biomedical Systems |
| ВР | Blood Pressure |
| CI | confidence interval |
| СМН | Cochran-Mantel-Haenszel |
| COPD | Chronic Obstructive Pulmonary Disease |
| CRO | Contract Research Organization |
| C-SSRS | Columbia-Suicidality Severity Rating Scale |
| DBP | diastolic blood pressure |
| DDI | Dopamine Decarboxylase Inhibitor |
| DL | Dose Level |
| DLCO | Carbon Monoxide Diffusion Capacity |
| DSMC | Data Safety Monitoring Committee |
| ECG | Electrocardiogram |
| ERS | European Respiratory Society |
| ET | Early Termination |
| FEV1 | Forced Expiratory Volume in 1 second |
| FVC | Forced Vital Capacity |
| Hb | hemoglobin |
| HR | Heart Rate |



| Abbreviation | Description |
|---|---|
| IEC | Independent Ethics Committee |
| IFU | Instructions for Use |
| IRB | Institutional Review Board |
| ITT | Intent-to-Treat |
| IWRS | Interactive Web Response System |
| LD | Levodopa |
| LS | least square |
| MAR | Missing At Random |
| MCMC | Markov Chain Monte Carlo |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MI | Multiple Imputation |
| MMSE | Mini Mental State Examination |
| MMRM | Mixed Model for Repeated Measures |
| PCS | potentially clinically significant values |
| PCSC | potentially clinically significant changes |
| PD | Parkinson's Disease |
| PDQ-39 | 39-Item Parkinson's Disease Questionnaire |
| PGI-C | Patient Global Impression of Change |
| PMM | Pattern Mixture Models |
| PRN | As needed |
| PT | Preferred Term |
| QUIP | Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease |
| QTcB | QT interval corrected using Bazett's formula |
| QTcF | QT interval corrected using Fridericia's formula |
| RR | Respiratory Rate |
| S&E | Schwab and England |
| SAP | Statistical Analysis Plan |



| Abbreviation | Description |
|--------------|-------------------------------------------|
| SBP | systolic blood pressure |
| SD | Standard Deviation |
| SEM | Standard Error of the Mean |
| SI | International System of Units |
| SOC | System Organ Class |
| SV | Screening Visit |
| TEAE | Treatment-Emergent Adverse Event |
| TLF | tables, listings, figure |
| TV | Treatment Visit |
| UPDRS | Unified Parkinson's Disease Rating Scale |
| WHO-DD | World Health Organization Drug Dictionary |



## Statistical Analysis Plan

#### 2. PURPOSE

The purpose of this statistical analysis plan (SAP) is to ensure that the data listings, summary tables and figures which will be produced, and the statistical methodologies that will be used, are complete and appropriate to allow valid conclusions regarding the study objectives.

This SAP describes the statistical analysis as it is foreseen at the time of planning the study. The SAP will serve as a compliment to the study protocol and supersedes it in case of differences. In case of major differences between the study protocol and SAP (e.g. changes in the analysis related to the primary endpoint) protocol amendment will be considered. The SAP may be updated during the conduct of the study and will be finalized before database lock. However, because this is an open-label study, the analyses defined after the first patient has been randomized to the study will be considered as exploratory.

#### 2.1. RESPONSIBILITIES

INC Research will perform the statistical analyses and are responsible for the production and quality control of all tables, figures and listings. Acorda (or its designee) will review and approve all statistical work done by INC Research as agreed between INC Research and Acorda.

### 2.2. TIMINGS OF ANALYSES

The primary analysis of safety and efficacy is planned after all patients complete the final study visit or terminate early from the study, and database is cleaned and locked.



## Statistical Analysis Plan

#### 3. STUDY OBJECTIVES AND STUDY DESIGN

#### 3.1. PRIMARY OBJECTIVE

To characterize the pulmonary safety, as assessed by spirometry (forced expiratory volume in 1 second [FEV1], forced vital capacity [FVC], and FEV1/ FVC ratio), over a 12-month period within the CVT-301-treated patients.

#### 3.2. SECONDARY OBJECTIVES

- To characterize the pulmonary safety, as assessed by spirometry (FEV1, FVC and FEV1/FVC ratio), over a 12-month period in the observational ('standard of care') cohort.
- To estimate the difference between the CVT-301-treated patients and the observational cohort on measures of pulmonary safety.
- To characterize the effects of CVT-301 on safety over a 12-month period: safety will be assessed by adverse event (AE) reports, physical examination, standard and orthostatic vital signs (blood pressure [BP], heart rate [HR], and respiratory rate [RR]), clinical laboratory tests, 12-lead electrocardiograms (ECGs), the Parkinson's Disease Impulsive-Compulsive Disorders Questionnaire (QUIP), the Epworth Sleepiness Scale, and the Columbia-Suicide Severity Rating Scale (C-SSRS).
- To evaluate the effect of CVT-301 on mean change from baseline in the UPDRS Part 4 measures of motor fluctuations (dyskinesias [Q32-35] and wearing off [Q36-39]) measured at baseline and at 6 and 12 months after the initiation of CVT-301 treatment.
- To characterize the occurrence and severity of examiner-rated dyskinesia following treatment of patients experiencing an OFF episode in the clinic over a 12-month period.
- To describe the effects of CVT-301 on Carbon Monoxide Diffusion Capacity (DLCO) over a 12-month period.

#### 3.3. EXPLORATORY EFFICACY OBJECTIVES

The following exploratory objectives related to the efficacy endpoints will primarily be assessed for the CVT-301-treated patients. The same objectives will be explored for the pool of CVT-301-naïve patients and patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies, if feasible.



## Statistical Analysis Plan

- Change from pre-dose in UPDRS Part 3 motor score at 10, 20, 30, and 60 minutes following treatment of patients experiencing an OFF episode.
- Time curves of the UPDRS response at 10, 20, 30 and 60 minutes will be evaluated descriptively
- Change from pre-dose in the average UPDRS Part 3 motor score at 10 to 60 minutes following treatment of patients experiencing an OFF episode.
- Proportion of patients with a ≥ 3, ≥ 6, and ≥ 11 point reduction in the UPDRS Part 3 motor score from pre-dose to post-dose, at 10, 20, 30, and 60 minutes.
- Proportion of patients achieving resolution of an OFF to an ON state within 60 minutes after study drug is administered in the clinic, maintaining the ON state at 60 minutes after study drug administration (per the examiner's subjective assessment).
- Total daily OFF time, total daily ON time without dyskinesia, total daily ON time with non-troublesome dyskinesia, and total daily ON time with troublesome dyskinesia, assessed by the patient and recorded in the patient diary.
- Change from baseline in 39-Item Parkinson's Disease Questionnaire (PDQ-39).
- Proportion of patients who improved based on the Patient Global Impression of Change (PGI-C) rating scale.
- Change from baseline in Schwab and England (S&E) Activities of Daily Living (ADL).
- Change from baseline in UPDRS Part 2 score.

#### 3.4. PATIENT SELECTION

The study population for this study is PD patients experiencing motor fluctuations (OFF episodes) that meet the following inclusion criteria and do not meet any of the following exclusion criteria.

Patients may have been previously enrolled in the CVT-301-002 or CVT-301-003 studies, or may be CVT-301-naïve i.e. no previous exposure to CVT-301. Patients previously enrolled in the CVT-301-002 and CVT-301-003 studies must have completed all of the CVT-301 study visits without any safety issues that would preclude participation in this study according to the investigator. Patients who withdrew from either of the CVT-301 studies prior to completion, for any reason, will not be eligible.



## Statistical Analysis Plan

#### 3.4.1. Inclusion Criteria

In order to be eligible to enter the study, patients must meet all of the following criteria:

- Has signed and dated an IRB/IEC-approved informed consent form before any protocol-specific screening procedures are performed.
- Is a male or female aged 30 to 85 years, inclusive. Women of child-bearing potential must use protocol-defined contraceptive measures (see Section 11.1.5) and must have a negative serum human chorionic gonadotropin (hCG) test at screening. These patients must be willing to remain on their current form of contraception for the duration of the study.
- Patients who have idiopathic PD (i.e., not induced by drugs or other diseases) as defined by fulfilling Steps 1 and 2 of the UK Brain Bank criteria, diagnosed after the age of 30 years.
- Patients who are classified as Stage 1 to 3 (in the ON state) on the modified Hoehn and Yahr scale for staging of PD severity.
- Patients who have experienced motor fluctuations for a minimum of 2 hours of average daily OFF time per waking day (excluding early morning OFF time) by self-report and confirmed by the PD Diary (on 3 consecutive days) during the screening period.
- Patients who are on a LD-containing therapy, not including Rytary (or equivalent), must be stable on oral LD-containing therapy for at least 2 weeks prior to SV1 with a LD/dopamine decarboxylase inhibitor (DDI)-containing regimen.
- Patients who are on a LD containing therapy, when including Rytary (or equivalent), should be on a stable dose for at least 6 weeks prior to SV1
- The frequency of L-dopa administrations must be at least 3 times during the waking day and a total daily LD dose of ≤1600 mg (exclusive of PRN LD-containing medications).
- Patients should be stable on other PD medications for at least 4 weeks prior to SV1.



## Statistical Analysis Plan

- Patients must have a ≥ 25% difference between UPDRS Part 3 scores recorded in their ON and OFF states at screening.
- Patients must have normal cognition as confirmed by a score of ≥ 25 on the MMSE.
- Patients must be able to perform a spirometry maneuver in the ON and OFF states, and must have a screening FEV1 ≥ 50% of predicted and an FEV1/FVC ratio >60% in the ON state at screening. (A pulmonologist will review the spirometry tracings/morphology of any patient with an FEV1 that is ≥ 50% to <60% of predicted or an FEV1/FVC ratio that is >60% to <70% in order to determine potential eligibility. All CVT-301-naïve patients with an FEV1/FVC ratio of >60% to <70% will be required to undergo a bronchodilator challenge and the results must be reviewed prior to entry into the study. Patients with an FEV1/FVC ratio that is >60% to <70% will complete spirometry before and after the administration of a bronchodilator in a pulmonary function laboratory. Testing will be performed in accordance with the 2005 ATS/European Respiratory Society [ERS] criteria prior to randomization. The results of the bronchodilator challenge will be reviewed by a pulmonologist prior to potential randomization.)

#### 3.4.2. Exclusion Criteria

Patients meeting any of the following exclusion criteria at screening will not be enrolled in the study:

- Patients who have dyskinesia of a severity that would significantly interfere with their ability to participate or perform study procedures.
- Pregnant or lactating females or females wishing to become pregnant.
- Patients who have any known contraindication to the use of LD, including a history of malignant melanoma or a history of narrow-angle glaucoma.
- Patients who have had previous surgery for PD (including but not limited to deep brain stimulation [DBS] or cell transplantation).
- Patients with a history of psychotic symptoms requiring treatment, or suicide ideation or attempt within the prior 12 months (stable regimens [for at least 4 weeks prior to SV1] of anti-depressant and certain low-dose atypical antipsychotic medications are permitted, in case they are indicated to treat symptoms other than psychotic symptoms).



# Statistical Analysis Plan

- Patients who have cancer with the exception of the following: basal cell carcinoma or successfully treated squamous cell carcinoma of the skin; cervical carcinoma in situ; prostatic carcinoma in situ; or other malignancies curatively treated and with no evidence of disease recurrence for at least 3 years.
- Patients taking certain prohibited medications (see Section 9.4.2).
- Patients with a history of drug or alcohol abuse within the prior 12 months.
- Patients with chronic obstructive pulmonary disease (COPD), asthma, or other chronic respiratory disease within the last 5 years.
- Patients with any contraindication to performing routine spirometry or who are unable to perform a spirometry maneuver (see Appendix 20 for a list of contraindications).
- Patients with a current history of *symptomatic* orthostatic hypotension despite adequate treatment.
- Patients with any condition that in the investigator's opinion would make patients unsuitable or interfere with their participation in the study. Potential issues of concern should be raised to the medical monitor during eligibility review.
- Patients who have any clinically significant abnormality or finding from examination, tests, or history that may compromise patient safety.
- Patients who have been treated with an investigational drug within 4 weeks or 5 half-lives (whichever is longer) prior to the beginning of the screening period (this includes investigational formulations of marketed products).
- Prior exposure to CVT-301.

#### 3.5. DETERMINATION OF SAMPLE SIZE

Approximately 350 CVT-301 treatment patients and 175 control patients will be enrolled in this study. It is assumed that the drop-out rate will be approximately 25%.

The primary objective of this study will be to characterize the pulmonary safety within the CVT-301-treated patients and the differences between the groups will be estimated as a secondary objective. However, for the secondary comparison of FEV1 change



## Statistical Analysis Plan

between the CVT-301 treatment group and the randomized observational cohort, the standard deviation of FEV1 change from baseline is expected to be 0.281 L, based on data from Study CVT-301-003. Assuming that there is no difference in the changes from baseline between the CVT-301-treated patients and the observational cohort, the study has the following power for the comparison between the 2 groups. The upper limit of the 95% confidence interval for the difference between the 2 groups in change from baseline in FEV1 will be less than 0.121 L with 90% power, assuming 188 and 86 patients completing the study in the CVT-301 treatment group and observational cohort, respectively. The sample size calculation was performed using nQuery Advisor, Version 7.0.

#### 3.6. TREATMENT ASSIGNMENT & BLINDING

This study is a 12-month, open-label, randomized, multicenter study which will evaluate the safety and effects of CVT-301 for the treatment of up to 5 OFF episodes per day in PD patients experiencing motor fluctuations (OFF episodes) and will include a concurrent observational cohort of PD patients managed using the usual standards of care. Patients may have been previously enrolled in the CVT-301-002 or CVT-301-003 studies, or may be CVT-301-naïve. Patients who were previously enrolled in the CVT-301-002 and CVT-301-003 studies will be assigned to the CVT-301 treatment group (CVT-301 at a target nominal respirable dose of 50 mg LD fine particle dose [FPD]), in this study. Patients who are CVT-301-naïve will be randomized in a 2:1 ratio to the CVT-301 treatment group (CVT-301 at a target nominal respirable dose of 50 mg LD FPD) or the observational cohort. Randomization can occur before the baseline DLCO has been performed. Note: Patients who were enrolled from the CVT-301-002 and CVT-301-003 studies under an earlier version of this protocol (Version 2) were assigned only to the CVT-301 treatment group. Randomization will be stratified by the patient's Hoehn and Yahr stage (<2.5 versus ≥2.5) to balance the severity of disease across each group and by screening spirometry (FEV1 <60% of predicted or FEV1/FVC ratio <70% versus FEV1  $\geq$ 60% of predicted and FEV1/FVC ratio  $\geq$ 70%).

Following completion of SV2 and prior to randomization, the patients' eligibility criteria will be reviewed by delegated staff. Upon confirmation of eligibility, the site will randomize an eligible patient using the Interactive Web Response System (IWRS). The study is an open-label study, so patients and clinical staff will not be blinded to study group assignment.

#### 3.7. ADMINISTRATION OF STUDY MEDICATION

Prior to the self-administration of inhaled study treatment, study staff will ensure that patients are adequately trained on the use of the inhaler according to the Instructions for Use (IFU). The IFU will be provided to each patient and will be part of the permanent study record.



## Statistical Analysis Plan

Since this is an open-label study, the patient, investigator, and study site personnel, the Sponsor, representatives of the Contract Research Organization (CRO) involved in monitoring, data management, or other aspects of the study, and Core Laboratories will be not blinded to the inhaled study treatment.

During inhaler training, patients will be instructed to use the inhalation system in accordance with the IFU which includes a breath hold of 5 seconds following each capsule inhalation. For the purposes of timing study assessments in the clinic, "Time 0" (T0) is defined as the time of completion of inhalation of the last capsule of inhaled study treatment administered (i.e., beginning of the final breath hold). In the event that a capsule needs to be reinhaled, T0 is at the end of the reinhalation administration.

During the treatment period, patients will self-administer inhaled study treatment (CVT-301 DL1, CVT-301 DL2) up to 5 times daily to treat OFF episodes during their waking day.

#### 3.8. STUDY PROCEDURES AND FLOWCHART

This study has 3 periods: screening period, treatment period, and follow-up period; and a total of 9 planned visits: 2 screening visits, 6 treatment visits, and 1 follow-up visit. For each patient, the planned treatment period will be approximately 52 weeks, and maximum anticipated study duration, including screening and follow-up, will be approximately 62 weeks.

The screening period, which takes place within 35 days prior to Day 1 of the treatment period, will have 2 separate visits: SV1 and SV2 must be separated by at least 4 days. The screening period may be extended an additional 7 days if repeat screening assessments are required.

Before patients return to the clinic for TV/OV1, they will be randomized to treatment. The treatment period includes 6 separate in-clinic visits over approximately 52 weeks. The first dose of study drug will be given in the clinic at TV/OV1. The subsequent visits during the treatment period take place as follows:

- TV/OV2: Week 4; 28±5 days after TV/OV1.
- TV/OV3: Week 12; 84±14 days after TV/OV1.
- TV/OV4: Week 24; 168±14 days after TV/OV1.
- TV/OV5: Week 36; 252±14 days after TV/OV1.




# Statistical Analysis Plan

• TV/OV6: Week 52; 364±14 days after TV/OV1.

Patients who terminate the study early will complete TV/OV6 and return for the Follow-up DLCO visit 4-5 weeks after TV/OV6.

Refer to Protocol Appendices 1 to 15 for tables of study assessments at each visit.

1003805

Acorda Therapeutics, Inc. CVT-301-005





| | S | V1 | S' | /2 | TV/OV1 | TV/OV2 | TV/OV3 | TV/OV4 | TV/OV5 | TV/OV6 |
|---|---|---|---|---|---|---|---|---|---|---|
| In Clinic Assessments | ON | OFF | ON | OFF | ON* | ON | ON | ON | ON | ON |
| MMSE | х | | | | | | | | | |
| UPDRS Part 1 | | | | | | | | | | |
| UPDRS Part 2 | | | | | Х | | | Х | | Х |
| UPDRS Part 3 | Х | Х | | | | X** | x** | x** | X** | X** |
| UPDRS Part 4 | | | | | Х | | | x*** | | x*** |
| C-SSRS | | | | | Х | х | Х | Х | х | х |
| Epworth Sleep Scale | | | | | Х | | | Х | | Х |
| QUIP | | | | | Х | | | Х | | х |
| PDQ-39 | | | | | х | | | Х | | х |
| PGI-C | | | | | | | | x*** | | x*** |
| S&E ADL | | | | | х | | | Х | | х |
| At home for patients | | | | | | | | | | |
| PD Diary (only treatment after screening) | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| ON/OFF logs (both groups) | Х | Х | | | | | | | | |
| Inhaled dosing (CVT-301 only) | | | | | х | х | х | х | х | х |

- \* For the CVT 301 arm these assessments are performed pre-dose
- \*\* Performed pre-dose, 10, 20, 30, and 60 min post dose (only performed in CVT 301 arm)
- \*\*\* CVT 301 arm only



## Statistical Analysis Plan

#### 4. ENDPOINTS

#### 4.1. PRIMARY ENDPOINT

The primary endpoints related to the primary objective of the study are the pulmonary safety measures, FEV1, FVC and FEV1/ FVC ratio, assessed over a 12 month period. FEV1, FVC and FEV1/FVC ratio will be recorded from the single "best test" (based on effort with highest summed FEV1 and FVC). Variables will include the absolute FEV1, FVC, and FEV1/FVC ratio and FEV1 and FVC expressed as % of predicted value. Changes from baseline (TV/OV1) for each variable will be calculated at each subsequent visit.

Percent Predicted = 100 \* (Observed) / Predicted, where predicted is calculated and provided to INC by Biomedical Systems (BMS).

#### 4.2. SECONDARY ENDPOINTS

The following endpoints related to the secondary objectives will be calculated.

- Standard safety endpoints; for definitions see Section 8 of this SAP
  - Adverse Event (AE) reports
  - Physical examination
  - Standard and orthostatic vital signs (BP, HR and RR)
  - Clinical laboratory tests (hematology, clinical chemistry, and additional laboratory parameters)
  - 12-lead ECGs (HR, PR, QRS, QT, QT interval corrected using Bazett's formula [QTcB] and QT interval corrected using Fridericia's formula [QTcF])
  - Parkinson's Disease Impulsive-Compulsive Disorders Questionnaire (QUIP)
  - Epworth Sleepiness Scale
  - Columbia-Suicide Severity Rating Scale (C-SSRS)
- Change from TV/OV1 (baseline) in the UPDRS Part 4 sum scores of dyskinesias (UPDRS items 32-35) and wearing-off (UPDRS items 36-39). The dyskinesia score will be calculated as the sum of the individual items 32-35 and the wearing-off score as sum of 36-39. Missing individual items will not be imputed and the sum score will be missing in case of 1 or more missing items.
- Occurrence and severity of examiner-rated dyskinesia following treatment of
  patients experiencing an OFF episode in the clinic. The occurrence will be based on
  the examiner's subjective assessment and no further derivation will be performed.
  Among the patients with reported dyskinesia, the severity will be classified as mild,
  moderate, severe or missing based on the examiner's subjective assessment and no
  further derivation will be performed. Only observed cases will be used for this
  endpoint and the visits with missing data will not be included in the analysis.




## Statistical Analysis Plan

• Carbon Monoxide Diffusion Capacity (DLCO) assessed over a 12 month period within the CVT 301 treated and the observational ('standard of care') cohorts. Variables will include the absolute DLCO values and DLCO expressed as % of predicted value.

#### 4.3. EXPLORATORY EFFICACY ENDPOINTS

The following endpoints related to the exploratory efficacy objectives will be calculated.

- Change from pre-dose in UPDRS Part 3 motor score at 10, 20, 30, and 60 minutes following treatment of patients experiencing an OFF episode.
  - o The UPDRS Part 3 total score will be calculated as the sum of the individual items of the UPDRS Part 3 questionnaire (UPDRS items 18-31) separately at each time point, i.e. the scores will range from 0 to 108. Missing individual items will be imputed using the 2 non-missing values at time points adjacent to the missing item on the same date. The maximum of the 2 adjacent values will be assigned as the score for the missing item. However, pre-dose values will not be assigned as post-dose values and if one of the adjacent values for a post-dose value is a pre-dose value, only 1 adjacent value will be used. The total score for UPDRS Part 3 assessments will be calculated after imputation of the missing item(s). Missing items at screening will not be imputed. If a pre-dose value is missing, the pre-dose value at the prior visit will be used. A missing TV/OV1 pre-dose value will be imputed using the last screening value in OFF state.
- Time curve of the UPDRS response shown as change from pre-dose in UPDRS Part 3 motor score to 10, 20, 30 and 60 minutes following treatment of patients experiencing an OFF episode in the clinic. The UPDRS Part 3 scores will be derived as described above.
- Change from pre-dose in the average UPDRS Part 3 score at 10 to 60 minutes following treatment of patients experiencing an OFF episode in the clinic. The change from pre-dose to the average of the 4 UPDRS Part 3 total scores (assessments scheduled at 10, 20, 30 and 60 minutes) will be used as the response variable in the statistical analysis.
- A ≥3, ≥6, and ≥11 point reduction in the UPDRS Part 3 motor score from pre-dose to post-dose, at 10 to 60 minutes following treatment in the clinic (cumulative and non-cumulative). The non-missing UPDRS Part 3 motor scores at each time point (10, 20, 30 and 60 minutes post-dose) are classified as a reduction of ≥3 points or not, reduction of ≥6 points or not and reduction of ≥11 points or not. Furthermore,



## Statistical Analysis Plan

for the purpose of the cumulative analysis, the time point (10, 20, 30 and 60 minutes post-dose) when the reduction of  $\ge 3$ ,  $\ge 6$  or  $\ge 11$  points occurs for the first time will be defined. The categorical scheduled time point is used in this analysis. The missing assessment regarding single items will be managed similarly as describe above. The missing values regarding visits will be managed by considering the missing visits as non-responses.

- Proportion of patients achieving resolution of an OFF to an ON state within 60 minutes after study drug is administered in the clinic and maintaining the ON at 60 minutes after study drug administration (per the examiner's subjective assessment). This endpoint will be based on the examiner's subjective assessment. In case the assessment of turning on within 60 minutes is missing but the assessment of maintaining the ON at 60 minutes has been done, the patient will be classified based on the available assessment. In case the assessment of maintenance of ON at 60 minutes is missing, the patient will be classified as having missing data.
- Change from baseline (3 consecutive days prior to TV1, or in case of missing data, the last 3 recorded days before TV1) in patient-recorded total daily OFF time, assessed by the patient and recorded in the PD Diary for 3 consecutive days prior to in-clinic visits (or in case of missing data, the last 3 recorded days before the visit). The validity of the PD diary entries will be checked prior to including a diary day in the summary calculations. Only valid diary days will be included in the diary summarizations. Change from baseline in total daily ON time without dyskinesia, total daily ON time with non-troublesome dyskinesia, and total daily ON time with troublesome dyskinesia will be calculated similarly.
  - A day will be considered as being valid if at least 80% of the entries during the day have been completed per instructions. That is, for each half hour period, only one entry among the responses (Asleep, OFF, ON without dyskinesia, ON with non-troublesome dyskinesia, or ON with troublesome dyskinesia) has been checked. The entry will not be used if no responses are checked or more than one response is checked. However, if the proportion of entries rejected due to multiple checked responses is large, sensitivity analysis will be performed by using the worst case out of the entries that had been checked. The worst case will be defined in the following order: OFF, ON with troublesome dyskinesia, ON with non-troublesome dyskinesia, ON without dyskinesia, Asleep. In case there are duplicate entries (i.e., multiple entries recorded with same date and time interval), the worst entry will be used for the date and time interval in question. The worst entry will be selected in the order defined above.
  - All diary data will be normalized to 16 awake hours per day. The daily OFF time will be extrapolated to a 16 hour period by determining the percentage



## Statistical Analysis Plan

of OFF time among accurately recorded entries, excluding Asleep time and missing/non-valid recordings, and by multiplying this percentage by 16 hours.

- Off Time / (Total time recorded Asleep Time missing time interval)
   x 16
- o The mean daily OFF time prior to each visit will be calculated as mean value of the valid days documented in the patient's diary prior to that visit. In case there are gaps within the 3 days preceding the visit, the last 3 recorded days before the visit will be used regardless of the gaps. If there are more than 3 valid days, only the last 3 days will be used. If there are only 1 or 2 valid days, the average of these days will be used.
- Change from TV/OV1 (baseline) in PDQ-39 sub-scores (mobility score, activities of daily living, bodily discomfort score, emotional wellbeing score, social support score, communication score, cognitive impairment score, and stigma score) and summary index score. The questionnaire provides scores on eight dimensions as outlined below:
  - o mobility (10 items, #1 to 10)
  - o activities of daily living (6 items, #11 to 16)
  - o emotional well-being (6 items, #17 to 22)
  - o stigma (4 items, #23 to 26)
  - o social support (3 items, #27 to 29)
  - o cognitions (4 items, #30 to 33)
  - o communication (3 items, #34 to 36)
  - o bodily discomfort (3 items, #37 to 39)

Items are scored from 0 (never) to 4 (always). Dimension scores are obtained by dividing the sum of the item scores by the maximum possible score for any given dimension and expressing this as a percentage. For example:

- o mobility = (sum of scores of #1 to 10)/(4 x 10) x 100
- o activities of daily living = (sum of scores of #11 to 16)/(4 x 6) x 100

For social support, if the response indicates that a patient does not have a spouse or partner for #28, social support can be calculated as [(sum of scores of #27 and 29)/(4 x 2) x 100].

A summary index is then calculated as the sum of the total score of the dimensions divided by the number of dimensions, i.e. (sum of dimension scores / 8). If any item score is missing, the relevant dimension score and the summary index will be missing.



- The PGI-C score. The non-missing values will be categorized as improvements (much improved, improved, a little improved) or non-improvements (no change, a little worse, worse, much worse).
- Change from TV/OV1 (baseline) Schwab and England (S&E) Activities of Daily Living (ADL). No further derivation will be done for the S&E scores.
- Change from TV/OV1 (baseline) in the UPDRS Part 2 score. The UPDRS Part 2 score will be calculated as the sum of the individual items of the UPDRS Part 2 questionnaire (UPDRS items 5-17). Missing individual items will not be imputed and the sum score will be missing in case of 1 or more missing items.



## Statistical Analysis Plan

#### 5. ANALYSIS SETS

### 5.1. ALL AVAILABLE POPULATION (AAP)

The AAP will include all patients who have consented for the study, including screening failures. Unless specified otherwise, the AAP will be used for patient listings and for the summary of patient disposition.

#### 5.2. SAFETY POPULATION

The Safety Population will include all randomized patients who received at least 1 dose of inhaled CVT-301 and patients from the Observational Cohort who came in for treatment visit 1. Patients will be analyzed according to study treatment that they received. The Safety Population will be used for all analyses of safety endpoints and summaries of patient demographics and baseline characteristics.

### 5.3. INTENT-TO-TREAT POPULATION (ITT)

The ITT population will include all patients from the safety population. Patients will be analyzed according to randomized treatment. The ITT Population will be used for all analyses of exploratory efficacy endpoints.

#### 5.4. PROTOCOL DEVIATIONS

A protocol deviation is any significant finding indicating that the study investigator or patient failed to adhere to the protocol requirements (e.g., drug noncompliance, failure to return for defined number of visits or within an acceptable visit window for completion of study assessments). The deviation may necessitate premature termination of the patient from the visit assessments, or from the study.

The deviations will be classified during a review process with the Sponsor and other study personnel (as appropriate) before database lock. The deviations will be classified as minor or major with/without impact on pulmonary assessments during the review process. All decisions regarding major deviations will also be discussed between the Sponsor, other study personnel (as appropriate), and the study statistician prior to commencing the final analysis on the locked database. The following deviations will be identified, but do not necessarily represent a complete list of potential deviations:

- Administration of PD medications after the usual morning dose of PD medication and before study drug administration
- Incorrect study drug administered at a visit
- Drug non-compliance including but not limited to unapproved dose modification
1003805

Acorda Therapeutics, Inc. CVT-301-005



## Statistical Analysis Plan

 Failure to return for defined study visits or within an acceptable visit window for completion of study assessments

The number of subjects with minor, major with/without impact on pulmonary assessments protocol deviations will be summarized by treatment groups and overall. All protocol deviations will be listed.



## Statistical Analysis Plan

#### 6. GENERAL ASPECTS FOR STATISTICAL ANALYSIS

#### 6.1. GENERAL METHODS

All patient data will be included in listings. All patients entered into the database will be included in patient data listings. The listings will be generally sorted by Patient ID (and by visit and by time point, if applicable), unless specified otherwise.

All applicable data will be summarized by treatment group (Observational Cohort or CVT-301) and overall in tables, unless specified otherwise. The CVT-301 group will be broken down into CVT-301-naïve patients and patients who were previously enrolled in the CVT-301-002 or CVT-301-003 studies. Where appropriate, data will be summarized by visit and/or time point in addition to treatment group. Unscheduled or repeat assessments will not be included in summary tables, but will be included in listings.

For the Observational Cohort, the "start of treatment" will be defined as attendance of TV/OV1, unless specified otherwise. Baseline will be defined as the assessments performed at TV/OV1. In case of missing data, the last non-missing screening assessment will be used as the baseline value.

Continuous variables will be summarized using the number of observations (n), mean, SD, median, minimum, and maximum. Standard error of the mean (SEM) will also be provided for summaries of UPDRS and other exploratory efficacy endpoints, if relevant. The same number of decimal places as in the raw data will be presented when reporting minimum and maximum, 1 more decimal place than in the raw data will be presented when reporting mean and median, and 2 more decimal places than in the raw data will be presented when reporting SD and SEM.

Descriptive statistics for categorical/qualitative data will include frequency counts and percentages. The total number of patients in the treatment group overall (N) will be used as the denominator for percent calculations, unless stated otherwise in the table shell. All percentages will be presented with one decimal point, unless specified otherwise. Percentages equal to 100 will be presented as 100% and percentages will not be presented for zero frequencies.

Significance testing will be 2-tailed using  $\alpha = 0.05$ , unless otherwise specified. All analyses and summaries will be produced using SAS® version 9.3 (or higher).

Deviations from the statistical plan will be reported in the clinical study report, including the rationale for use.



## Statistical Analysis Plan

#### 6.2. KEY DEFINITIONS

#### Age

Age, as an integer, will be calculated using the date of birth and the date of informed consent.

Age = int ((date of informed consent- date of birth)/365.25)

#### Body Mass Index (BMI)

BMI will be calculated as follows and rounded to 1 decimal place:

BMI  $(kg/m^2)$  = weight (kg) /  $[height (m)]^2$ 

#### Parkinson's Disease History

The following parameters will be calculated for the PD history:

Time since diagnosis of PD (months) = Date of Screening Visit 1 (M/Y) - Date of diagnosis (M/Y)

Duration of levodopa treatment (months) = Date of Screening Visit 1 (M/Y) - Start date of levodopa treatment (M/Y)

Time since onset of wearing off episodes (months) = Date of Screening Visit 1 (M/Y) - Date of onset of wearing off episodes (M/Y)

If the month is missing, the first month of the year will be used.

### Change from pre-dose to post-dose

The change from pre-dose to post-dose within each visit will be calculated for each post-dose assessment as:

Change from Pre-dose to Post-dose = Post-dose value - Pre-dose value

#### Percent change from pre-dose to post-dose

The percent change from pre-dose to post-dose within each visit will be calculated for each post-dose assessment as:

Percent Change from Pre-dose to Post-dose =



## Statistical Analysis Plan

(Post-dose value - Pre-dose value)\*100/Pre-dose value

#### Baseline

For CVT-301 patients, baseline is defined as the last non-missing assessment before the first dose of study drug, unless specified otherwise. For the Observational Cohort, baseline is defined as TV/OV1, or, in the case of missing data, the last non-missing assessment before TV/OV1, unless specified otherwise. However, for all patients who were included in the CVT 301-002 or CVT-301-003 studies, TV/OV1 of the CVT-301-005 study will be used as baseline.

#### Change from baseline

The change from baseline will be calculated for each post-baseline assessment as:

Change from Baseline = Post-baseline value - Baseline value

#### Percent change from baseline

The percent change from baseline will be calculated for specified post-baseline assessments as:

Percent Change from Baseline = (Post-baseline value - Baseline value)\*100/Baseline value

DLCO predicted and DLCO predicted, adjusted for hemoglobin (Hb)

#### DLCO predicted

DLCO predicted will be calculated by Miller equation. (Miller A, Thornton JC, Warshaw R, Anderson H, Teirstein AS, Selikoff IJ. Single breath diffusing capacity in a representative of Michigan, a large industrial state. Am Rev Resp Dis 1983; 127: 270-277).

- Men predicted DLCO = 12.9113 (0.229 x age) + (0.418 x height in)
- Women predicted DLCO = 2.2382 (0.1111 x age) + (0.4068 x height in)

Where age is the age at baseline, height is measured in inches.

#### DLCO Predicted, adjusted for Hb

DLCO predicted adjusted for Hb is calculated using the Cotes method, according to the 2005 ATS/ERS guidelines for DLCO.

CVT-301-005




## Statistical Analysis Plan

- DLCO predicted, adjusted for Hb in adult men: DLCO predicted for Hb = DLCO predicted 1.7\* Hb / (10.22 + Hb)
- DLCO predicted, adjusted for Hb in adult women: DLCO predicted for Hb = DLCO predicted 1.7 \*Hb / (9.38 + Hb)

Where  $DLCO_{predicted}$  is the DLCO calculated from Miller equation; Hb = hemoglobin, measured in g/dL. The Hb closest to the date/time of DLCO taken will be used.

#### Percent predicted of FEV1 and FVC

The percent predicted of FEV1 and FVC will be calculated using the following equation.

Percent Predicted = 100 \* (Observed) / Predicted

where observed value is the value provided by TechEd, and the predicted value is the predicted value that provided by BMS and is the values closest to the date of observed value taken. The details are listed in table below.

| DLCO <sub>predicted</sub> , percent predicted of | Value selection for Hb, predicted FEV1 and FVC |
|---|---|
| FEV1 and FVC | |
| Screening (prior to randomization) | From TV/OV1 or the value closest to the date of DLCO |
| | assessment if the value at TV/OV1 is missing |
| TV/OV3, within 2 weeks prior to 3 | From TV/OV3 or the value closest to the date of DLCO |
| | assessment if the value at TV/OV3 is missing |
| TV/OV4, within 2 weeks prior to 6 | From TV/OV4 or the value closest to the date of DLCO |
| | assessment if the value at TV/OV4 is missing |
| TV/OV5, within 2 weeks prior to 9 | From TV/OV5 or the value closest to the date of DLCO |
| | assessment if the value at TV/OV5 is missing |
| TV/OV6, within 2 weeks prior to 12 | From TV/OV6 or the value closest to the date of DLCO |
| | assessment if the value at TV/OV6 is missing |
| 4 to 5 weeks after TV/OV6 | The latest non-missing Hb that closest to the date of |
| | DLCO assessment taken. |

#### 6.3. **MISSING DATA**

Several different methods to handle the missing data will be used.

For calculation of the UPDRS part 3 scores, the missing single UPDRS items will be imputed as described in Section 4.3.



## Statistical Analysis Plan

- For the primary analysis of spirometry and selected explorative efficacy endpoints, likelihood-based modeling approach will be used to handle incomplete data. For this purpose, Mixed Model for Repeated Measures (MMRM) will be applied, see Section 8.1.
- Sensitivity analysis for spirometry and selected explorative efficacy endpoints will be conducted using the Multiple Imputation (MI) approach, i.e. by replacing each missing value with a set of plausible values that represent the uncertainty about the right value to impute, see Section 8.1.
- For the binary explorative efficacy endpoints, sensitivity analyses will be conducted using worst case imputation, where visits with missing data are counted as non-resolved (primary method), see Section 9.1.
- For AEs, the overall incidence of TEAEs, normalized for duration of exposure will be calculated to account for the shorter follow-up time in patients who discontinue the study prematurely, see Section 8.4.

The Safety and ITT populations will be used for the analysis of the primary, secondary and exploratory endpoints. The patients with no post-baseline data will not contribute to the analyses performed with the MMRM approach, but they do contribute to the sensitivity analyses using the MI approach. Due to this, no additional population, like a modified ITT population including only the patients with post-baseline will be defined.

#### 6.4. VISIT WINDOWS

The visits recorded in database will be used for all analyses. There is no plan to re-assign visits based on actual visit dates.

For the patients who discontinue the study prematurely, a set of assessments is scheduled to be performed at the Early Termination (ET) visit (PDQ-39, UPDRS Part 2, UPDRS Part 4, S&E ADL score and safety assessments). CVT 301 treated patients will also perform the UPDRS Part 3 assessments at 10, 20, 30, and 60 minutes post dose as well as the PGI-C. The following rules will be used to analyze the data collected at the ET visit:

- For the PDQ-39, PGI-C, UPDRS Part 2, UPDRS Part 3, UPDRS Part 4 and S&E ADL score, the data from the ET visit will be re-assigned to TV/OV6 in case there is no TV/OV6 assessment.
- In case there are PD diary assessments performed during the three days before the ET visit, these assessments will be re-assigned to the first visit at which the PD diary assessments were scheduled but are missing due to the premature withdrawal.



## Statistical Analysis Plan

- The safety assessment assessments performed at the ET visit will be re-assigned to the first time point at which the corresponding safety assessments were scheduled but are missing due to the premature withdrawal.
- Any other data collected at the ET visit will not be used.

#### 6.5. POOLING OF SITES

Not applicable.

#### 6.6. SUBGROUPS

At least the following subgroup analyses have been pre-planned. The subgroup analyses will be performed for selected efficacy endpoints (at least the Change from pre-dose in UPDRS Part 3 motor score at 30 minutes post-dose and the mean daily OFF time). Selected baseline data will be presented for the subgroups as well.

- Patients with baseline PD severity < 2.5 points on the Hoehn & Yahr scale versus patients with baseline PD severity ≥ 2.5 points on the Hoehn & Yahr scale
- Patients who are dyskinetic before TV/OV1 versus non-dyskinetic patients. The
  classification will be done based on the Parkinson's disease diary data. The
  patients who have recorded at least 1 hour of dyskinesia (either ON with nontroublesome dyskinesia or ON with troublesome dyskinesia) on at least 2 days
  before TV/OV1 will be classified as dyskinetic
- Patient with the baseline daily levodopa dose less than or equal to the median versus the patients with the baseline daily levodopa dose higher than the median
- Patients who have less than 4.5 hours of PD diary mean daily OFF time before TV/OV1 versus patients who have 4.5 hours or more of OFF time
- Patients with FEV1 <60% of predicted or FEV1/FVC ratio <70% at baseline versus patients with FEV1 ≥60% of predicted and FEV1/FVC ratio ≥70%
- Non-elderly (<65 years) versus elderly (≥65 years) patients</li>
- Female versus male patients.



## Statistical Analysis Plan

# 7. DEMOGRAPHIC, OTHER BASELINE CHARACTERISTICS AND MEDICATION

#### 7.1. PATIENT DISPOSITION AND WITHDRAWALS

The patient disposition table will summarize the following and will be presented for each treatment group, as applicable, and overall. The percentages will be calculated based on the number of randomized patients, unless otherwise specified). The randomized set will include all randomized patients as well as those from CVT-301-002 and CVT-301-003 studies who were assigned to the CVT 301 treatment group.

- The number of patients screened (i.e. the number of patients in the AAP population)
- The number of patients who failed screening
- The number (%) of patients randomized into the study (% calculated from the AAP population)
- The number (%) of patients in the different study populations (Safety and ITT populations)
- The number (%) of patients who completed the study (based on end-of-study case record page)
- The number (%) of patients who withdrew from the study and associated reasons (% calculated from the Safety population)

#### 7.2. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Demographics and baseline characteristics will be summarized descriptively for the Safety population by treatment group and overall. The following variables will be summarized:

- Demographics (age (continuous), age categorized as <65 years versus ≥65 years, gender, ethnicity, race, height, weight, BMI, country)
- Smoking history (current, former, never, Number of Years Smoked and Number of Cigarettes/Day)
- Cognitive status (MMSE)
- Average number of daily OFF episodes experienced from the Screening ON/OFF Log. The screening ON/OFF log data collected on 3 days prior to TV/OV1 will be used as baseline. If the data are only available on 1 or 2 days prior to TV/OV1, the available data will be used as baseline. If there is no data prior to TV/OV1, the data collected on 3 days prior to SV2 will be used as baseline.



## Statistical Analysis Plan

- Proportion of patients who changed the timing of their usual levodopa medication and proportion of patients who took an extra dose of levodopa or other PD medication from the Screening ON/OFF Log. The screening ON/OFF log data collected on 3 days prior to TV/OV1 will be used as baseline. If the data are only available on 1 or 2 days prior to TV/OV1, the available data will be used as baseline. If there is no data prior to TV/OV1, the data collected on 3 days prior to SV2 will be used as baseline.
- Average daily OFF time, ON time Without Dyskinesia, ON time with troublesome and non-troublesome dyskinesia (from PD diary before TV/OV1)
- Proportion of patients with total daily OFF time <4.5 hours or ≥4.5 hours (from PD diary before TV/OV1)
- Distribution of average daily OFF time in 30-minute intervals (00:00 00:30, 00:30 01:00, ...). The percentage based on the total daily OFF time will also be presented and is calculated as the average of total OFF time collected three days prior to TV1 and is normalized to 16 awake hours per day.
- PD history (time since diagnosis of PD, duration of levodopa treatment, time since onset of wearing off episodes)
- Total daily levodopa dose, number of levodopa doses per day
- PD disease severity (Modified Hoehn and Yahr Staging in "ON" State)
- UPDRS Part 3 Motor score in ON/OFF (from screening assessment); the change from OFF to ON state in UPDRS part 3 Motor score at the Screening will also be classified as ≥6 points, or ≥11 points reduction.
- Baseline Dyskinesia (Dyskinetic before TV/OV1, Non-dyskinetic before TV/OV1).
   The classification will be done based on the Parkinson's disease diary data. The patients who have recorded at least 1 hour of dyskinesia (either ON with non-troublesome dyskinesia or ON with troublesome dyskinesia) on at least 2 days before TV will be classified as dyskinetic.
- Proportion of patients with FEV1 <60% of predicted or FEV1/FVC ratio <70% at baseline versus FEV1 ≥60% of predicted and FEV1/FVC ratio ≥70% (based on the randomization strata).
- Screening spirometry data: FEV1, FVC, and FEV1/FVC ratio, presented for each motor status, ON or OFF, separately.

Demographics and PD disease data will also be summarized by subgroups (Patients with baseline PD severity < 2.5 points on the Hoehn & Yahr scale versus  $\geq$  2.5 points; Patients who are dyskinetic before TV/OV1 versus non-dyskinetic; Patient with the baseline less than or equal to the median versus above median; Patients who have less than 4.5 hours of PD diary mean daily OFF time before TV/OV1 versus 4.5 hours or more; Patients with FEV1 <60% of predicted or FEV1/FVC ratio <70% at baseline versus FEV1  $\geq$ 60% of predicted and FEV1/FVC ratio  $\geq$ 70%, Non-elderly (<65 years) versus elderly ( $\geq$ 65 years) patients, Female versus Male patients).



## Statistical Analysis Plan

#### 7.3. MEDICAL HISTORY

Medical history data will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 17.0. The medical history data will be summarized with frequencies and percentages of patients with at least one medical history item, and patient frequencies and percentages on the system organ class (SOC) and preferred term (PT) levels. The events will also be summarized. The table, using the Safety population, will be sorted by overall descending frequency of SOC and then, within a SOC, by overall descending frequency of PT.

#### 7.4. MEDICATION

All medications will be classified using the Anatomical Therapeutic Chemical (ATC) classification codes and preferred drug names from the World Health Organization Drug Dictionary (WHO-DD), Q1March2014.

For the medications recorded on CRF page "Prior and Concomitant Medications", medications with a stop date before the first date of study drug dosing or TV/OV1 for the observational cohort will be considered prior medications. Medications with start date or stop date on or after the first date of study drug dosing will be considered concomitant medications.

Tables will be generated for the Safety Population. Summaries of baseline PD treatment medications (medications which start with ATC code N04) will be presented in tabular form using the ATC Level 4 and preferred term. Other prior medications and concomitant medications will be presented in tabular form using the ATC Level 1, ATC Level 2, and PT. Frequencies and percentages will be presented by treatment group and overall. The counts of medications will also be summarized. The tables will be sorted by overall descending frequency of ATC Level(s) and then, within an ATC Level, by overall descending frequency of PT.

If the medication start date is incomplete, then it will be imputed as follows for the purpose of determining concomitance only:

- If the start date is completely missing, the start date will be equal to the first dose date. However, if the stop date is not missing and is before the first dose date, then the stop date will be used instead.
- If the start day is missing, the first day of the month will be used.
- If the start day and month are missing, then the first day of the first month (January) will be used.

If the medication stop date is partial, then it will be imputed as follows for the purpose of determining concomitance only:



- If the stop date is completely missing and the medication is not ongoing, the stop date will be equal to the last dose date or date of completion/withdrawal, whichever is the latest.
- If the stop day is missing, the last day of the month will be used.
- If the stop day and month are missing, then the last day of the last month (December) will be used.



## Statistical Analysis Plan

#### 8. SAFETY

The population used for safety analyses will be the Safety Population. The analyses are outlined below.

#### 8.1. SPIROMETRY

Spirometry will be performed by trained and qualified staff at each study site. Spirometry data obtained in the study site will reviewed by a central spirometry laboratory (Biomedical Systems, Inc.) which will provide a quality over read of all evaluations based on acceptability and repeatability metrics in accordance with ATS criteria. FEV1, FVC and FEV1/FVC ratio will be recorded from the single "best test" (based on effort with highest summed FEV1 and FVC). Variables will include the absolute FEV1, FVC, and FEV1/FVC ratio and FEV1 and FVC expressed as % of predicted value.

The variables from pulmonary laboratory will include the FEV1, FVC, FEV1/FVC ratio, DLCO, IVC, SVC and VA. FEV1 and FVC expressed as % of predicted value, predicted DLCO, hemoglobin (Hb) adjusted predicted DLCO, and DLCO expressed as % of these predicted values will be calculated per the method in section 6.2. The following analysis will be performed:

All the parameters collected at the pulmonary laboratory as well as the % of predicted DLCO and % of Hb adjusted predicted DLCO DLCO will be summarized descriptively by treatment group and overall.

- Change from baseline to other visits for each parameter. The summary for FEV1 will also be provided by smoker status.
- Number and percentage of patients with FEV1/FVC < 60% and <70% by Visit
- DLCO data will also be provided to indicate whether specific determinations met American Thoracic Society (ATS) quality criteria. The proportion of DLCO/spirometry data measurements meeting or not meeting ATS quality criteria will be summarized by treatment group and overall.
- Categories of changes (<-50%, -50% -<-40%, -40% -<-30%, , -30% -<-20%, , -20% -<-10%, -10% -<-10%, 10% -<20%, 20% -<30%, 30% -<40%, 40% -<50%, >=50%) from baseline for FEV1, FEV, FEV1/FVC ratio and DLCO by visit. The summary for FEV1 will also be provided by smoker status.

The descriptive summaries will be repeated for the subset of assessments meeting the ATS quality criteria.



## Statistical Analysis Plan

Another subset analysis will be performed by excluding the DLCO data from patients with a very high intra-individual variability. For the purpose of this analysis, all patients who have a co-efficient of variation (CV) value >7.5% for FEV1 will be excluded. The CV will be calculated for each patient as standard deviation divided by the mean. The screening visit FEV1 data (assessed in ON state) and arrival values at subsequent visits will be used for the calculation.

In addition to the descriptive statistics, the changes in the FEV1, FEV1/FVC ratio, and DLCO values within each treatment group and differences between the treatment groups will be estimated with MMRM. The model will include the treatment group (CVT-301 or observational cohort), visit (visits at 1, 3, 6, 9, and 12 months), the stratification variables (Hoehn and Yahr stage and screening FEV1 and/or FEV1/FVC) and the interaction between the treatment group and visit as fixed factors. The baseline spirometry value will be included as a covariate. An unstructured covariance structure will be applied for MMRM. In case the model will not converge with the unstructured covariance structure, the heterogeneous compound symmetry (CSH) or heterogeneous Toeplitz structure (TOEPH) will be used instead. If the unstructured covariance structure will be used, the denominator degrees of freedom will be computed using the Kenward-Roger method. In case of other covariance structures, the BETWITHIN option will be used for the denominator degrees of freedom. The least square (LS) mean, standard error, and LS mean difference between CVT-301 and observational cohort at each visit; along with the 95% confidence interval (CI) will be provided in a table. Treatment difference will be assessed with a 2-sided alpha level of 0.05, unless specified otherwise.

The SAS code planned for the analysis is outlined below.

The Safety population will be used for the primary analysis.



## Statistical Analysis Plan

#### Sensitivity analyses of the spirometry data

The following sensitivity analysis will be performed for the FEV1, FVC/FEV1 and DLCO assessments.

MI analysis: MI techniques based on Pattern Mixture Models (PMM) will be applied (Ratitch et al., 2011) as a further sensitivity analysis in the Safety population. This methodology will structure data based on missing data patterns. The method will be based on a missingness pattern having a monotone structure, i.e. if among the observations over time one data value is missing, all other values after this missing value will also be treated as missing. For patients with intermittent missing values, before performing MI based on the PMM, it will be necessary to create a monotone missingness pattern. Intermittent missing values will be imputed using the Markov Chain Monte Carlo (MCMC) methodology which assumes a multivariate normal distribution over all variables included in the imputation model. The MI procedure in SAS will be used for this purpose and this first MI step is planned to be repeated 100 times, creating several different datasets with a monotone missing data structure. Seed value of 201508 will be used in the MI procedure. The imputation is based on the missing at random (MAR) assumption, i.e. the missing data are assumed to follow the same model as the other patients in their respective treatment arm that have complete data.

After this, the remaining missing data can be imputed using a method for monotone missingness, also based on the MAR assumption. Thus, for each of the created datasets with a monotone missing data pattern, the MI procedure in SAS will used to impute missing values based on a sequential procedure reflecting the monotone missing data pattern. Patients with the first missing value occurring at visit at Month 1 will have their missing Month 1 value replaced by an imputed value from a regression model with treatment group, baseline spirometry value and the stratification factors as explanatory variables. In the next step, patients with their Month 3 value missing will have their missing Month 3 value replaced by an imputed value from a regression model with treatment group, baseline spirometry value, stratification factors and the Month 1 value as explanatory variables. Similar procedure will be used to replace the missing values at Month 6, 9 and 12.

The imputed datasets generated with the approach described above do contain only non-missing values and are used as input in the model for the primary endpoint. MMRM models similar as described above will thus be run on each of the generated imputed datasets and the difference between the treatment groups will be estimated. The MMRM model will be similar to the primary analysis. Finally, the MIANALYZE procedure in SAS will be applied to combine the results from these several datasets to derive an overall estimate of the within-group changes and



## Statistical Analysis Plan

treatment differences. Estimates and corresponding 95% confidence intervals will be calculated.

The following summary will be performed on the neurology sites data.

- Change from baseline to other visits for each parameter. The baseline is defined as the TV/OV1 Arrival value. If the TV/OV1 Arrival value is missing, the last available value in ON state before the first dose of study drug will be used. The summary for FEV1 will also be provided by smoker status.
- Number and percentage of patients with FEV1/FVC < 60% and <70% by visit</li>
- Spirometry data will also be provided to indicate whether specific determinations met American Thoracic Society (ATS) quality criteria. The proportion of DLCO/spirometry data measurements meeting or not meeting ATS quality criteria will be summarized by treatment group and overall. The summary will also be performed for ON state measurements, OFF state measurements, and all measurements, separately. The reasons for not meeting ATS quality criteria will be summarized, as data allow.
- Categories of changes (<-50%, -50% -<-40%, -40% -<-30%, , -30% -<-20%, , -20% -<-10%, -10% -<-10%, 10% -<20%, 20% -<30%, 30% -<40%, 40% -<50%, >=50%) from baseline for FEV1, FEV, FEV1/FVC ratio and DLCO by visit. The summary for FEV1 will also be provided by smoker status.

#### 8.2. EXTENT OF EXPOSURE

The following information will be summarized for CVT-301 treated subjects:

- The number of patients with dose change
- Duration of exposure (days)
- Total exposure to study treatment, expressed as person years (sum of exposure to study treatment over all CVT - 301 treated patients)
- Total number of doses and capsules taken, by visit and overall. Average number of daily doses and number of capsules, by visit and overall
- Proportion of days with 5, 4, 3, 2, 1 or 0 doses administered
- Proportion of patients using 5, 4, 3, 2, 1 or 0 doses/day at least once

In addition, these in-clinic data will be summarized by treatment group and visit:

- Standard morning dose of LD-containing medications to in-clinic OFF (mins)
- In-clinic OFF to start of study drug inhalation (mins)
- Standard morning dose of LD-containing medications to start of study drug inhalation (mins)



## Statistical Analysis Plan

• Duration of study drug inhalation (mins), calculated as (Completion time of last inhalation - Time of start of first capsule inhalation).

Furthermore, the distribution of time of intake of study medication (00:00 - 00:30, 00:30 - 01:00, ...) as percentage of the total number of study medication intakes will be displayed during the whole treatment period. This data will be collected on the Inhaled Dosing Log.

All study drug data will be listed. A listing will also be provided to show how many times each patient will take study drug and the capsules taken for each day.

#### 8.3. TREATMENT COMPLIANCE

Patients will be instructed to administer inhaled study drug up to 5 times each day during the treatment period. In-clinic administration of study drug will be supervised by study personnel, and at-home diary data will be reviewed to ensure patient compliance. Since there are no fixed scheduled doses for each day, compliance will not be calculated for this study; alternatively, study drug use will be evaluated based on the inhaled medication treatment log by summarizing the proportion of days with >5, 5, 4, 3, 2, 1 or 0 doses administered.

#### 8.4. ADVERSE EVENTS

All AEs will be coded using the MedDRA version 17.0.

Treatment-emergent adverse events (TEAEs) are defined as all AEs that start after the patient receives the first dose of study drug. For the observational cohort, TEAE will be defined as events that occur during/after TV/OV1. Events will be classified as drug-related if the AE is classified as possibly, probably, or definitely related to study drug.

Events with a missing start time, but with a start date equal to the date of first dose of study drug will be considered treatment-emergent. If the AE start date is incomplete, then it will be imputed as follows for the purpose of determining TEAE:

- If the start date is completely missing, the start date will be equal to the first dose date. However, if the stop date is not missing and is before the first dose date, then the stop date will be used instead.
- If the start day is missing, the first day of the month will be used.
- If the start day and month are missing, then the first day of the first month (January) will be used.

The original date and time will be shown on all listings of AEs. Listings will be provided for all AEs, serious AEs, AEs leading to study drug discontinuation, AEs leading to dose

CVT-301-005 Final Version 2.0

Acorda Therapeutics, Inc.



## Statistical Analysis Plan

reduction, and deaths.

TEAEs will be summarized by SOC and PT for each treatment group and overall total. TEAEs with onset after the treatment period are attributed to the treatment group and dose level during the treatment period. Both event and patient counts, where applicable, will be summarized. The counts will be complemented by percentages will be calculated for the patient counts unless otherwise specified. In addition, the incidence of TEAEs, normalized for duration of exposure will be presented (number of TEAEs divided by the total exposure to CVT 301 or observation, measured as patient years).

- An overall summary of the number and percentage of patients reporting TEAEs and the number of TEAE events, drug-related TEAEs, severe TEAEs, serious TEAEs, TEAEs leading to dose interruption, TEAEs leading to study drug discontinuation, TEAEs leading to dose reduction and TEAEs leading to death
- TEAEs by SOC and PT, both as event and patient counts
- TEAEs by PT, both as event and patient counts
- Drug-related TEAEs by SOC and PT, both as event and patient counts
- Severe TEAEs by SOC and PT, both as event and patient counts
- Drug-related TEAEs by SOC, PT and severity, as event counts; percentages will be calculated for the event count out of total number of events
- Drug-related TEAEs by SOC, PT and relationship, as event counts; percentages will be calculated for the event count out of total number of events
- Serious TEAEs by SOC and PT, both as event and patient counts
- TEAEs leading to study drug interruption, both as event and patient counts
- TEAEs leading to study drug withdrawal, both as event and patient counts
- TEAEs leading to dose reduction, both as event and patient counts
- Most common AEs, both as event and patient counts, most common TEAEs is defined any AE preferred term occurred in greater than 10% total patients.
- Time to first onset of most common AEs, classified as 0-1 months, >1-3 months, >3-6 months, >6-9 months and after 9 months, where the date of TEAE onset will be used as the time point for classification.

The tables will be sorted by overall descending frequency of SOC and then, within a SOC, by overall descending frequency of PT based on the patient count for the Total column. If only event count is presented, the sorting will be done based on the event count.

#### 8.5. LABORATORY EVALUATIONS

Laboratory samples for hematology and clinical chemistry will be analyzed by a central

1003805 Acorda Therapeutics, Inc. CVT-301-005




## Statistical Analysis Plan

laboratory (located in the United Kingdom for EU sites and the United States for US sites) to ensure consistent interpretation of results. In the event of an unexplained clinically significant abnormal laboratory test value, the test should be repeated immediately and followed up until it has returned to the normal range and/or an adequate explanation of the abnormality is found.

All parameters will be converted to consistent units according to the International System of Units (SI) before summarization. The following will be summarized by treatment group and overall:

- Actual values and change from baseline, if applicable, at each visit for each parameter (for handling of data from the ET visit, see Section 6.4)
- Number and percentage of patients with normal or "abnormal" (i.e., out of reference range) labs at each visit for each parameter
- Number and percentage of patients with potentially clinically significant (PCS) lab values at each visit for each parameter
- Number and percentage of patients with potentially clinically significant changes (PCSC) in lab values at each post-baseline visit for each parameter

PCS and PCSC will be identified for specific laboratory parameters as outlined in the following table.



## Statistical Analysis Plan

| Laboratory<br>Parameter | Units | Criteria for PCS Values (Actual values) | | Criteria for PCSC values<br>(Changes from baseline<br>values) | |
|---|---|---|---|---|---|
| | | High | Low | % increase | % decrease |
| Hemoglobin | g/L | > 10 above ULN | >20 below LLN | NA | 25% |
| Hematocrit | L/L | >0.04 above ULN | >0.05 below LLN | NA | 25% |
| WBC | GI/L | >5 above ULN | >1 below LLN | 100% | 50% |
| Neutrophils | GI/L | NA | <0.5xLLN | 100% | 50% |
| Neutrophils | % | NA | <0.5xLLN | 100% | 50% |
| Lymphocytes | GI/L | NA | <0.5xLLN | 100% | 50% |
| Lymphocytes | % | NA | <0.5xLLN | 100% | 50% |
| Total bilirubin | µmol/L | >1.5xULN | NA | 300% | NA |
| Total protein | g/L | >15 above ULN | >15 below LLN | 200% | 60% |
| Albumin | g/L | >5 above ULN | >5 below LLN | NA | 60% |
| AST | U/L | >3xULN | NA | 300% | NA |
| ALT | U/L | >3xULN | NA | 300% | NA |
| Alkaline | U/L | >3xULN | NA | 300% | NA |
| Phosphatase | | | | | |
| GGT | U/L | >3xULN | NA | 300% | NA |
| Creatinine | µmol/L | >1.5xULN | NA | 200% | NA |
| Urea | mmol/L | >2.5xULN | NA | 300% | NA |
| Uric Acid | µmol/L | >3xULN | NA | 300% | NA |
| Sodium | mmol/L | >5 above ULN | >5 below LLN | 10% | 10% |
| Potassium | mmol/L | >1 above ULN | >0.5 below LLN | 25% | 20% |
| Carbon dioxide | mmol/L | >40 | <16 | 25% | 25% |
| Calcium | mmol/L | >2.99 | <1.78 | 30% | 30% |
| Glucose (fasting)* | mmol/L | >11.1 | <2.8 | 300% | 40% |

ULN = Upper limit of normal range, LLN = Lower limit of normal range

Baseline is defined as the visit 3 assessment. If the visit 3 assessment is missing, the last non-missing screening assessment will be used as baseline. \* fasting defined as  $\geq 4$  hr from prior meal

The tables showing the normal/abnormal values, PCS values and PCSCs will be done both as summaries of all data and as shift tables (i.e., classified by the baseline status).

Values which fall outside the central laboratory normal range will be flagged as "L" - below normal range, or "H" - above normal range, on the data listings. PCS and PCSC values will also be flagged. All repeated values will be presented on the data listings but not included in the summaries showing data by visit.

#### 8.6. VITAL SIGNS

Standard vital sign measurements will include RR, systolic and diastolic BP (SBP, DBP), and HR. At SV1 (or SV2) and each of the subsequent study visits, and in the event of a clinically significant finding that could be suggestive of symptomatic orthostatic



## Statistical Analysis Plan

hypotension (e.g., dizziness, lightheadedness, or other AE), orthostatic vital signs will be performed. Orthostatic vital sign measurements will include SBP, DBP, and HR.

The following will be summarized:

- Change from baseline to other visit for each parameter. The baseline is defined as the TV/OV1. If TV/OV1 is missing, the last non-missing screening assessment will be used as baseline.
- Actual values and change from pre-dose to post-dose time points at TV/OV1 by time point for each parameter for CVT-301 treated patients
- Number and percentage of patients with PCS values at each applicable visit and time point for each standard vital sign parameter
- Number and percentage of patients with PCSC values at each applicable visit and time point for each standard vital sign parameter
- Number and percentage of patients with Orthostatic hypotension at each applicable visit

PCS and PCSC for standard vital sign will be identified as outlined in the following table.

| Vital Sign | Units | Criteria for PCS Values<br>(Actual values) | | Criteria for PCSC values<br>(Change from Baseline or<br>pre-dose values *) | |
|---|---|---|---|---|---|
| | | High | Low | increase | decrease |
| Pulse rate | bpm | >120 | <40 | 100 | 50 |
| Respiration Rate | brpm | >32 | <8 | 50 | NA |
| Systolic Blood | mmHg | >200 | <85 | 60 | 20 |
| Pressure (supine) | | | | | |
| Diastolic Blood | mmHg | >120 | <40 | | 0.2x |
| pressure (supine) | | | | | |

<sup>\*</sup>Pre-dose values will be used for corresponding post-dose values assessment at TV/OV1. Otherwise baseline values are used.

Orthostatic hypotension will be defined as a reduction in SBP of 20 mmHg or more, and/or a reduction in DBP of 10 mmHg or more, for the standing measurement compared to the supine/semi-supine measurement.

#### 8.7. ELECTROCARDIOGRAM

Standard 12-lead ECGs will be obtained after the patient has rested in a supine position for at least 5 minutes. Electrocardiograms will be measured using an ECG machine that automatically calculates the HR and measures PR, QRS, QT, QT interval corrected using Bazett's formula (QTcB) and QT interval corrected using Fridericia's formula (QTcF).



## Statistical Analysis Plan

The following will be summarized:

- Change from baseline to other visit for each parameter. The baseline is defined
  as the TV/OV1 value. If TV/OV1 value is missing, the last non-missing screening
  assessment will be used as baseline.
- Number and percentage of patients with PCS values at each applicable visit for each parameter
- Number and percentage of patients with PCSC values at each applicable visit for each parameter

PCS and PCSC will be identified as outlined in the following table.

| ECG | Units | Criteria for PCS Values | | Criteria for PCSC values (Change from | |
|---|---|---|---|---|---|
| | | (Actual values) | | Baseline) | |
| | | High | Low | increase | decrease |
| PR interval | msec | >300 | NA | >25% for baseline ≥200 | NA |
| | | | | >50% for baseline <200 | |
| QRS interval | msec | >200 | NA | >25% for baseline ≥100 | NA |
| | | | | >50% for baseline <100 | |
| QTcB | msec | >500 | NA | >15% for baseline ≥440 | NA |
| | | | | >30% for baseline <440 | |
| | | | | >30 msec increase | |
| | | | | >60 msec increase | |
| | | | | Change>30 and value>500 | |
| | | | | Change>60 and value>500 | |
| QTcF | msec | >500 | NA | >15% for baseline ≥440 | NA |
| | | | | >30% for baseline <440 | |
| | | | | >30 msec increase | |
| | | | | >60 msec increase | |
| | | | | >Change>30 and value>500 | |
| | | | | Change>60 and value>500 | |
| Heart Rate | bpm | >120 | <35 | NA | NA |

#### 8.8. PHYSICAL EXAMINATION

A complete physical examination (head, eyes, ears, nose, and throat [HEENT], heart, lungs, abdomen, skin, cervical and axillary lymph nodes, neurological, and musculoskeletal systems) will be performed at screening. Genital, rectal, and breast examination may be excluded if not clinically indicated.

The following will be summarized:

 Total number and percentage of patients reporting abnormal clinically significant physical examination results



## Statistical Analysis Plan

#### 8.9. COLUMBIA-SUICIDALITY SEVERITY RATING SCALE

The C-SSRS is a measure of suicidal ideation and behavior. The rating scale has 4 general categories: suicidal ideation, intensity of ideation, suicidal behavior, and actual attempts. All C-SSRS data will be listed. The frequency and percentage of patients with each response for suicidal ideation, intensity of ideation, and suicidal behavior items will be summarized as appropriate by treatment group and overall.

A shift from baseline table will be constructed to assess any changes in the subjects' suicidal ideation and behavior during the treatment period.

#### 8.10. EPWORTH SLEEPINESS SCALE

The Epworth Sleepiness Scale is used to determine the level of daytime sleepiness. There are 8 situations listed for which patients rate their likelihood of dozing or sleeping (0=would never doze or sleep, 1=slight chance of dozing or sleeping, 2=moderate chance of dozing or sleeping, and 3=high chance of dozing or sleeping). The total score is the sum of 8 item scores and can range between 0 and 24. In case of missing item scores, the missing value will be replaced by the average of non-missing scores at the same visit from the same patient. In case all item scores are missing, the total score will be set as missing. The higher total score indicates the higher level of daytime sleepiness. A score of 10 or more is considered sleepy, and a score of 18 or more is very sleepy.

All Epworth Sleepiness Scale data will be listed. The total score and change from baseline will be summarized by treatment group and overall (for handling of data from the ET visit, see Section 6.4).

# 8.11. QUESTIONNAIRE FOR IMPULSIVE-COMPULSIVE DISORDERS IN PARKINSON'S DISEASE

The QUIP is an instrument used to measure the extent of impulsive and compulsive behaviors in PD patients. The QUIP has 3 sections: Section 1 assesses any impulsive control disorder (gambling, sexual, buying, and eating disorders); Section 2 assesses other compulsive behaviors (punding, hobbyism, and walkabout); and Section 3 assesses compulsive medication use.

The frequency and percentage of patients with positive response for each of the item within each section will be summarized by visit treatment group and overall. The assessment of positive response for each item will be based on the table below.

1003805 Acorda Therapeutics, Inc. CVT-301-005




## Statistical Analysis Plan

| Section and Item | Number of items with positive response |
|-------------------------------|----------------------------------------|
| A. Impulse Control Disorders | |
| Compulsive gambling | any 2 of the 5 gambling items |
| Compulsive sexual behavior | any 1 of the 5 sexual behavior items |
| Compulsive buying | any 1 of the 5 buying items |
| Compulsive eating | any 2 of the 5 eating items |
| B. Other Compulsive Behaviors | |
| Hobbyism | item #1A |
| Punding | item #1B |
| Walkabout | item #1C |
| C. Compulsive Medication Use | items #1 and #4 |

#### **8.12. UPDRS PART 4**

Changes from baseline to the subsequent visits in UPDRS Part 4 sum scores (dyskinesia sum score, wearing-off sum score) will be analyzed using a similar MMRM as for the UPDRS Part 3 scores (described below) to estimate the within-group changes. Otherwise, the data will be presented with descriptive statistics only classified by visit for CVT treated patients. The observed cases will be used in the analysis and summaries.

#### 8.13. EXAMINER-RATED DYSKINESIA

The occurrence and severity will be tabulated by treatment group and visit. The observed cases will be used in the summaries. No formal statistical methods will be used.



## Statistical Analysis Plan

#### 9. EXPLORATORY EFFICACY

#### 9.1. EXPLORATORY EFFICACY ENDPOINT AND ANALYSIS

The ITT population will be used for the exploratory efficacy analysis. Patients will be analyzed according to randomized treatment. The within group changes from baseline in continuous efficacy variables will be estimated using an MMRM. No between group differences will be calculated, unless otherwise specified. The model will include visit and the stratification variables (Hoehn and Yahr stage and screening FEV1 and/or FEV1/FVC) as fixed factors. The baseline value will be used as a covariate. For variables which do not have a pretreatment baseline assessment, OFF-state baseline UPDRS Part 3 score will be used as the baseline covariate. An unstructured covariance structure will be applied for the MMRM. In case the model will not converge with the unstructured covariance structure, compound symmetry will be used instead. For all patients, categorical data will be evaluated descriptively. Each visit will be evaluated separately for the categorical endpoints. The exploratory efficacy endpoints and associated analyses are as follows. For the detailed definition of the endpoints, see Section 4.3.

- Change from pre-dose in UPDRS Part 3 motor score at 10, 20, 30, and 60 minutes and the average of the motor score at 10-60 following treatment of patients experiencing an OFF episode in the clinic. Change from pre-dose in the average UPDRS Part 3 score at 10 to 60 minutes is calculated as the mean of change of UPDRS Part III total score from pre-dose to each time point post-dose if UPDRS Part III total score is available for at least 2 time points post-dose. The scheduled post-dose UPDRS Part III assessments are at 10, 20, 30, 60 minutes post-dose, respectively. If there is more than 2 time points post-dose with missing UPDRS Part III total score, the change of UPDRS Part III total score from pre-dose to 10 to 60 minutes post-dose will be missing. A MMRM model as defined above will be used.
- Time curve of the UPDRS response shown as change from pre-dose in UPDRS Part 3 motor score to 10, 20, 30 and 60 minutes following treatment of patients experiencing an OFF episode in the clinic. A separate MMRM model will be fitted for each of the time points.
- A ≥3, ≥6, and ≥11 point reduction in the UPDRS Part 3 motor score from pre-dose to post-dose, at 10 to 60 minutes following treatment in the clinic (cumulative and non-cumulative). For the non-cumulative analysis, the proportions of patients with a reduction will be tabulated by treatment group, visit and time point. For the cumulative analysis, the cumulative proportions of patients who achieved the first reduction before or at the time point in question will be tabulated by visit and time point.



## Statistical Analysis Plan

- Resolution of an OFF to an ON state within 60 minutes after study drug is administered in the clinic and maintaining the ON at 60 minutes after study drug administration (per the examiner's subjective assessment). This endpoint will be based on the examiner's subjective assessment. The proportions of patients will be summarized descriptively for each CVT-301 treated patients. The missing values will be counted as non-resolved.
- Change from baseline (3 consecutive days prior to TV1) in patient-recorded total daily OFF time, assessed by the patient and recorded in the PD Diary for 3 consecutive days prior to the visit. Similar methods as for primary endpoint will be used. However, the baseline daily OFF time will be used as a covariate in the MMRM model instead of the OFF-state baseline UPDRS part 3 score. Only valid diary days will be included in the diary summarizations. In addition, change from baseline in total daily ON time without dyskinesia, total daily ON time with non-troublesome dyskinesia, and total daily ON time with troublesome dyskinesia.
- The PGI-C score. The proportions of patients who improved (much improved, improved or a little improved) will be tabulated by visit for CVT-301 treated patients. This summary will be complemented by the distribution of each response category (much improved, improved, a little improved, no change, a little worse, worse, much worse) tabulated by the treatment group.
- Changes from TV/OV1 in endpoints based on S&E ADL score, UPDRS Part 2 score, and PDQ-39 sub-scores. An ANCOVA model with the treatment group and stratification variables as fixed factors and the TV/OV1 value as a covariate will be used to estimate the treatment differences. Otherwise, the data will be presented with descriptive statistics only classified by treatment group and visit. The observed cases will be used in the analysis and summaries.

#### Sensitivity analyses of the exploratory efficacy data

The following sensitivity analysis will be performed for the UPDRS Part 3 motor scores at 30 minutes post-dose and daily OFF time exploratory efficacy endpoints.

• MI analysis: MI techniques based on Pattern Mixture Models (PMM) will be applied (Ratitch et al., 2011) as a further sensitivity analysis in the ITT population. This methodology will structure data based on missing data patterns. The method will be based on a missingness pattern having a monotone structure, i.e. if among the observations over time one data value is missing, all other values after this missing value will also be treated as missing. For patients with intermittent missing values, before performing MI based on the PMM, it will be necessary to create a monotone missingness pattern. Intermittent missing values will be imputed using the Markov Chain Monte Carlo (MCMC) methodology which assumes a multivariate normal



## Statistical Analysis Plan

distribution over all variables included in the imputation model. The MI procedure in SAS will be used for this purpose and this first MI step is planned to be repeated 100 times, creating several different datasets with a monotone missing data structure. Seed value of 201508 will be used in the MI procedure. The imputation is based on the missing at random (MAR) assumption, i.e. the missing data are assumed to follow the same model as the other patients in their respective treatment arm that have complete data.

After this, the remaining missing data can be imputed using a method for monotone missingness, also based on the MAR assumption. Thus, for each of the created datasets with a monotone missing data pattern, the MI procedure in SAS will used to impute missing values based on a sequential procedure reflecting the monotone missing data pattern. Patients with the first missing value occurring at visit at Month 1 will have their missing Month 1 value replaced by an imputed value from a regression model with baseline value and the stratification factors as explanatory variables. In the next step, patients with their Month 3 value missing will have their missing Month 3 value replaced by an imputed value from a regression mode with baseline spirometry value, stratification factors and the Month 1 value as explanatory variables. Similar procedure will be used to replace the missing values at Month 6, 9 and 12.

The imputed datasets generated with the approach described above do contain only non-missing values and are used as input in the model for the exploratory efficacy endpoint. MMRM models similar as described above will thus be run on each of the generated imputed datasets. Finally, the MIANALYZE procedure in SAS will be applied to combine the results from these several datasets to derive an overall estimate of the within-group changes.



## Statistical Analysis Plan

#### 10. INTERIM ANALYSES

Safety data will be reviewed by a Data Safety Monitoring Committee (DSMC) that will include relevant medical experts (including a neurologist and pulmonologist), an independent statistician, and additional representatives (as will be defined in the DSMC Charter). Safety data, including but not limited to AEs, spirometry, vital signs, and ECG data will be reviewed. The safety review will be documented in a DSMC Charter prior to the start of the study. In the event that potential safety issues are identified, the committee may recommend modification of the study design or study termination, which will be communicated promptly with investigators, IRBs, IECs, and regulatory agencies, in accordance with legal and regulatory requirements.

Data summary, which will not affect study conduct, may be prepared to support regulatory submission.



## Statistical Analysis Plan

## 11. CHANGE FROM ANALYSIS PLANNED IN PROTOCOL

There are no changes from the analyses planned in the protocol.



## Statistical Analysis Plan

#### 12. PROGRAMMING CONSIDERATIONS

All tables, listings, figures (TLFs), and statistical analyses will be generated using SAS® for Windows, Release 9.3 (SAS® Institute Inc., Cary, NC, USA) or higher. Computergenerated table, listing and figure output produced by INC Research will adhere to the following specifications.

#### 12.1. GENERAL CONSIDERATIONS

- One SAS program can create several outputs.
- One output file can contain several outputs.
- Output files will be delivered in Word format.
- Numbering of TFLs will follow ICH E3 guidance

#### 12.2. TABLE, LISTING, AND FIGURE FORMAT

#### 12.2.1. General

- All TLFs will be produced in landscape format, unless otherwise specified.
- All TLFs will be produced using the Courier New font, size 8
- The data displays for all TLFs will have a 1.5-inch binding margin on top of a landscape oriented page and a minimum 1-inch margin on the other 3 sides.
- Headers and footers for figures will be in Courier New font, size 8.
- Legends will be used for all figures with more than 1 variable, group, or item displayed.
- TLFs will be in black and white (no color), unless otherwise specified. For spirometry graphs, separate colors will be used for ON (red circles) and OFF (blue triangles) State data.
- Specialized text styles, such as bolding, italics, borders, shading, and superscripted and subscripted text, will not be used in the TLFs, unless otherwise specified.
- Only standard keyboard characters will be used in the TLFs. Special characters, such as non-printable control characters, printer-specific, or font-specific characters, will not be used.
- Mixed case will be used for all titles, column headers, and programmer-supplied formats, as appropriate.

#### 12.2.2. Headers

All output should have the following header at the top left of each page:



## Statistical Analysis Plan

Civitas Therapeutics, Inc.

- All output should have Page n of N at the top or bottom right corner of each page.
  TLFs should be internally paginated in relation to the total length (i.e., the page
  number should appear sequentially as page n of N, where N is the total number of
  pages in the table).
- The date and time (date and time output was generated) should appear along with program name and location as the last footer on each page.

### 12.2.3. Display Titles

• Each TLF should be identified by the designation and a numeral. (i.e., Table 14.1.1). The title is centered. The title and table designation are single spaced. A solid line spanning the margins will separate the display titles from the column headers. There will be 1 blank line between the last title and the solid line.

#### 12.2.4. Column Headers

- Column headings should be displayed immediately below the solid line described above.
- Analysis set sizes will be presented for each treatment group in the column heading as (N=xx) (or in the row headings if applicable). This is distinct from the 'n' used for the descriptive statistics representing the number of patients in the analysis set.
- The order of treatments in the tables will be Placebo first, followed by CVT-301 and a total column (if applicable in tables).

#### 12.2.5. Body of the Data Display

#### 12.2.5.1. General Conventions

Data in columns of a table or listing should be formatted as follows:

- alphanumeric values are left-justified;
- whole numbers (e.g., counts) are right-justified; and
- numbers containing fractional portions are decimal aligned.

#### 12.2.5.2. Table Conventions

- Units will be included where available
- Unless otherwise specified, the estimated mean and median for a set of values should be printed out to 1 more significant digit than the original values, and



## Statistical Analysis Plan

standard deviations should be printed out to 2 more significant digits than the original values. The minimum and maximum should report the same significant digits as the original values. For example, for systolic blood pressure:

| N | XX |
|---------|-------|
| Mean | XXX.X |
| Std Dev | X.XX |
| Median | XXX.X |
| Minimum | XXX, |
| Maximum | XXX |

- P-values should be output in the format: "0.xxx", where xxx is the value rounded to 3 decimal places. Any p-value less than 0.001 will be presented as <0.001. If the p-value is returned as >0.999 then present as >0.999.
- Percentage values should be printed to one decimal place, in parentheses with no spaces, one space after the count, e.g., 7 (12.8%), 13 (5.4%). For a value that rounds down to 0.0, display it as "<0.1". Unless otherwise noted, for all percentages, the number of patients in the analysis set for the treatment group who have an observation will be the denominator. Percentages after zero counts should not be displayed and percentages equating to 100% should be presented as 100%, without any decimal places.

#### 12.2.5.3. Listing Conventions

- Listings will be sorted for presentation in order of patient number, visit/collection day, and visit/collection time.
- Dates should be printed in SAS® DATE9.format ("ddMMMyyyy": 01JUL2000). Missing portions of dates should be represented on patient listings as dashes (--JUL2000).
- All observed time values must be presented using a 24-hour clock HH:MM or HH:MM:SS format (e.g., 11:26:45, or 11:26).

#### 12.2.6. Footnotes

- A solid line spanning the margins will separate the body of the data display from the footnotes.
- All footnotes will be left justified with single-line spacing immediately below the solid line underneath the data display.

1003805

Acorda Therapeutics, Inc. CVT-301-005 Final Version 2.0



## Statistical Analysis Plan

• The last line of the footnote section will be a standard source line that indicates the name of the program used to produce the data display, date and time the program was run.



## Statistical Analysis Plan

### 13. QUALITY CONTROL

SAS programs are developed to produce clinical trial output such as analysis data sets, summary tables, data listings, figures or statistical analyses. INC Research SOP 03.010.00 and 03.013.00 provide an overview of the development of such SAS programs.

INC Research SOP 03.009.00 describes the quality control procedures that are performed for all SAS programs and output. Quality control is defined here as the operational techniques and activities undertaken to verify that the SAS programs produce the proper clinical trial output by checking for their logic, efficiency and commenting and by review of the produced output.

CVT-301-005




## Statistical Analysis Plan

## 14. INDEX OF TABLES

| Table 14.1.1.1 | Number of Subjects Enrolled and Study Termination (All Available Population) |
|---|---|
| Table 14.1.1.2 | Number of Subjects in Each Population by Study Center All Subjects |
| Table 14.1.2.1 | Summary of Protocol Deviation Randomized Set |
| Table | Demographic and Baseline Characteristics (Safety Population) |
| 14.1.3.1.1 | |
| Table | Demographic and Baseline Characteristics (ITT Population) |
| 14.1.3.1.2 | |
| Table | Demographic and Baseline Characteristics by Baseline PD Severity (ITT |
| 14.1.3.1.3 | Population) |
| Table | Demographic and Baseline Characteristics by Baseline Dyskinesia (ITT |
| 14.1.3.1.4 | Population) |
| Table | Demographic and Baseline Characteristics by Baseline Daily Levodopa Dose (ITT |
| 14.1.3.1.5 | Population) |
| Table | Demographic and Baseline Characteristics by PD Diary Mean Daily OFF Time |
| 14.1.3.1.6 | during Screening (ITT Population) |
| Table | Demographic and Baseline Characteristics by Screening Spirometry (ITT |
| 14.1.3.1.7 | Population) |
| Table | Demographic and Baseline Characteristics by Age Group (ITT Population) |
| 14.1.3.1.8 | |
| Table | Demographic and Baseline Characteristics by Gender (ITT Population) |
| 14.1.3.1.9 | |
| Table | Parkinson's Disease History (Safety Population) |
| 14.1.3.2.1 | |
| Table | Parkinson's Disease History (ITT Population) |
| 14.1.3.2.2 | |
| Table | Parkinson's Disease History by Baseline PD Severity (ITT Population) |
| 14.1.3.2.3 | |
| Table | Parkinson's Disease History by Baseline Dyskinesia (ITT Population) |
| 14.1.3.2.4 | |
| Table | Parkinson's Disease History by Baseline Daily Levodopa Dose (ITT Population) |
| 14.1.3.2.5 | |
| Table | Parkinson's Disease History by PD Diary Mean Daily OFF Time during Screening |
| 14.1.3.2.6 | (ITT Population) |
| Table | Parkinson's Disease History by Screening Spirometry (ITT Population) |
| 14.1.3.2.7 | D. L. D. W. L. L. C. (ITT D. L.) |
| Table | Parkinson's Disease History by Age Group (ITT Population) |
| 14.1.3.2.8 | Deddinger). Discour History by Conday (ITT D. 1911) |
| Table | Parkinson's Disease History by Gender (ITT Population) |
| 14.1.3.2.9 | Madified Hasher and Value Chaming in "ONI" Chate (Cafate Daniel Line) |
| Table | Modified Hoehn and Yahr Staging in "ON" State (Safety Population) |
| 14.1.3.2.10 | Madified Hasher and Value Chaming in "ONI" Chata (ITT Danielation) |
| Table | Modified Hoehn and Yahr Staging in "ON" State (ITT Population) |
| 14.1.3.2.11 | Distribution of Average Daily OFF Time (C-f-ty Decoletion) |
| Table | Distribution of Average Daily OFF Time (Safety Population) |



| 14.1.3.2.12 | |
|---|---|
| Table | Distribution of cumulative Average Daily OFF Time (Safety Population) |
| 14.1.3.2.13 | biscribation of camatative riverage barry of thine (surety repatation) |
| Table 14.1.3.3 | Medical History (Safety Population) |
| Table 14.1.4.1 | Prior Medications (Safety Population) |
| Table 14.1.4.2 | Concomitant Medications (Safety Population) |
| Table 14.1.4.3 | Parkinson's disease Treatment Medications at Baseline (ITT Population) |
| Table 14.2.1.1 | Exploratory Efficacy Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 10 Minutes Post-dose by Visit (ITT Population) |
| Table 14.2.1.2 | Exploratory Efficacy Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 20 Minutes Post-dose by Visit (ITT Population) |
| Table | Exploratory Efficacy Analysis: Change from Pre-dose in the UPDRS Part 3 Score at |
| 14.2.1.3.1 | 30 Minutes Post-dose by Visit (ITT Population) |
| Table | Sensitivity Analysis: Change from Pre-dose in the UPDRS Part 3 Score at 30 |
| 14.2.1.3.2 | Minutes Post-dose by Visit (ITT Population) |
| Table | Exploratory Efficacy Subgroup Analysis: Change from Pre-dose in the UPDRS Part |
| 14.2.1.3.3 | 3 Score at 30 Minutes Post-dose by Visit by Baseline PD Severity (ITT Population) |
| Table | Exploratory Efficacy Subgroup Analysis: Change from Pre-dose in the UPDRS Part |
| 14.2.1.3.4 | 3 Score at 30 Minutes Post-dose by Visit by Baseline Dyskinesia (ITT Population) |
| Table | Exploratory Efficacy Subgroup Analysis: Change from Pre-dose in the UPDRS Part |
| 14.2.1.3.5 | 3 Score at 30 Minutes Post-dose by Visit by Baseline Daily Levodopa Dose (ITT |
| | Population) |
| Table | Exploratory Efficacy Subgroup Analysis: Change from Pre-dose in the UPDRS Part |
| 14.2.1.3.6 | 3 Score at 30 Minutes Post-dose by Visit by PD Diary Mean Daily OFF Time during |
| | Screening (ITT Population) |
| Table | Exploratory Efficacy Exploratory Efficacy Subgroup Analysis: Change from Pre- |
| 14.2.1.3.7 | dose in the UPDRS Part 3 Score at 30 Minutes Post-dose by Visit by Screening |
| 11.2.11.5.7 | Spirometry (ITT Population) |
| Table | Exploratory Efficacy Exploratory Efficacy Subgroup Analysis: Mean Change from |
| 14.2.1.3.8 | Pre-dose in the UPDRS Part 3 Score at 30 Minutes Post-dose by Visit by Age Group |
| 14.2.1.3.0 | (ITT Population) |
| Table | Exploratory Efficacy Exploratory Efficacy Subgroup Analysis: Mean Change from |
| 14.2.1.3.9 | Pre-dose in the UPDRS Part 3 Score at 30 Minutes Post-dose by Visit by Gender |
| 14.2.1.3.7 | (ITT Population) |
| Table 14.2.1.4 | Exploratory Efficacy Analysis: Change from Pre-dose in the UPDRS Part 3 Score at |
| 14.2.1.4 | 60 Minutes Post-dose by Visit (ITT Population) |
| Table 14.2.1.5 | Exploratory Efficacy Analysis: Change from Pre-dose in the Average UPDRS Part |
| 14500 17.2.1.3 | 3 Score at 10 to 60 Minutes Post-dose by Visit (ITT Population) |
| Table 14.2.2.1 | Exploratory Efficacy Analysis: Change from Pre-dose in UPDRS Part 3 Score to 10, |
| | 20, 30, 60 minutes Post-dose by Visit (ITT Population) |
| Table 14.2.2.2 | Exploratory Efficacy Analysis: Change from Pre-Dose to 10, 20, 30, 60 minutes |
| | Post-dose in UPDRS Part 3 Score by Visit and Timepoint (ITT Population) |
| Table 14.2.2.3 | Exploratory Efficacy Analysis: Change from Pre-Dose to 10, 20, 30, 60 minutes |
| | Post-dose in UPDRS Part 3 Score by Timepoint and Visit (ITT Population) |
| Table 14.2.3.1 | Exploratory Efficacy Analysis Subjects with a >= 3 Reduction from Pre-dose to |
| . 45.6 . 1.2.5.1 | _ injuries and _ inju |



| | Post-dose in the UPDRS Part 3 Score by Visit (ITT Population) |
|---|---|
| Table 14.2.3.2 | Exploratory Efficacy Analysis Subjects with a >= 3 Reduction from Pre-dose to |
| 14.2.3.2 | Post-dose in the UPDRS Part 3 Score by Visit With Percentages Based on N (ITT |
| | Population) |
| Table 14.2.3.3 | Exploratory Efficacy Analysis Subjects with a >=6 Reduction from Pre-dose to |
| 145(6 1 1.2.3.3 | Post-dose in the UPDRS Part 3 Score by Visit (ITT Population) |
| Table 14.2.3.4 | Exploratory Efficacy Analysis Subjects with a >=6 Reduction from Pre-dose to |
| 1 4546 1 112151 1 | Post-dose in the UPDRS Part 3 Score by Visit With Percentages Based on N (ITT |
| | Population) |
| Table 14.2.3.5 | Exploratory Efficacy Analysis Subjects with a >=11 Reduction from Pre-dose to |
| | Post-dose in the UPDRS Part 3 Score by Visit (ITT Population) |
| Table 14.2.3.6 | Exploratory Efficacy Analysis Subjects with a >=11 Reduction from Pre-dose to |
| | Post-dose in the UPDRS Part 3 Score by Visit With Percentages Based on N (ITT |
| | Population) |
| Table 14.2.4.1 | Exploratory Efficacy Analysis: Subjects Achieving Resolution of an OFF to an ON |
| | State within 60 Minutes by Visit Worst Case Imputation [a] (ITT Population) |
| Table | Exploratory Efficacy Analysis: Mean of Total Daily OFF Time by Visit (ITT |
| 14.2.5.1.1 | Population) |
| Table | Sensitivity Analysis: Mean of Total Daily OFF Time by Visit MI analysis with Missing |
| 14.2.5.1.2 | At Random Assumption (ITT Population |
| Table | Exploratory Efficacy Subgroup Analysis: Mean of Total Daily OFF Time by Visit by |
| 14.2.5.1.3 | Baseline PD Severity (ITT Population) |
| Table | Exploratory Efficacy Subgroup Analysis: Mean of Total Daily OFF Time by Visit by |
| 14.2.5.1.4 | Baseline Dyskinesia (ITT Population) Exploratory Efficacy Subgroup Analysis: Mean of Total Daily OFF Time by Visit by |
| Table<br>14.2.5.1.5 | Baseline Daily Levodopa Dose (ITT Population) |
| Table | Exploratory Efficacy Subgroup Analysis: Mean of Total Daily OFF Time by Visit by |
| 14.2.5.1.6 | PD Diary Mean Daily OFF Time during Screening (ITT Population) |
| Table | Exploratory Efficacy Subgroup Analysis: Mean of Total Daily OFF Time by Visit by |
| 14.2.5.1.7 | Screening Spirometry (ITT Population) |
| Table | Exploratory Efficacy Subgroup Analysis: Mean of Total Daily OFF Time by Visit by |
| 14.2.5.1.8 | Age Group (ITT Population) |
| Table | Exploratory Efficacy Subgroup Analysis: Mean of Total Daily OFF Time by Visit by |
| 14.2.5.1.9 | Gender (ITT Population) |
| Table 14.2.5.2 | Exploratory Efficacy Analysis: Mean of Total Daily ON Time without Dyskinesia by |
| | Visit (ITT Population) |
| Table 14.2.5.3 | Exploratory Efficacy Analysis: Mean of Total Daily ON Time with non-Troublesome |
| | Dyskinesia by Visit (ITT Population) |
| Table 14.2.5.4 | Exploratory Efficacy Analysis: Mean of Total Daily ON Time with Troublesome |
| | Dyskinesia by Visit (ITT Population) |
| Table 14.2.6.1 | Exploratory Efficacy Analysis: Subjects Global Impression of Change (PGI-C) by |
| T. I.I. 440.74 | Visit Worst Case Imputation [a] (ITT Population) |
| Table 14.2.7.1 | Exploratory Efficacy Analysis: UPDRS Part 2 Score at TV4/OV4 (ITT Population) |
| Table 14.2.7.2 | Exploratory Efficacy Analysis: UPDRS Part 2 Score at TV6/OV6 (ITT Population) |
| Table 14.2.8.1 | Exploratory Efficacy Analysis: Schwab and England (S&E) Activities of Daily |
| | Living (ADL) Score at TV4/OV4 (ITT Population) |

CVT-301-005 Final Version 2.0



| Table 14.2.8.2 | Exploratory Efficacy Analysis: Schwab and England (S&E) Activities of Daily Living |
|---|---|
| Table 14.2.0.1 | (ADL) Score at TV6/OV6 (ITT Population) |
| Table 14.2.9.1 | Exploratory Efficacy Analysis: 39 Item Parkinson's disease Questionnaire (PDQ-39) Sub-scores and Summary Index Score at TV4/OV4 (ITT Population) |
| Table 14.2.9.2 | Exploratory Efficacy Analysis: 39 Item Parkinson's disease Questionnaire (PDQ-39) |
| | Sub-scores and Summary Index Score at TV6/OV6 (ITT Population) |
| Table 14.3.1.1 | Extent of Exposure: Overall (Safety Population) |
| Table 14.3.1.2 | In-Clinic Study Drug Administration (Safety Population) |
| Table 14.3.1.3 | Distribution of Time of Study Drug Administration (Safety Population) |
| Table 14.3.2.1 | Treatment-emergent adverse events -Overall Summary (Safety Population) |
| Table | Treatment-emergent adverse events by System Organ Class and Preferred Term |
| 14.3.2.2.1 | (Safety Population) |
| Table | Treatment-emergent adverse events by Preferred Term (Safety Population) |
| 14.3.2.2.2 | |
| Table | Number of Treatment-Emergent Adverse Events per Subject-year by System |
| 14.3.2.2.3 | Organ Class and Preferred Term (Safety Population) |
| Table 14.3.2.3 | Drug-Related Treatment-emergent adverse events by System Organ Class, |
| | Preferred Term and Severity (Safety Population) |
| Table 14.3.2.4 | Drug -Related Treatment-emergent adverse events by System Organ Class, |
| | Preferred Term and Relationship (Safety Population) |
| Table 14.3.2.5 | Drug-related Treatment-emergent adverse events by System Organ Class and |
| | Preferred Term (Safety Population) |
| Table 14.3.2.6 | Serious Treatment-emergent adverse events by System Organ Class and Preferred |
| | Term (Safety Population) |
| Table 14.3.2.7 | Listing of Serious Adverse Events |
| Table 14.3.2.8 | Listing of Adverse Events Leading to Death |
| Table 14.3.2.9 | Severe Treatment-emergent adverse events by System Organ Class and Preferred |
| | Term (Safety Population) |
| Table | Listing of Severe Treatment-Emergent Adverse Events |
| 14.3.2.10 | |
| Table | Treatment-emergent adverse events Leading to Study Drug Interruption by |
| 14.3.2.11 | System Organ Class and Preferred Term (Safety Population) |
| Table | Listing of Adverse Events Leading to Study Drug Interruption |
| 14.3.2.12 | |
| Table | Treatment-emergent adverse events Leading to Study Drug Discontinuation by |
| 14.3.2.13 | System Organ Class and Preferred Term (Safety Population) |
| Table | Listing of Adverse Events Leading to Study Drug Discontinuation |
| 14.3.2.14 | |
| Table | Treatment-emergent adverse events Leading to Dose Reduction by System Organ |
| 14.3.2.15 | Class and Preferred Term (Safety Population) |
| Table | Listing of Adverse Events Leading to Dose Reduction |
| 14.3.2.16 | Hart Community of the C |
| Table | Most Common Treatment-Emergent Adverse Events (Preferred Term Occurred in |
| 14.3.2.17 | >10% of Over Patients) by System Organ Class and Preferred Term (Safety |
| Tilli | Population) |
| Table | Listing of Most Common Treatment-Emergent Adverse Events |



| 14.3.2.18 | |
|---|---|
| Table | Time to first Onset of most Common Treatment-Emergent Adverse Events |
| 14.3.2.19 | (Preferred Term Occurred in >10% of Over Patients) (Safety Population) |
| Table 14.3.4.1 | Clinical Laboratory Results: PCS and PCSC Criteria |
| Table | Summary of Clinical Laboratory Results: Hematology (Safety Population) |
| 14.3.4.1.1.1 | carriery or extinour =azor atory research remaining (earlies) repaired only |
| Table | Summary of Clinical Laboratory Results: Hematology Abnormal Values (Safety |
| 14.3.4.1.1.2 | Population) |
| Table | Summary of Clinical Laboratory Results: Hematology Abnormal Values -Shift from |
| 14.3.4.1.1.3 | Baseline (Safety Population) |
| Table | Summary of Clinical Laboratory Results: Hematology PCS Values -Shift from |
| 14.3.4.1.1.4 | Baseline (Safety Population) |
| Table | Summary of Clinical Laboratory Results: Hematology PCSC Values -Shift from |
| 14.3.4.1.1.5 | Baseline (Safety Population) |
| Table | Clinical Laboratory Results - Hematology PCS and PCSC Values (Safety Population) |
| 14.3.4.1.1.6 | timeat Euboratory Results Trematotogy Fest and Feste Values (surety Fopulation) |
| Table | Summary of Clinical Laboratory Results: Chemistry (Safety Population) |
| 14.3.4.1.2.1 | Summary of eliment Euboratory Results. Chemistry (surety ropulation) |
| Table | Summary of Clinical Laboratory Results: Chemistry Abnormal Values (Safety |
| 14.3.4.1.2.2 | Population) |
| Table | Summary of Clinical Laboratory Results: Chemistry Abnormal Values -Shift from |
| 14.3.4.1.2.3 | Baseline (Safety Population) |
| Table | Summary of Clinical Laboratory Results: Chemistry PCS Values -Shift from |
| 14.3.4.1.2.4 | Baseline (Safety Population) |
| Table | Summary of Clinical Laboratory Results: Chemistry PCSC Values -Shift from |
| 14.3.4.1.2.5 | Baseline (Safety Population) |
| Table | Clinical Laboratory Results - Chemistry PCS and PCSC Values (Safety Population) |
| 14.3.4.1.2.6 | Stilled Edbordery Results Stillingtry Feb and Febr Falaes (surety Februarion) |
| Table 14.3.4.2 | Vital Signs: PCS and PCSC Criteria |
| Table | Summary of Vital Signs: Actual Values and Change from Baseline across Visits |
| 14.3.4.2.1 | (Safety Population) |
| Table | Summary of Vital Signs: Actual Values and Change from Pre-dose at TV1 (Safety |
| 14.3.4.2.2 | Population) |
| Table | Summary of Standard Vital Signs: PCS and PCSC Values by Visit (Safety |
| 14.3.4.2.3 | Population) |
| Table | Summary of Standard Vital Signs: PCS and PCSC Values by Scheduled Timepoint at |
| 14.3.4.2.4 | TV1 (Safety Population) |
| Table | Standard Vital Signs: PCS and PCSC Values |
| 14.3.4.2.5 | <b>3</b> |
| Table | Summary of Vital Signs: Orthostatic Hypotension by Visit (Safety Population) |
| 14.3.4.2.6 | and the second of the second o |
| Table | Summary of Vital Signs: Orthostatic Hypotension by Scheduled Timepoint at TV1 |
| 14.3.4.2.7 | (Safety Population) |
| Table | Orthostatic Vital Signs |
| 14.3.4.2.8 | |
| Table 14.3.4.3 | 12-Lead ECG:PCS and PCSC Criteria |
| 145(6 1 1.5. 1.5 | 12 2000 2001 00 010 1 000 0110010 |

| T-1-1- | Commence of 42 Lond ECC - Actual Values and Change agree Visite (Cofety |
|---|---|
| Table<br>14.3.4.3.1 | Summary of 12-Lead ECG: Actual Values and Change across Visits (Safety Population) |
| Table | Summary of 12-Lead ECG: PCS and PCSC Values (Safety Population) |
| 14.3.4.3.2 | Summary of 12-Lead Led. Les and Lese values (Safety Lopulation) |
| Table | 12-Lead Electrocardiogram (ECG): PCS and PCSC Values |
| 14.3.4.3.3 | 12 2000 2000 000 010 (200) FF 05 and F 050 values |
| Table 14.3.4.4 | Physical Examination (Safety Population) |
| Table | Summary of Spirometry(Pulmonary Function Facility): Actual Values and Change |
| 14.3.4.5.1.1 | from Baseline for FEV1 and FVC by Visit (Safety Population) |
| Table | Summary of Spirometry(Pulmonary Function Facility): Actual Values and Change |
| 14.3.4.5.1.2 | from Baseline for FEV1 and FVC by Visit Using Subset of Assessments Meeting the |
| | ATS Quality Criteria (Safety Population) |
| Table | Summary of Spirometry(Pulmonary Function Facility: Actual Values and Change |
| 14.3.4.5.1.3 | from Baseline for FEV1 and FVC by Visit Excluding Patients with Co-efficient of |
| | Variation (CV) of FEV1 >7.5% (Safety Population) |
| Table | MMRM Analysis of Spirometry Data (Pulmonary Function Facility): Change from |
| 14.3.4.5.1.4 | Baseline for FEV1 by Visit (Safety Population) |
| Table | MMRM Analysis of Spirometry Data (Pulmonary Function Facility): Change from |
| 14.3.4.5.1.5 | Baseline for FEV1 by Visit Using Subset of Assessments Meeting the ATS Quality |
| | Criteria (Safety Population) |
| Table | MMRM Analysis of Spirometry Data (Pulmonary Function Facility): Change from |
| 14.3.4.5.1.6 | Baseline for FEV1 by Visit Excluding Patients with Co-efficient of Variation (CV) |
| | of FEV1 >7.5% (Safety Population) |
| Table | Sensitivity Analysis Using MMRM: Change from Baseline for FEV1 by Visit MI |
| 14.3.4.5.1.7 | analysis with Missing At Random Assumption (Safety Population) |
| Table | Summary of Spirometry (Pulmonary Function Facility): Actual Values and Change |
| 14.3.4.5.1.8 | from Baseline for Calculated DLco Parameters by Visit (Safety Population) |
| Table | Summary of Spirometry (Pulmonary Function Facility): Actual Values and Change |
| 14.3.4.5.1.9 | from Baseline for Calculated DLco Parameters by Visit Using Subset of |
| | Assessments Meeting the ATS Quality Criteria (Safety Population) |
| Table | Summary of Spirometry (Pulmonary Function Facility): Actual Values and Change |
| 14.3.4.5.1.10 | from Baseline for Calculated DLco Parameters by Visit Excluding Patients with |
| | Co-efficient of Variation (CV) of FEV1 >7.5% (Safety Population) |
| Table | MMRM Analysis of Spirometry Data (Pulmonary Function Facility): Change from |
| 14.3.4.5.1.11 | Baseline for DLCO by Visit (Safety Population) |
| Table | MMRM Analysis of Spirometry Data (Pulmonary Function Facility): Change from |
| 14.3.4.5.1.12 | Baseline for DLCO by Visit Using Subset of Assessments Meeting the ATS Quality |
| | Criteria (Safety Population) |
| Table | MMRM Analysis of Spirometry Data (Pulmonary Function Facility): Change from |
| 14.3.4.5.1.13 | Baseline for DLCO by Visit Excluding Patients with Co-efficient of Variation (CV) |
| | of FEV1 >7.5% (Safety Population) |
| Table | Sensitivity Analysis Using MMRM: Change from Baseline for DLCO by Visit MI |
| 14.3.4.5.1.14 | analysis with Missing At Random Assumption (Safety Population) |
| Table | Summary of Spirometry (Pulmonary Function Facility): Categories of Change from |
| 14.3.4.5.1.15 | Baseline for FEV1 and FVC by Visit (Safety Population) |
| Table | Summary of Spirometry (Pulmonary Function Facility): Categories of Change from |

CVT-301-005 Final Version 2.0



| 14.3.4.5.1.16 | Baseline for DLCO by Visit (Safety Population) |
|---|---|
| Table | Summary of Spirometry (Pulmonary Function Facility): Actual Values and Change |
| 14.3.4.5.1.17 | |
| | from Baseline for FEV1 by Visit and by Smoker Status (Safety Population) |
| Table | Summary of Spirometry (Pulmonary Function Facility): Categories of Percent |
| 14.3.4.5.1.18 | Change from Baseline for FEV1 by Visit and Smoker Status (Safety Population) |
| Table | Summary of Spirometry: (Pulmonary Function Facility):): Actual Values and |
| 14.3.4.5.2.1 | Change from Baseline for FEV1/FVC by Visit (Safety Population) |
| Table | Summary of Spirometry: (Pulmonary Function Facility):): Actual Values and |
| 14.3.4.5.2.2 | Change from Baseline for FEV1/FVC by Visit Using Subset of Assessments Meeting |
| | the ATS Quality Criteria (Safety Population) |
| Table | Summary of Spirometry: (Pulmonary Function Facility):): Actual Values and |
| 14.3.4.5.2.3 | Change from Baseline for FEV1/FVC by Visit Excluding Patients with Co-efficient |
| | of Variation (CV) of FEV1 >7.5% (Safety Population) |
| Table | MMRM Analysis of Spirometry Data (Pulmonary Function Facility):): Change from |
| 14.3.4.5.2.4 | Baseline for FEV1/FVC by Visit (Safety Population) |
| Table | MMRM Analysis of Spirometry Data (Pulmonary Function Facility):): Change from |
| 14.3.4.5.2.5 | Baseline for FEV1/FVC by Visit Using Subset of Assessments Meeting the ATS |
| 14.3.4.3.2.3 | Quality Criteria (Safety Population) |
| Table | MMRM Analysis of Spirometry Data (Pulmonary Function Facility):): Change from |
| 14.3.4.5.2.6 | Baseline for FEV1/FVC by Visit Excluding Patients with Co-efficient of Variation |
| 14.3.4.3.2.0 | |
| T-LI- | (CV) of FEV1 >7.5% (Safety Population) |
| Table | Sensitivity Analysis Using MMRM: Change from Baseline for FEV1/FVC by Visit MI |
| 14.3.4.5.2.7 | analysis with Missing At Random Assumption (ITT Population) |
| Table | Summary of Spirometry(Pulmonary Function Facility): Categories of Change from |
| 14.3.4.5.2.8 | Baseline for FEV1/FVC by Visit (Safety Population) |
| Table | Summary of Spirometry (Pulmonary Function Facility): Summary of FEV1/FVC < |
| 14.3.4.5.3.1 | 60% and <70% by Visit (Safety Population) |
| Table | Summary of Spirometry (Pulmonary Function Facility): Summary of FEV1/FVC < |
| 14.3.4.5.3.2 | 60% and <70% by Visit Using Subset of Assessments Meeting the ATS Quality |
| | Criteria (Safety Population) |
| Table | Summary of Spirometry (Pulmonary Function Facility): Summary of FEV1/FVC < |
| 14.3.4.5.3.3 | 60% and <70% by Visit Excluding Patients with Co-efficient of Variation (CV) of |
| | FEV1 >7.5% (Safety Population) |
| Table | Spirometry(Pulmonary Function Facility): 70% or Smaller FEV1/FVC Values and |
| 14.3.4.5.4 | >=200 Reduction from Pre-dose |
| Table | Summary of Spirometry(Pulmonary Function Facility): Measurements Meeting ATS |
| 14.3.4.5.5 | Quality Criteria (Safety Population) |
| Table | Summary of Spirometry(Neurology Office): Actual Values and Change from |
| 14.3.4.5.6 | Baseline for FEV1 and FVC by Visit (Safety Population) |
| Table | Summary of Spirometry (Neurology Office): Actual Values and Change from |
| 14.3.4.5.7 | Baseline for FEV1/FVC by Visit (Safety Population) |
| Table | Summary of Spirometry (Neurology Office): Summary of FEV1/FVC < 60% and |
| 14.3.4.5.8 | <70%by Visit (Safety Population) |
| Table | Spirometry(Neurology Office):70% or Smaller FEV1/FVC Values by Visit |
| 14.3.4.5.9 | |
| Table | Summary of Spirometry(Neurology Office): Measurements Meeting ATS Quality |



| 14.3.4.5.10 | Criteria (Safety Population) |
|---|---|
| Table | Summary of Spirometry (Pulmonary Function Facility): Categories of Change from |
| 14.3.4.5.11 | Baseline for FEV1 and FVC by Visit (Safety Population |
| Table | Summary of Spirometry (Pulmonary Function Facility): Categories of Change from |
| 14.3.4.5.12 | Baseline for FEV1/FVC by Visit (Safety Population) |
| Table | Summary of Spirometry (Neurology Office): Actual Values and Change from |
| 14.3.4.5.13 | Baseline for FEV1 by Visit and by Smoker Status (Safety Population) |
| Table | Summary of Spirometry (Neurology Office): Categories of Percent Change from |
| 14.3.4.5.14 | Baseline for FEV1 by Visit and Smoker Status (Safety Population) |
| Table | Summary of Columbia-Suicide Severity Rating Scale (C-SSRS) (Safety Population) |
| 14.3.4.6.1 | |
| Table | Shift from Baseline in Columbia-Suicide Severity Rating Scale (C-SSRS) (Safety |
| 14.3.4.6.2 | Population) |
| Table 14.3.4.7 | Summary of Epworth Sleepiness Scale Total Score: Actual Values and Change |
| | from Baseline by Visit (Safety Population) |
| Table 14.3.4.8 | Summary of Questionnaire for Impulsive-Compulsive Disorders in Parkinson's |
| | (QUIP) by Visit (Safety Population) |
| Table | MMRM Analysis of UPDRS Part 4: Change from Baseline in the UPDRS Part 4 Score |
| 14.3.4.9.1 | at TV4 (Safety Population) |
| Table | MMRM Analysis of UPDRS Part 4 Dyskinesias Score: Change from Baseline in the |
| 14.3.4.9.2 | UPDRS Part 4 Score at TV4 (Safety Population) |
| Table | MMRM Analysis of UPDRS Part 4 Fluctuations Score: Change from Baseline in the |
| 14.3.4.9.3 | UPDRS Part 4 Score at TV4 (Safety Population) |
| Table | Summary of UPDRS Part 4: Actual Values and Change from Baseline by Visit |
| 14.3.4.9.4 | (Safety Population) |
| Table | Summary of UPDRS Part 4 Dyskinesias Score: Actual Values and Change from |
| 14.3.4.9.5 | Baseline by Visit (Safety Population) |
| Table | Summary of UPDRS Part 4 Fluctuations Score: Actual Values and Change from |
| 14.3.4.9.6 | Baseline by Visit (Safety Population) |
| Table | Dyskinesia: Occurrence and Severity (In-clinic) by Visit (ITT Population) |
| 14.3.4.10 | |



Statistical Analysis Plan

## 15. INDEX OF LISTINGS

| Listing 16.2.1 | Patient Disposition |
|---|---|
| Listing 16.2.2.1 | Protocol Deviations |
| Listing 16.2.3.1 | Inclusion Criteria not Met at Screening |
| Listing 16.2.3.2 | Exclusion Criteria Met at Screening |
| Listing 16.2.3.3 | Analysis Populations |
| Listing 16.2.4.1 | Demographics |
| Listing 16.2.4.2 | Medical History |
| Listing 16.2.4.3 | Parkinson's Disease History |
| Listing 16.2.4.4 | Smoking History |
| Listing 16.2.4.5 | ON and OFF Concordance Testing at Screening |
| Listing 16.2.4.6 | Modified Hoehn and Yahr Staging in "ON" State at Screening |
| Listing 16.2.4.7 | Mini Mental State Examination (MMSE) at Screening |
| Listing 16.2.4.8 | Parkinson's Disease Diary Data at Screening: Derived Time |
| Listing 16.2.4.9 | Screening ON/OFF Log |
| Listing 16.2.4.10 | Randomization |
| Listing 16.2.4.11.1 | Prior and Concomitant Medications |
| Listing 16.2.4.11.2 | Parkinson's disease Treatment Medications at Baseline |
| Listing 16.2.4.12 | Baseline Pulmonary Assessment Part 2 - Pulmonary History |
| Listing 16.2.4.13 | Baseline Pulmonary Assessment Part 3 - Assessments of Symptoms |
| Listing 16.2.5.1.1 | Study Drug Administration: in Clinic and at Home |
| Listing 16.2.5.1.2 | Study Drug Administration: Derived Variables (in Clinic) |
| Listing 16.2.5.1.3 | Study Drug Administration: Derived Variables (Overall) |
| Listing 16.2.5.1.4 | Study Drug Administration: Derived Variables (Overall by Visit) |
| Listing 16.2.5.1.5 | Listing of Study Drug Dose Change |
| Listing 16.2.5.2 | Study Drug Kit Dispensation |
| Listing 16.2.5.3 | Daily Levodopa Dose |
| Listing 16.2.6.1.1 | Unified Parkinson's Disease Rating Scale (UPDRS) Part 3 |
| Listing 16.2.6.1.2 | Unified Parkinson's Disease Rating Scale (UPDRS) Part 3: Derived |
| | Variables |
| Listing 16.2.6.2.1 | Clinic Assessment |
| Listing 16.2.6.2.2 | Parkinson's Disease Diary Data |
| Listing 16.2.6.2.3.1 | Parkinson's Disease Diary Data - Derived Variable by Dairy Date |
| Listing 16.2.6.2.3.2 | Parkinson's Disease Diary Data - Derived Variable by Visit |
| Listing 16.2.6.2.4 | Patient's Global Impression of Change (PGI-C) |
| Listing 16.2.6.2.5 | Impact of Parkinson's OFF Episodes |
| Listing 16.2.6.3.1 | Unified Parkinson's Disease Rating Scale (UPDRS) Part 2 |
| Listing 16.2.6.3.2 | Listing of S&E Activities of Daily Living |
| Listing 16.2.6.3.3 | 39 Item Parkinson's Disease Questionnaire (PDQ-39) |
| Listing 16.2.7.1 | Adverse Events |
| Listing 16.2.8.1.1 | Clinical Laboratory Results - Hematology |
| Listing 16.2.8.1.2 | Clinical Laboratory Results - Chemistry |
| Listing 16.2.8.1.3 | Serum Pregnancy Test - Positive Only |
| Listing 16.2.8.2.1 | Vital Signs |



| 14.0.0.0 | 101 151 ( 150) |
|---|---|
| Listing 16.2.8.2.2 | 12-Lead Electrocardiogram (ECG) |
| Listing 16.2.8.2.3 | Physical Examination |
| Listing 16.2.8.2.4.1 | Spirometry( Neurology Office) |
| Listing 16.2.8.2.4.2 | Spirometry( Neurology Office) Measurements Not Meeting ATS Quality |
| | Criteria |
| Listing 16.2.8.2.4.3 | Spirometry(Pulmonary Function Facility): DLCO Parameters |
| Listing 16.2.8.2.4.4 | Spirometry(Pulmonary Function Facility): Spirometry/DLCO Measurements |
| | Not Meeting ATS Quality Criteria |
| Listing 16.2.8.2.5.1 | Columbia-Suicide Severity Rating Scale (C-SSRS) |
| Listing 16.2.8.2.5.2 | Columbia-Suicide Severity Rating Scale (C-SSRS) - Subject Answered 'Yes' |
| | to any Questions |
| Listing 16.2.8.2.6 | Epworth Sleepiness Scale |
| Listing 16.2.8.2.7 | Questionnaire for Impulsive-Compulsive Disorders in Parkinson's (QUIP) |
| Listing 16.2.8.2.8.1 | Unified Parkinson's Disease Rating Scale (UPDRS) Part 4 |
| Listing 16.2.8.2.8.2 | Unified Parkinson's Disease Rating Scale (UPDRS) Part 4: Derived |
| | Variables |
| Listing 16.2.8.2.9 | Telephone Contact: Challenges with Inhaler or Capsules Data |

1003805

Acorda Therapeutics, Inc. CVT-301-005 Final Version 2.0



## Statistical Analysis Plan

## 16. INDEX OF FIGURES

Not Applicable.

## **Abuse Assessment Methodology and Adverse Event Terms**

A pre-NDA meeting was held with the Agency on 28 September 2016 (see FDA pre-NDA Meeting Minutes) to gain agreement on the adequacy of the nonclinical and clinical program and content and format and assessment of abuse potential for the 505(b)(2) NDA for CVT-301. In the CVT-301 Pre-NDA Meeting Package submitted to IND 115750 in Sequence 086 on 25 August 2016, Acorda provided a Draft Abuse Potential Assessment report and indicated that abuse related adverse event terms were assessed based on the terms published by Love and Sun (2013) for the completed clinical studies and for the clinical study reports and Integrated Summary of Safety for the ongoing clinical studies. In the CVT-301 pre-NDA Meeting minutes regarding question 4a, "Does the Division agree with the plan for assessment and reporting of abuse potential?" The Division indicated in the FDA Response to Question 4a, point 5, that the following AE terms were of particular interest:

- "5. Because abuse of levodopa is mainly known in the population of patients with PD, your Abuse Potential Assessment Report, in which you plan to include the analysis of published literature, should include the following items:
  - Populations: analysis should to be performed separately for PD patients and healthy subjects
  - For the PD study population, the following adverse events are of particular interest: abuse, misuse, withdrawal, dependence, dopamine dysregulation syndrome, hedonistic homeostatic dysregulation, euphoria, high, overdose, misuse, diversion, hoarding of medication, neuroleptic malignant syndrome, hyperpyrexia and confusion, rebound
- 6. Search and analysis of adverse events from your clinical data and the post-marketing data for levodopa formulations in publically available data bases should include and use the same search terms listed above in point 5."

In 2016 the International Society for Central Nervous System Clinical Trials and Methodology (ISCTM) recommended a list of 41 adverse event terms for assessment of abuse potential (Setnik 2016). Subsequent to the Pre-NDA meeting the FDA also issued a new Final Guidance, FDA Guidance for Industry: Assessment of Abuse Potential of Drugs (January 2017) that included 19 adverse event terms for assessment of abuse potential. Therefore, based on the FDA recommendations and more recent publications, Acorda has modified its methodology for assessment of abuse potential based on the list of 213 adverse event terms published by Love and Sun (2013). Instead, Acorda is using a shorter more focused composite list of 73 adverse event terms including the 15 terms recommended by FDA in the CVT-301 FDA pre-NDA Meeting Minutes (October 2016), the 19 terms from the new FDA Guidance for Industry: Assessment of Abuse Potential of Drugs (January 2017) and the 41 terms recommended by ISCTM (Setnik 2016). Note, two terms (euphoria and drug withdrawal) are repeated in two of the lists. All of these terms except hedonistic hemostatic dysregulation have been converted into MedDRA, Version 19.0 Preferred Terms (PT). Because there was no MedDRA conversion term for the verbatim term hedonistic hemostatic dysregulation it was included in the composite list of 73 MedDRA terms. The MedDRA PT may provide abuse-related information about a drug, and

were used for assessment of abuse related adverse events in the CVT-301 clinical studies and Integrated Summary of Safety. The verbatim adverse event terms and MedDRA PT are provided in Table 1.

# Table 1: Drug Adverse Event Terms for Abuse Potential Assessment of CVT-301 Safety Data

# 15 Adverse Event Terms From CVT-301 Pre-NDA Meeting Minutes, page 5, FDA Response to Question 4b, Item 5 (October 2016)

Abuse, misuse, withdrawal, dependence, dopamine dysregulation syndrome, hedonistic homeostatic dysregulation, euphoria, high, overdose, diversion, hoarding of medication, neuroleptic malignant syndrome, hyperpyrexia, confusion, rebound

# 19 Adverse Event Terms From FDA Guidance for Industry: Assessment of Abuse Potential of Drugs (January 2017)

Euphoric mood, elevated mood, feeling abnormal, feeling drunk, feeling of relaxation, dizziness, thinking abnormal, hallucination, inappropriate affect, somnolence, mood disorders and disturbances, psychosis, aggression, confusion, disorientation, drug tolerance, habituation, drug withdrawal syndrome, substance related disorders

# 41 Adverse Event Terms From Setnik, B. A Consensus List Proposal For Adverse Events Related To Abuse And Dependence Potential (Setnik 2016)

Abnormal behavior, abnormal thinking, agitation, cognition disorder, concentration impaired, concentration loss, confusion and disorientation, confusional state, delirium, delusional disorder unspecified type, detachment, disturbance in attention, elation inappropriate, elevated mood, emotional disorder, euphoria/euphoric mood, exhilaration inappropriate, feeling abnormal, feeling drunk, feeling happy inappropriately, flight of ideas, hallucination(visual and auditory), inappropriate affect, inappropriate, elation, inappropriate, laughter, inappropriate mood, elevation, irritability, memory impairment, mental disorder

#### MedDRA Preferred Terms based on the composite list of 73 Adverse Event Terms

Abnormal behavior, acute psychosis, aggression, agitation, cognitive disorder, confusional state, delirium, delirium tremens, delusional disorder unspecified type, delusional perception, dependence, disorientation, dissociation, disturbance in attention, dizziness, dopamine dysregulation syndrome, drug abuse, drug abuser, drug dependence, drug diversion, drug tolerance, drug withdrawal convulsions, drug withdrawal syndrome, elevated mood, emotional disorder, euphoric mood, feeling abnormal, feeling drunk, feeling of relaxation, flight of ideas, hallucination, hallucination auditory, hallucination gustatory, hallucination mixed, hallucination olfactory, hallucination synanesthetic, hallucination tactile, hallucination visual, hedonistic homeostatic dysregulation<sup>a</sup>, hyperpyrexia, inappropriate affect, intentional overdose, intentional product misuse, irritability, medication overuse headache, memory impairment, mental disorder, mental impairment, mood altered, mood swings, neuroleptic malignant syndrome, overdose, paranoia, parkinsonism hyperpyrexia syndrome, psychosis, psychotic disorder, reactive psychosis, rebound psychosis, rebound tachycardia, sedation, sensory disturbance, somnolence, stupor, substance abuse, substance abuse psychotic disorder, substance abuser, substance dependence, substance-induced mood disorder, substance-induced psychotic disorder, thinking abnormal, thought withdrawal, withdrawal hypertension, withdrawal syndrome

#### References

Acorda Therapeutics, Inc., CVT-301 Type B Pre-NDA FDA Meeting Minutes dated 27 October 2016.

FDA Guidance for Industry: Assessment of Abuse Potential of Drugs January 2017.

Setnik, B. A consensus list proposal for adverse events related to abuse and dependence potential, February 16, 2016, International society for CNS clinical trials and methodology (ISCTM) 12th Annual Scientific Meeting, The Fairmont, Washington, DC, February 16, 2016.

Love LA, Sun S. Proposed query to capture abuse-related adverse events. Paper presented at the annual meeting of the College on Problems of Drug Dependence. San Diego, CA: June 15-20, 2013.

There is no MedDRA PT for "hedonistic hemostatic dysregulation" listed in the pre-NDA Meeting Minutes, page 5, FDA Response to Question 4b, Item 5 (October 2016) and it was included in the list of MedDRA PT for completeness.